CLINICAL TRIAL: NCT03278067
Title: Post-authorisation Passive Enhanced Safety Surveillance of Seasonal Influenza Vaccines: Pilot Study in England 2017/18
Brief Title: Post-authorisation Passive Enhanced Safety Surveillance of Seasonal Influenza Vaccines: Pilot Study in England
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: 207781
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Influenza, Human
Keywords: England; Adverse Event of Interest; Seasonal influenza vaccines; Pilot study; Prospective passive enhanced safety surveillance
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — Not applicable (no sample)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vaccinated_Fluarix Tetra Group: Volunteered subjects who received GlaxoSmithKline's (GSK's) influenza vaccination (Fluarix Tetra) in 10 volunteer GP practices between 01 September and 30 November 2017.
  Interventions: Other: Enhanced vaccine safety surveillance
- Vaccinated_Non GSK Group: Volunteered subjects who received non-GSK influenza vaccination in 10 volunteer GP practices between 01 September and 30 November 2017.
  Interventions: Other: Enhanced vaccine safety surveillance
- Vaccinated_Unknown Group: Volunteered subjects who received influenza vaccination (GSK or non-GSK not known) in 10 volunteer GP practices between 01 September and 30 November 2017.
  Interventions: Other: Enhanced vaccine safety surveillance

INTERVENTIONS:
Other: Enhanced vaccine safety surveillance — Routinely collected primary care data from up to ten general practices to support passive surveillance. Additionally, this passive surveillance will be enhanced by the use of a customized card-based ADR reporting system.
  Other Names: Data collection

SUMMARY:
This pilot study, to be conducted in the 2017/2018 influenza season, is a safety surveillance study using passive surveillance enhanced with a reporting card system to report adverse events of interest (AEIs) after Flu vaccination.

DETAILED DESCRIPTION:
This is the third pilot study following, EPI-FLU-045 VS UK [NCT02567721] and EPI-FLU-046 VS UK [NCT02893878] studies, carried out in the 2 previous influenza seasons (2015/2016 and 2016/2017). This study will collect data about vaccination status and adverse events following influenza immunisation (AEFI) on a weekly basis, from 01 September 2017 onwards, using a customized Adverse Drug Reaction (ADR) Cards and data from Electronic Health Records system for a period of approximately 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who receive influenza vaccination among the 10 participating GP practices between 1 September and 30 November 2017 are eligible for inclusion in the analysis.

Exclusion Criteria:

* Registered patients who have explicitly opted out of data sharing will be excluded from the analysis.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Registered patients in up to 10 general practices in UK immunized against seasonal influenza at the beginning of 2017/18 season.
Sampling Method: Non-Probability Sample
Enrollment: 23939 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Surrey, United Kingdom

REFERENCES:
- [Derived] de Lusignan S, Damaso S, Ferreira F, Byford R, McGee C, Pathirannehelage S, Shende V, Yonova I, Schmidt A, Schuind A, Dos Santos G. Brand-specific enhanced safety surveillance of GSK's Fluarix Tetra seasonal influenza vaccine in England: 2017/2018 season. Hum Vaccin Immunother. 2020 Aug 2;16(8):1762-1771. doi: 10.1080/21645515.2019.1705112. Epub 2020 Mar 2. PMID 32118513

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One study General Practitioner (GP2) did not follow the procedure as per protocol in distributing, handling of the returned cards and the unused Adverse Drug Reaction (ADR) cards, therefore the data from that GP were excluded from the analysis.
Groups:
- Vaccinated_Unknown Brand Group: Volunteered subjects who received influenza vaccination (GSK or non-GSK brand not known) in 10 volunteer GP practices between 01 September and 30 November 2017
Period: Overall Study
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Started | 16433 | 3310 | 4196
Completed | 16433 | 3310 | 4196
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participant flow data were only collected for the overall group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group | Total
Number analyzed (Participants) | 16433 | 3310 | 4196 | 23939
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (16.3) | 23.6 (27.4) | 52.2 (28.0) | 57.67 (25.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9177 | 1696 | 2330 | 13203
  Male | 7256 | 1614 | 1866 | 10736
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 393 | 63 | 98 | 554
  Black | 84 | 26 | 17 | 127
  White | 11697 | 2121 | 2880 | 16698
  Mixed | 57 | 21 | 23 | 101
  Other | 25 | 3 | 15 | 43
  Missing | 4177 | 1076 | 1163 | 6416

OUTCOME MEASURES:

1. Primary Outcome: Weekly Incidence Rates of Any Adverse Events of Interest (AEIs) Reported Via Adverse Drug Reaction (ADR) Card, by Vaccine Group
Description: The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on the Weekly Vaccinated cohort which included all subjects who were vaccinated with a seasonal influenza vaccine during the week of interest and were registered in electronic health record (EHR), using card-based ADR reporting system during the safety follow-up (FU) period (from vaccination up to 7 days post-vaccination).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35: number analyzed (Participants) | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 1 | 1 | 3
  Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Week 37 | 10.10 [8.53 to 11.84] | 0.00 [0.00 to 70.76] | 12.50 [1.55 to 38.35]
  Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Week 38 | 7.69 [5.94 to 9.77] | 14.29 [0.00 to 90.97] | 12.50 [1.50 to 38.73]
  Week 39: number analyzed (Participants) | 16387 | 94 | 24
  Week 39 | 7.97 [7.16 to 8.84] | 0.00 [0.00 to 3.85] | 4.17 [0.11 to 21.12]
  Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Week 40 | 8.22 [4.92 to 12.73] | 4.75 [2.74 to 7.60] | 0.00 [0.00 to 11.22]
  Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Week 41 | 6.40 [4.45 to 8.86] | 3.25 [1.08 to 7.37] | 1.79 [0.05 to 9.55]
  Week 42: number analyzed (Participants) | 910 | 401 | 17
  Week 42 | 3.74 [1.74 to 6.93] | 1.25 [0.36 to 3.06] | 0.00 [0.00 to 19.51]
  Week 43: number analyzed (Participants) | 496 | 378 | 22
  Week 43 | 4.64 [1.86 to 9.38] | 2.65 [0.69 to 6.81] | 0.00 [0.00 to 15.44]
  Week 44: number analyzed (Participants) | 750 | 2946 | 30
  Week 44 | 4.40 [1.33 to 10.39] | 3.66 [0.70 to 10.72] | 0.00 [0.00 to 11.57]
  Week 45: number analyzed (Participants) | 453 | 402 | 546
  Week 45 | 3.75 [1.64 to 7.25] | 2.24 [0.20 to 8.71] | 1.92 [0.62 to 4.41]
  Week 46: number analyzed (Participants) | 350 | 264 | 19
  Week 46 | 4.29 [1.59 to 9.10] | 1.89 [0.08 to 9.13] | 0.00 [0.00 to 17.65]
  Week 47: number analyzed (Participants) | 258 | 157 | 41
  Week 47 | 1.55 [0.22 to 5.19] | 0.64 [0.02 to 3.50] | 0.00 [0.00 to 8.60]
  Week 48: number analyzed (Participants) | 145 | 100 | 10
  Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

2. Primary Outcome: Cumulative Incidence Rates of Any AEIs Reported Via ADR Card, by Vaccine Group
Description: The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on the Cumulative vaccinated cohort which included all subjects who were vaccinated with a seasonal influenza vaccine at any point from study start, up to end of the week of interest and were registered in EHR, using card-based ADR reporting system during the safety FU period (from vaccination up to 7 days post-vaccination).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Week 35-37 | 10.09 [8.52 to 11.84] | 0.00 [0.00 to 60.24] | 10.53 [1.30 to 33.14]
  Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Week 35-38 | 8.83 [7.25 to 10.63] | 9.09 [0.08 to 47.67] | 11.43 [3.20 to 26.74]
  Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Week 35-39 | 8.45 [7.37 to 9.64] | 0.95 [0.02 to 5.19] | 8.47 [2.81 to 18.68]
  Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Week 35-40 | 8.41 [7.29 to 9.63] | 3.85 [2.14 to 6.33] | 5.56 [1.83 to 12.49]
  Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Week 35-41 | 8.15 [7.00 to 9.43] | 3.59 [1.96 to 5.98] | 4.11 [1.52 to 8.73]
  Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Week 35-42 | 7.87 [6.68 to 9.19] | 2.79 [1.49 to 4.74] | 3.68 [1.36 to 7.84]
  Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Week 35-43 | 7.75 [6.54 to 9.12] | 2.76 [1.38 to 4.90] | 3.24 [1.20 to 6.93]
  Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Week 35-44 | 7.59 [6.36 to 8.97] | 2.97 [1.29 to 5.75] | 2.79 [1.03 to 5.97]
  Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Week 35-45 | 7.48 [6.25 to 8.86] | 2.85 [1.32 to 5.30] | 2.31 [1.16 to 4.10]
  Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Week 35-46 | 7.41 [6.13 to 8.86] | 2.75 [1.14 to 5.52] | 2.22 [1.11 to 3.94]
  Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Week 35-47 | 7.31 [6.03 to 8.78] | 2.64 [1.05 to 5.39] | 2.05 [1.03 to 3.64]
  Week 35-48 | 7.25 [5.95 to 8.73] | 2.55 [1.01 to 5.23] | 2.01 [1.01 to 3.58]

3. Primary Outcome: Weekly Incidence Rates of Fever/Pyrexia Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Fever/pyrexia = all subjects with a fever/pyrexia read code recorded were considered as having fever/pyrexia, regardless of what temperature had been recorded. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35: number analyzed (Participants) | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 1 | 1 | 3
  Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Week 37 | 0.45 [0.20 to 0.85] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Week 38 | 0.51 [0.15 to 1.26] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Week 39: number analyzed (Participants) | 16387 | 94 | 24
  Week 39 | 0.46 [0.20 to 0.92] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Week 40 | 0.34 [0.12 to 0.77] | 1.19 [0.09 to 4.96] | 0.00 [0.00 to 11.22]
  Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Week 41 | 0.36 [0.13 to 0.79] | 0.59 [0.07 to 2.12] | 0.00 [0.00 to 6.38]
  Week 42: number analyzed (Participants) | 910 | 401 | 17
  Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 19.51]
  Week 43: number analyzed (Participants) | 496 | 378 | 22
  Week 43 | 0.40 [0.05 to 1.47] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 15.44]
  Week 44: number analyzed (Participants) | 750 | 464 | 30
  Week 44 | 0.27 [0.02 to 1.20] | 0.43 [0.05 to 1.55] | 0.00 [0.00 to 11.57]
  Week 45: number analyzed (Participants) | 453 | 402 | 546
  Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.38 [0.01 to 2.12]
  Week 46: number analyzed (Participants) | 350 | 264 | 19
  Week 46 | 0.57 [0.03 to 2.58] | 0.00 [0.00 to 1.39] | 0.00 [0.00 to 17.65]
  Week 47: number analyzed (Participants) | 258 | 157 | 41
  Week 47 | 0.39 [0.00 to 2.82] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Week 48: number analyzed (Participants) | 145 | 100 | 10
  Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

4. Primary Outcome: Cumulative Incidence Rates of Fever/Pyrexia Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Fever/pyrexia = all subjects with a fever/pyrexia read code recorded were considered as having fever/pyrexia, regardless of what temperature had been recorded. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Week 35-37 | 0.45 [0.20 to 0.85] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Week 35-38 | 0.48 [0.26 to 0.80] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 10.00]
  Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Week 35-39 | 0.47 [0.24 to 0.83] | 0.00 [0.00 to 3.45] | 0.00 [0.00 to 6.06]
  Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Week 35-40 | 0.45 [0.25 to 0.73] | 0.90 [0.03 to 4.68] | 0.00 [0.00 to 4.02]
  Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Week 35-41 | 0.44 [0.27 to 0.68] | 0.77 [0.16 to 2.23] | 0.00 [0.00 to 2.49]
  Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Week 35-42 | 0.41 [0.24 to 0.65] | 0.51 [0.08 to 1.67] | 0.00 [0.00 to 2.24]
  Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Week 35-43 | 0.41 [0.24 to 0.64] | 0.38 [0.05 to 1.38] | 0.00 [0.00 to 1.97]
  Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Week 35-44 | 0.40 [0.24 to 0.63] | 0.40 [0.09 to 1.08] | 0.00 [0.00 to 1.70]
  Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Week 35-45 | 0.39 [0.23 to 0.62] | 0.33 [0.07 to 0.94] | 0.21 [0.01 to 1.16]
  Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Week 35-46 | 0.39 [0.23 to 0.64] | 0.30 [0.06 to 0.87] | 0.20 [0.01 to 1.12]
  Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Week 35-47 | 0.39 [0.23 to 0.63] | 0.28 [0.06 to 0.83] | 0.19 [0.00 to 1.04]
  Week 35-48 | 0.39 [0.23 to 0.62] | 0.27 [0.05 to 0.80] | 0.18 [0.00 to 1.02]

5. Primary Outcome: Weekly Incidence Rates of Local Symptoms Reported Via ADR Card, by Vaccine Group
Description: Local symptoms include local erythema. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35: number analyzed (Participants) | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 1 | 1 | 3
  Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Week 37 | 1.87 [0.78 to 3.72] | 0.00 [0.00 to 70.76] | 6.25 [0.16 to 30.23]
  Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Week 38 | 1.61 [0.84 to 2.79] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Week 39: number analyzed (Participants) | 16387 | 94 | 24
  Week 39 | 1.90 [1.23 to 2.79] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Week 40 | 1.95 [0.77 to 4.02] | 0.30 [0.00 to 1.82] | 0.00 [0.00 to 11.22]
  Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Week 41 | 1.45 [0.93 to 2.15] | 0.89 [0.15 to 2.82] | 0.00 [0.00 to 6.38]
  Week 42: number analyzed (Participants) | 910 | 401 | 17
  Week 42 | 0.55 [0.09 to 1.78] | 0.50 [0.06 to 1.79] | 0.00 [0.00 to 19.51]
  Week 43: number analyzed (Participants) | 496 | 378 | 22
  Week 43 | 0.40 [0.04 to 1.50] | 0.79 [0.06 to 3.28] | 0.00 [0.00 to 15.44]
  Week 44: number analyzed (Participants) | 750 | 2946 | 30
  Week 44 | 1.20 [0.25 to 3.43] | 0.65 [0.08 to 2.28] | 0.00 [0.00 to 11.57]
  Week 45: number analyzed (Participants) | 453 | 402 | 546
  Week 45 | 0.66 [0.05 to 2.76] | 0.50 [0.00 to 3.52] | 0.00 [0.00 to 1.40]
  Week 46: number analyzed (Participants) | 350 | 264 | 19
  Week 46 | 1.43 [0.20 to 4.82] | 1.14 [0.09 to 4.61] | 0.00 [0.00 to 17.65]
  Week 47: number analyzed (Participants) | 258 | 157 | 41
  Week 47 | 1.16 [0.06 to 5.45] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Week 48: number analyzed (Participants) | 145 | 100 | 10
  Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

6. Primary Outcome: Cumulative Incidence Rates of Local Symptoms Reported Via ADR Card, by Vaccine Group
Description: Local symptoms include local erythema. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Week 35-37 | 1.86 [0.78 to 3.72] | 0.00 [0.00 to 60.24] | 5.26 [0.13 to 26.03]
  Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Week 35-38 | 1.73 [0.99 to 2.81] | 0.00 [0.00 to 28.49] | 2.86 [0.07 to 14.92]
  Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Week 35-39 | 1.80 [1.14 to 2.71] | 0.00 [0.00 to 3.45] | 1.69 [0.02 to 10.67]
  Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Week 35-40 | 1.83 [1.17 to 2.71] | 0.23 [0.01 to 1.25] | 1.11 [0.02 to 6.81]
  Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Week 35-41 | 1.78 [1.20 to 2.54] | 0.51 [0.04 to 2.05] | 0.68 [0.01 to 4.24]
  Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Week 35-42 | 1.70 [1.19 to 2.36] | 0.51 [0.06 to 1.89] | 0.61 [0.01 to 3.64]
  Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Week 35-43 | 1.66 [1.17 to 2.28] | 0.58 [0.06 to 2.17] | 0.54 [0.01 to 3.14]
  Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Week 35-44 | 1.63 [1.17 to 2.21] | 0.59 [0.08 to 2.05] | 0.47 [0.01 to 2.73]
  Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Week 35-45 | 1.61 [1.16 to 2.17] | 0.58 [0.12 to 1.65] | 0.21 [0.00 to 1.82]
  Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Week 35-46 | 1.60 [1.17 to 2.14] | 0.63 [0.13 to 1.83] | 0.20 [0.00 to 1.74]
  Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Week 35-47 | 1.59 [1.17 to 2.12] | 0.60 [0.12 to 1.74] | 0.19 [0.00 to 1.59]
  Week 35-48 | 1.58 [1.16 to 2.10] | 0.58 [0.12 to 1.68] | 0.18 [0.00 to 1.57]

7. Primary Outcome: Weekly Incidence Rates of General Non-specific Symptoms Reported Via ADR Card, by Vaccine Group
Description: General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, headache, irritability, and malaise. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Any, Week 37 | 3.89 [3.16 to 4.74] | 0.00 [0.00 to 70.76] | 6.25 [0.03 to 39.17]
  Any, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Any, Week 38 | 2.97 [2.02 to 4.19] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Any, Week 39: number analyzed (Participants) | 4116 | 94 | 24
  Any, Week 39 | 2.94 [2.41 to 3.55] | 0.00 [0.00 to 3.85] | 4.17 [0.11 to 21.12]
  Any, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Any, Week 40 | 2.43 [1.76 to 3.27] | 1.48 [0.36 to 4.00] | 0.00 [0.00 to 11.22]
  Any, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Any, Week 41 | 1.75 [1.18 to 2.50] | 1.18 [0.19 to 3.76] | 0.00 [0.00 to 6.38]
  Any, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Any, Week 42 | 1.54 [0.53 to 3.43] | 0.25 [0.01 to 1.38] | 0.00 [0.00 to 19.51]
  Any, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Any, Week 43 | 1.81 [0.54 to 4.39] | 1.06 [0.08 to 4.36] | 0.00 [0.00 to 15.44]
  Any, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Any, Week 44 | 1.60 [0.67 to 3.18] | 1.29 [0.09 to 5.42] | 0.00 [0.00 to 11.57]
  Any, Week 45: number analyzed (Participants) | 453 | 402 | 261
  Any, Week 45 | 1.10 [0.19 to 3.43] | 1.00 [0.15 to 3.24] | 0.38 [0.01 to 2.12]
  Any, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Any, Week 46 | 0.57 [0.03 to 2.58] | 0.76 [0.01 to 5.22] | 0.00 [0.00 to 17.65]
  Any, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Any, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]
  Drowsiness, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Drowsiness, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Drowsiness, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Drowsiness, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Drowsiness, Week 37 | 1.05 [0.62 to 1.68] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Drowsiness, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Drowsiness, Week 38 | 0.81 [0.29 to 1.76] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Drowsiness, Week 39: number analyzed (Participants) | 4116 | 94 | 24
  Drowsiness, Week 39 | 0.63 [0.32 to 1.12] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Drowsiness, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Drowsiness, Week 40 | 0.68 [0.37 to 1.14] | 0.30 [0.01 to 1.64] | 0.00 [0.00 to 11.22]
  Drowsiness, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Drowsiness, Week 41 | 0.48 [0.20 to 0.98] | 0.59 [0.07 to 2.12] | 0.00 [0.00 to 6.38]
  Drowsiness, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Drowsiness, Week 42 | 0.33 [0.02 to 1.52] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 19.51]
  Drowsiness, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Drowsiness, Week 43 | 0.81 [0.01 to 5.29] | 0.26 [0.01 to 1.47] | 0.00 [0.00 to 15.44]
  Drowsiness, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Drowsiness, Week 44 | 0.27 [0.02 to 1.18] | 0.43 [0.01 to 2.52] | 0.00 [0.00 to 11.57]
  Drowsiness, Week 45: number analyzed (Participants) | 453 | 402 | 261
  Drowsiness, Week 45 | 0.22 [0.00 to 1.58] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.40]
  Drowsiness, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Drowsiness, Week 46 | 0.00 [0.00 to 1.05] | 0.38 [0.00 to 2.63] | 0.00 [0.00 to 17.65]
  Drowsiness, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Drowsiness, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Drowsiness, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Drowsiness, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]
  Fatigue, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Fatigue, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Fatigue, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Fatigue, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Fatigue, Week 37 | 2.11 [1.58 to 2.76] | 0.00 [0.00 to 70.76] | 6.25 [0.03 to 39.17]
  Fatigue, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Fatigue, Week 38 | 1.79 [1.16 to 2.65] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Fatigue, Week 39: number analyzed (Participants) | 4116 | 94 | 24
  Fatigue, Week 39 | 1.58 [1.22 to 2.01] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Fatigue, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Fatigue, Week 40 | 1.12 [0.54 to 2.05] | 0.59 [0.01 to 3.61] | 0.00 [0.00 to 11.22]
  Fatigue, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Fatigue, Week 41 | 1.09 [0.65 to 1.71] | 0.30 [0.01 to 1.64] | 0.00 [0.00 to 6.38]
  Fatigue, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Fatigue, Week 42 | 0.77 [0.08 to 2.92] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 19.51]
  Fatigue, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Fatigue, Week 43 | 0.81 [0.14 to 2.53] | 0.53 [0.04 to 2.19] | 0.00 [0.00 to 15.44]
  Fatigue, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Fatigue, Week 44 | 0.53 [0.15 to 1.36] | 0.65 [0.10 to 2.08] | 0.00 [0.00 to 11.57]
  Fatigue, Week 45: number analyzed (Participants) | 453 | 402 | 261
  Fatigue, Week 45 | 0.88 [0.15 to 2.77] | 0.50 [0.02 to 2.39] | 0.38 [0.01 to 2.12]
  Fatigue, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Fatigue, Week 46 | 0.57 [0.03 to 2.58] | 0.00 [0.00 to 1.39] | 0.00 [0.00 to 17.65]
  Fatigue, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Fatigue, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Fatigue, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Fatigue, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]
  Headache, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Headache, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Headache, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Headache, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Headache, Week 37 | 2.19 [1.65 to 2.85] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Headache, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Headache, Week 38 | 1.79 [0.90 to 3.18] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Headache, Week 39: number analyzed (Participants) | 4116 | 94 | 24
  Headache, Week 39 | 1.68 [1.22 to 2.25] | 0.00 [0.00 to 3.85] | 4.17 [0.11 to 21.12]
  Headache, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Headache, Week 40 | 1.41 [0.88 to 2.14] | 0.89 [0.06 to 3.80] | 0.00 [0.00 to 11.22]
  Headache, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Headache, Week 41 | 0.91 [0.51 to 1.49] | 0.89 [0.15 to 2.82] | 0.00 [0.00 to 6.38]
  Headache, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Headache, Week 42 | 0.77 [0.24 to 1.82] | 0.25 [0.01 to 1.38] | 0.00 [0.00 to 19.51]
  Headache, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Headache, Week 43 | 1.21 [0.27 to 3.36] | 0.79 [0.06 to 3.28] | 0.00 [0.00 to 15.44]
  Headache, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Headache, Week 44 | 1.33 [0.52 to 2.78] | 0.65 [0.10 to 2.08] | 0.00 [0.00 to 11.57]
  Headache, Week 45: number analyzed (Participants) | 453 | 402 | 261
  Headache, Week 45 | 0.88 [0.07 to 3.62] | 0.75 [0.07 to 2.91] | 0.38 [0.01 to 2.12]
  Headache, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Headache, Week 46 | 0.29 [0.00 to 2.15] | 0.38 [0.00 to 2.63] | 0.00 [0.00 to 17.65]
  Headache, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Headache, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Headache, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Headache, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]
  Irritability, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Irritability, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Irritability, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Irritability, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Irritability, Week 37 | 0.36 [0.14 to 0.76] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Irritability, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Irritability, Week 38 | 0.26 [0.09 to 0.56] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Irritability, Week 39: number analyzed (Participants) | 4116 | 94 | 24
  Irritability, Week 39 | 0.34 [0.12 to 0.76] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Irritability, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Irritability, Week 40 | 0.15 [0.03 to 0.43] | 0.00 [0.00 to 1.09] | 0.00 [0.00 to 11.22]
  Irritability, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Irritability, Week 41 | 0.12 [0.01 to 0.44] | 0.00 [0.00 to 1.09] | 0.00 [0.00 to 6.38]
  Irritability, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Irritability, Week 42 | 0.11 [0.00 to 0.80] | 0.25 [0.01 to 1.38] | 0.00 [0.00 to 19.51]
  Irritability, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Irritability, Week 43 | 0.20 [0.00 to 1.34] | 0.26 [0.01 to 1.47] | 0.00 [0.00 to 15.44]
  Irritability, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Irritability, Week 44 | 0.00 [0.00 to 0.49] | 0.43 [0.01 to 2.52] | 0.00 [0.00 to 11.57]
  Irritability, Week 45: number analyzed (Participants) | 453 | 402 | 261
  Irritability, Week 45 | 0.22 [0.00 to 1.58] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.40]
  Irritability, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Irritability, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 1.39] | 0.00 [0.00 to 17.65]
  Irritability, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Irritability, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Irritability, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Irritability, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]
  Malaise, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Malaise, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Malaise, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Malaise, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Malaise, Week 37 | 0.04 [0.00 to 0.25] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Malaise, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Malaise, Week 38 | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Malaise, Week 39: number analyzed (Participants) | 4116 | 94 | 24
  Malaise, Week 39 | 0.00 [0.00 to 0.09] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Malaise, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Malaise, Week 40 | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 1.09] | 0.00 [0.00 to 11.22]
  Malaise, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Malaise, Week 41 | 0.00 [0.00 to 0.22] | 0.00 [0.00 to 1.09] | 0.00 [0.00 to 6.38]
  Malaise, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Malaise, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 19.51]
  Malaise, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Malaise, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 15.44]
  Malaise, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Malaise, Week 44 | 0.00 [0.00 to 0.49] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 11.57]
  Malaise, Week 45: number analyzed (Participants) | 453 | 402 | 261
  Malaise, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.40]
  Malaise, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Malaise, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 1.39] | 0.00 [0.00 to 17.65]
  Malaise, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Malaise, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Malaise, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Malaise, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

8. Primary Outcome: Cumulative Incidence Rates of General Non-specific Symptoms Reported Via ADR Card, by Vaccine Group
Description: General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, headache, irritability, and malaise. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Any, Week 35-37 | 3.89 [3.15 to 4.74] | 0.00 [0.00 to 60.24] | 5.26 [0.06 to 29.55]
  Any, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Any, Week 35-38 | 3.41 [2.58 to 4.40] | 0.00 [0.00 to 28.49] | 2.86 [0.02 to 18.52]
  Any, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Any, Week 35-39 | 3.20 [2.47 to 4.07] | 0.00 [0.00 to 3.45] | 3.39 [0.41 to 11.71]
  Any, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Any, Week 35-40 | 3.06 [2.39 to 3.85] | 1.13 [0.37 to 2.62] | 2.22 [0.27 to 7.80]
  Any, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Any, Week 35-41 | 2.89 [2.24 to 3.67] | 1.15 [0.34 to 2.80] | 1.37 [0.17 to 4.86]
  Any, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Any, Week 35-42 | 2.81 [2.14 to 3.60] | 0.85 [0.27 to 2.00] | 1.23 [0.15 to 4.36]
  Any, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Any, Week 35-43 | 2.77 [2.10 to 3.59] | 0.90 [0.21 to 2.44] | 1.08 [0.13 to 3.85]
  Any, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Any, Week 35-44 | 2.71 [2.04 to 3.54] | 0.99 [0.19 to 2.96] | 0.93 [0.11 to 3.32]
  Any, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Any, Week 35-45 | 2.67 [2.00 to 3.47] | 0.99 [0.27 to 2.50] | 0.63 [0.13 to 1.83]
  Any, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Any, Week 35-46 | 2.62 [1.95 to 3.45] | 0.97 [0.22 to 2.68] | 0.61 [0.13 to 1.76]
  Any, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Any, Week 35-47 | 2.58 [1.91 to 3.41] | 0.91 [0.20 to 2.56] | 0.56 [0.12 to 1.63]
  Any, Week 35-48 | 2.56 [1.89 to 3.38] | 0.88 [0.20 to 2.48] | 0.55 [0.11 to 1.60]
  Drowsiness, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Drowsiness, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Drowsiness, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Drowsiness, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Drowsiness, Week 35-37 | 1.05 [0.62 to 1.68] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Drowsiness, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Drowsiness, Week 35-38 | 0.92 [0.49 to 1.59] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 10.00]
  Drowsiness, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Drowsiness, Week 35-39 | 0.79 [0.42 to 1.36] | 0.00 [0.00 to 3.45] | 0.00 [0.00 to 6.06]
  Drowsiness, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Drowsiness, Week 35-40 | 0.77 [0.43 to 1.28] | 0.23 [0.01 to 1.25] | 0.00 [0.00 to 4.02]
  Drowsiness, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Drowsiness, Week 35-41 | 0.74 [0.41 to 1.23] | 0.38 [0.08 to 1.12] | 0.00 [0.00 to 2.49]
  Drowsiness, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Drowsiness, Week 35-42 | 0.71 [0.38 to 1.21] | 0.25 [0.05 to 0.74] | 0.00 [0.00 to 2.24]
  Drowsiness, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Drowsiness, Week 35-43 | 0.71 [0.36 to 1.26] | 0.26 [0.07 to 0.66] | 0.00 [0.00 to 1.97]
  Drowsiness, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Drowsiness, Week 35-44 | 0.69 [0.34 to 1.24] | 0.30 [0.06 to 0.89] | 0.00 [0.00 to 1.70]
  Drowsiness, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Drowsiness, Week 35-45 | 0.68 [0.34 to 1.21] | 0.25 [0.04 to 0.78] | 0.00 [0.00 to 0.77]
  Drowsiness, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Drowsiness, Week 35-46 | 0.66 [0.33 to 1.19] | 0.26 [0.04 to 0.90] | 0.00 [0.00 to 0.74]
  Drowsiness, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Drowsiness, Week 35-47 | 0.65 [0.32 to 1.17] | 0.25 [0.03 to 0.86] | 0.00 [0.00 to 0.69]
  Drowsiness, Week 35-48 | 0.65 [0.32 to 1.16] | 0.24 [0.03 to 0.83] | 0.00 [0.00 to 0.67]
  Fatigue, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Fatigue, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Fatigue, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Fatigue, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Fatigue, Week 35-37 | 2.11 [1.58 to 2.76] | 0.00 [0.00 to 60.24] | 5.26 [0.06 to 29.55]
  Fatigue, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Fatigue, Week 35-38 | 1.94 [1.46 to 2.54] | 0.00 [0.00 to 28.49] | 2.86 [0.02 to 18.52]
  Fatigue, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Fatigue, Week 35-39 | 1.78 [1.37 to 2.28] | 0.00 [0.00 to 3.45] | 1.69 [0.01 to 12.12]
  Fatigue, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Fatigue, Week 35-40 | 1.66 [1.27 to 2.13] | 0.45 [0.01 to 2.35] | 1.11 [0.01 to 7.73]
  Fatigue, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Fatigue, Week 35-41 | 1.59 [1.20 to 2.06] | 0.38 [0.03 to 1.54] | 0.68 [0.02 to 3.76]
  Fatigue, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Fatigue, Week 35-42 | 1.54 [1.14 to 2.02] | 0.25 [0.03 to 0.95] | 0.61 [0.02 to 3.37]
  Fatigue, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Fatigue, Week 35-43 | 1.51 [1.13 to 1.98] | 0.32 [0.03 to 1.21] | 0.54 [0.01 to 2.97]
  Fatigue, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Fatigue, Week 35-44 | 1.46 [1.09 to 1.92] | 0.40 [0.06 to 1.30] | 0.47 [0.01 to 2.56]
  Fatigue, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Fatigue, Week 35-45 | 1.45 [1.09 to 1.88] | 0.41 [0.14 to 0.95] | 0.42 [0.05 to 1.51]
  Fatigue, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Fatigue, Week 35-46 | 1.43 [1.05 to 1.89] | 0.37 [0.11 to 0.91] | 0.40 [0.05 to 1.45]
  Fatigue, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Fatigue, Week 35-47 | 1.40 [1.03 to 1.86] | 0.35 [0.10 to 0.87] | 0.37 [0.05 to 1.34]
  Fatigue, Week 35-48 | 1.39 [1.02 to 1.85] | 0.34 [0.10 to 0.84] | 0.37 [0.04 to 1.32]
  Headache, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Headache, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Headache, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Headache, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Headache, Week 35-37 | 2.19 [1.64 to 2.85] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Headache, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Headache, Week 35-38 | 1.98 [1.25 to 2.97] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 10.00]
  Headache, Week 35-39: number analyzed (Participants) | 9313 | 105 | 1
  Headache, Week 35-39 | 1.85 [1.24 to 2.64] | 0.00 [0.00 to 3.45] | 1.69 [0.04 to 9.09]
  Headache, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Headache, Week 35-40 | 1.77 [1.24 to 2.44] | 0.68 [0.08 to 2.44] | 1.11 [0.03 to 6.04]
  Headache, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Headache, Week 35-41 | 1.66 [1.16 to 2.29] | 0.77 [0.14 to 2.32] | 0.68 [0.01 to 4.40]
  Headache, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Headache, Week 35-42 | 1.60 [1.12 to 2.21] | 0.59 [0.13 to 1.69] | 0.61 [0.01 to 4.02]
  Headache, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Headache, Week 35-43 | 1.59 [1.11 to 2.20] | 0.64 [0.12 to 1.95] | 0.54 [0.00 to 3.67]
  Headache, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Headache, Week 35-44 | 1.57 [1.10 to 2.19] | 0.64 [0.12 to 1.93] | 0.47 [0.00 to 3.34]
  Headache, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Headache, Week 35-45 | 1.55 [1.09 to 2.15] | 0.66 [0.17 to 1.73] | 0.42 [0.05 to 1.51]
  Headache, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Headache, Week 35-46 | 1.53 [1.06 to 2.12] | 0.63 [0.14 to 1.78] | 0.40 [0.05 to 1.45]
  Headache, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Headache, Week 35-47 | 1.50 [1.04 to 2.09] | 0.60 [0.13 to 1.70] | 0.37 [0.05 to 1.34]
  Headache, Week 35-48 | 1.49 [1.03 to 2.08] | 0.58 [0.13 to 1.64] | 0.37 [0.04 to 1.32]
  Irritability, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Irritability, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Irritability, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Irritability, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Irritability, Week 35-37 | 0.36 [0.14 to 0.76] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Irritability, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Irritability, Week 35-38 | 0.31 [0.14 to 0.60] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 10.00]
  Irritability, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Irritability, Week 35-39 | 0.32 [0.17 to 0.56] | 0.00 [0.00 to 3.45] | 0.00 [0.00 to 6.06]
  Irritability, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Irritability, Week 35-40 | 0.29 [0.16 to 0.47] | 0.00 [0.00 to 0.83] | 0.00 [0.00 to 4.02]
  Irritability, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Irritability, Week 35-41 | 0.27 [0.15 to 0.45] | 0.00 [0.00 to 0.47] | 0.00 [0.00 to 2.49]
  Irritability, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Irritability, Week 35-42 | 0.26 [0.14 to 0.45] | 0.08 [0.00 to 0.47] | 0.00 [0.00 to 2.24]
  Irritability, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Irritability, Week 35-43 | 0.26 [0.13 to 0.46] | 0.13 [0.01 to 0.48] | 0.00 [0.00 to 1.97]
  Irritability, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Irritability, Week 35-44 | 0.24 [0.12 to 0.44] | 0.20 [0.02 to 0.82] | 0.00 [0.00 to 1.70]
  Irritability, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Irritability, Week 35-45 | 0.24 [0.13 to 0.42] | 0.16 [0.01 to 0.71] | 0.00 [0.00 to 0.77]
  Irritability, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Irritability, Week 35-46 | 0.24 [0.12 to 0.42] | 0.15 [0.01 to 0.67] | 0.00 [0.00 to 0.74]
  Irritability, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Irritability, Week 35-47 | 0.23 [0.12 to 0.41] | 0.14 [0.01 to 0.64] | 0.00 [0.00 to 0.69]
  Irritability, Week 35-48 | 0.23 [0.12 to 0.41] | 0.14 [0.01 to 0.62] | 0.00 [0.00 to 0.67]
  Malaise, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Malaise, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Malaise, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Malaise, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Malaise, Week 35-37 | 0.04 [0.00 to 0.25] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Malaise, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Malaise, Week 35-38 | 0.02 [0.00 to 0.12] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 10.00]
  Malaise, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Malaise, Week 35-39 | 0.01 [0.00 to 0.07] | 0.00 [0.00 to 3.45] | 0.00 [0.00 to 6.06]
  Malaise, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Malaise, Week 35-40 | 0.01 [0.00 to 0.06] | 0.00 [0.00 to 0.83] | 0.00 [0.00 to 4.02]
  Malaise, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Malaise, Week 35-41 | 0.01 [0.00 to 0.05] | 0.00 [0.00 to 0.47] | 0.00 [0.00 to 2.49]
  Malaise, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Malaise, Week 35-42 | 0.01 [0.00 to 0.05] | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 2.24]
  Malaise, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Malaise, Week 35-43 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.24] | 0.00 [0.00 to 1.97]
  Malaise, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Malaise, Week 35-44 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 1.70]
  Malaise, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Malaise, Week 35-45 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 0.77]
  Malaise, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Malaise, Week 35-46 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 0.74]
  Malaise, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Malaise, Week 35-47 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 0.69]
  Malaise, Week 35-48 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 0.67]

9. Primary Outcome: Weekly Incidence Rates of Respiratory/Miscellaneous Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Respiratory/miscellaneous adverse events include any respiratory/miscellaneous adverse events, conjunctivitis, coryza, cough, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhoea and wheezing. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Any, Week 37 | 5.76 [4.81 to 6.83] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Any, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Any, Week 38 | 3.88 [2.99 to 4.95] | 14.29 [0.00 to 90.97] | 6.25 [0.16 to 30.23]
  Any, Week 39: number analyzed (Participants) | 16387 | 94 | 24
  Any, Week 39 | 4.23 [3.63 to 4.89] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Any, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Any, Week 40 | 4.57 [2.77 to 7.05] | 2.67 [0.48 to 8.06] | 0.00 [0.00 to 11.22]
  Any, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Any, Week 41 | 3.32 [2.19 to 4.81] | 2.07 [0.75 to 4.49] | 0.00 [0.00 to 6.38]
  Any, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Any, Week 42 | 2.09 [0.95 to 3.94] | 0.50 [0.06 to 1.79] | 0.00 [0.00 to 19.51]
  Any, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Any, Week 43 | 2.62 [0.83 to 6.10] | 1.85 [0.66 to 4.07] | 0.00 [0.00 to 15.44]
  Any, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Any, Week 44 | 2.40 [0.64 to 6.09] | 2.16 [0.63 to 5.25] | 0.00 [0.00 to 11.57]
  Any, Week 45: number analyzed (Participants) | 453 | 402 | 261
  Any, Week 45 | 1.77 [0.54 to 4.23] | 1.00 [0.01 to 6.97] | 1.92 [0.62 to 4.41]
  Any, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Any, Week 46 | 1.43 [0.41 to 3.52] | 1.14 [0.01 to 7.76] | 0.00 [0.00 to 17.65]
  Any, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Any, Week 47 | 1.55 [0.22 to 5.19] | 0.64 [0.02 to 3.50] | 0.00 [0.00 to 8.60]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

10. Primary Outcome: Cumulative Incidence Rates of Respiratory/Miscellaneous Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Respiratory/miscellaneous adverse events include any respiratory/miscellaneous adverse events, conjunctivitis, coryza, cough, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhoea and wheezing. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Any, Week 35-37 | 5.76 [4.81 to 6.83] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Any, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Any, Week 35-38 | 4.77 [3.99 to 5.65] | 9.09 [0.08 to 47.67] | 2.86 [0.05 to 16.10]
  Any, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Any, Week 35-39 | 4.53 [3.96 to 5.16] | 0.95 [0.02 to 5.19] | 1.69 [0.04 to 9.09]
  Any, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Any, Week 35-40 | 4.54 [3.88 to 5.27] | 2.26 [0.44 to 6.66] | 1.11 [0.03 to 6.04]
  Any, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Any, Week 35-41 | 4.38 [3.71 to 5.14] | 2.18 [0.80 to 4.71] | 0.68 [0.01 to 4.40]
  Any, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Any, Week 35-42 | 4.23 [3.53 to 5.03] | 1.61 [0.58 to 3.50] | 0.61 [0.01 to 4.02]
  Any, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Any, Week 35-43 | 4.18 [3.44 to 5.02] | 1.67 [0.84 to 2.95] | 0.54 [0.00 to 3.67]
  Any, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Any, Week 35-44 | 4.09 [3.35 to 4.94] | 1.78 [0.96 to 2.99] | 0.47 [0.00 to 3.34]
  Any, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Any, Week 35-45 | 4.02 [3.28 to 4.88] | 1.65 [0.83 to 2.91] | 1.26 [0.46 to 2.72]
  Any, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Any, Week 35-46 | 3.97 [3.19 to 4.86] | 1.60 [0.80 to 2.85] | 1.21 [0.45 to 2.62]
  Any, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Any, Week 35-47 | 3.93 [3.16 to 4.82] | 1.55 [0.77 to 2.77] | 1.12 [0.41 to 2.42]
  Any, Week 35-48 | 3.89 [3.12 to 4.79] | 1.49 [0.73 to 2.69] | 1.10 [0.40 to 2.38]

11. Primary Outcome: Weekly Incidence Rates of Gastrointestinal Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhea, nausea, and vomiting. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Any, Week 37 | 2.03 [1.29 to 3.03] | 0.00 [0.00 to 70.76] | 6.25 [0.03 to 39.17]
  Any, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Any, Week 38 | 1.65 [0.95 to 2.65] | 14.29 [0.00 to 90.97] | 0.00 [0.00 to 20.59]
  Any, Week 39: number analyzed (Participants) | 16387 | 94 | 24
  Any, Week 39 | 1.34 [0.81 to 2.08] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Any, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Any, Week 40 | 1.36 [0.80 to 2.16] | 1.19 [0.32 to 3.01] | 0.00 [0.00 to 11.22]
  Any, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Any, Week 41 | 1.15 [0.62 to 1.94] | 0.59 [0.07 to 2.12] | 0.00 [0.00 to 6.38]
  Any, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Any, Week 42 | 0.66 [0.19 to 1.63] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 19.51]
  Any, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Any, Week 43 | 0.40 [0.04 to 1.61] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 15.44]
  Any, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Any, Week 44 | 0.40 [0.08 to 1.16] | 0.43 [0.01 to 2.52] | 0.00 [0.00 to 11.57]
  Any, Week 45: number analyzed (Participants) | 453 | 402 | 261
  Any, Week 45 | 1.32 [0.22 to 4.18] | 1.00 [0.15 to 3.24] | 0.38 [0.01 to 2.12]
  Any, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Any, Week 46 | 0.86 [0.06 to 3.72] | 0.00 [0.00 to 1.39] | 0.00 [0.00 to 17.65]
  Any, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Any, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

12. Primary Outcome: Cumulative Incidence Rates of Gastrointestinal Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhea, nausea and, vomiting. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Any, Week 35-37 | 2.03 [1.29 to 3.03] | 0.00 [0.00 to 60.24] | 5.26 [0.06 to 29.55]
  Any, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Any, Week 35-38 | 1.83 [1.33 to 2.44] | 9.09 [0.08 to 47.67] | 2.86 [0.02 to 18.52]
  Any, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Any, Week 35-39 | 1.61 [1.11 to 2.26] | 0.95 [0.02 to 5.19] | 1.69 [0.01 to 12.12]
  Any, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Any, Week 35-40 | 1.57 [1.15 to 2.07] | 1.13 [0.37 to 2.62] | 1.11 [0.01 to 7.73]
  Any, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Any, Week 35-41 | 1.51 [1.12 to 1.99] | 0.90 [0.35 to 1.87] | 0.68 [0.02 to 3.76]
  Any, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Any, Week 35-42 | 1.46 [1.09 to 1.91] | 0.59 [0.24 to 1.23] | 0.61 [0.02 to 3.37]
  Any, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Any, Week 35-43 | 1.42 [1.05 to 1.88] | 0.45 [0.16 to 1.01] | 0.54 [0.01 to 2.97]
  Any, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Any, Week 35-44 | 1.37 [1.01 to 1.81] | 0.44 [0.10 to 1.22] | 0.47 [0.01 to 2.56]
  Any, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Any, Week 35-45 | 1.37 [1.03 to 1.78] | 0.54 [0.21 to 1.12] | 0.42 [0.05 to 1.51]
  Any, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Any, Week 35-46 | 1.36 [1.02 to 1.76] | 0.48 [0.17 to 1.07] | 0.40 [0.05 to 1.45]
  Any, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Any, Week 35-47 | 1.34 [1.00 to 1.74] | 0.46 [0.16 to 1.03] | 0.37 [0.05 to 1.34]
  Any, Week 35-48 | 1.32 [0.99 to 1.73] | 0.44 [0.15 to 1.00] | 0.37 [0.04 to 1.32]

13. Primary Outcome: Weekly Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial edema, and hypersensitivity reactions. The weekly incidence rates expressed as the percentage of subjects, of AEIs were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Any, Week 37 | 0.65 [0.01 to 4.33] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Any, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Any, Week 38 | 0.55 [0.07 to 1.92] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Any, Week 39: number analyzed (Participants) | 16387 | 94 | 24
  Any, Week 39 | 0.36 [0.03 to 1.54] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Any, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Any, Week 40 | 0.39 [0.06 to 1.28] | 0.59 [0.01 to 3.61] | 0.00 [0.00 to 11.22]
  Any, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Any, Week 41 | 0.24 [0.05 to 0.70] | 0.59 [0.07 to 2.12] | 0.00 [0.00 to 6.38]
  Any, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Any, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 19.51]
  Any, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Any, Week 43 | 0.20 [0.00 to 1.37] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 15.44]
  Any, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Any, Week 44 | 0.27 [0.02 to 1.20] | 0.65 [0.01 to 3.77] | 0.00 [0.00 to 11.57]
  Any, Week 45: number analyzed (Participants) | 453 | 402 | 261
  Any, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.38 [0.01 to 2.12]
  Any, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Any, Week 46 | 0.29 [0.00 to 2.10] | 0.00 [0.00 to 1.39] | 0.00 [0.00 to 17.65]
  Any, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Any, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

14. Primary Outcome: Cumulative Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial edema, and hypersensitivity reactions. The cumulative incidence rates expressed as the percentage of subjects, of AEIs were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Any, Week 35-37 | 0.65 [0.01 to 4.33] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Any, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Any, Week 35-38 | 0.60 [0.03 to 2.83] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 10.00]
  Any, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Any, Week 35-39 | 0.49 [0.03 to 2.23] | 0.00 [0.00 to 3.45] | 0.00 [0.00 to 6.06]
  Any, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Any, Week 35-40 | 0.48 [0.03 to 2.05] | 0.45 [0.01 to 2.35] | 0.00 [0.00 to 4.02]
  Any, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Any, Week 35-41 | 0.45 [0.04 to 1.81] | 0.51 [0.04 to 2.05] | 0.00 [0.00 to 2.49]
  Any, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Any, Week 35-42 | 0.42 [0.03 to 1.73] | 0.34 [0.04 to 1.26] | 0.00 [0.00 to 2.24]
  Any, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Any, Week 35-43 | 0.41 [0.03 to 1.67] | 0.26 [0.03 to 0.97] | 0.00 [0.00 to 1.97]
  Any, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Any, Week 35-44 | 0.40 [0.04 to 1.58] | 0.35 [0.03 to 1.43] | 0.00 [0.00 to 1.70]
  Any, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Any, Week 35-45 | 0.39 [0.04 to 1.54] | 0.29 [0.02 to 1.24] | 0.21 [0.01 to 1.16]
  Any, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Any, Week 35-46 | 0.39 [0.03 to 1.55] | 0.26 [0.02 to 1.17] | 0.20 [0.01 to 1.12]
  Any, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Any, Week 35-47 | 0.38 [0.03 to 1.53] | 0.25 [0.01 to 1.11] | 0.19 [0.00 to 1.04]
  Any, Week 35-48 | 0.38 [0.03 to 1.51] | 0.24 [0.01 to 1.08] | 0.18 [0.00 to 1.02]

15. Primary Outcome: Weekly Incidence Rates of Rash Adverse Events Reported Via ADR Card, by Vaccine Group
Description: The weekly incidence rates expressed as the percentage of subjects, of AEIs were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35: number analyzed (Participants) | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 1 | 1 | 3
  Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Week 37 | 0.53 [0.23 to 1.04] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Week 38 | 0.29 [0.10 to 0.67] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Week 39: number analyzed (Participants) | 16387 | 94 | 24
  Week 39 | 0.19 [0.08 to 0.38] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Week 40 | 0.44 [0.20 to 0.83] | 0.00 [0.00 to 1.09] | 0.00 [0.00 to 11.22]
  Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Week 41 | 0.12 [0.01 to 0.44] | 0.30 [0.01 to 1.64] | 0.00 [0.00 to 6.38]
  Week 42: number analyzed (Participants) | 910 | 401 | 17
  Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 19.51]
  Week 43: number analyzed (Participants) | 496 | 378 | 22
  Week 43 | 0.40 [0.03 to 1.69] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 15.44]
  Week 44: number analyzed (Participants) | 750 | 2946 | 30
  Week 44 | 0.40 [0.02 to 1.80] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 11.57]
  Week 45: number analyzed (Participants) | 453 | 402 | 546
  Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.40]
  Week 46: number analyzed (Participants) | 350 | 264 | 19
  Week 46 | 0.29 [0.00 to 2.08] | 0.00 [0.00 to 1.39] | 0.00 [0.00 to 17.65]
  Week 47: number analyzed (Participants) | 258 | 157 | 41
  Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Week 48: number analyzed (Participants) | 145 | 100 | 10
  Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

16. Primary Outcome: Cumulative Incidence Rates of Rash Adverse Events Reported Via ADR Card, by Vaccine Group
Description: as for outcome 2
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Week 35-37 | 0.53 [0.23 to 1.04] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Week 35-38 | 0.40 [0.17 to 0.80] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 10.00]
  Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Week 35-39 | 0.31 [0.17 to 0.53] | 0.00 [0.00 to 3.45] | 0.00 [0.00 to 6.06]
  Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Week 35-40 | 0.33 [0.22 to 0.48] | 0.00 [0.00 to 0.83] | 0.00 [0.00 to 4.02]
  Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Week 35-41 | 0.31 [0.20 to 0.44] | 0.13 [0.00 to 0.71] | 0.00 [0.00 to 2.49]
  Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Week 35-42 | 0.29 [0.19 to 0.41] | 0.08 [0.00 to 0.47] | 0.00 [0.00 to 2.24]
  Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Week 35-43 | 0.29 [0.20 to 0.41] | 0.06 [0.00 to 0.36] | 0.00 [0.00 to 1.97]
  Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Week 35-44 | 0.30 [0.21 to 0.41] | 0.05 [0.00 to 0.28] | 0.00 [0.00 to 1.70]
  Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Week 35-45 | 0.29 [0.20 to 0.40] | 0.04 [0.00 to 0.23] | 0.00 [0.00 to 0.77]
  Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Week 35-46 | 0.29 [0.20 to 0.40] | 0.04 [0.00 to 0.21] | 0.00 [0.00 to 0.74]
  Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Week 35-47 | 0.28 [0.20 to 0.39] | 0.04 [0.00 to 0.20] | 0.00 [0.00 to 0.69]
  Week 35-48 | 0.28 [0.20 to 0.39] | 0.03 [0.00 to 0.19] | 0.00 [0.00 to 0.67]

17. Primary Outcome: Weekly Incidence Rates of Musculoskeletal Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Musculoskeletal adverse events include any musculoskeletal adverse events, arthropathy, and muscle aches/myalgia. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Any, Week 37 | 3.65 [2.94 to 4.47] | 0.00 [0.00 to 70.76] | 6.25 [0.16 to 30.23]
  Any, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Any, Week 38 | 2.82 [2.12 to 3.67] | 0.00 [0.00 to 40.96] | 6.25 [0.01 to 45.43]
  Any, Week 39: number analyzed (Participants) | 16387 | 94 | 24
  Any, Week 39 | 2.55 [2.04 to 3.14] | 0.00 [0.00 to 3.85] | 4.17 [0.11 to 21.12]
  Any, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Any, Week 40 | 2.19 [1.60 to 2.92] | 1.19 [0.02 to 7.15] | 0.00 [0.00 to 11.22]
  Any, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Any, Week 41 | 1.99 [1.37 to 2.79] | 0.00 [0.00 to 1.09] | 0.00 [0.00 to 6.38]
  Any, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Any, Week 42 | 1.54 [0.59 to 3.23] | 0.25 [0.01 to 1.38] | 0.00 [0.00 to 19.51]
  Any, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Any, Week 43 | 2.82 [1.31 to 5.26] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 15.44]
  Any, Week 44: number analyzed (Participants) | 750 | 464 | 30
  Any, Week 44 | 1.60 [0.39 to 4.27] | 1.08 [0.02 to 6.23] | 0.00 [0.00 to 11.57]
  Any, Week 45: number analyzed (Participants) | 453 | 402 | 546
  Any, Week 45 | 1.32 [0.26 to 3.91] | 0.25 [0.01 to 1.38] | 0.38 [0.01 to 2.12]
  Any, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Any, Week 46 | 0.86 [0.17 to 2.52] | 0.38 [0.00 to 2.63] | 0.00 [0.00 to 17.65]
  Any, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Any, Week 47 | 0.39 [0.00 to 2.82] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

18. Primary Outcome: Cumulative Incidence Rates of Musculoskeletal Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Musculoskeletal adverse events include any musculoskeletal adverse events, arthropathy, and muscle aches/myalgia. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Any, Week 35-37 | 3.65 [2.94 to 4.47] | 0.00 [0.00 to 60.24] | 5.26 [0.13 to 26.03]
  Any, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Any, Week 35-38 | 3.21 [2.56 to 3.98] | 0.00 [0.00 to 28.49] | 5.71 [0.61 to 20.03]
  Any, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Any, Week 35-39 | 2.92 [2.35 to 3.58] | 0.00 [0.00 to 3.45] | 5.08 [1.06 to 14.15]
  Any, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Any, Week 35-40 | 2.79 [2.32 to 3.32] | 0.90 [0.03 to 4.68] | 3.33 [0.69 to 9.43]
  Any, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Any, Week 35-41 | 2.69 [2.21 to 3.23] | 0.51 [0.04 to 2.05] | 2.05 [0.42 to 5.91]
  Any, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Any, Week 35-42 | 2.61 [2.12 to 3.18] | 0.42 [0.05 to 1.57] | 1.84 [0.38 to 5.28]
  Any, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Any, Week 35-43 | 2.62 [2.12 to 3.19] | 0.32 [0.03 to 1.21] | 1.62 [0.34 to 4.67]
  Any, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Any, Week 35-44 | 2.57 [2.08 to 3.13] | 0.49 [0.04 to 2.04] | 1.40 [0.26 to 4.21]
  Any, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Any, Week 35-45 | 2.53 [2.05 to 3.10] | 0.45 [0.03 to 1.94] | 0.84 [0.14 to 2.67]
  Any, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Any, Week 35-46 | 2.50 [2.01 to 3.06] | 0.45 [0.03 to 1.99] | 0.81 [0.14 to 2.56]
  Any, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Any, Week 35-47 | 2.46 [1.98 to 3.02] | 0.42 [0.02 to 1.90] | 0.75 [0.14 to 2.27]
  Any, Week 35-48 | 2.44 [1.96 to 3.00] | 0.41 [0.02 to 1.84] | 0.73 [0.13 to 2.24]

19. Primary Outcome: Weekly Incidence Rates of Neurological Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Neurological adverse events include any neurological adverse events, Bell's palsy, Guillain-Barre Syndrome, peripheral tremor and seizure/febrile convulsions. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Any, Week 37 | 0.28 [0.11 to 0.58] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Any, Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Any, Week 38 | 0.26 [0.10 to 0.53] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Any, Week 39: number analyzed (Participants) | 16387 | 94 | 24
  Any, Week 39 | 0.17 [0.04 to 0.44] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Any, Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Any, Week 40 | 0.00 [0.00 to 0.18] | 0.30 [0.00 to 1.82] | 0.00 [0.00 to 11.22]
  Any, Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Any, Week 41 | 0.18 [0.03 to 0.59] | 0.30 [0.01 to 1.64] | 1.79 [0.05 to 9.55]
  Any, Week 42: number analyzed (Participants) | 910 | 401 | 17
  Any, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 19.51]
  Any, Week 43: number analyzed (Participants) | 496 | 378 | 22
  Any, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 15.44]
  Any, Week 44: number analyzed (Participants) | 750 | 2946 | 30
  Any, Week 44 | 0.13 [0.00 to 1.05] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 11.57]
  Any, Week 45: number analyzed (Participants) | 453 | 402 | 546
  Any, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.40]
  Any, Week 46: number analyzed (Participants) | 350 | 264 | 19
  Any, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 1.39] | 0.00 [0.00 to 17.65]
  Any, Week 47: number analyzed (Participants) | 258 | 157 | 41
  Any, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 10
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

20. Primary Outcome: Cumulative Incidence Rates of Neurological Adverse Events Reported Via ADR Card, by Vaccine Group
Description: Neurological adverse events include any neurological adverse events, Bell's palsy, Guillain-Barre Syndrome, peripheral tremor and seizure/febrile convulsions. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Any, Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Any, Week 35-37 | 0.28 [0.11 to 0.58] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Any, Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Any, Week 35-38 | 0.27 [0.15 to 0.45] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 10.00]
  Any, Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Any, Week 35-39 | 0.23 [0.12 to 0.39] | 0.00 [0.00 to 3.45] | 0.00 [0.00 to 6.06]
  Any, Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Any, Week 35-40 | 0.18 [0.09 to 0.34] | 0.23 [0.01 to 1.25] | 0.00 [0.00 to 4.02]
  Any, Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Any, Week 35-41 | 0.18 [0.10 to 0.31] | 0.26 [0.02 to 1.03] | 0.68 [0.02 to 3.76]
  Any, Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Any, Week 35-42 | 0.17 [0.09 to 0.29] | 0.17 [0.02 to 0.63] | 0.61 [0.02 to 3.37]
  Any, Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Any, Week 35-43 | 0.17 [0.09 to 0.28] | 0.13 [0.01 to 0.48] | 0.54 [0.01 to 2.97]
  Any, Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Any, Week 35-44 | 0.16 [0.09 to 0.28] | 0.10 [0.01 to 0.41] | 0.47 [0.01 to 2.56]
  Any, Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Any, Week 35-45 | 0.16 [0.09 to 0.27] | 0.08 [0.01 to 0.35] | 0.21 [0.01 to 1.16]
  Any, Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Any, Week 35-46 | 0.16 [0.08 to 0.27] | 0.07 [0.00 to 0.33] | 0.20 [0.01 to 1.12]
  Any, Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Any, Week 35-47 | 0.15 [0.08 to 0.26] | 0.07 [0.00 to 0.32] | 0.19 [0.00 to 1.04]
  Any, Week 35-48 | 0.15 [0.08 to 0.26] | 0.07 [0.00 to 0.31] | 0.18 [0.00 to 1.02]

21. Primary Outcome: Weekly Incidence Rates of SAEs Reported Via ADR Card by Vaccine Group
Description: The weekly incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card;
  * The numerator was the number of subjects from the denominator who reported any SAEs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine.
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35: number analyzed (Participants) | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 1 | 1 | 3
  Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 37: number analyzed (Participants) | 2466 | 3 | 16
  Week 37 | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 20.59]
  Week 38: number analyzed (Participants) | 2730 | 7 | 16
  Week 38 | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 20.59]
  Week 39: number analyzed (Participants) | 4116 | 94 | 24
  Week 39 | 0.00 [0.00 to 0.09] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 14.25]
  Week 40: number analyzed (Participants) | 2055 | 337 | 31
  Week 40 | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 1.09] | 0.00 [0.00 to 11.22]
  Week 41: number analyzed (Participants) | 1657 | 338 | 56
  Week 41 | 0.00 [0.00 to 0.22] | 0.00 [0.00 to 1.09] | 0.00 [0.00 to 6.38]
  Week 42: number analyzed (Participants) | 910 | 401 | 17
  Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 19.51]
  Week 43: number analyzed (Participants) | 496 | 378 | 22
  Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 15.44]
  Week 44: number analyzed (Participants) | 750 | 464 | 30
  Week 44 | 0.00 [0.00 to 0.49] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 11.57]
  Week 45: number analyzed (Participants) | 453 | 402 | 261
  Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.40]
  Week 46: number analyzed (Participants) | 350 | 264 | 19
  Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 1.39] | 0.00 [0.00 to 17.65]
  Week 47: number analyzed (Participants) | 258 | 157 | 41
  Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 8.60]
  Week 48: number analyzed (Participants) | 145 | 100 | 10
  Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 30.85]

22. Primary Outcome: Cumulative Incidence Rates of SAEs Reported Via ADR Card by Vaccine Group
Description: The cumulative incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card;
  * The numerator was the number of subjects from the denominator who reported any SAEs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine.
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017.
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  Week 35-37: number analyzed (Participants) | 2467 | 4 | 19
  Week 35-37 | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 17.65]
  Week 35-38: number analyzed (Participants) | 5197 | 11 | 35
  Week 35-38 | 0.00 [0.00 to 0.07] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 10.00]
  Week 35-39: number analyzed (Participants) | 9313 | 105 | 59
  Week 35-39 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 3.45] | 0.00 [0.00 to 6.06]
  Week 35-40: number analyzed (Participants) | 11368 | 442 | 90
  Week 35-40 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.83] | 0.00 [0.00 to 4.02]
  Week 35-41: number analyzed (Participants) | 13025 | 780 | 146
  Week 35-41 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.47] | 0.00 [0.00 to 2.49]
  Week 35-42: number analyzed (Participants) | 13935 | 1181 | 163
  Week 35-42 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 2.24]
  Week 35-43: number analyzed (Participants) | 14431 | 1559 | 185
  Week 35-43 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.24] | 0.00 [0.00 to 1.97]
  Week 35-44: number analyzed (Participants) | 15181 | 2023 | 215
  Week 35-44 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 1.70]
  Week 35-45: number analyzed (Participants) | 15634 | 2425 | 476
  Week 35-45 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 0.77]
  Week 35-46: number analyzed (Participants) | 15984 | 2689 | 495
  Week 35-46 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 0.74]
  Week 35-47: number analyzed (Participants) | 16242 | 2846 | 536
  Week 35-47 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 0.69]
  Week 35-48 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 0.67]

23. Primary Outcome: Weekly Incidence Rates of Any AEIs Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 3.38 [1.37 to 6.84] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 1.63 [0.02 to 10.28] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.52 [0.00 to 3.94] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 1.97 [0.07 to 9.78] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 33.33 [0.00 to 100] | 14.29 [3.05 to 36.34] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 1.06 [0.02 to 5.93] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.99 [0.00 to 10.54] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 7.14 [0.02 to 44.90] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 11.11 [0.19 to 51.19] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 1.25 [0.03 to 6.77] | 1.46 [0.30 to 4.22]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18-65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18-65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18-65 years, Week 37 | 9.87 [6.92 to 13.55] | 0.00 [0.00 to 84.19] | 22.22 [2.81 to 60.01]
  18-65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18-65 years, Week 38 | 7.45 [4.89 to 10.79] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18-65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18-65 years, Week 39 | 8.48 [7.08 to 10.06] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18-65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18-65 years, Week 40 | 8.37 [4.12 to 14.76] | 6.78 [1.88 to 16.46] | 0.00 [0.00 to 33.63]
  18-65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18-65 years, Week 41 | 4.88 [2.78 to 7.88] | 4.44 [1.22 to 10.99] | 0.00 [0.00 to 30.85]
  18-65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18-65 years, Week 42 | 3.67 [1.25 to 8.20] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18-65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18-65 years, Week 43 | 4.59 [1.48 to 10.46] | 6.03 [2.46 to 12.04] | 0.00 [0.00 to 24.71]
  18-65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18-65 years, Week 44 | 3.83 [1.31 to 8.54] | 8.97 [0.36 to 37.68] | 0.00 [0.00 to 36.94]
  18-65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18-65 years, Week 45 | 2.25 [0.60 to 5.75] | 1.82 [0.00 to 93.05] | 5.88 [0.72 to 19.68]
  18-65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18-65 years, Week 46 | 4.93 [1.73 to 10.77] | 8.00 [0.74 to 28.24] | 0.00 [0.00 to 60.24]
  18-65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18-65 years, Week 47 | 2.74 [0.36 to 9.27] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18-65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18-65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 10.27 [8.88 to 11.79] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 7.90 [6.31 to 9.74] | 16.67 [0.00 to 91.51] | 20.00 [1.06 to 65.28]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 7.74 [6.52 to 9.12] | 0.00 [0.00 to 70.76] | 5.88 [0.15 to 28.69]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 8.15 [5.16 to 12.10] | 2.44 [0.06 to 12.86] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 7.43 [5.38 to 9.96] | 6.33 [2.09 to 14.16] | 33.33 [0.00 to 99.94]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 3.85 [1.67 to 7.46] | 6.15 [1.70 to 15.01] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 4.74 [1.88 to 9.68] | 3.70 [0.00 to 98.52] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 4.88 [1.08 to 13.29] | 7.81 [0.00 to 63.88] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 5.41 [2.08 to 11.19] | 16.22 [0.00 to 99.95] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 3.51 [0.58 to 10.84] | 2.70 [0.00 to 99.94] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 3.70 [0.00 to 99.88] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

24. Primary Outcome: Cumulative Incidence Rates of Any AEIs Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 2.59 [0.63 to 6.88] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 2.29 [0.33 to 7.54] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 1.71 [0.25 to 5.63] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 1.38 [0.15 to 5.09] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 1.51 [0.26 to 4.71] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 1.32 [0.20 to 4.30] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 1.19 [0.18 to 3.94] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 1.13 [0.16 to 3.75] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 1.10 [0.16 to 3.67] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 3.70 [0.00 to 39.49] | 7.32 [0.90 to 24.00] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 3.45 [0.00 to 35.58] | 4.29 [0.36 to 16.39] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 2.94 [0.00 to 26.56] | 3.19 [0.28 to 12.23] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 2.86 [0.00 to 25.94] | 2.52 [0.21 to 9.89] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 2.44 [0.00 to 20.29] | 1.88 [0.24 to 6.46] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 2.38 [0.00 to 19.99] | 1.59 [0.07 to 7.48] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 2.13 [0.00 to 17.04] | 1.37 [0.05 to 6.77] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 2.13 [0.00 to 17.04] | 1.31 [0.05 to 6.49] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 2.08 [0.00 to 16.23] | 1.25 [0.04 to 6.39] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 2.63 [0.01 to 18.97] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 2.22 [0.02 to 14.79] | 7.14 [0.04 to 41.49] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 1.82 [0.01 to 12.25] | 3.23 [0.01 to 24.14] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 1.69 [0.02 to 10.77] | 2.08 [0.02 to 13.45] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 1.64 [0.02 to 10.46] | 1.64 [0.01 to 11.31] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 1.61 [0.02 to 10.31] | 1.16 [0.01 to 8.31] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 1.43 [0.02 to 9.07] | 1.20 [0.15 to 4.28] | 1.23 [0.25 to 3.55]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 1.32 [0.01 to 8.53] | 1.12 [0.14 to 4.00] | 1.22 [0.25 to 3.52]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 1.22 [0.01 to 8.11] | 1.09 [0.13 to 3.89] | 1.20 [0.25 to 3.45]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 1.16 [0.01 to 7.70] | 1.09 [0.13 to 3.87] | 1.20 [0.25 to 3.45]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 9.87 [6.92 to 13.55] | 0.00 [0.00 to 84.19] | 22.22 [2.81 to 60.01]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 8.56 [6.27 to 11.34] | 0.00 [0.00 to 70.76] | 13.33 [1.66 to 40.46]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 8.52 [7.40 to 9.75] | 0.00 [0.00 to 45.93] | 10.00 [1.23 to 31.70]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 8.49 [7.19 to 9.94] | 6.15 [1.70 to 15.01] | 6.90 [0.85 to 22.77]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 7.97 [6.82 to 9.23] | 5.16 [2.25 to 9.92] | 5.13 [0.63 to 17.32]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 7.64 [6.47 to 8.95] | 3.09 [1.34 to 6.00] | 4.65 [0.57 to 15.81]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 7.51 [6.29 to 8.88] | 4.00 [2.26 to 6.51] | 3.57 [0.44 to 12.31]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 7.29 [6.02 to 8.73] | 4.86 [3.07 to 7.26] | 3.13 [0.38 to 10.84]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 7.09 [5.82 to 8.52] | 4.53 [2.89 to 6.72] | 4.08 [1.12 to 10.12]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 7.00 [5.66 to 8.54] | 4.84 [3.21 to 6.96] | 3.92 [1.08 to 9.74]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 6.89 [5.57 to 8.42] | 4.53 [3.01 to 6.52] | 3.42 [0.94 to 8.52]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 6.79 [5.46 to 8.33] | 4.32 [2.87 to 6.22] | 3.31 [0.91 to 8.25]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 10.26 [8.87 to 11.78] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 9.04 [7.70 to 10.54] | 12.50 [0.10 to 60.63] | 10.00 [0.88 to 34.70]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 8.49 [7.30 to 9.80] | 9.09 [0.21 to 41.85] | 8.11 [1.70 to 21.91]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 8.43 [7.22 to 9.77] | 3.85 [0.47 to 13.21] | 6.12 [1.28 to 16.87]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 8.31 [7.08 to 9.68] | 5.34 [2.18 to 10.70] | 7.69 [2.14 to 18.54]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 8.04 [6.77 to 9.47] | 5.61 [2.83 to 9.82] | 7.02 [1.95 to 17.00]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 7.95 [6.66 to 9.39] | 5.05 [2.56 to 8.85] | 6.67 [1.85 to 16.20]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 7.81 [6.57 to 9.21] | 5.57 [3.11 to 9.11] | 6.25 [1.73 to 15.24]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 7.76 [6.52 to 9.16] | 6.61 [6.61 to 9.61] | 4.76 [0.69 to 15.23]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 7.71 [6.45 to 9.14] | 6.27 [4.13 to 9.05] | 4.44 [0.54 to 15.14]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 7.63 [6.35 to 9.08] | 6.11 [4.06 to 8.76] | 4.30 [0.52 to 14.72]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 7.59 [6.31 to 9.05] | 5.82 [3.87 to 8.35] | 4.21 [0.49 to 14.59]

25. Primary Outcome: Weekly Incidence Rates of Fever/Pyrexia Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Fever/pyrexia = all subjects with a fever/pyrexia read code recorded were considered as having fever/pyrexia, regardless of what temperature had been recorded. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 1.45 [0.30 to 4.18] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.91] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 0.49 [0.01 to 2.71] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 4.76 [0.03 to 29.74] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.85] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.59] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.49 [0.01 to 2.69]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 0.56 [0.15 to 1.42] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 0.81 [0.13 to 2.66] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 0.57 [0.24 to 1.11] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 0.54 [0.05 to 2.16] | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 1.04 [0.02 to 1.39] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.04] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 0.46 [0.01 to 2.96] | 0.00 [0.00 to 3.13] | 0.00 [0.00 to 24.71]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 0.32 [0.01 to 1.77] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.28]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 0.45 [0.00 to 3.36] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 0.68 [0.00 to 4.94] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 0.40 [0.16 to 0.83] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 0.38 [0.15 to 0.78] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 30.85]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 0.41 [0.12 to 1.01] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 19.51]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 0.23 [0.05 to 0.67] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 0.40 [0.09 to 1.11] | 2.53 [0.31 to 8.85] | 0.00 [0.00 to 70.76]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 0.00 [0.00 to 0.67] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 0.36 [0.00 to 2.44] | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 0.23 [0.01 to 1.29] | 1.56 [0.00 to 64.84] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 0.88 [0.01 to 6.20] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

26. Primary Outcome: Cumulative Incidence Rates of Fever/Pyrexia Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Fever/pyrexia = all subjects with a fever/pyrexia read code recorded were considered as having fever/pyrexia, regardless of what temperature had been recorded. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 1.11 [0.14 to 3.88] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.76 [0.06 to 3.15] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.51 [0.02 to 2.44] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.41 [0.01 to 2.18] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.43 [0.04 to 1.68] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.38 [0.03 to 1.53] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.34 [0.03 to 1.41] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.32 [0.02 to 1.34] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.31 [0.02 to 1.31] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 2.44 [0.03 to 14.54] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 1.43 [0.01 to 9.35] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 1.06 [0.01 to 7.27] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.84 [0.01 to 5.77] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.47 [0.00 to 3.56] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.32 [0.00 to 2.62] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.27 [0.00 to 2.31] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.26 [0.00 to 2.22] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.25 [0.00 to 2.15] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.41 [0.01 to 2.26]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.41 [0.01 to 2.24]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.40 [0.01 to 2.20]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.40 [0.01 to 2.20]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 0.56 [0.15 to 1.42] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 0.70 [0.22 to 1.64] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 0.63 [0.26 to 1.29] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 16.84]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 0.62 [0.28 to 1.17] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 11.94]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 0.57 [0.29 to 1.02] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 9.03]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 0.53 [0.26 to 0.97] | 0.00 [0.00 to 1.41] | 0.00 [0.00 to 8.22]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 0.53 [0.25 to 0.97] | 0.00 [0.00 to 0.98] | 0.00 [0.00 to 6.38]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 0.51 [0.25 to 0.94] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 5.60]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 0.49 [0.24 to 0.90] | 0.00 [0.00 to 0.72] | 0.00 [0.00 to 3.69]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 0.49 [0.22 to 0.94] | 0.00 [0.00 to 0.66] | 0.00 [0.00 to 3.55]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 0.50 [0.24 to 0.91] | 0.00 [0.00 to 0.62] | 0.00 [0.00 to 3.10]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 0.49 [0.24 to 0.89] | 0.00 [0.00 to 0.59] | 0.00 [0.00 to 3.00]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 0.40 [0.16 to 0.83] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 0.39 [0.21 to 0.65] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 16.84]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 0.40 [0.22 to 0.66] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 9.49]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 0.37 [0.22 to 0.58] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 7.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 0.37 [0.24 to 0.55] | 1.53 [0.19 to 5.41] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 0.35 [0.22 to 0.53] | 1.02 [0.12 to 3.64] | 0.00 [0.00 to 6.27]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 0.35 [0.22 to 0.54] | 0.72 [0.09 to 2.58] | 0.00 [0.00 to 5.96]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 0.35 [0.21 to 0.53] | 0.88 [0.18 to 2.55] | 0.00 [0.00 to 5.60]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 0.34 [0.21 to 0.52] | 0.79 [0.16 to 2.30] | 0.00 [0.00 to 4.30]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 0.34 [0.21 to 0.54] | 0.72 [0.15 to 2.10] | 0.00 [0.00 to 4.02]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 0.34 [0.20 to 0.54] | 0.68 [0.14 to 1.97] | 0.00 [0.00 to 3.89]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 0.34 [0.20 to 0.53] | 0.65 [0.13 to 1.88] | 0.00 [0.00 to 3.81]

27. Primary Outcome: Weekly Incidence Rates of Local Symptoms Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Local symptoms include local erythema. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.91] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.85] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.59] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 3.06 [1.93 to 4.60] | 0.00 [0.00 to 84.19] | 11.11 [0.19 to 51.19]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 3.03 [1.36 to 5.75] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 2.12 [1.26 to 3.33] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 3.10 [0.67 to 8.64] | 1.69 [0.04 to 9.09] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 1.26 [0.55 to 2.47] | 2.22 [0.27 to 7.80] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 0.85 [0.06 to 3.52] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 0.46 [0.01 to 2.96] | 1.72 [0.11 to 7.43] | 0.00 [0.00 to 24.71]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 2.24 [0.76 to 5.02] | 1.28 [0.03 to 6.94] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.28]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 2.24 [0.30 to 7.65] | 4.00 [0.49 to 13.71] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 2.05 [0.10 to 9.40] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 1.38 [0.31 to 3.85] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 0.97 [0.53 to 1.63] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 30.85]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 1.80 [1.19 to 2.60] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 19.51]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 1.31 [0.44 to 2.97] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 1.59 [0.91 to 2.56] | 1.27 [0.03 to 6.85] | 0.00 [0.00 to 70.76]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 0.37 [0.00 to 2.82] | 3.08 [0.37 to 10.68] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 0.36 [0.00 to 2.55] | 1.23 [0.00 to 73.92] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 0.47 [0.02 to 2.39] | 3.13 [0.00 to 46.96] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 1.35 [0.09 to 5.79] | 5.41 [0.00 to 99.64] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 2.70 [0.00 to 99.94] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

28. Primary Outcome: Cumulative Incidence Rates of Local Symptoms Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Local symptoms include local erythema. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.17] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.50]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.49]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.46]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.46]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 3.06 [1.93 to 4.60] | 0.00 [0.00 to 84.19] | 11.11 [0.19 to 51.19]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 3.04 [1.83 to 4.73] | 0.00 [0.00 to 70.76] | 6.67 [0.17 to 31.95]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 2.61 [1.61 to 3.97] | 0.00 [0.00 to 45.93] | 5.00 [0.10 to 26.11]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 2.70 [1.52 to 4.42] | 1.54 [0.04 to 8.28] | 3.45 [0.05 to 19.42]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 2.49 [1.48 to 3.92] | 1.94 [0.40 to 5.55] | 2.56 [0.05 to 14.20]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 2.37 [1.44 to 3.67] | 1.16 [0.24 to 3.35] | 2.33 [0.06 to 12.41]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 2.29 [1.39 to 3.52] | 1.33 [0.43 to 3.08] | 1.79 [0.05 to 9.55]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 2.28 [1.44 to 3.43] | 1.32 [0.49 to 2.86] | 1.56 [0.04 to 8.40]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 2.19 [1.38 to 3.30] | 1.18 [0.43 to 2.55] | 1.02 [0.02 to 5.93]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 2.19 [1.41 to 3.25] | 1.43 [0.62 to 2.81] | 0.98 [0.02 to 5.69]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 2.19 [1.43 to 3.20] | 1.34 [0.58 to 2.63] | 0.85 [0.02 to 4.96]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 2.16 [1.41 to 3.16] | 1.28 [0.55 to 2.51] | 0.83 [0.01 to 4.93]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 1.38 [0.31 to 3.85] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 1.17 [0.47 to 2.42] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 16.84]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 1.44 [0.82 to 2.34] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 9.49]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 1.42 [0.87 to 2.16] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 7.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 1.44 [0.94 to 2.10] | 0.76 [0.02 to 4.18] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 1.37 [0.93 to 1.94] | 1.53 [0.32 to 4.41] | 0.00 [0.00 to 6.27]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 1.34 [0.92 to 1.89] | 1.44 [0.39 to 3.66] | 0.00 [0.00 to 5.96]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 1.30 [0.90 to 1.83] | 1.76 [0.65 to 3.79] | 0.00 [0.00 to 5.60]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 1.31 [0.90 to 1.83] | 2.12 [0.92 to 4.13] | 0.00 [0.00 to 4.30]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 1.29 [0.89 to 1.81] | 2.17 [1.00 to 4.08] | 0.00 [0.00 to 4.02]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 1.28 [0.88 to 1.79] | 2.04 [0.94 to 3.83] | 0.00 [0.00 to 3.89]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 1.27 [0.88 to 1.78] | 1.94 [0.89 to 3.65] | 0.00 [0.00 to 3.81]

29. Primary Outcome: Weekly Incidence Rates of General Non-specific Symptoms Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, headache, irritability, and malaise. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.91] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 0.49 [0.01 to 2.71] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 9.52 [1.17 to 30.38] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.85] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.99 [0.00 to 10.54] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.49 [0.01 to 2.69]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 3.76 [2.09 to 6.18] | 0.00 [0.00 to 84.19] | 11.11 [0.03 to 62.14]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 3.26 [1.90 to 5.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 3.75 [2.61 to 5.18] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 2.56 [1.55 to 3.98] | 3.39 [0.41 to 11.71] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 1.42 [0.65 to 2.67] | 2.22 [0.27 to 7.80] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 2.54 [0.87 to 5.70] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 0.46 [0.00 to 3.13] | 1.72 [0.11 to 7.43] | 0.00 [0.00 to 24.71]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 1.60 [0.48 to 3.84] | 5.13 [0.23 to 22.68] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 0.90 [0.09 to 3.43] | 1.82 [0.00 to 93.05] | 0.00 [0.00 to 10.28]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 0.45 [0.00 to 3.36] | 4.00 [0.00 to 40.02] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 3.98 [3.11 to 5.01] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 2.87 [2.06 to 3.88] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 30.85]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 2.54 [1.78 to 3.51] | 0.00 [0.00 to 70.76] | 5.88 [0.15 to 28.69]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 2.38 [1.49 to 3.59] | 2.44 [0.06 to 12.86] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 1.98 [1.17 to 3.13] | 2.53 [0.31 to 8.85] | 0.00 [0.00 to 70.76]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 0.92 [0.11 to 3.23] | 1.54 [0.04 to 8.28] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 2.92 [1.11 to 6.13] | 2.47 [0.00 to 93.58] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 1.63 [0.53 to 3.74] | 1.56 [0.00 to 64.84] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 1.35 [0.11 to 5.51] | 5.41 [0.03 to 33.24] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 0.88 [0.01 to 6.20] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

30. Primary Outcome: Cumulative Incidence Rates of General Non-specific Symptoms Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, headache, irritability, and malaise. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- 2Vaccinated_Non GSK Group: Volunteered subjects who received non-GSK influenza vaccination in 10 volunteer GP practices between 01 September and 30 November 2017
Arm/Group | Vaccinated_Fluarix Tetra Group | 2Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.11 [0.00 to 0.78] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.09 [0.00 to 0.70] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.09 [0.00 to 0.62] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.08 [0.00 to 0.58] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.08 [0.00 to 0.56] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 4.88 [0.60 to 16.53] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 2.86 [0.34 to 10.06] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 2.13 [0.26 to 7.48] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 1.68 [0.20 to 5.94] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.94 [0.07 to 3.94] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.96 [0.02 to 5.20] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.82 [0.02 to 4.69] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.79 [0.02 to 4.50] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.75 [0.01 to 4.41] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.41 [0.01 to 2.26]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.41 [0.01 to 2.24]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.40 [0.01 to 2.20]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.40 [0.01 to 2.20]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 3.76 [2.09 to 6.18] | 0.00 [0.00 to 84.19] | 11.11 [0.03 to 62.14]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 3.49 [2.10 to 5.41] | 0.00 [0.00 to 70.76] | 6.67 [0.04 to 38.91]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 3.61 [2.61 to 4.85] | 0.00 [0.00 to 45.93] | 5.00 [0.03 to 30.57]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 3.40 [2.60 to 4.37] | 3.08 [0.37 to 10.68] | 3.45 [0.05 to 19.42]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 3.11 [2.30 to 4.11] | 2.58 [0.71 to 6.48] | 2.56 [0.06 to 13.56]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 3.07 [2.29 to 4.02] | 1.54 [0.42 to 3.91] | 2.33 [0.05 to 12.95]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 2.95 [2.17 to 3.92] | 1.60 [0.59 to 3.45] | 1.79 [0.03 to 10.14]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 2.87 [2.10 to 3.83] | 2.21 [1.06 to 4.02] | 1.56 [0.02 to 9.62]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 2.79 [2.05 to 3.71] | 2.17 [1.09 to 3.84] | 1.02 [0.03 to 5.55]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 2.70 [1.95 to 3.65] | 2.33 [1.25 to 3.95] | 0.98 [0.02 to 5.34]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 2.63 [1.89 to 3.57] | 2.18 [1.17 to 3.70] | 0.85 [0.02 to 4.67]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 2.60 [1.85 to 3.53] | 2.08 [1.11 to 3.53] | 0.83 [0.02 to 4.52]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 3.98 [3.11 to 5.01] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 3.40 [2.73 to 4.19] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 16.84]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 3.04 [2.29 to 3.95] | 0.00 [0.00 to 28.49] | 2.70 [0.07 to 14.16]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 2.92 [2.19 to 3.83] | 1.92 [0.05 to 10.26] | 2.04 [0.05 to 10.85]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 2.81 [2.11 to 3.67] | 2.29 [0.47 to 6.55] | 1.92 [0.05 to 10.26]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 2.70 [1.98 to 3.59] | 2.04 [0.56 to 5.14] | 1.75 [0.04 to 9.39]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 2.71 [1.98 to 3.61] | 2.17 [0.80 to 4.65] | 1.67 [0.04 to 8.94]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 2.66 [1.94 to 3.56] | 2.05 [0.83 to 4.18] | 1.56 [0.04 to 8.40]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 2.63 [1.92 to 3.52] | 2.38 [1.09 to 4.47] | 1.19 [0.02 to 7.24]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 2.61 [1.89 to 3.51] | 2.17 [1.00 to 4.08] | 1.11 [0.01 to 7.09]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 2.58 [1.86 to 3.49] | 2.04 [0.91 to 3.89] | 1.08 [0.01 to 6.96]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 2.57 [1.85 to 3.47] | 1.94 [0.84 to 3.79] | 1.05 [0.01 to 6.88]

31. Primary Outcome: Weekly Incidence Rates of Respiratory/Miscellaneous Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Respiratory/miscellaneous adverse events include any respiratory/miscellaneous adverse events, conjunctivitis, coryza, cough, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhoea and wheezing. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 2.90 [1.07 to 6.20] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 1.63 [0.02 to 10.28] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.52 [0.00 to 3.94] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 1.97 [0.07 to 9.78] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 33.33 [0.00 to 100] | 9.52 [1.17 to 30.38] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 1.06 [0.02 to 5.93] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.59] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 7.14 [0.02 to 44.90] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 11.11 [0.19 to 51.19] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 1.46 [0.30 to 4.22]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 5.98 [3.78 to 8.93] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 3.38 [2.06 to 5.20] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 4.66 [3.43 to 6.18] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 3.24 [2.01 to 4.91] | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 2.52 [1.45 to 4.06] | 2.22 [0.27 to 7.80] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 1.69 [0.61 to 3.69] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 1.83 [0.30 to 5.81] | 5.17 [1.92 to 10.92] | 0.00 [0.00 to 24.71]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 1.60 [0.52 to 3.69] | 1.28 [0.03 to 6.94] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 1.80 [0.46 to 4.69] | 1.82 [0.00 to 93.05] | 5.88 [0.72 to 19.68]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 1.35 [0.21 to 4.35] | 6.00 [0.00 to 54.61] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 2.74 [0.36 to 9.27] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 5.71 [4.66 to 6.91] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 4.17 [3.29 to 5.20] | 16.67 [0.00 to 91.51] | 10.00 [0.25 to 44.50]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 4.00 [2.98 to 5.25] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 19.51]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 5.30 [2.90 to 8.81] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 3.87 [2.34 to 5.97] | 3.80 [0.79 to 10.70] | 0.00 [0.00 to 70.76]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 2.38 [0.86 to 5.17] | 1.54 [0.04 to 8.28] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 3.28 [1.32 to 6.67] | 1.23 [0.00 to 73.92] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 3.02 [0.48 to 9.57] | 6.25 [0.14 to 30.86] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 1.80 [0.29 to 5.74] | 8.11 [0.00 to 99.99] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 1.75 [0.12 to 7.34] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 3.70 [0.00 to 99.88] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

32. Primary Outcome: Cumulative Incidence Rates of Respiratory/Miscellaneous Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Respiratory/miscellaneous adverse events include any respiratory/miscellaneous adverse events, conjunctivitis, coryza, cough, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhoea and wheezing. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 2.22 [0.58 to 5.73] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 2.04 [0.32 to 6.56] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 1.54 [0.25 to 4.89] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 1.24 [0.15 to 4.43] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 1.40 [0.25 to 4.31] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 1.23 [0.20 to 3.94] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 1.11 [0.17 to 3.60] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 1.05 [0.16 to 3.42] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 1.02 [0.16 to 3.35] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 3.70 [0.00 to 39.49] | 4.88 [0.60 to 16.53] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 3.45 [0.00 to 35.58] | 2.86 [0.34 to 10.06] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 2.94 [0.00 to 26.56] | 2.13 [0.26 to 7.48] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 2.86 [0.00 to 25.94] | 1.68 [0.20 to 5.94] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 2.44 [0.00 to 20.29] | 1.41 [0.26 to 4.26] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 2.38 [0.00 to 19.99] | 0.96 [0.08 to 3.79] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 2.13 [0.00 to 17.04] | 0.82 [0.06 to 3.47] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 2.13 [0.00 to 17.04] | 0.79 [0.06 to 3.32] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 2.08 [0.00 to 16.23] | 0.75 [0.05 to 3.29] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 2.63 [0.01 to 18.97] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 2.22 [0.02 to 14.79] | 7.14 [0.04 to 41.49] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 1.82 [0.01 to 12.25] | 3.23 [0.01 to 24.14] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 1.69 [0.02 to 10.77] | 2.08 [0.02 to 13.45] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 1.64 [0.02 to 10.46] | 1.64 [0.01 to 11.31] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 1.61 [0.02 to 10.31] | 1.16 [0.01 to 8.31] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 1.43 [0.02 to 9.07] | 0.60 [0.00 to 5.27] | 1.23 [0.25 to 3.55]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 1.32 [0.01 to 8.53] | 0.56 [0.00 to 4.82] | 1.22 [0.25 to 3.52]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 546
  13 - 17 years, Week 35-47 | 1.22 [0.01 to 8.11] | 0.55 [0.00 to 4.69] | 1.20 [0.25 to 3.45]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 546
  13 - 17 years, Week 35-48 | 1.16 [0.01 to 7.70] | 0.54 [0.00 to 4.66] | 1.20 [0.25 to 3.45]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 5.98 [3.78 to 8.93] | 0.0 [0.0 to 84.19] | 0.0 [0.0 to 33.63]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 4.56 [3.03 to 6.56] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 4.61 [3.81 to 5.53] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 16.84]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 4.34 [3.70 to 5.06] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 11.94]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 4.07 [3.51 to 4.70] | 1.29 [0.16 to 4.58] | 0.00 [0.00 to 9.03]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 3.90 [3.28 to 4.59] | 0.77 [0.09 to 2.76] | 0.00 [0.00 to 8.22]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 3.80 [3.19 to 4.50] | 2.13 [0.93 to 4.16] | 0.00 [0.00 to 6.38]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 3.67 [3.08 to 4.34] | 1.99 [0.91 to 3.74] | 0.00 [0.00 to 5.60]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 3.60 [3.03 to 4.23] | 1.97 [0.95 to 3.59] | 2.04 [0.14 to 8.50]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 3.51 [2.96 to 4.13] | 2.33 [1.25 to 3.95] | 1.96 [0.13 to 8.26]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 3.49 [2.98 to 4.06] | 2.18 [1.17 to 3.70] | 1.71 [0.11 to 7.37]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 3.44 [2.93 to 4.00] | 2.08 [1.11 to 3.53] | 1.65 [0.12 to 6.86]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 5.71 [4.66 to 6.90] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38 | 4.91 [4.23 to 5.67] | 12.50 [0.10 to 60.63] | 5.00 [0.13 to 24.87]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 4.52 [3.80 to 5.34] | 9.09 [0.21 to 41.85] | 2.70 [0.07 to 14.16]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 4.66 [3.75 to 5.71] | 1.92 [0.05 to 10.26] | 2.04 [0.05 to 10.85]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 4.56 [3.64 to 5.65] | 3.05 [0.84 to 7.63] | 1.92 [0.05 to 10.26]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 4.43 [3.48 to 5.56] | 2.55 [0.83 to 5.85] | 1.75 [0.04 to 9.39]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 4.40 [3.43 to 5.55] | 2.17 [0.80 to 4.65] | 1.67 [0.04 to 8.94]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 4.34 [3.40 to 5.45] | 2.93 [1.42 to 5.33] | 1.56 [0.04 to 8.40]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 2946 | 546
  >65 years, Week 35-45 | 4.28 [3.34 to 5.40] | 3.44 [1.84 to 5.81] | 1.19 [0.02 to 7.24]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 4.26 [3.30 to 5.39] | 3.13 [1.68 to 5.30] | 1.11 [0.01 to 7.09]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 4.21 [3.25 to 5.36] | 3.17 [1.74 to 5.26] | 1.08 [0.01 to 6.96]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 4.19 [3.23 to 5.34] | 3.02 [1.66 to 5.01] | 1.05 [0.01 to 6.88]

33. Primary Outcome: Weekly Incidence Rates of Gastrointestinal Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhoea, nausea and vomiting. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.97 [0.12 to 3.45] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.91] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.85] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.99 [0.00 to 10.54] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 1.25 [0.03 to 6.77] | 0.49 [0.01 to 2.69]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 1.95 [0.56 to 4.80] | 0.00 [0.00 to 84.19] | 11.11 [0.03 to 62.14]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 1.63 [0.59 to 3.56] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 1.77 [0.70 to 3.63] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 1.62 [0.46 to 4.04] | 3.39 [0.41 to 11.71] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 0.94 [0.35 to 2.05] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 0.85 [0.12 to 2.86] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 0.00 [0.00 to 1.68] | 0.00 [0.00 to 3.13] | 0.00 [0.00 to 24.71]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 0.32 [0.00 to 2.44] | 1.28 [0.03 to 6.94] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.65] | 1.82 [0.00 to 93.05] | 0.00 [0.00 to 10.28]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 2.08 [0.98 to 3.85] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 1.68 [1.10 to 2.44] | 16.67 [0.00 to 91.51] | 0.00 [0.00 to 30.85]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 1.12 [0.73 to 1.66] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 19.51]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 1.23 [0.52 to 2.45] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 1.29 [0.59 to 2.43] | 2.53 [0.31 to 8.85] | 0.00 [0.00 to 70.76]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 0.55 [0.09 to 1.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 0.73 [0.06 to 2.90] | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 0.47 [0.06 to 1.67] | 1.56 [0.00 to 64.84] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 2.70 [0.54 to 7.83] | 2.70 [0.00 to 93.12] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 2.63 [0.20 to 10.66] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

34. Primary Outcome: Cumulative Incidence Rates of Gastrointestinal Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhea, nausea, and vomiting. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.74 [0.09 to 2.65] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.51 [0.04 to 2.11] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.34 [0.02 to 1.63] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.28 [0.01 to 1.46] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.22 [0.00 to 1.24] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.19 [0.00 to 1.12] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.17 [0.00 to 1.04] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.16 [0.00 to 0.99] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.16 [0.00 to 0.97] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.32 [0.00 to 2.62] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.27 [0.00 to 2.31] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.26 [0.00 to 2.22] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.25 [0.00 to 2.15] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.60 [0.02 to 3.31] | 0.41 [0.01 to 2.26]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.56 [0.01 to 3.09] | 0.41 [0.01 to 2.24]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.55 [0.01 to 3.01] | 0.40 [0.01 to 2.20]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.54 [0.01 to 2.99] | 0.40 [0.01 to 2.20]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 1.95 [0.56 to 4.80] | 0.00 [0.00 to 84.19] | 11.11 [0.03 to 62.14]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 1.77 [0.60 to 4.01] | 0.00 [0.00 to 70.76] | 6.67 [0.04 to 38.91]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 1.77 [0.84 to 3.26] | 0.00 [0.00 to 45.93] | 5.00 [0.03 to 30.57]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 1.74 [0.99 to 2.82] | 3.08 [0.37 to 10.68] | 3.45 [0.05 to 19.42]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 1.63 [0.95 to 2.58] | 1.29 [0.16 to 4.58] | 2.56 [0.06 to 13.56]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 1.57 [0.93 to 2.47] | 0.77 [0.09 to 2.76] | 2.33 [0.05 to 12.95]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 1.50 [0.87 to 2.40] | 0.53 [0.06 to 1.91] | 1.79 [0.03 to 10.14]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 1.43 [0.81 to 2.32] | 0.66 [0.14 to 1.92] | 1.56 [0.02 to 9.62]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 1.37 [0.77 to 2.24] | 0.79 [0.21 to 2.00] | 1.02 [0.03 to 5.55]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 1.32 [0.73 to 2.17] | 0.72 [0.20 to 1.83] | 0.98 [0.02 to 5.34]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 1.28 [0.71 to 2.12] | 0.67 [0.18 to 1.71] | 0.85 [0.02 to 4.67]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 1.26 [0.70 to 2.09] | 0.64 [0.17 to 1.63] | 0.83 [0.02 to 4.52]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 2.07 [0.98 to 3.84] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 1.87 [1.45 to 2.37] | 12.50 [0.10 to 60.63] | 0.00 [0.00 to 16.84]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 1.55 [1.15 to 2.04] | 9.09 [0.21 to 41.85] | 0.00 [0.00 to 9.49]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 1.50 [1.11 to 1.97] | 1.92 [0.05 to 10.26] | 0.00 [0.00 to 7.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 1.47 [1.10 to 1.93] | 2.29 [0.47 to 6.55] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 1.42 [1.07 to 1.83] | 1.53 [0.32 to 4.41] | 0.00 [0.00 to 6.27]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 1.40 [1.06 to 1.81] | 1.08 [0.22 to 3.13] | 0.00 [0.00 to 5.96]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 1.35 [1.04 to 1.73] | 1.17 [0.32 to 2.98] | 0.00 [0.00 to 5.60]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 1.38 [1.09 to 1.73] | 1.32 [0.43 to 3.06] | 0.00 [0.00 to 4.30]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 1.40 [1.09 to 1.77] | 1.20 [0.39 to 2.79] | 0.00 [0.00 to 4.02]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 1.38 [1.08 to 1.75] | 1.13 [0.37 to 2.62] | 0.00 [0.00 to 3.89]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 1.38 [1.07 to 1.74] | 1.08 [0.35 to 2.50] | 0.00 [0.00 to 3.81]

35. Primary Outcome: Weekly Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial oedema and hypersensitivity reactions. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.91] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.85] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.59] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 0.56 [0.01 to 3.49] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 0.70 [0.06 to 2.79] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 0.71 [0.05 to 3.00] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 0.27 [0.03 to 0.97] | 3.39 [0.41 to 11.71] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 0.31 [0.01 to 1.85] | 1.11 [0.03 to 6.04] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.04] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 0.00 [0.00 to 1.68] | 0.00 [0.00 to 3.13] | 0.00 [0.00 to 24.71]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 0.00 [0.00 to 1.17] | 3.85 [0.18 to 17.30] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 6.49] | 2.94 [0.07 to 15.33]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 0.45 [0.00 to 3.36] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 0.69 [0.01 to 4.78] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 0.49 [0.08 to 1.58] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 30.85]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 0.19 [0.02 to 0.74] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 19.51]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 0.46 [0.03 to 2.06] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 0.20 [0.01 to 0.94] | 1.27 [0.03 to 6.85] | 0.00 [0.00 to 70.76]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 0.00 [0.00 to 0.67] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 0.36 [0.00 to 2.55] | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 0.47 [0.02 to 2.39] | 0.00 [0.00 to 5.60] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

36. Primary Outcome: Cumulative Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial edema, and hypersensitivity reactions. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35- 40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35- 40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.17] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.50]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.49]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.46]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.46]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 0.56 [0.01 to 3.49] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 0.63 [0.03 to 2.94] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 0.67 [0.04 to 2.90] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 16.84]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 0.59 [0.05 to 2.39] | 3.08 [0.37 to 10.68] | 0.00 [0.00 to 11.94]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 0.55 [0.06 to 2.08] | 1.94 [0.40 to 5.55] | 0.00 [0.00 to 9.03]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 0.51 [0.05 to 1.97] | 1.16 [0.24 to 3.35] | 0.00 [0.00 to 8.22]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 0.49 [0.05 to 1.91] | 0.80 [0.17 to 2.32] | 0.00 [0.00 to 6.38]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 0.46 [0.04 to 1.82] | 1.32 [0.49 to 2.86] | 0.00 [0.00 to 5.60]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 0.44 [0.04 to 1.76] | 1.18 [0.43 to 2.55] | 1.02 [0.03 to 5.55]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 0.44 [0.04 to 1.80] | 1.08 [0.40 to 2.33] | 0.98 [0.02 to 5.34]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 0.43 [0.03 to 1.76] | 1.01 [0.37 to 2.18] | 0.85 [0.02 to 4.67]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 0.42 [0.03 to 1.73] | 0.96 [0.35 to 2.08] | 0.83 [0.02 to 4.52]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 0.69 [0.01 to 4.78] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 0.59 [0.03 to 2.82] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 16.84]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 0.42 [0.02 to 1.91] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 9.49]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 0.42 [0.02 to 1.92] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 7.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 0.40 [0.03 to 1.71] | 0.76 [0.02 to 4.18] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 0.37 [0.02 to 1.63] | 0.51 [0.01 to 2.81] | 0.00 [0.00 to 6.27]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 0.37 [0.03 to 1.57] | 0.36 [0.01 to 1.99] | 0.00 [0.00 to 5.96]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 0.38 [0.03 to 1.49] | 0.29 [0.01 to 1.62] | 0.00 [0.00 to 5.60]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 0.37 [0.03 to 1.46] | 0.26 [0.01 to 1.47] | 0.00 [0.00 to 4.30]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 0.36 [0.03 to 1.45] | 0.24 [0.01 to 1.34] | 0.00 [0.00 to 4.02]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 0.36 [0.03 to 1.43] | 0.23 [0.01 to 1.25] | 0.00 [0.00 to 3.89]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 0.36 [0.03 to 1.43] | 0.22 [0.01 to 1.19] | 0.00 [0.00 to 3.81]

37. Primary Outcome: Weekly Incidence Rates of Rash Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: as for outcome 23
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.91] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.85] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.59] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 0.28 [0.00 to 1.80] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 0.47 [0.07 to 1.58] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 0.35 [0.11 to 0.82] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 0.54 [0.15 to 1.38] | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.04] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 0.92 [0.08 to 3.71] | 0.00 [0.00 to 3.13] | 0.00 [0.00 to 24.71]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 0.64 [0.06 to 2.51] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.28]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 0.45 [0.00 to 3.27] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 0.63 [0.28 to 1.22] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 0.22 [0.04 to 0.68] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 30.85]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 0.11 [0.02 to 0.36] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 19.51]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 0.38 [0.12 to 0.89] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 0.20 [0.02 to 0.71] | 1.27 [0.03 to 6.85] | 0.00 [0.00 to 70.76]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 0.00 [0.00 to 0.67] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 0.23 [0.01 to 1.29] | 0.00 [0.00 to 5.60] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

38. Primary Outcome: Cumulative Incidence Rates of Rash Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: as for outcome 24
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.17] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.50]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.49]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.46]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.46]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 0.28 [0.00 to 1.80] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 0.38 [0.12 to 0.89] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 0.37 [0.18 to 0.66] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 16.84]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 0.40 [0.22 to 0.67] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 11.94]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 0.34 [0.19 to 0.57] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 9.03]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 0.32 [0.18 to 0.52] | 0.00 [0.00 to 1.41] | 0.00 [0.00 to 8.22]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 0.34 [0.20 to 0.55] | 0.00 [0.00 to 0.98] | 0.00 [0.00 to 6.38]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 0.36 [0.22 to 0.57] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 5.60]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 0.35 [0.21 to 0.55] | 0.00 [0.00 to 0.72] | 0.00 [0.00 to 3.69]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 0.35 [0.21 to 0.54] | 0.00 [0.00 to 0.66] | 0.00 [0.00 to 3.55]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 0.34 [0.21 to 0.53] | 0.00 [0.00 to 0.62] | 0.00 [0.00 to 3.10]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 0.34 [0.21 to 0.52] | 0.00 [0.00 to 0.59] | 0.00 [0.00 to 3.00]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 0.63 [0.28 to 1.22] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 0.42 [0.18 to 0.82] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 16.84]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 0.29 [0.13 to 0.56] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 9.49]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 0.30 [0.16 to 0.54] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 7.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 0.29 [0.15 to 0.50] | 0.76 [0.02 to 4.18] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 0.27 [0.15 to 0.47] | 0.51 [0.01 to 2.81] | 0.00 [0.00 to 6.27]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 0.27 [0.14 to 0.45] | 0.36 [0.01 to 1.99] | 0.00 [0.00 to 5.96]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 0.26 [0.15 to 0.43] | 0.29 [0.01 to 1.62] | 0.00 [0.00 to 5.60]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 0.26 [0.15 to 0.42] | 0.26 [0.01 to 1.47] | 0.00 [0.00 to 4.30]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 0.26 [0.14 to 0.42] | 0.24 [0.01 to 1.34] | 0.00 [0.00 to 4.02]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 0.25 [0.14 to 0.42] | 0.23 [0.01 to 1.25] | 0.00 [0.00 to 3.89]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 0.25 [0.14 to 0.41] | 0.22 [0.01 to 1.19] | 0.00 [0.00 to 3.81]

39. Primary Outcome: Weekly Incidence Rates of Musculoskeletal Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Musculoskeletal adverse events include any musculoskeletal adverse events, arthropathy, and muscle aches/myalgia. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.91] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.85] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.59] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.49 [0.01 to 2.69]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 4.59 [3.10 to 6.51] | 0.00 [0.00 to 84.19] | 11.11 [0.19 to 51.19]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 2.91 [1.89 to 4.27] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 2.76 [1.88 to 3.89] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 2.56 [1.55 to 3.98] | 5.08 [1.06 to 14.15] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 1.57 [0.76 to 2.88] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 1.69 [0.36 to 4.79] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 3.67 [1.60 to 7.10] | 0.00 [0.00 to 3.13] | 0.00 [0.00 to 24.71]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 1.28 [0.25 to 3.78] | 3.85 [0.18 to 17.30] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 0.90 [0.09 to 3.43] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.28]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 1.35 [0.24 to 4.12] | 2.00 [0.00 to 21.99] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 0.68 [0.00 to 4.94] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 3.29 [2.50 to 4.24] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 2.81 [2.04 to 3.78] | 0.00 [0.00 to 45.93] | 10.00 [0.00 to 75.66]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 2.47 [1.82 to 3.27] | 0.00 [0.00 to 70.76] | 5.88 [0.15 to 28.69]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 2.00 [0.99 to 3.58] | 2.44 [0.06 to 12.86] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 2.28 [1.18 to 3.95] | 0.00 [0.00 to 4.56] | 0.00 [0.00 to 70.76]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 1.47 [0.49 to 3.33] | 1.54 [0.04 to 8.28] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 2.19 [0.81 to 4.71] | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 1.86 [0.16 to 7.37] | 3.13 [0.00 to 88.31] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 1.80 [0.09 to 8.23] | 2.70 [0.00 to 99.67] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

40. Primary Outcome: Cumulative Incidence Rates of Musculoskeletal Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Musculoskeletal adverse events include any musculoskeletal adverse events, arthropathy, and muscle aches/myalgia. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.17] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [lower limit 0.00]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.41 [0.01 to 2.26]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.41 [0.01 to 2.24]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.40 [0.01 to 2.20]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.40 [0.01 to 2.20]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 4.59 [3.10 to 6.51] | 0.00 [0.00 to 84.19] | 11.11 [0.19 to 51.19]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 3.68 [2.63 to 4.99] | 0.00 [0.00 to 70.76] | 6.67 [0.17 to 31.95]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 3.24 [2.55 to 4.06] | 0.00 [0.00 to 45.93] | 5.00 [0.10 to 26.11]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 3.11 [2.57 to 3.71] | 4.62 [0.96 to 12.90] | 3.45 [0.05 to 19.42]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 2.88 [2.39 to 3.45] | 1.94 [0.40 to 5.55] | 2.56 [0.05 to 14.20]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 2.79 [2.24 to 3.45] | 1.16 [0.24 to 3.35] | 2.33 [0.06 to 12.41]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 2.83 [2.28 to 3.48] | 0.80 [0.17 to 2.32] | 1.79 [0.05 to 9.55]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 2.74 [2.15 to 3.45] | 1.32 [0.49 to 2.86] | 1.56 [0.04 to 8.40]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 2.67 [2.11 to 3.33] | 1.18 [0.43 to 2.55] | 1.02 [0.02 to 5.93]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 2.61 [2.07 to 3.26] | 1.25 [0.51 to 2.57] | 0.98 [0.02 to 5.69]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 2.57 [2.04 to 3.19] | 1.17 [0.45 to 2.47] | 0.85 [0.02 to 4.96]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 2.53 [2.00 to 3.14] | 1.12 [0.41 to 2.41] | 0.83 [0.01 to 4.93]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 3.29 [2.50 to 4.24] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 3.04 [2.48 to 3.70] | 0.00 [0.00 to 36.94] | 5.00 [0.01 to 35.33]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 2.80 [2.21 to 3.50] | 0.00 [0.00 to 28.49] | 5.41 [0.66 to 18.19]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 2.66 [2.14 to 3.27] | 1.92 [0.05 to 10.26] | 4.08 [0.50 to 13.98]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 2.61 [2.09 to 3.23] | 0.76 [0.02 to 4.18] | 3.85 [0.47 to 13.21]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 2.55 [2.02 to 3.16] | 1.02 [0.12 to 3.64] | 3.51 [0.43 to 12.11]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 2.54 [2.01 to 3.16] | 0.72 [0.09 to 2.58] | 3.33 [0.41 to 11.53]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 2.51 [2.04 to 3.05] | 1.17 [0.32 to 2.98] | 3.13 [0.35 to 11.09]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 2.49 [2.01 to 3.05] | 1.32 [0.43 to 3.06] | 2.38 [0.15 to 10.17]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 2.46 [1.98 to 3.02] | 1.20 [0.30 to 3.22] | 2.22 [0.12 to 9.92]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 2.44 [1.96 to 3.00] | 1.13 [0.24 to 3.21] | 2.15 [0.11 to 9.70]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 2.42 [1.94 to 2.99] | 1.08 [0.22 to 3.13] | 2.11 [0.11 to 9.58]

41. Primary Outcome: Weekly Incidence Rates of Neurological Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Neurological adverse events include any neurological adverse events, Bell's palsy, Guillain-Barre Syndrome, peripheral tremor and seizure/febrile convulsions. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.91] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.85] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.59] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 0.28 [0.03 to 1.00] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 0.35 [0.04 to 1.25] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 0.14 [0.00 to 0.86] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 0.00 [0.00 to 0.50] | 1.69 [0.04 to 9.09] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 0.16 [0.00 to 0.93] | 1.11 [0.03 to 6.04] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.04] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 0.00 [0.00 to 1.68] | 0.00 [0.00 to 3.13] | 0.00 [0.00 to 24.71]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 0.00 [0.00 to 1.17] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.28]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 0.29 [0.09 to 0.67] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 0.22 [0.05 to 0.59] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 30.85]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 0.19 [0.06 to 0.44] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 19.51]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 0.00 [0.00 to 0.28] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 0.20 [0.00 to 1.21] | 0.00 [0.00 to 4.56] | 33.33 [0.00 to 99.94]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 0.00 [0.00 to 0.67] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 0.23 [0.00 to 1.90] | 0.00 [0.00 to 5.60] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

42. Primary Outcome: Cumulative Incidence Rates of Neurological Adverse Events Reported Via ADR Card, by Vaccine and Age Group
Description: AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Neurological adverse events include any neurological adverse events, Bell's palsy, Guillain-Barre Syndrome, peripheral tremor and seizure/febrile convulsions. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.17] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.50]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.49]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.46]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.46]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 0.28 [0.03 to 1.00] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 0.32 [0.07 to 0.89] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 0.23 [0.07 to 0.57] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 16.84]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 0.19 [0.05 to 0.51] | 1.54 [0.04 to 8.28] | 0.00 [0.00 to 11.94]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 0.18 [0.05 to 0.45] | 1.29 [0.16 to 4.58] | 0.00 [0.00 to 9.03]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 0.17 [0.05 to 0.43] | 0.77 [0.09 to 2.76] | 0.00 [0.00 to 8.22]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 0.16 [0.04 to 0.41] | 0.53 [0.06 to 1.91] | 0.00 [0.00 to 6.38]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 0.15 [0.04 to 0.39] | 0.44 [0.05 to 1.59] | 0.00 [0.00 to 5.60]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 0.15 [0.04 to 0.38] | 0.39 [0.05 to 1.41] | 0.00 [0.00 to 3.69]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 0.14 [0.04 to 0.36] | 0.36 [0.04 to 1.29] | 0.00 [0.00 to 3.55]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 0.14 [0.04 to 0.36] | 0.34 [0.04 to 1.21] | 0.00 [0.00 to 3.10]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 0.13 [0.04 to 0.35] | 0.32 [0.04 to 1.15] | 0.00 [0.00 to 3.00]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 0.29 [0.09 to 0.67] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 0.25 [0.11 to 0.48] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 16.84]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 0.22 [0.12 to 0.39] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 9.49]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 0.19 [0.09 to 0.33] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 7.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 0.19 [0.10 to 0.31] | 0.00 [0.00 to 2.78] | 1.92 [0.00 to 15.59]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 0.18 [0.09 to 0.30] | 0.00 [0.00 to 1.86] | 1.75 [0.00 to 13.94]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 0.17 [0.09 to 0.29] | 0.00 [0.00 to 1.32] | 1.67 [0.00 to 13.08]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 0.17 [0.09 to 0.29] | 0.00 [0.00 to 1.08] | 1.56 [0.01 to 11.81]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 0.17 [0.09 to 0.29] | 0.00 [0.00 to 0.97] | 1.19 [0.00 to 9.68]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 0.17 [0.09 to 0.29] | 0.00 [0.00 to 0.88] | 1.11 [0.00 to 9.22]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 0.17 [0.09 to 0.28] | 0.00 [0.00 to 0.83] | 1.08 [0.00 to 8.81]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 0.16 [0.09 to 0.28] | 0.00 [0.00 to 0.79] | 1.05 [0.00 to 8.66]

43. Primary Outcome: Weekly Incidence Rates of Serious Adverse Events (SAEs) Reported Via ADR Card, by Vaccine and Age Group
Description: SAE data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. The weekly incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any SAEs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 5
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 1
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 191 | 4
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.91] | 0.00 [0.00 to 60.24]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 203 | 13
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 24.71]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 113 | 5
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 3.21] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 8
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 36.94]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 20 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 4
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 29 | 11
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 28.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 24 | 4
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 0
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] |
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 94 | 0
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.85] |
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 101 | 0
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.59] |
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 52 | 2
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 84.19]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 10
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 1
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 31
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 5
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 37 | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 38: number analyzed (Participants) | 859 | 1 | 6
  18 - 65 years, Week 38 | 0.00 [0.00 to 0.43] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 3 | 5
  18 - 65 years, Week 39 | 0.00 [0.00 to 0.26] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 52.18]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 59 | 9
  18 - 65 years, Week 40 | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 90 | 10
  18 - 65 years, Week 41 | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 42: number analyzed (Participants) | 354 | 104 | 4
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.04] | 0.00 [0.00 to 3.48] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 43: number analyzed (Participants) | 218 | 116 | 13
  18 - 65 years, Week 43 | 0.00 [0.00 to 1.68] | 0.00 [0.00 to 3.13] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 78 | 8
  18 - 65 years, Week 44 | 0.00 [0.00 to 1.17] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 36.94]
  18 - 65 years, Week 45: number analyzed (Participants) | 222 | 55 | 34
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.28]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 50 | 4
  18 - 65 years, Week 46 | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 60.24]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 38 | 15
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 4
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 37: number analyzed (Participants) | 1734 | 1 | 7
  >65 years, Week 37 | 0.00 [0.00 to 0.21] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 40.96]
  >65 years, Week 38: number analyzed (Participants) | 1848 | 6 | 10
  >65 years, Week 38 | 0.00 [0.00 to 0.20] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 30.85]
  >65 years, Week 39: number analyzed (Participants) | 2673 | 3 | 17
  >65 years, Week 39 | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 19.51]
  >65 years, Week 40: number analyzed (Participants) | 1301 | 41 | 12
  >65 years, Week 40 | 0.00 [0.00 to 0.28] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 26.46]
  >65 years, Week 41: number analyzed (Participants) | 1009 | 79 | 3
  >65 years, Week 41 | 0.00 [0.00 to 0.36] | 0.00 [0.00 to 4.56] | 0.00 [0.00 to 70.76]
  >65 years, Week 42: number analyzed (Participants) | 546 | 65 | 5
  >65 years, Week 42 | 0.00 [0.00 to 0.67] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 52.18]
  >65 years, Week 43: number analyzed (Participants) | 274 | 81 | 3
  >65 years, Week 43 | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 70.76]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 4
  >65 years, Week 44 | 0.00 [0.00 to 0.85] | 0.00 [0.00 to 5.60] | 0.00 [0.00 to 60.24]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 20
  >65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 16.84]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 6
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 45.93]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 3
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 70.76]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 2
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 84.19]

44. Primary Outcome: Cumulative Incidence Rates of SAEs Reported Via ADR Card, by Vaccine and Age Group
Description: SAE data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. The cumulative incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any SAEs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 6
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 45.93]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 7
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 40.96]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 584 | 11
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 28.49]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 727 | 16
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 930 | 29
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 11.94]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1059 | 31
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 11.22]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1172 | 36
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 9.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1244 | 44
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 8.04]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1273 | 48
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 7.40]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 20 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.84] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 41 | 4
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 70 | 15
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 21.80]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 94 | 19
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 119 | 19
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 213 | 19
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 314 | 19
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.17] | 0.00 [0.00 to 17.65]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 366 | 21
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 16.11]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 381 | 31
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 11.22]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 400 | 31
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.92] | 0.00 [0.00 to 11.22]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 2
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 33
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 33
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.58]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 34
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 10.28]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 39
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 9.03]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 244
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.50]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 246
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.49]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 251
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.46]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 251
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.46]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 2 | 9
  18 - 65 years, Week 35-37 | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 33.63]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1578 | 3 | 15
  18 - 65 years, Week 35-38 | 0.00 [0.00 to 0.23] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 21.80]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2993 | 6 | 20
  18 - 65 years, Week 35-39 | 0.00 [0.00 to 0.12] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 16.84]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3734 | 65 | 29
  18 - 65 years, Week 35-40 | 0.00 [0.00 to 0.10] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 11.94]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4369 | 155 | 39
  18 - 65 years, Week 35-41 | 0.00 [0.00 to 0.08] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 9.03]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4723 | 259 | 43
  18 - 65 years, Week 35-42 | 0.00 [0.00 to 0.08] | 0.00 [0.00 to 1.41] | 0.00 [0.00 to 8.22]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4941 | 375 | 56
  18 - 65 years, Week 35-43 | 0.00 [0.00 to 0.07] | 0.00 [0.00 to 0.98] | 0.00 [0.00 to 6.38]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5254 | 453 | 64
  18 - 65 years, Week 35-44 | 0.00 [0.00 to 0.07] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 5.60]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5476 | 508 | 98
  18 - 65 years, Week 35-45 | 0.00 [0.00 to 0.07] | 0.00 [0.00 to 0.72] | 0.00 [0.00 to 3.69]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5699 | 558 | 102
  18 - 65 years, Week 35-46 | 0.00 [0.00 to 0.06] | 0.00 [0.00 to 0.66] | 0.00 [0.00 to 3.55]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5845 | 596 | 117
  18 - 65 years, Week 35-47 | 0.00 [0.00 to 0.06] | 0.00 [0.00 to 0.62] | 0.00 [0.00 to 3.10]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5933 | 625 | 121
  18 - 65 years, Week 35-48 | 0.00 [0.00 to 0.06] | 0.00 [0.00 to 0.59] | 0.00 [0.00 to 3.00]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  >65 years, Week 35-37: number analyzed (Participants) | 1735 | 2 | 10
  >65 years, Week 35-37 | 0.00 [0.00 to 0.21] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 30.85]
  >65 years, Week 35-38: number analyzed (Participants) | 3583 | 8 | 20
  >65 years, Week 35-38 | 0.00 [0.00 to 0.10] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 16.84]
  >65 years, Week 35-39: number analyzed (Participants) | 6256 | 11 | 37
  >65 years, Week 35-39 | 0.00 [0.00 to 0.06] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 9.49]
  >65 years, Week 35-40: number analyzed (Participants) | 7557 | 52 | 49
  >65 years, Week 35-40 | 0.00 [0.00 to 0.05] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 7.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8566 | 131 | 52
  >65 years, Week 35-41 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 2.78] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-42: number analyzed (Participants) | 9112 | 196 | 57
  >65 years, Week 35-42 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 6.27]
  >65 years, Week 35-43: number analyzed (Participants) | 9386 | 277 | 60
  >65 years, Week 35-43 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 5.96]
  >65 years, Week 35-44: number analyzed (Participants) | 9816 | 341 | 64
  >65 years, Week 35-44 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 5.60]
  >65 years, Week 35-45: number analyzed (Participants) | 10038 | 378 | 84
  >65 years, Week 35-45 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 4.30]
  >65 years, Week 35-46: number analyzed (Participants) | 10152 | 415 | 90
  >65 years, Week 35-46 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 0.88] | 0.00 [0.00 to 4.02]
  >65 years, Week 35-47: number analyzed (Participants) | 10258 | 442 | 93
  >65 years, Week 35-47 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 0.83] | 0.00 [0.00 to 3.89]
  >65 years, Week 35-48: number analyzed (Participants) | 10310 | 464 | 95
  >65 years, Week 35-48 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 3.81]

45. Primary Outcome: Weekly Incidence Rates of Any AEIs Reported Via ADR Card, by Vaccine Group and United Kingdom Chief Medical Officer (UK CMO)-Specified Risk Status
Description: as for outcome 1
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 9.94 [8.24 to 11.87] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 7.56 [5.85 to 9.58] | 14.29 [0.00 to 90.97] | 15.38 [1.47 to 48.44]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 7.79 [6.95 to 8.69] | 0.00 [0.00 to 4.06] | 4.17 [0.11 to 21.12]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 8.14 [4.89 to 12.57] | 5.14 [2.97 to 8.22] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 6.43 [4.46 to 8.92] | 3.67 [1.08 to 8.82] | 2.78 [0.07 to 14.53]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 4.13 [1.91 to 7.68] | 1.42 [0.35 to 3.82] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 4.72 [2.00 to 9.26] | 2.15 [0.66 to 5.09] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 4.41 [1.31 to 10.49] | 2.92 [0.61 to 8.30] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 3.69 [1.48 to 7.50] | 2.32 [0.05 to 12.57] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 2.60 [0.72 to 6.52] | 0.87 [0.00 to 6.67] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 1.42 [0.26 to 4.32] | 0.73 [0.02 to 4.06] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 12.78 [7.63 to 19.67] |  | 50.00 [0.00 to 100]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 9.70 [5.40 to 15.75] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 10.00 [6.17 to 15.10] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 9.14 [4.45 to 16.21] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 6.10 [1.66 to 15.01] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 3.92 [0.34 to 14.93] | 5.77 [0.44 to 22.18] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 4.35 [0.91 to 12.18] | 9.43 [2.00 to 25.09] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 4.05 [0.64 to 12.73] | 2.00 [0.10 to 9.21] | 2.29 [0.75 to 5.27]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 9.88 [2.59 to 24.02] | 8.57 [1.80 to 23.06] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 2.17 [0.01 to 16.04] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

46. Primary Outcome: Cumulative Incidence Rates of Any AEIs Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 2
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 9.94 [8.23 to 11.87] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 8.70 [7.07 to 10.56] | 9.09 [0.08 to 47.67] | 7.14 [0.68 to 25.29]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 8.30 [7.13 to 9.59] | 1.00 [0.03 to 5.45] | 5.77 [1.21 to 15.95]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 8.27 [7.09 to 9.57] | 4.14 [2.39 to 6.61] | 3.80 [0.70 to 11.27]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 8.04 [6.86 to 9.36] | 3.94 [2.11 to 6.65] | 3.48 [0.88 to 9.02]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 7.79 [6.57 to 9.16] | 3.11 [1.57 to 5.47] | 3.08 [0.70 to 8.37]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 7.69 [6.44 to 9.09] | 2.88 [1.38 to 5.25] | 2.78 [0.61 to 7.71]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 7.53 [6.28 to 8.94] | 2.89 [1.24 to 5.66] | 2.31 [0.45 to 6.76]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 7.43 [6.19 to 8.83] | 2.81 [1.19 to 5.54] | 1.85 [0.31 to 5.77]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 7.34 [6.07 to 8.78] | 2.62 [0.98 to 5.58] | 1.75 [0.28 to 5.54]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 7.26 [5.97 to 8.72] | 2.51 [0.91 to 5.45] | 1.53 [0.27 to 4.71]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 7.20 [5.91 to 8.67] | 2.43 [0.88 to 5.28] | 1.48 [0.25 to 4.61]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 12.78 [7.63 to 19.67] |  | 50.00 [0.00 to 100]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 11.07 [7.75 to 15.20] |  | 28.57 [3.67 to 70.96]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 10.50 [7.61 to 14.02] | 0.00 [0.00 to 52.18] | 28.57 [3.67 to 70.96]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 10.21 [7.67 to 13.25] | 0.00 [0.00 to 11.22] | 18.18 [1.26 to 58.58]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 9.52 [7.05 to 12.50] | 0.00 [0.00 to 5.21] | 6.45 [0.79 to 21.42]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 8.74 [6.60 to 11.30] | 0.00 [0.00 to 3.05] | 6.06 [0.74 to 20.23]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 8.52 [6.46 to 10.98] | 1.75 [0.36 to 5.04] | 4.88 [0.60 to 16.53]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 8.28 [6.26 to 10.68] | 3.57 [1.55 to 6.92] | 4.76 [0.58 to 16.16]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 8.03 [6.11 to 10.32] | 3.09 [1.49 to 5.60] | 2.69 [1.09 to 5.47]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 8.14 [6.25 to 10.38] | 3.62 [1.94 to 6.11] | 2.63 [1.06 to 5.35]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 7.94 [6.10 to 10.13] | 3.43 [1.84 to 5.79] | 2.55 [1.03 to 5.19]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 7.77 [5.90 to 9.99] | 3.29 [1.76 to 5.56] | 2.55 [1.03 to 5.17]

47. Primary Outcome: Weekly Incidence Rates of Fever/Pyrexia Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 3
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 0.39 [0.17 to 0.76] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 0.43 [0.13 to 1.05] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 24.71]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 0.48 [0.21 to 0.91] | 0.00 [0.00 to 4.06] | 0.00 [0.00 to 14.25]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 0.27 [0.09 to 0.62] | 1.29 [0.12 to 4.97] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 0.40 [0.15 to 0.87] | 0.67 [0.08 to 2.39] | 0.00 [0.00 to 9.74]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 0.00 [0.00 to 0.45] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 0.45 [0.05 to 1.63] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 0.29 [0.02 to 1.34] | 0.49 [0.06 to 1.75] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 0.37 [0.00 to 2.71] | 0.00 [0.00 to 1.60] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 0.47 [0.00 to 3.37] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 1.50 [0.18 to 5.33] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 1.82 [0.30 to 5.77] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 0.29 [0.01 to 1.63] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 1.14 [0.02 to 6.55] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 0.00 [0.00 to 2.22] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 6.72] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.46 [0.01 to 2.53]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 1.23 [0.00 to 9.48] | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

48. Primary Outcome: Cumulative Incidence Rates of Fever/Pyrexia Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 4
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 0.39 [0.17 to 0.76] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 0.41 [0.24 to 0.65] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 12.34]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 0.44 [0.24 to 0.74] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 6.85]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 0.41 [0.24 to 0.66] | 0.97 [0.04 to 4.78] | 0.00 [0.00 to 4.56]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 0.41 [0.26 to 0.61] | 0.84 [0.19 to 2.34] | 0.00 [0.00 to 3.16]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 0.38 [0.24 to 0.58] | 0.56 [0.10 to 1.79] | 0.00 [0.00 to 2.80]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 0.38 [0.24 to 0.58] | 0.43 [0.06 to 1.50] | 0.00 [0.00 to 2.53]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 0.38 [0.24 to 0.57] | 0.44 [0.11 to 1.20] | 0.00 [0.00 to 2.11]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 0.37 [0.23 to 0.56] | 0.38 [0.08 to 1.09] | 0.00 [0.00 to 1.69]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 0.37 [0.23 to 0.56] | 0.34 [0.07 to 1.01] | 0.00 [0.00 to 1.60]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 0.37 [0.23 to 0.56] | 0.32 [0.06 to 0.96] | 0.00 [0.00 to 1.40]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 0.37 [0.23 to 0.55] | 0.31 [0.06 to 0.94] | 0.00 [0.00 to 1.35]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 1.50 [0.18 to 5.33] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 1.68 [0.36 to 4.74] |  | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 0.94 [0.20 to 2.69] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 0.98 [0.24 to 2.64] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 28.49]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 0.82 [0.19 to 2.27] | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 11.22]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 0.75 [0.16 to 2.14] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 0.72 [0.15 to 2.08] | 0.00 [0.00 to 2.13] | 0.00 [0.00 to 8.60]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 0.68 [0.13 to 2.01] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 8.41]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 0.64 [0.12 to 1.91] | 0.00 [0.00 to 1.13] | 0.38 [0.01 to 2.12]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 0.67 [0.11 to 2.18] | 0.00 [0.00 to 1.02] | 0.38 [0.01 to 2.08]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 0.65 [0.10 to 2.10] | 0.00 [0.00 to 0.97] | 0.36 [0.01 to 2.02]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 0.64 [0.10 to 2.06] | 0.00 [0.00 to 0.93] | 0.36 [0.01 to 2.01]

49. Primary Outcome: Weekly Incidence Rates of Local Symptoms Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 5
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 1.67 [0.58 to 3.73] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 1.33 [0.65 to 2.40] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 24.71]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 1.77 [1.24 to 2.46] | 0.00 [0.00 to 4.06] | 0.00 [0.00 to 14.25]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 1.70 [0.72 to 3.39] | 0.32 [0.00 to 2.12] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 1.54 [0.98 to 2.30] | 1.00 [0.14 to 3.40] | 0.00 [0.00 to 9.74]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 0.61 [0.10 to 1.96] | 0.57 [0.07 to 2.07] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 0.45 [0.05 to 1.67] | 0.61 [0.04 to 2.66] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 0.88 [0.13 to 2.95] | 0.49 [0.06 to 1.75] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 0.79 [0.07 to 3.18] | 0.66 [0.00 to 4.57] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 0.74 [0.09 to 2.70] | 0.44 [0.00 to 3.38] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 0.94 [0.05 to 4.24] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 5.26 [1.54 to 12.59] |  | 25.00 [0.00 to 100]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 6.06 [2.82 to 11.16] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 3.24 [1.06 to 7.38] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 4.57 [1.62 to 9.92] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 0.61 [0.00 to 4.32] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 0.00 [0.00 to 6.98] | 1.92 [0.05 to 10.26] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 4.35 [0.91 to 12.18] | 1.89 [0.05 to 10.07] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 1.68]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 3.70 [0.08 to 40] | 5.71 [0.70 to 19.16] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 2.17 [0.01 to 16.04] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

50. Primary Outcome: Cumulative Incidence Rates of Local Symptoms Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 6
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 1.67 [0.58 to 3.72] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 1.49 [0.78 to 2.57] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 12.34]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 1.61 [1.02 to 2.42] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 6.85]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 1.63 [1.05 to 2.41] | 0.24 [0.01 to 1.35] | 0.00 [0.00 to 4.56]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 1.62 [1.10 to 2.29] | 0.56 [0.04 to 2.40] | 0.00 [0.00 to 3.16]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 1.55 [1.10 to 2.13] | 0.56 [0.05 to 2.26] | 0.00 [0.00 to 2.80]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 1.52 [1.08 to 2.07] | 0.58 [0.05 to 2.32] | 0.00 [0.00 to 2.53]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 1.49 [1.07 to 2.01] | 0.56 [0.07 to 1.99] | 0.00 [0.00 to 2.11]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 1.47 [1.06 to 1.98] | 0.57 [0.11 to 1.73] | 0.00 [0.00 to 1.69]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 1.45 [1.05 to 1.96] | 0.56 [0.09 to 1.81] | 0.00 [0.00 to 1.60]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 1.45 [1.05 to 1.95] | 0.53 [0.08 to 1.72] | 0.00 [0.00 to 1.40]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 1.44 [1.04 to 1.93] | 0.51 [0.08 to 1.66] | 0.00 [0.00 to 1.35]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 5.26 [1.54 to 12.59] |  | 25.00 [0.00 to 100]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 5.70 [2.72 to 10.36] |  | 14.29 [0.04 to 71.51]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 4.39 [1.96 to 8.34] | 0.00 [0.00 to 52.18] | 14.29 [0.04 to 71.51]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 4.43 [2.31 to 7.59] | 0.00 [0.00 to 11.22] | 9.09 [0.00 to 65.53]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 3.79 [2.04 to 6.37] | 0.00 [0.00 to 5.21] | 3.23 [0.00 to 33.66]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 3.48 [1.94 to 5.72] | 0.00 [0.00 to 3.05] | 3.03 [0.00 to 26.51]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 3.32 [1.89 to 5.37] | 0.58 [0.01 to 3.22] | 2.44 [0.01 to 17.96]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 3.38 [2.04 to 5.24] | 0.89 [0.11 to 3.19] | 2.38 [0.01 to 17.83]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 3.18 [1.93 to 4.92] | 0.62 [0.07 to 2.21] | 0.38 [0.00 to 5.26]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 3.21 [2.16 to 4.59] | 1.11 [0.30 to 2.83] | 0.38 [0.00 to 4.72]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 3.18 [2.14 to 4.52] | 1.06 [0.29 to 2.68] | 0.36 [0.00 to 4.34]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 3.11 [2.09 to 4.44] | 1.01 [0.28 to 2.57] | 0.36 [0.00 to 4.33]

51. Primary Outcome: Weekly Incidence Rates of General Non-specific Symptoms Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, headache, irritability and malaise. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 3.86 [3.11 to 4.72] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 2.96 [2.02 to 4.19] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 24.71]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 2.78 [2.18 to 3.49] | 0.00 [0.00 to 4.06] | 4.17 [0.11 to 21.12]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 2.39 [1.75 to 3.19] | 1.61 [0.31 to 4.76] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 1.74 [0.95 to 2.92] | 1.33 [0.18 to 4.53] | 0.00 [0.00 to 9.74]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 1.70 [0.59 to 3.80] | 0.28 [0.01 to 1.58] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 2.02 [0.63 to 4.79] | 0.92 [0.06 to 3.98] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 1.76 [0.74 to 3.52] | 0.97 [0.09 to 3.76] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 1.06 [0.19 to 3.22] | 0.99 [0.06 to 4.45] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 0.37 [0.00 to 2.71] | 0.44 [0.00 to 3.38] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 4.51 [1.67 to 9.56] |  | 25.00 [0.00 to 99.42]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 3.03 [0.99 to 6.93] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 4.71 [1.62 to 10.38] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 2.86 [0.76 to 7.27] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 1.83 [0.23 to 6.42] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 0.00 [0.00 to 6.98] | 1.92 [0.05 to 10.26] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 3.77 [0.17 to 17.08] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 1.35 [0.01 to 9.52] | 1.00 [0.00 to 15.27] | 0.46 [0.01 to 2.53]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 1.23 [0.00 to 9.48] | 2.86 [0.07 to 14.92] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

52. Primary Outcome: Cumulative Incidence Rates of General Non-specific Symptoms Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 8
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 3.86 [3.11 to 4.72] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 3.39 [2.57 to 4.38] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 12.34]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 3.12 [2.36 to 4.04] | 0.00 [0.00 to 3.62] | 1.92 [0.05 to 10.26]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 2.99 [2.29 to 3.84] | 1.22 [0.37 to 2.91] | 1.27 [0.03 to 6.85]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 2.84 [2.15 to 3.67] | 1.27 [0.33 to 3.30] | 0.87 [0.01 to 5.18]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 2.77 [2.07 to 3.61] | 0.94 [0.25 to 2.41] | 0.77 [0.01 to 4.74]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 2.74 [2.04 to 3.61] | 0.94 [0.20 to 2.67] | 0.69 [0.01 to 4.39]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 2.69 [1.98 to 3.57] | 0.94 [0.18 to 2.86] | 0.58 [0.00 to 3.95]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 2.65 [1.95 to 3.51] | 0.95 [0.20 to 2.71] | 0.46 [0.00 to 3.33]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 2.61 [1.91 to 3.48] | 0.90 [0.16 to 2.77] | 0.44 [0.00 to 3.19]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 2.57 [1.87 to 3.44] | 0.85 [0.15 to 2.63] | 0.38 [0.00 to 2.86]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 2.55 [1.86 to 3.42] | 0.82 [0.15 to 2.54] | 0.37 [0.00 to 2.79]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 4.51 [1.67 to 9.56] |  | 25.00 [0.00 to 99.42]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 3.69 [1.86 to 6.51] |  | 14.29 [0.35 to 58.19]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 4.23 [2.22 to 7.23] | 0.00 [0.00 to 52.18] | 14.29 [0.35 to 58.19]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 3.94 [2.30 to 6.24] | 0.00 [0.00 to 11.22] | 9.09 [0.05 to 50.77]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 3.58 [1.95 to 5.98] | 0.00 [0.00 to 5.21] | 3.23 [0.08 to 16.70]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 3.29 [1.78 to 5.51] | 0.00 [0.00 to 3.05] | 3.03 [0.08 to 15.76]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 3.14 [1.71 to 5.26] | 0.58 [0.01 to 3.22] | 2.44 [0.06 to 12.86]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 2.96 [1.57 to 5.02] | 1.34 [0.28 to 3.86] | 2.38 [0.06 to 12.57]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 2.86 [1.59 to 4.72] | 1.23 [0.34 to 3.13] | 0.77 [0.09 to 2.75]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 2.76 [1.49 to 4.66] | 1.39 [0.45 to 3.22] | 0.75 [0.09 to 2.69]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 2.67 [1.43 to 4.54] | 1.32 [0.43 to 3.05] | 0.73 [0.09 to 2.61]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 2.61 [1.39 to 4.45] | 1.27 [0.41 to 2.93] | 0.73 [0.09 to 2.60]

53. Primary Outcome: Weekly Incidence Rates of Respiratory/Miscellaneous Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 9
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 5.62 [4.72 to 6.63] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38 | 3.86 [2.98 to 4.91] | 14.29 [0.00 to 90.97] | 7.69 [0.19 to 36.03]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 4.03 [3.26 to 4.91] | 0.00 [0.00 to 4.06] | 0.00 [0.00 to 14.25]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 4.68 [2.70 to 7.49] | 2.89 [0.64 to 8.00] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 3.35 [2.14 to 4.97] | 2.33 [0.79 to 5.27] | 0.00 [0.00 to 9.74]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 2.31 [1.05 to 4.37] | 0.57 [0.07 to 2.04] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 2.92 [0.97 to 6.65] | 1.53 [0.50 to 3.54] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 2.50 [0.55 to 6.92] | 1.95 [0.53 to 4.90] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 1.32 [0.35 to 3.40] | 1.32 [0.01 to 9.00] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 0.74 [0.05 to 3.22] | 0.44 [0.00 to 3.38] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 1.42 [0.26 to 4.32] | 0.73 [0.02 to 4.06] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 8.27 [4.20 to 14.32] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 4.24 [1.72 to 8.55] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 6.47 [2.73 to 12.64] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 3.43 [1.27 to 7.31] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 3.05 [1.00 to 6.97] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 0.00 [0.00 to 6.98] | 3.85 [0.30 to 15.08] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 1.45 [0.01 to 10.55] | 3.77 [0.46 to 12.98] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 4.05 [0.64 to 12.73] | 0.00 [0.00 to 3.62] | 2.29 [0.75 to 5.27]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 3.70 [0.77 to 10.44] | 5.71 [0.70 to 19.16] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 2.17 [0.01 to 16.04] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

54. Primary Outcome: Cumulative Incidence Rates of Respiratory/Miscellaneous Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 10
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 5.61 [4.71 to 6.62] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 4.69 [3.96 to 5.53] | 9.09 [0.08 to 47.67] | 3.57 [0.08 to 18.86]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 4.40 [3.75 to 5.13] | 1.00 [0.03 to 5.45] | 1.92 [0.05 to 10.26]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 4.45 [3.71 to 5.30] | 2.43 [0.53 to 6.77] | 1.27 [0.03 to 6.85]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 4.32 [3.56 to 5.18] | 2.39 [0.94 to 4.93] | 0.87 [0.01 to 5.18]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 4.19 [3.41 to 5.09] | 1.79 [0.69 to 3.74] | 0.77 [0.01 to 4.74]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 4.15 [3.34 to 5.08] | 1.73 [0.81 to 3.22] | 0.69 [0.01 to 4.39]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 4.07 [3.27 to 4.99] | 1.78 [0.91 to 3.13] | 0.58 [0.00 to 3.95]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 3.99 [3.20 to 4.92] | 1.71 [0.79 to 3.23] | 0.46 [0.00 to 3.33]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 3.93 [3.12 to 4.89] | 1.59 [0.71 to 3.05] | 0.44 [0.00 to 3.19]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 3.90 [3.09 to 4.85] | 1.54 [0.69 to 2.96] | 0.38 [0.00 to 2.86]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 3.87 [3.06 to 4.82] | 1.49 [0.66 to 2.87] | 0.37 [0.00 to 2.79]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 8.27 [4.20 to 14.32] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 6.04 [3.59 to 9.43] |  | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 6.27 [3.96 to 9.35] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 5.66 [3.70 to 8.24] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 28.49]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 5.22 [3.64 to 7.22] | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 11.22]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 4.79 [3.37 to 6.59] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 4.57 [3.25 to 6.23] | 1.17 [0.14 to 4.16] | 0.00 [0.00 to 8.60]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 4.39 [3.15 to 5.94] | 1.79 [0.49 to 4.51] | 0.00 [0.00 to 8.41]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 4.37 [3.26 to 5.72] | 1.23 [0.34 to 3.13] | 1.92 [0.63 to 4.43]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 4.33 [3.31 to 5.56] | 1.67 [0.62 to 3.60] | 1.88 [0.61 to 4.33]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 4.26 [3.26 to 5.46] | 1.58 [0.58 to 3.41] | 1.82 [0.60 to 4.21]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 4.17 [3.19 to 5.34] | 1.52 [0.56 to 3.28] | 1.82 [0.59 to 4.19]

55. Primary Outcome: Weekly Incidence Rates of Gastrointestinal Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 11
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 2.01 [1.33 to 2.93] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 1.64 [0.89 to 2.75] | 14.29 [0.00 to 90.97] | 0.00 [0.00 to 24.71]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 1.27 [0.80 to 1.92] | 0.00 [0.00 to 4.06] | 0.00 [0.00 to 14.25]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 1.44 [0.87 to 2.23] | 1.29 [0.35 to 3.26] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 1.14 [0.58 to 2.01] | 0.67 [0.08 to 2.39] | 0.00 [0.00 to 9.74]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 0.73 [0.21 to 1.82] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 0.45 [0.04 to 1.77] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 0.44 [0.09 to 1.28] | 0.24 [0.00 to 1.50] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 1.58 [0.27 to 4.95] | 0.66 [0.00 to 4.57] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 1.12 [0.07 to 4.86] | 0.00 [0.00 to 1.60] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 2.26 [0.23 to 8.42] |  | 25.00 [0.00 to 99.42]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 1.82 [0.21 to 6.56] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 2.06 [0.68 to 4.71] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 0.57 [0.01 to 3.31] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 1.22 [0.03 to 6.81] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 1.89 [0.05 to 10.07] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 2.00 [0.10 to 9.21] | 0.46 [0.01 to 2.53]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

56. Primary Outcome: Cumulative Incidence Rates of Gastrointestinal Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhea, nausea, and vomiting. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 2.01 [1.33 to 2.93] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 1.82 [1.39 to 2.33] | 9.09 [0.08 to 47.67] | 0.00 [0.00 to 12.34]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 1.58 [1.12 to 2.15] | 1.00 [0.03 to 5.45] | 0.00 [0.00 to 6.85]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 1.55 [1.17 to 2.02] | 1.22 [0.40 to 2.82] | 0.00 [0.00 to 4.56]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 1.50 [1.12 to 1.96] | 0.98 [0.35 to 2.17] | 0.00 [0.00 to 3.16]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 1.45 [1.09 to 1.90] | 0.66 [0.23 to 1.46] | 0.00 [0.00 to 2.80]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 1.42 [1.06 to 1.86] | 0.50 [0.16 to 1.20] | 0.00 [0.00 to 2.53]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 1.37 [1.02 to 1.80] | 0.44 [0.10 to 1.25] | 0.00 [0.00 to 2.11]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 1.38 [1.05 to 1.77] | 0.48 [0.17 to 1.06] | 0.00 [0.00 to 1.69]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 1.37 [1.05 to 1.77] | 0.43 [0.13 to 1.02] | 0.00 [0.00 to 1.60]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 1.35 [1.03 to 1.75] | 0.41 [0.12 to 0.97] | 0.00 [0.00 to 1.40]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 1.34 [1.02 to 1.73] | 0.39 [0.12 to 0.94] | 0.00 [0.00 to 1.35]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 2.26 [0.23 to 8.42] |  | 25.00 [0.00 to 99.42]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 2.01 [0.38 to 6.01] |  | 14.29 [0.35 to 58.19]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 2.04 [0.66 to 4.71] | 0.00 [0.00 to 52.18] | 14.29 [0.35 to 58.19]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 1.72 [0.58 to 3.91] | 0.00 [0.00 to 11.22] | 9.09 [0.05 to 50.77]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 977 | 31
  Not at risk, Week 35-41 | 1.64 [0.64 to 3.41] | 0.00 [0.00 to 5.21] | 3.23 [0.08 to 16.70]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 1.50 [0.57 to 3.19] | 0.00 [0.00 to 3.05] | 3.03 [0.08 to 15.76]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 1.43 [0.54 to 3.05] | 0.00 [0.00 to 2.13] | 2.44 [0.06 to 12.86]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 1.35 [0.49 to 2.96] | 0.45 [0.01 to 2.46] | 2.38 [0.06 to 12.57]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 1.27 [0.45 to 2.80] | 0.93 [0.19 to 2.68] | 0.77 [0.09 to 2.75]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 1.19 [0.41 to 2.69] | 0.84 [0.17 to 2.42] | 0.75 [0.09 to 2.69]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 1.16 [0.39 to 2.61] | 0.79 [0.16 to 2.30] | 0.73 [0.09 to 2.61]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 1.13 [0.39 to 2.55] | 0.76 [0.16 to 2.20] | 0.73 [0.09 to 2.60]

57. Primary Outcome: Weekly Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial edema, and hypersensitivity reactions. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 0.64 [0.01 to 4.30] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 0.51 [0.05 to 1.93] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 24.71]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 0.29 [0.02 to 1.34] | 0.00 [0.00 to 4.06] | 0.00 [0.00 to 14.25]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 0.43 [0.06 to 1.40] | 0.64 [0.01 to 4.22] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 0.20 [0.04 to 0.60] | 0.67 [0.08 to 2.39] | 0.00 [0.00 to 9.74]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 0.00 [0.00 to 0.45] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 0.22 [0.00 to 1.52] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 0.29 [0.02 to 1.34] | 0.24 [0.00 to 1.50] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 0.37 [0.00 to 2.68] | 0.00 [0.00 to 1.60] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 0.75 [0.01 to 5.16] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 1.21 [0.15 to 4.31] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 1.18 [0.17 to 3.93] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 0.00 [0.00 to 2.09] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 0.61 [0.01 to 3.69] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 3.77 [0.17 to 17.08] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.46 [0.01 to 2.53]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

58. Primary Outcome: Cumulative Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial edema, and hypersensitivity reactions. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 0.64 [0.01 to 4.30] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 0.57 [0.02 to 2.84] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 12.34]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 0.45 [0.02 to 2.15] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 6.85]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 0.45 [0.03 to 1.99] | 0.49 [0.01 to 2.67] | 0.00 [0.00 to 4.56]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 0.42 [0.03 to 1.77] | 0.56 [0.04 to 2.40] | 0.00 [0.00 to 3.16]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 0.39 [0.03 to 1.68] | 0.38 [0.03 to 1.51] | 0.00 [0.00 to 2.80]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 0.38 [0.03 to 1.63] | 0.29 [0.02 to 1.16] | 0.00 [0.00 to 2.53]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 0.38 [0.03 to 1.54] | 0.28 [0.02 to 1.22] | 0.00 [0.00 to 2.11]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 0.37 [0.03 to 1.50] | 0.24 [0.01 to 1.12] | 0.00 [0.00 to 1.69]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 0.37 [0.03 to 1.52] | 0.21 [0.01 to 1.06] | 0.00 [0.00 to 1.60]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 0.36 [0.03 to 1.50] | 0.20 [0.01 to 1.01] | 0.00 [0.00 to 1.40]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 0.36 [0.03 to 1.49] | 0.20 [0.01 to 0.97] | 0.00 [0.00 to 1.35]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 0.75 [0.01 to 5.16] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 1.01 [0.18 to 3.13] |  | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 1.10 [0.21 to 3.29] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 0.86 [0.12 to 2.89] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 28.49]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 0.82 [0.15 to 2.52] | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 11.22]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 0.75 [0.12 to 2.39] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 0.72 [0.11 to 2.31] | 0.00 [0.00 to 2.13] | 0.00 [0.00 to 8.60]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 0.68 [0.10 to 2.23] | 0.89 [0.11 to 3.19] | 0.00 [0.00 to 8.41]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 0.64 [0.09 to 2.11] | 0.62 [0.07 to 2.21] | 0.38 [0.01 to 2.12]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 0.60 [0.09 to 2.01] | 0.56 [0.07 to 2.00] | 0.38 [0.01 to 2.08]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 0.58 [0.08 to 1.94] | 0.53 [0.06 to 1.89] | 0.36 [0.01 to 2.02]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 0.56 [0.08 to 1.89] | 0.51 [0.06 to 1.82] | 0.36 [0.01 to 2.01]

59. Primary Outcome: Weekly Incidence Rates of Rash Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 1
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 0.51 [0.23 to 1.00] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 0.23 [0.08 to 0.53] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 24.71]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 0.16 [0.06 to 0.35] | 0.00 [0.00 to 4.06] | 0.00 [0.00 to 14.25]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 0.48 [0.22 to 0.91] | 0.00 [0.00 to 1.18] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 0.13 [0.02 to 0.48] | 0.33 [0.01 to 1.84] | 0.00 [0.00 to 9.74]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 0.00 [0.00 to 0.45] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 0.45 [0.03 to 1.87] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 0.44 [0.03 to 2.00] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 1.60] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 0.75 [0.01 to 4.87] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 1.21 [0.10 to 4.88] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 0.59 [0.05 to 2.42] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 0.00 [0.00 to 2.09] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 0.00 [0.00 to 2.22] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 6.72] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 1.68]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 1.23 [0.01 to 8.69] | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

60. Primary Outcome: Cumulative Incidence Rates of Rash Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 2
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 0.51 [0.23 to 1.00] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 0.37 [0.16 to 0.72] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 12.34]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 0.28 [0.15 to 0.47] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 6.85]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 0.31 [0.21 to 0.46] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 4.56]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 0.29 [0.19 to 0.42] | 0.14 [0.00 to 0.78] | 0.00 [0.00 to 3.16]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 0.27 [0.18 to 0.39] | 0.09 [0.00 to 0.52] | 0.00 [0.00 to 2.80]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 0.28 [0.19 to 0.40] | 0.07 [0.00 to 0.40] | 0.00 [0.00 to 2.53]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 0.29 [0.19 to 0.41] | 0.06 [0.00 to 0.31] | 0.00 [0.00 to 2.11]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 0.28 [0.19 to 0.40] | 0.05 [0.00 to 0.26] | 0.00 [0.00 to 1.69]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 0.27 [0.18 to 0.39] | 0.04 [0.00 to 0.24] | 0.00 [0.00 to 1.60]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 0.27 [0.18 to 0.38] | 0.04 [0.00 to 0.23] | 0.00 [0.00 to 1.40]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 0.27 [0.18 to 0.38] | 0.04 [0.00 to 0.22] | 0.00 [0.00 to 1.35]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 0.75 [0.01 to 4.87] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 1.01 [0.21 to 2.91] |  | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 0.78 [0.21 to 2.02] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 0.62 [0.18 to 1.53] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 28.49]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 0.51 [0.15 to 1.26] | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 11.22]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 0.47 [0.14 to 1.14] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 0.45 [0.14 to 1.07] | 0.00 [0.00 to 2.13] | 0.00 [0.00 to 8.60]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 0.42 [0.13 to 1.02] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 8.41]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 0.40 [0.12 to 0.96] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 1.41]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 0.45 [0.16 to 0.97] | 0.00 [0.00 to 1.02] | 0.00 [0.00 to 1.38]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 0.43 [0.16 to 0.94] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 1.34]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 0.42 [0.16 to 0.92] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 1.33]

61. Primary Outcome: Weekly Incidence Rates of Musculoskeletal Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 17
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 3.51 [2.79 to 4.37] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 2.81 [2.03 to 3.78] | 0.00 [0.00 to 40.96] | 7.69 [0.00 to 57.26]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 2.41 [1.90 to 3.02] | 0.00 [0.00 to 4.06] | 4.17 [0.11 to 21.12]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 2.02 [1.37 to 2.88] | 1.29 [0.01 to 8.32] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 1.94 [1.20 to 2.96] | 0.00 [0.00 to 1.22] | 0.00 [0.00 to 9.74]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 1.70 [0.66 to 3.56] | 0.28 [0.01 to 1.58] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 2.70 [1.36 to 4.75] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 1.76 [0.42 to 4.74] | 0.97 [0.01 to 5.90] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 1.32 [0.17 to 4.62] | 0.33 [0.00 to 2.45] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 0.37 [0.01 to 2.19] | 0.00 [0.00 to 1.60] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 0.47 [0.00 to 3.37] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 6.02 [2.38 to 12.21] |  | 25.00 [0.00 to 100]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 3.03 [0.99 to 6.93] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 4.12 [1.40 to 9.18] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 4.00 [1.42 to 8.69] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 41 | 4.00 [1.42 to 8.69] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 3.92 [0.34 to 14.93] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 1.89 [1.89 to 10.07] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 1.35 [0.01 to 9.52] | 0.00 [0.00 to 3.62] | 0.46 [0.01 to 2.53]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 2.47 [0.07 to 12.65] | 2.86 [0.07 to 14.92] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

62. Primary Outcome: Cumulative Incidence Rates of Musculoskeletal Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 18
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 3.51 [2.78 to 4.37] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 3.14 [2.41 to 4.03] | 0.00 [0.00 to 28.49] | 3.57 [0.01 to 24.71]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 2.82 [2.20 to 3.57] | 0.00 [0.00 to 3.62] | 3.85 [0.47 to 13.21]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 2.68 [2.19 to 3.25] | 0.97 [0.02 to 5.30] | 2.53 [0.31 to 8.85]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 2.59 [2.08 to 3.18] | 0.56 [0.04 to 2.40] | 1.74 [0.17 to 6.55]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 2.53 [2.01 to 3.15] | 0.47 [0.04 to 1.88] | 1.54 [0.15 to 5.92]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 2.54 [2.02 to 3.14] | 0.36 [0.03 to 1.45] | 1.39 [0.12 to 5.49]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 2.50 [2.00 to 3.09] | 0.50 [0.03 to 2.19] | 1.16 [0.08 to 4.94]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 2.47 [1.97 to 3.06] | 0.48 [0.02 to 2.24] | 0.93 [0.05 to 4.23]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 2.43 [1.93 to 3.01] | 0.43 [0.02 to 2.12] | 0.87 [0.04 to 4.08]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 2.40 [1.91 to 2.98] | 0.41 [0.02 to 2.01] | 0.76 [0.05 to 3.40]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 2.38 [1.89 to 2.96] | 0.39 [0.02 to 1.94] | 0.74 [0.04 to 3.35]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 6.02 [2.38 to 12.21] |  | 25.00 [0.00 to 100]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 4.36 [2.34 to 7.34] |  | 14.29 [0.04 to 71.51]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 4.23 [2.26 to 7.15] | 0.00 [0.00 to 52.18] | 14.29 [0.04 to 71.51]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 4.18 [2.41 to 6.71] | 0.00 [0.00 to 11.22] | 9.09 [0.00 to 65.53]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 3.89 [2.35 to 6.02] | 0.00 [0.00 to 5.21] | 3.23 [0.00 to 33.66]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 3.57 [2.21 to 5.44] | 0.00 [0.00 to 3.05] | 3.03 [0.00 to 26.51]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 3.59 [2.28 to 5.36] | 0.00 [0.00 to 2.13] | 2.44 [0.01 to 17.96]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 3.38 [2.18 to 4.99] | 0.45 [0.01 to 2.46] | 2.38 [0.01 to 17.83]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 3.26 [2.14 to 4.75] | 0.31 [0.01 to 1.71] | 0.77 [0.04 to 3.45]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 3.21 [2.19 to 4.53] | 0.56 [0.07 to 2.00] | 0.75 [0.06 to 3.14]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 3.10 [2.08 to 4.45] | 0.53 [0.06 to 1.89] | 0.73 [0.06 to 2.93]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 3.04 [2.01 to 4.38] | 0.51 [0.06 to 1.82] | 0.73 [0.06 to 2.92]

63. Primary Outcome: Weekly Incidence Rates of Neurological Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 19
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 0.21 [0.07 to 0.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 0.23 [0.08 to 0.51] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 24.71]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 0.19 [0.05 to 0.50] | 0.00 [0.00 to 4.06] | 0.00 [0.00 to 14.25]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 0.00 [0.00 to 0.20] | 0.32 [0.00 to 2.12] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 0.20 [0.03 to 0.66] | 0.33 [0.01 to 1.84] | 2.78 [0.07 to 14.53]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 0.00 [0.00 to 0.45] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 0.00 [0.00 to 0.83] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 0.15 [0.00 to 1.16] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 1.60] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 1.50 [0.18 to 5.33] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 0.61 [0.01 to 4.01] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 0.00 [0.00 to 2.09] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 0.00 [0.00 to 2.22] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 6.72] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 1.68]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

64. Primary Outcome: Cumulative Incidence Rates of Neurological Adverse Events Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 20
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 0.21 [0.07 to 0.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 0.22 [0.11 to 0.40] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 12.34]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 0.21 [0.09 to 0.40] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 6.85]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 0.17 [0.07 to 0.34] | 0.24 [0.01 to 1.35] | 0.00 [0.00 to 4.56]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 0.17 [0.09 to 0.31] | 0.28 [0.02 to 1.20] | 0.87 [0.02 to 5.09]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 0.16 [0.08 to 0.30] | 0.19 [0.02 to 0.76] | 0.77 [0.01 to 4.61]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 0.16 [0.08 to 0.29] | 0.14 [0.01 to 0.58] | 0.69 [0.01 to 4.07]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 0.16 [0.08 to 0.29] | 0.11 [0.01 to 0.49] | 0.58 [0.01 to 3.18]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 0.15 [0.07 to 0.28] | 0.10 [0.00 to 0.45] | 0.46 [0.01 to 2.55]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 0.15 [0.07 to 0.27] | 0.09 [0.00 to 0.42] | 0.44 [0.01 to 2.41]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 0.15 [0.07 to 0.27] | 0.08 [0.00 to 0.40] | 0.38 [0.01 to 2.11]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 0.15 [0.07 to 0.27] | 0.08 [0.00 to 0.39] | 0.37 [0.01 to 2.04]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 1.50 [0.18 to 5.33] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 1.01 [0.13 to 3.49] |  | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 0.47 [0.04 to 1.84] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 0.37 [0.03 to 1.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 28.49]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 0.31 [0.02 to 1.26] | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 11.22]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 0.28 [0.02 to 1.15] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 0.27 [0.02 to 1.08] | 0.00 [0.00 to 2.13] | 0.00 [0.00 to 8.60]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 0.25 [0.02 to 1.03] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 8.41]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 0.24 [0.02 to 0.97] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 1.41]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 0.22 [0.02 to 0.90] | 0.00 [0.00 to 1.02] | 0.00 [0.00 to 1.38]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 0.22 [0.02 to 0.88] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 1.34]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 0.21 [0.02 to 0.86] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 1.33]

65. Primary Outcome: Weekly Incidence Rates of SAEs Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: The weekly incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any SAEs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 37: number analyzed (Participants) | 2333 | 3 | 12
  At risk, Week 37 | 0.00 [0.00 to 0.16] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 26.46]
  At risk, Week 38: number analyzed (Participants) | 2565 | 7 | 13
  At risk, Week 38 | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 24.71]
  At risk, Week 39: number analyzed (Participants) | 3776 | 89 | 24
  At risk, Week 39 | 0.00 [0.00 to 0.10] | 0.00 [0.00 to 4.06] | 0.00 [0.00 to 14.25]
  At risk, Week 40: number analyzed (Participants) | 1880 | 311 | 27
  At risk, Week 40 | 0.00 [0.00 to 0.20] | 0.00 [0.00 to 1.18] | 0.00 [0.00 to 12.77]
  At risk, Week 41: number analyzed (Participants) | 1493 | 300 | 36
  At risk, Week 41 | 0.00 [0.00 to 0.25] | 0.00 [0.00 to 1.22] | 0.00 [0.00 to 9.74]
  At risk, Week 42: number analyzed (Participants) | 823 | 351 | 15
  At risk, Week 42 | 0.00 [0.00 to 0.45] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 21.80]
  At risk, Week 43: number analyzed (Participants) | 445 | 326 | 14
  At risk, Week 43 | 0.00 [0.00 to 0.83] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 23.16]
  At risk, Week 44: number analyzed (Participants) | 681 | 411 | 29
  At risk, Week 44 | 0.00 [0.00 to 0.54] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 11.94]
  At risk, Week 45: number analyzed (Participants) | 379 | 302 | 43
  At risk, Week 45 | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 8.22]
  At risk, Week 46: number analyzed (Participants) | 269 | 229 | 13
  At risk, Week 46 | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 1.60] | 0.00 [0.00 to 24.71]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 33
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 10.58]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 9
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 33.63]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 37 | 0.00 [0.00 to 2.74] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 0 | 3
  Not at risk, Week 38 | 0.00 [0.00 to 2.21] |  | 0.00 [0.00 to 70.76]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 5 | 0
  Not at risk, Week 39 | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 52.18] |
  Not at risk, Week 40: number analyzed (Participants) | 175 | 26 | 4
  Not at risk, Week 40 | 0.00 [0.00 to 2.09] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 60.24]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 38 | 20
  Not at risk, Week 41 | 0.00 [0.00 to 2.22] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 16.84]
  Not at risk, Week 42: number analyzed (Participants) | 87 | 50 | 2
  Not at risk, Week 42 | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 7.11] | 0.00 [0.00 to 84.19]
  Not at risk, Week 43: number analyzed (Participants) | 51 | 52 | 8
  Not at risk, Week 43 | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 36.94]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 53 | 1
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 6.72] | 0.00 [0.00 to 97.50]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 218
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 1.68]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 35 | 6
  Not at risk, Week 46 | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 45.93]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 20 | 8
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 36.94]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 1
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 97.50]

66. Primary Outcome: Cumulative Incidence Rates of SAEs Reported Via ADR Card, by Vaccine Group and UK CMO-specified Risk Status
Description: The cumulative incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any SAEs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16387 | 2946 | 546
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 3
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76]
  At risk, Week 35-37: number analyzed (Participants) | 2334 | 4 | 15
  At risk, Week 35-37 | 0.00 [0.00 to 0.16] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 21.80]
  At risk, Week 35-38: number analyzed (Participants) | 4899 | 11 | 28
  At risk, Week 35-38 | 0.00 [0.00 to 0.08] | 0.00 [0.00 to 28.49] | 0.00 [0.00 to 12.34]
  At risk, Week 35-39: number analyzed (Participants) | 8675 | 100 | 52
  At risk, Week 35-39 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 6.85]
  At risk, Week 35-40: number analyzed (Participants) | 10555 | 411 | 79
  At risk, Week 35-40 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 4.56]
  At risk, Week 35-41: number analyzed (Participants) | 12048 | 711 | 115
  At risk, Week 35-41 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.52] | 0.00 [0.00 to 3.16]
  At risk, Week 35-42: number analyzed (Participants) | 12871 | 1062 | 130
  At risk, Week 35-42 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 2.80]
  At risk, Week 35-43: number analyzed (Participants) | 13316 | 1388 | 144
  At risk, Week 35-43 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.27] | 0.00 [0.00 to 2.53]
  At risk, Week 35-44: number analyzed (Participants) | 13997 | 1799 | 173
  At risk, Week 35-44 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.20] | 0.00 [0.00 to 2.11]
  At risk, Week 35-45: number analyzed (Participants) | 14376 | 2101 | 216
  At risk, Week 35-45 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 1.69]
  At risk, Week 35-46: number analyzed (Participants) | 14645 | 2330 | 229
  At risk, Week 35-46 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.16] | 0.00 [0.00 to 1.60]
  At risk, Week 35-47: number analyzed (Participants) | 14857 | 2467 | 262
  At risk, Week 35-47 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 1.40]
  At risk, Week 35-48: number analyzed (Participants) | 14971 | 2551 | 271
  At risk, Week 35-48 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 1.35]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 4
  Not at risk, Week 35-37 | 0.00 [0.00 to 2.74] |  | 0.00 [0.00 to 60.24]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 0 | 7
  Not at risk, Week 35-38 | 0.00 [0.00 to 1.23] |  | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 5 | 7
  Not at risk, Week 35-39 | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 40.96]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 31 | 11
  Not at risk, Week 35-40 | 0.00 [0.00 to 0.45] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 28.49]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 69 | 31
  Not at risk, Week 35-41 | 0.00 [0.00 to 0.38] | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 11.22]
  Not at risk, Week 35-42: number analyzed (Participants) | 1064 | 119 | 33
  Not at risk, Week 35-42 | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-43: number analyzed (Participants) | 1115 | 171 | 41
  Not at risk, Week 35-43 | 0.00 [0.00 to 0.33] | 0.00 [0.00 to 2.13] | 0.00 [0.00 to 8.60]
  Not at risk, Week 35-44: number analyzed (Participants) | 1184 | 224 | 42
  Not at risk, Week 35-44 | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 8.41]
  Not at risk, Week 35-45: number analyzed (Participants) | 1258 | 324 | 260
  Not at risk, Week 35-45 | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 1.41]
  Not at risk, Week 35-46: number analyzed (Participants) | 1339 | 359 | 266
  Not at risk, Week 35-46 | 0.00 [0.00 to 0.28] | 0.00 [0.00 to 1.02] | 0.00 [0.00 to 1.38]
  Not at risk, Week 35-47: number analyzed (Participants) | 1385 | 379 | 274
  Not at risk, Week 35-47 | 0.00 [0.00 to 0.27] | 0.00 [0.00 to 0.97] | 0.00 [0.00 to 1.34]
  Not at risk, Week 35-48: number analyzed (Participants) | 1416 | 395 | 275
  Not at risk, Week 35-48 | 0.00 [0.00 to 0.26] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 1.33]

67. Secondary Outcome: Weekly Incidence Rates of Any AEIs Recorded in Electronic Health Record (EHR), by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from General Practitioners (GPs). The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on the Weekly Vaccinated cohort which included all subjects who were vaccinated with a seasonal influenza vaccine during the week of interest and were registered in EHR (combining routine data collection and card-based ADR reporting system) during the safety follow-up period (from vaccination up to 7 days post-vaccination).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Week 35: number analyzed (Participants) | 0 | 0 | 1
  Week 35 |  |  | 0.00 [0.00 to 97.50]
  Week 36: number analyzed (Participants) | 1 | 1 | 61
  Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.64 [0.00 to 15.62]
  Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Week 37 | 11.63 [9.72 to 13.77] | 0.00 [0.00 to 52.18] | 1.28 [0.40 to 3.00]
  Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Week 38 | 10.01 [7.49 to 13.03] | 10.00 [0.00 to 74.36] | 1.48 [0.64 to 2.89]
  Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Week 39 | 10.03 [8.81 to 11.36] | 1.89 [0.23 to 6.65] | 2.26 [0.90 to 4.64]
  Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Week 40 | 9.97 [6.19 to 14.98] | 7.31 [4.79 to 10.60] | 1.54 [0.46 to 3.74]
  Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Week 41 | 8.58 [6.13 to 11.61] | 5.54 [2.93 to 9.41] | 0.50 [0.06 to 1.86]
  Week 42: number analyzed (Participants) | 912 | 412 | 241
  Week 42 | 5.26 [2.93 to 8.62] | 2.18 [1.00 to 4.11] | 1.66 [0.21 to 5.75]
  Week 43: number analyzed (Participants) | 499 | 382 | 164
  Week 43 | 6.01 [2.73 to 11.23] | 4.45 [2.19 to 7.95] | 1.83 [0.38 to 5.25]
  Week 44: number analyzed (Participants) | 750 | 471 | 561
  Week 44 | 6.00 [2.35 to 12.24] | 5.94 [1.76 to 14.05] | 0.36 [0.04 to 1.28]
  Week 45: number analyzed (Participants) | 455 | 403 | 350
  Week 45 | 6.59 [3.97 to 10.20] | 3.23 [0.38 to 11.32] | 4.00 [2.04 to 6.98]
  Week 46: number analyzed (Participants) | 350 | 577 | 97
  Week 46 | 7.43 [3.88 to 12.65] | 1.56 [0.13 to 6.27] | 3.09 [0.24 to 12.26]
  Week 47: number analyzed (Participants) | 258 | 158 | 199
  Week 47 | 4.26 [1.74 to 8.55] | 3.16 [1.04 to 7.23] | 1.51 [0.16 to 5.60]
  Week 48: number analyzed (Participants) | 145 | 100 | 42
  Week 48 | 0.00 [0.00 to 2.51] | 5.00 [1.06 to 13.81] | 0.00 [0.00 to 8.41]

68. Secondary Outcome: Weekly Incidence Rates of Fever/Pyrexia Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Fever/pyrexia = all subjects with a fever/pyrexia read code recorded were considered as having fever/pyrexia, regardless of what temperature had been recorded. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Week 35: number analyzed (Participants) | 0 | 0 | 1
  Week 35 |  |  | 0.00 [0.00 to 97.50]
  Week 36: number analyzed (Participants) | 1 | 1 | 61
  Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Week 37 | 0.45 [0.20 to 0.85] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Week 38 | 0.54 [0.19 to 1.23] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Week 39 | 0.51 [0.21 to 1.04] | 0.00 [0.00 to 3.42] | 0.21 [0.00 to 1.50]
  Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Week 40 | 0.44 [0.11 to 1.19] | 1.46 [0.41 to 3.63] | 0.00 [0.00 to 0.63]
  Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Week 41 | 0.36 [0.13 to 0.78] | 0.58 [0.07 to 2.09] | 0.00 [0.00 to 0.92]
  Week 42: number analyzed (Participants) | 912 | 412 | 241
  Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Week 43: number analyzed (Participants) | 499 | 382 | 164
  Week 43 | 0.40 [0.05 to 1.46] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Week 44: number analyzed (Participants) | 750 | 471 | 561
  Week 44 | 0.27 [0.02 to 1.20] | 0.42 [0.05 to 1.53] | 0.00 [0.00 to 0.66]
  Week 45: number analyzed (Participants) | 455 | 403 | 350
  Week 45 | 0.22 [0.00 to 1.60] | 0.00 [0.00 to 0.91] | 0.29 [0.01 to 1.58]
  Week 46: number analyzed (Participants) | 350 | 577 | 97
  Week 46 | 0.57 [0.03 to 2.58] | 0.17 [0.00 to 1.71] | 0.00 [0.00 to 3.73]
  Week 47: number analyzed (Participants) | 258 | 158 | 199
  Week 47 | 0.39 [0.00 to 2.82] | 0.63 [0.01 to 4.02] | 0.00 [0.00 to 1.84]
  Week 48: number analyzed (Participants) | 145 | 100 | 42
  Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]

69. Secondary Outcome: Weekly Incidence Rates of Local Symptoms Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Local symptoms include local erythema. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Week 35: number analyzed (Participants) | 0 | 0 | 1
  Week 35 |  |  | 0.00 [0.00 to 97.50]
  Week 36: number analyzed (Participants) | 1 | 1 | 61
  Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Week 37 | 1.91 [0.82 to 3.74] | 0.00 [0.00 to 52.18] | 0.21 [0.01 to 1.18]
  Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Week 38 | 1.63 [0.89 to 2.75] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Week 39 | 1.94 [1.31 to 2.77] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Week 40 | 1.94 [0.77 to 4.02] | 0.29 [0.00 to 1.78] | 0.00 [0.00 to 0.63]
  Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Week 41 | 1.44 [0.93 to 2.14] | 0.87 [0.16 to 2.69] | 0.00 [0.00 to 0.92]
  Week 42: number analyzed (Participants) | 912 | 412 | 241
  Week 42 | 0.55 [0.09 to 1.78] | 0.49 [0.06 to 1.74] | 0.00 [0.00 to 1.52]
  Week 43: number analyzed (Participants) | 499 | 382 | 164
  Week 43 | 0.40 [0.04 to 1.49] | 0.79 [0.06 to 3.25] | 0.00 [0.00 to 2.22]
  Week 44: number analyzed (Participants) | 750 | 471 | 561
  Week 44 | 1.20 [0.25 to 3.43] | 0.64 [0.08 to 2.26] | 0.00 [0.00 to 0.66]
  Week 45: number analyzed (Participants) | 455 | 403 | 350
  Week 45 | 0.88 [0.15 to 2.76] | 0.50 [0.00 to 3.52] | 0.00 [0.00 to 1.05]
  Week 46: number analyzed (Participants) | 350 | 577 | 97
  Week 46 | 1.43 [0.20 to 4.82] | 0.52 [0.01 to 3.35] | 0.00 [0.00 to 3.73]
  Week 47: number analyzed (Participants) | 258 | 158 | 199
  Week 47 | 1.16 [0.06 to 5.45] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Week 48: number analyzed (Participants) | 145 | 100 | 42
  Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]

70. Secondary Outcome: Weekly Incidence Rates of General Non-specific Symptoms Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, headache, irritability, and malaise. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Any, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Any, Week 37 | 4.01 [3.23 to 4.92] | 0.00 [0.00 to 52.18] | 0.21 [0.00 to 1.80]
  Any, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Any, Week 38 | 3.19 [2.35 to 4.23] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Any, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Any, Week 39 | 3.30 [2.61 to 4.12] | 0.94 [0.02 to 5.14] | 0.41 [0.05 to 1.48]
  Any, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Any, Week 40 | 2.72 [2.06 to 3.52] | 2.34 [0.64 to 5.88] | 0.00 [0.00 to 0.63]
  Any, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Any, Week 41 | 1.98 [1.37 to 2.77] | 1.17 [0.21 to 3.57] | 0.00 [0.00 to 0.92]
  Any, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Any, Week 42 | 1.64 [0.58 to 3.64] | 0.49 [0.06 to 1.74] | 0.00 [0.00 to 1.52]
  Any, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Any, Week 43 | 2.00 [0.73 to 4.36] | 1.05 [0.08 to 4.32] | 0.00 [0.00 to 2.22]
  Any, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Any, Week 44 | 1.87 [0.74 to 3.85] | 1.70 [0.20 to 6.03] | 0.00 [0.00 to 0.66]
  Any, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Any, Week 45 | 1.54 [0.33 to 4.38] | 1.49 [0.27 to 4.57] | 1.43 [0.47 to 3.30]
  Any, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Any, Week 46 | 1.14 [0.31 to 2.91] | 0.35 [0.00 to 3.20] | 0.00 [0.00 to 3.73]
  Any, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Any, Week 47 | 0.39 [0.01 to 2.41] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Drowsiness, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Drowsiness, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Drowsiness, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Drowsiness, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Drowsiness, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Drowsiness, Week 37 | 1.05 [0.62 to 1.68] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Drowsiness, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Drowsiness, Week 38 | 0.80 [0.29 to 1.75] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Drowsiness, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Drowsiness, Week 39 | 0.63 [0.32 to 1.12] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Drowsiness, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Drowsiness, Week 40 | 0.68 [0.37 to 1.14] | 0.29 [0.01 to 1.62] | 0.00 [0.00 to 0.63]
  Drowsiness, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Drowsiness, Week 41 | 0.54 [0.25 to 1.02] | 0.58 [0.07 to 2.09] | 0.00 [0.00 to 0.92]
  Drowsiness, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Drowsiness, Week 42 | 0.33 [0.02 to 1.52] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Drowsiness, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Drowsiness, Week 43 | 0.80 [0.01 to 5.27] | 0.26 [0.01 to 1.45] | 0.00 [0.00 to 2.22]
  Drowsiness, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Drowsiness, Week 44 | 0.27 [0.02 to 1.18] | 0.42 [0.01 to 2.49] | 0.00 [0.00 to 0.66]
  Drowsiness, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Drowsiness, Week 45 | 0.22 [0.00 to 1.58] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Drowsiness, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Drowsiness, Week 46 | 0.00 [0.00 to 1.05] | 0.17 [0.00 to 1.61] | 0.00 [0.00 to 3.73]
  Drowsiness, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Drowsiness, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Drowsiness, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Drowsiness, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Fatigue, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Fatigue, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Fatigue, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Fatigue, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Fatigue, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Fatigue, Week 37 | 2.19 [1.65 to 2.85] | 0.00 [0.00 to 52.18] | 0.21 [0.00 to 1.80]
  Fatigue, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Fatigue, Week 38 | 1.89 [1.33 to 2.59] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Fatigue, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Fatigue, Week 39 | 1.80 [1.40 to 2.27] | 0.00 [0.00 to 3.42] | 0.21 [0.00 to 1.29]
  Fatigue, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Fatigue, Week 40 | 1.17 [0.60 to 2.03] | 0.58 [0.01 to 3.53] | 0.00 [0.00 to 0.63]
  Fatigue, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Fatigue, Week 41 | 1.20 [0.73 to 1.85] | 0.29 [0.01 to 1.61] | 0.00 [0.00 to 0.92]
  Fatigue, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Fatigue, Week 42 | 0.77 [0.08 to 2.91] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Fatigue, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Fatigue, Week 43 | 0.80 [0.14 to 2.52] | 0.52 [0.04 to 2.17] | 0.00 [0.00 to 2.22]
  Fatigue, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Fatigue, Week 44 | 0.67 [0.22 to 1.55] | 0.64 [0.10 to 2.06] | 0.00 [0.00 to 0.66]
  Fatigue, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Fatigue, Week 45 | 1.10 [0.19 to 3.42] | 0.50 [0.02 to 2.38] | 0.29 [0.01 to 1.58]
  Fatigue,Week 46: number analyzed (Participants) | 350 | 577 | 97
  Fatigue,Week 46 | 1.14 [0.31 to 2.91] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Fatigue,Week 47: number analyzed (Participants) | 258 | 158 | 199
  Fatigue,Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Fatigue,Week 48: number analyzed (Participants) | 145 | 100 | 42
  Fatigue,Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Headache, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Headache, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Headache, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Headache, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Headache, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Headache, Week 37 | 2.27 [1.61 to 3.11] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Headache, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Headache, Week 38 | 1.92 [1.11 to 3.08] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Headache, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Headache, Week 39 | 1.92 [1.29 to 2.73] | 0.94 [0.02 to 5.14] | 0.21 [0.00 to 1.15]
  Headache, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Headache, Week 40 | 1.60 [1.02 to 2.40] | 1.46 [0.07 to 6.71] | 0.00 [0.00 to 0.63]
  Headache, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Headache, Week 41 | 0.96 [0.55 to 1.55] | 0.87 [0.16 to 2.69] | 0.00 [0.00 to 0.92]
  Headache, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Headache, Week 42 | 0.88 [0.22 to 2.35] | 0.24 [0.01 to 1.34] | 0.00 [0.00 to 1.52]
  Headache, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Headache, Week 43 | 1.40 [0.43 to 3.37] | 0.79 [0.06 to 3.25] | 0.00 [0.00 to 2.22]
  Headache, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Headache, Week 44 | 1.47 [0.61 to 2.94] | 1.06 [0.26 to 2.85] | 0.00 [0.00 to 0.66]
  Headache, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Headache, Week 45 | 1.32 [0.17 to 4.59] | 0.99 [0.16 to 3.22] | 1.43 [0.47 to 3.30]
  Headache, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Headache, Week 46 | 0.29 [0.00 to 2.15] | 0.17 [0.00 to 1.61] | 0.00 [0.00 to 3.73]
  Headache, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Headache, Week 47 | 0.39 [0.01 to 2.41] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Headache, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Headache, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Irritability, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Irritability, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Irritability, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Irritability, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Irritability, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Irritability, Week 37 | 0.41 [0.19 to 0.74] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Irritability, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Irritability, Week 38 | 0.25 [0.09 to 0.55] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Irritability, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Irritability, Week 39 | 0.36 [0.11 to 0.88] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Irritability, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Irritability, Week 40 | 0.15 [0.03 to 0.43] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Irritability, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Irritability, Week 41 | 0.12 [0.01 to 0.43] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Irritability, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Irritability, Week 42 | 0.11 [0.00 to 0.79] | 0.24 [0.01 to 1.34] | 0.00 [0.00 to 1.52]
  Irritability, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Irritability, Week 43 | 0.20 [0.00 to 1.33] | 0.26 [0.01 to 1.45] | 0.00 [0.00 to 2.22]
  Irritability, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Irritability, Week 44 | 0.00 [0.00 to 0.49] | 0.42 [0.01 to 2.49] | 0.00 [0.00 to 0.66]
  Irritability, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Irritability, Week 45 | 0.44 [0.00 to 3.14] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Irritability, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Irritability, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Irritability, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Irritability, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Irritability, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Irritability, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Malaise, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Malaise, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Malaise, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Malaise, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Malaise, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Malaise, Week 37 | 0.04 [0.00 to 0.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Malaise, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Malaise, Week 38 | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Malaise, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Malaise, Week 39 | 0.00 [0.00 to 0.09] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Malaise, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Malaise, Week 40 | 0.05 [0.00 to 0.28] | 0.29 [0.01 to 1.62] | 0.00 [0.00 to 0.63]
  Malaise, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Malaise, Week 41 | 0.06 [0.00 to 0.37] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Malaise, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Malaise, Week 42 | 0.00 [0.00 to 0.40] | 0.24 [0.01 to 1.34] | 0.00 [0.00 to 1.52]
  Malaise, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Malaise, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Malaise, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Malaise, Week 44 | 0.00 [0.00 to 0.49] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Malaise, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Malaise, Week 45 | 0.00 [0.00 to 0.81] | 0.25 [0.00 to 1.77] | 0.00 [0.00 to 1.05]
  Malaise, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Malaise, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Malaise, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Malaise, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Malaise, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Malaise, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]

71. Secondary Outcome: Weekly Incidence Rates of Respiratory/Miscellaneous Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Respiratory/miscellaneous adverse events include any respiratory/miscellaneous adverse events, conjunctivitis, coryza, cough, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhoea and wheezing. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.64 [0.00 to 15.62]
  Any, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Any, Week 37 | 6.45 [5.26 to 7.80] | 0.00 [0.00 to 52.18] | 0.64 [0.07 to 2.39]
  Any, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Any, Week 38 | 4.86 [3.59 to 6.42] | 10.00 [0.00 to 74.36] | 0.55 [0.03 to 2.54]
  Any, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Any, Week 39 | 4.98 [4.33 to 5.69] | 0.94 [0.02 to 5.14] | 1.23 [0.34 to 3.12]
  Any, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Any, Week 40 | 5.30 [3.29 to 8.02] | 4.09 [2.26 to 6.77] | 1.03 [0.37 to 2.23]
  Any, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Any, Week 41 | 4.68 [3.48 to 6.15] | 3.79 [2.03 to 6.39] | 0.25 [0.00 to 1.66]
  Any, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Any, Week 42 | 2.52 [1.40 to 4.15] | 0.73 [0.15 to 2.13] | 1.66 [0.21 to 5.75]
  Any, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Any, Week 43 | 2.81 [0.88 to 6.58] | 2.88 [1.17 to 5.84] | 0.00 [0.00 to 2.22]
  Any, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Any, Week 44 | 3.07 [1.08 to 6.74] | 3.61 [1.41 to 7.45] | 0.36 [0.04 to 1.28]
  Any, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Any, Week 45 | 2.20 [0.63 to 5.41] | 1.24 [0.05 to 6.01] | 2.29 [0.99 to 4.45]
  Any, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Any, Week 46 | 2.86 [1.09 to 6.01] | 0.69 [0.02 to 3.73] | 0.00 [0.00 to 3.73]
  Any, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Any, Week 47 | 2.71 [0.51 to 8.06] | 1.27 [0.15 to 4.50] | 1.51 [0.16 to 5.60]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Any, Week 48 | 0.00 [0.00 to 2.51] | 2.00 [0.24 to 7.04] | 0.00 [0.00 to 8.41]
  Conjunctivitis, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Conjunctivitis, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Conjunctivitis, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Conjunctivitis, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Conjunctivitis, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Conjunctivitis, Week 37 | 0.24 [0.09 to 0.53] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Conjunctivitis, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Conjunctivitis, Week 38 | 0.51 [0.18 to 1.14] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Conjunctivitis, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Conjunctivitis, Week 39 | 0.32 [0.17 to 0.55] | 0.00 [0.00 to 3.42] | 0.21 [0.00 to 1.56]
  Conjunctivitis, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Conjunctivitis, Week 40 | 0.34 [0.14 to 0.70] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Conjunctivitis, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Conjunctivitis, Week 41 | 0.42 [0.09 to 1.19] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Conjunctivitis, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Conjunctivitis, Week 42 | 0.11 [0.00 to 0.79] | 0.24 [0.01 to 1.34] | 0.41 [0.00 to 3.24]
  Conjunctivitis, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Conjunctivitis, Week 43 | 0.20 [0.00 to 1.33] | 0.26 [0.01 to 1.45] | 0.00 [0.00 to 2.22]
  Conjunctivitis, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Conjunctivitis, Week 44 | 0.53 [0.11 to 1.53] | 0.21 [0.00 to 1.46] | 0.18 [0.00 to 0.99]
  Conjunctivitis, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Conjunctivitis, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.57 [0.07 to 2.05]
  Conjunctivitis, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Conjunctivitis, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Conjunctivitis, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Conjunctivitis, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Conjunctivitis, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Conjunctivitis, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Coryza, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Coryza, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Coryza, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Coryza, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Coryza, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Coryza, Week 37 | 1.38 [0.75 to 2.32] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Coryza, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Coryza, Week 38 | 0.94 [0.50 to 1.62] | 0.00 [0.00 to 30.85] | 0.18 [0.00 to 1.36]
  Coryza, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Coryza, Week 39 | 1.24 [0.85 to 1.75] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Coryza, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Coryza, Week 40 | 1.02 [0.63 to 1.56] | 1.46 [0.48 to 3.38] | 0.00 [0.00 to 0.63]
  Coryza, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Coryza, Week 41 | 1.26 [0.70 to 2.10] | 0.29 [0.01 to 1.61] | 0.00 [0.00 to 0.92]
  Coryza, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Coryza, Week 42 | 0.44 [0.12 to 1.12] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Coryza, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Coryza, Week 43 | 0.60 [0.04 to 2.61] | 0.79 [0.16 to 2.31] | 0.00 [0.00 to 2.22]
  Coryza, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Coryza, Week 44 | 0.67 [0.11 to 2.15] | 0.42 [0.05 to 1.53] | 0.00 [0.00 to 0.66]
  Coryza, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Coryza, Week 45 | 0.44 [0.00 to 3.14] | 0.25 [0.00 to 1.77] | 0.29 [0.01 to 1.58]
  Coryza, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Coryza, Week 46 | 0.86 [0.14 to 2.76] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Coryza, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Coryza, Week 47 | 0.78 [0.08 to 2.99] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Coryza, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Coryza, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Cough, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Cough, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Cough, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Cough, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.64 [0.00 to 15.62]
  Cough, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Cough, Week 37 | 2.31 [1.64 to 3.16] | 0.00 [0.00 to 52.18] | 0.64 [0.07 to 2.39]
  Cough, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Cough, Week 38 | 1.96 [1.36 to 2.72] | 0.00 [0.00 to 30.85] | 0.18 [0.00 to 1.36]
  Cough, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Cough, Week 39 | 2.31 [1.87 to 2.81] | 0.94 [0.02 to 5.14] | 1.03 [0.19 to 3.09]
  Cough, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Cough, Week 40 | 1.65 [0.74 to 3.18] | 2.63 [1.13 to 5.16] | 0.85 [0.22 to 2.25]
  Cough, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Cough, Week 41 | 2.04 [1.17 to 3.29] | 2.04 [0.82 to 4.16] | 0.25 [0.00 to 1.66]
  Cough, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Cough, Week 42 | 1.10 [0.53 to 2.01] | 0.24 [0.00 to 2.15] | 0.41 [0.00 to 3.45]
  Cough, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Cough, Week 43 | 1.20 [0.26 to 3.40] | 1.83 [0.74 to 3.74] | 0.00 [0.00 to 2.22]
  Cough, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Cough, Week 44 | 1.33 [0.59 to 2.58] | 2.12 [0.63 to 5.12] | 0.00 [0.00 to 0.66]
  Cough, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Cough, Week 45 | 1.32 [0.24 to 4.00] | 0.99 [0.06 to 4.42] | 0.86 [0.18 to 2.48]
  Cough, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Cough, Week 46 | 2.29 [0.91 to 4.69] | 0.35 [0.00 to 3.20] | 0.00 [0.00 to 3.73]
  Cough, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Cough, Week 47 | 1.55 [0.15 to 5.98] | 0.00 [0.00 to 2.31] | 1.01 [0.05 to 4.78]
  Cough, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Cough, Week 48 | 0.00 [0.00 to 2.51] | 2.00 [0.24 to 7.04] | 0.00 [0.00 to 8.41]
  Epistaxis, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Epistaxis, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Epistaxis, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Epistaxis, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Epistaxis, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Epistaxis, Week 37 | 0.08 [0.00 to 0.48] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Epistaxis, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Epistaxis, Week 38 | 0.04 [0.00 to 0.27] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Epistaxis, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Epistaxis, Week 39 | 0.12 [0.02 to 0.39] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Epistaxis, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Epistaxis, Week 40 | 0.15 [0.02 to 0.50] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Epistaxis, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Epistaxis, Week 41 | 0.06 [0.00 to 0.37] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Epistaxis, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Epistaxis, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Epistaxis, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Epistaxis, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Epistaxis, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Epistaxis, Week 44 | 0.27 [0.03 to 0.96] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Epistaxis, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Epistaxis, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Epistaxis, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Epistaxis, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Epistaxis, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Epistaxis, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Epistaxis, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Epistaxis, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Hoarseness, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Hoarseness, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Hoarseness, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Hoarseness, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Hoarseness, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Hoarseness, Week 37 | 1.09 [0.72 to 1.59] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Hoarseness, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Hoarseness, Week 38 | 0.83 [0.46 to 1.40] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Hoarseness, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Hoarseness, Week 39 | 0.53 [0.34 to 0.81] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Hoarseness, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Hoarseness, Week 40 | 0.49 [0.23 to 0.89] | 0.29 [0.01 to 1.62] | 0.00 [0.00 to 0.63]
  Hoarseness, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Hoarseness, Week 41 | 0.54 [0.12 to 1.53] | 0.58 [0.07 to 2.09] | 0.00 [0.00 to 0.92]
  Hoarseness, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Hoarseness, Week 42 | 0.22 [0.02 to 0.86] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Hoarseness, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Hoarseness, Week 43 | 0.80 [0.15 to 2.43] | 0.26 [0.01 to 1.45] | 0.00 [0.00 to 2.22]
  Hoarseness, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Hoarseness, Week 44 | 0.27 [0.02 to 1.20] | 0.21 [0.00 to 1.25] | 0.00 [0.00 to 0.66]
  Hoarseness, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Hoarseness, Week 45 | 0.66 [0.00 to 4.69] | 0.00 [0.00 to 0.91] | 0.29 [0.01 to 1.58]
  Hoarseness, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Hoarseness, Week 46 | 0.29 [0.00 to 1.91] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Hoarseness, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Hoarseness, Week 47 | 0.39 [0.00 to 2.82] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Hoarseness, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Hoarseness, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Nasal congestion, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Nasal congestion, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Nasal congestion, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Nasal congestion, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Nasal congestion, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Nasal congestion, Week 37 | 1.34 [0.92 to 1.87] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Nasal congestion, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Nasal congestion, Week 38 | 0.91 [0.51 to 1.49] | 0.00 [0.00 to 30.85] | 0.18 [0.00 to 1.36]
  Nasal congestion, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Nasal congestion, Week 39 | 0.95 [0.62 to 1.39] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Nasal congestion, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Nasal congestion, Week 40 | 0.88 [0.37 to 1.74] | 0.58 [0.04 to 2.49] | 0.00 [0.00 to 0.63]
  Nasal congestion, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Nasal congestion, Week 41 | 0.48 [0.21 to 0.94] | 0.87 [0.16 to 2.69] | 0.00 [0.00 to 0.92]
  Nasal congestion, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Nasal congestion, Week 42 | 0.44 [0.02 to 2.19] | 0.00 [0.00 to 0.89] | 0.41 [0.00 to 3.20]
  Nasal congestion, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Nasal congestion, Week 43 | 0.20 [0.00 to 1.37] | 0.79 [0.16 to 2.28] | 0.00 [0.00 to 2.22]
  Nasal congestion, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Nasal congestion, Week 44 | 0.27 [0.03 to 0.96] | 0.21 [0.00 to 1.46] | 0.00 [0.00 to 0.66]
  Nasal congestion, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Nasal congestion, Week 45 | 0.88 [0.14 to 2.81] | 0.25 [0.00 to 1.77] | 0.29 [0.01 to 1.58]
  Nasal congestion, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Nasal congestion, Week 46 | 0.86 [0.12 to 2.94] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Nasal congestion, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Nasal congestion, Week 47 | 0.78 [0.05 to 3.40] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Nasal congestion, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Nasal congestion, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Oropharyngeal pain, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Oropharyngeal pain, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Oropharyngeal pain, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Oropharyngeal pain, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Oropharyngeal pain, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Oropharyngeal pain, Week 37 | 2.27 [1.64 to 3.06] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Oropharyngeal pain, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Oropharyngeal pain, Week 38 | 1.38 [0.79 to 2.22] | 0.00 [0.00 to 30.85] | 0.18 [0.00 to 1.28]
  Oropharyngeal pain, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Oropharyngeal pain, Week 39 | 1.58 [1.22 to 2.01] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Oropharyngeal pain, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Oropharyngeal pain, Week 40 | 1.02 [0.48 to 1.91] | 0.29 [0.00 to 1.78] | 0.17 [0.00 to 1.48]
  Oropharyngeal pain, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Oropharyngeal pain, Week 41 | 1.20 [0.54 to 2.29] | 0.87 [0.16 to 2.69] | 0.00 [0.00 to 0.92]
  Oropharyngeal pain, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Oropharyngeal pain, Week 42 | 0.44 [0.07 to 1.43] | 0.24 [0.00 to 2.05] | 0.41 [0.00 to 3.14]
  Oropharyngeal pain, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Oropharyngeal pain, Week 43 | 0.60 [0.05 to 2.44] | 0.52 [0.04 to 2.17] | 0.00 [0.00 to 2.22]
  Oropharyngeal pain, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Oropharyngeal pain, Week 44 | 0.93 [0.22 to 2.56] | 0.64 [0.01 to 3.72] | 0.18 [0.00 to 0.99]
  Oropharyngeal pain, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Oropharyngeal pain, Week 45 | 0.88 [0.03 to 4.37] | 0.50 [0.00 to 3.52] | 0.57 [0.07 to 2.05]
  Oropharyngeal pain, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Oropharyngeal pain, Week 46 | 0.29 [0.00 to 1.91] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Oropharyngeal pain, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Oropharyngeal pain, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.50 [0.00 to 3.77]
  Oropharyngeal pain, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Oropharyngeal pain, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Rhinorrhoea, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Rhinorrhoea, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Rhinorrhoea, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Rhinorrhoea, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Rhinorrhoea, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Rhinorrhoea, Week 37 | 3.28 [2.18 to 4.74] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Rhinorrhoea, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Rhinorrhoea, Week 38 | 2.43 [1.71 to 3.35] | 10.00 [0.00 to 74.36] | 0.00 [0.00 to 0.68]
  Rhinorrhoea, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Rhinorrhoea, Week 39 | 2.26 [1.68 to 2.97] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Rhinorrhoea, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Rhinorrhoea, Week 40 | 2.43 [1.31 to 4.10] | 1.17 [0.22 to 3.53] | 0.00 [0.00 to 0.63]
  Rhinorrhoea, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Rhinorrhoea, Week 41 | 1.92 [1.19 to 2.92] | 1.75 [0.64 to 3.79] | 0.00 [0.00 to 0.92]
  Rhinorrhoea, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Rhinorrhoea, Week 42 | 0.99 [0.33 to 2.27] | 0.49 [0.06 to 1.74] | 0.00 [0.00 to 1.52]
  Rhinorrhoea, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Rhinorrhoea, Week 43 | 2.00 [0.48 to 5.36] | 1.57 [0.58 to 3.39] | 0.00 [0.00 to 2.22]
  Rhinorrhoea, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Rhinorrhoea, Week 44 | 1.47 [0.37 to 3.86] | 1.06 [0.25 to 2.89] | 0.00 [0.00 to 0.66]
  Rhinorrhoea, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Rhinorrhoea, Week 45 | 1.32 [0.38 to 3.24] | 0.50 [0.00 to 3.52] | 0.86 [0.18 to 2.48]
  Rhinorrhoea, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Rhinorrhoea, Week 46 | 1.14 [0.27 to 3.12] | 0.17 [0.00 to 1.61] | 0.00 [0.00 to 3.73]
  Rhinorrhoea, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Rhinorrhoea, Week 47 | 1.16 [0.06 to 5.45] | 0.63 [0.02 to 3.48] | 0.00 [0.00 to 1.84]
  Rhinorrhoea, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Rhinorrhoea, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Wheezing, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Wheezing, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Wheezing, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Wheezing, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Wheezing, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Wheezing, Week 37 | 0.93 [0.59 to 1.40] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Wheezing, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Wheezing, Week 38 | 0.58 [0.29 to 1.02] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Wheezing, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Wheezing, Week 39 | 0.41 [0.24 to 0.67] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Wheezing, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Wheezing, Week 40 | 0.63 [0.25 to 1.33] | 0.29 [0.01 to 1.62] | 0.00 [0.00 to 0.63]
  Wheezing, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Wheezing, Week 41 | 0.30 [0.08 to 0.78] | 0.58 [0.07 to 2.09] | 0.00 [0.00 to 0.92]
  Wheezing, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Wheezing, Week 42 | 0.22 [0.01 to 1.06] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Wheezing, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Wheezing, Week 43 | 0.20 [0.00 to 1.46] | 0.52 [0.04 to 2.17] | 0.00 [0.00 to 2.22]
  Wheezing, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Wheezing, Week 44 | 0.27 [0.03 to 0.96] | 1.06 [0.20 to 3.19] | 0.00 [0.00 to 0.66]
  Wheezing, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Wheezing, Week 45 | 0.22 [0.00 to 1.58] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Wheezing, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Wheezing, Week 46 | 0.00 [0.00 to 1.05] | 0.35 [0.04 to 1.25] | 0.00 [0.00 to 3.73]
  Wheezing, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Wheezing, Week 47 | 0.39 [0.01 to 2.44] | 0.63 [0.01 to 3.88] | 0.00 [0.00 to 1.84]
  Wheezing, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Wheezing, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]

72. Secondary Outcome: Weekly Incidence Rates of Gastrointestinal Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhoea, nausea, and vomiting. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Any, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Any, Week 37 | 2.11 [1.30 to 3.22] | 0.00 [0.00 to 52.18] | 0.21 [0.00 to 1.80]
  Any, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Any, Week 38 | 1.81 [1.08 to 2.84] | 10.00 [0.00 to 74.36] | 0.00 [0.00 to 0.68]
  Any, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Any, Week 39 | 1.51 [0.99 to 2.19] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Any, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Any, Week 40 | 1.46 [0.88 to 2.27] | 1.17 [0.32 to 2.97] | 0.00 [0.00 to 0.63]
  Any, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Any, Week 41 | 1.26 [0.63 to 2.24] | 0.58 [0.07 to 2.09] | 0.00 [0.00 to 0.92]
  Any, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Any, Week 42 | 1.10 [0.46 to 2.18] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Any, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Any, Week 43 | 0.80 [0.22 to 2.04] | 0.00 [0.00 to 0.96] | 0.61 [0.00 to 4.42]
  Any, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Any, Week 44 | 0.67 [0.22 to 1.55] | 0.42 [0.01 to 2.49] | 0.00 [0.00 to 0.66]
  Any, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Any, Week 45 | 1.98 [0.63 to 4.60] | 0.99 [0.15 to 3.23] | 0.86 [0.18 to 2.48]
  Any, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Any, Week 46 | 1.43 [0.18 to 5.01] | 0.17 [0.00 to 1.48] | 1.03 [0.01 to 6.91]
  Any, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Any, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Decreased appetite, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Decreased appetite, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Decreased appetite, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Decreased appetite, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Decreased appetite, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Decreased appetite, Week 37 | 0.73 [0.43 to 1.15] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Decreased appetite, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Decreased appetite, Week 38 | 0.47 [0.25 to 0.81] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Decreased appetite, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Decreased appetite, Week 39 | 0.46 [0.19 to 0.94] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Decreased appetite, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Decreased appetite, Week 40 | 0.34 [0.12 to 0.75] | 1.17 [0.32 to 2.97] | 0.00 [0.00 to 0.63]
  Decreased appetite, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Decreased appetite, Week 41 | 0.48 [0.13 to 1.23] | 0.29 [0.01 to 1.61] | 0.00 [0.00 to 0.92]
  Decreased appetite, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Decreased appetite, Week 42 | 0.22 [0.01 to 0.95] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Decreased appetite, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Decreased appetite, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Decreased appetite, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Decreased appetite, Week 44 | 0.13 [0.00 to 1.01] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Decreased appetite, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Decreased appetite, Week 45 | 0.66 [0.09 to 2.22] | 0.25 [0.00 to 1.77] | 0.00 [0.00 to 1.05]
  Decreased appetite, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Decreased appetite, Week 46 | 0.57 [0.04 to 2.38] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Decreased appetite, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Decreased appetite, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Decreased appetite, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Decreased appetite, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Diarrhoea, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Diarrhoea, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Diarrhoea, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Diarrhoea, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Diarrhoea, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Diarrhoea, Week 37 | 0.97 [0.58 to 1.54] | 0.00 [0.00 to 52.18] | 0.21 [0.00 to 1.80]
  Diarrhoea, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Diarrhoea, Week 38 | 0.76 [0.46 to 1.18] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Diarrhoea, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Diarrhoea, Week 39 | 0.68 [0.45 to 0.98] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Diarrhoea, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Diarrhoea, Week 40 | 0.68 [0.25 to 1.47] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Diarrhoea, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Diarrhoea, Week 41 | 0.66 [0.28 to 1.30] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Diarrhoea, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Diarrhoea, Week 42 | 0.44 [0.12 to 1.12] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Diarrhoea, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Diarrhoea, Week 43 | 0.40 [0.04 to 1.55] | 0.00 [0.00 to 0.96] | 0.61 [0.00 to 4.42]
  Diarrhoea, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Diarrhoea, Week 44 | 0.27 [0.01 to 1.27] | 0.21 [0.00 to 1.25] | 0.00 [0.00 to 0.66]
  Diarrhoea, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Diarrhoea, Week 45 | 0.66 [0.05 to 2.70] | 0.25 [0.01 to 1.37] | 0.29 [0.01 to 1.58]
  Diarrhoea, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Diarrhoea, Week 46 | 0.86 [0.07 to 3.46] | 0.00 [0.00 to 0.64] | 1.03 [0.01 to 6.91]
  Diarrhoea, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Diarrhoea, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Diarrhoea, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Diarrhoea, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Nausea, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Nausea, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Nausea, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Nausea, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Nausea, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Nausea, Week 37 | 0.97 [0.49 to 1.72] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Nausea, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Nausea, Week 38 | 1.05 [0.43 to 2.14] | 10 [0 to 74.36] | 0.00 [0.00 to 0.68]
  Nausea, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Nausea, Week 39 | 0.78 [0.35 to 1.50] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Nausea, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Nausea, Week 40 | 0.53 [0.23 to 1.05] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Nausea, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Nausea, Week 41 | 0.54 [0.25 to 1.02] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Nausea, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Nausea, Week 42 | 0.33 [0.02 to 1.47] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Nausea, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Nausea, Week 43 | 0.40 [0.04 to 1.61] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Nausea, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Nausea, Week 44 | 0.53 [0.15 to 1.36] | 0.21 [0.00 to 1.25] | 0.00 [0.00 to 0.66]
  Nausea, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Nausea, Week 45 | 0.88 [0.12 to 3.05] | 0.50 [0.02 to 2.38] | 0.29 [0.01 to 1.58]
  Nausea, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Nausea, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Nausea, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Nausea, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Nausea, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Nausea, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Vomiting, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Vomiting, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Vomiting, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Vomiting, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Vomiting, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Vomiting, Week 37 | 0.12 [0.02 to 0.38] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Vomiting, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Vomiting, Week 38 | 0.22 [0.08 to 0.48] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Vomiting, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Vomiting, Week 39 | 0.19 [0.08 to 0.38] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Vomiting, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Vomiting, Week 40 | 0.05 [0.00 to 0.28] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Vomiting, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Vomiting, Week 41 | 0.30 [0.05 to 0.92] | 0.29 [0.01 to 1.61] | 0.00 [0.00 to 0.92]
  Vomiting, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Vomiting, Week 42 | 0.33 [0.03 to 1.37] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Vomiting, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Vomiting, Week 43 | 0.20 [0.00 to 1.32] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Vomiting, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Vomiting, Week 44 | 0.13 [0.00 to 1.05] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Vomiting, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Vomiting, Week 45 | 0.44 [0.01 to 2.73] | 0.00 [0.00 to 0.91] | 0.57 [0.07 to 2.05]
  Vomiting, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Vomiting, Week 46 | 0.00 [0.00 to 1.05] | 0.17 [0.00 to 1.48] | 0.00 [0.00 to 3.73]
  Vomiting, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Vomiting, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Vomiting, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Vomiting, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]

73. Secondary Outcome: Weekly Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial edema, and hypersensitivity reactions. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Any, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Any, Week 37 | 0.69 [0.01 to 4.09] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Any, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Any, Week 38 | 0.58 [0.07 to 2.10] | 0.00 [0.00 to 30.85] | 0.18 [0.00 to 1.06]
  Any, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Any, Week 39 | 0.41 [0.04 to 1.65] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Any, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Any, Week 40 | 0.44 [0.05 to 1.59] | 0.58 [0.01 to 3.53] | 0.00 [0.00 to 0.63]
  Any, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Any, Week 41 | 0.24 [0.05 to 0.69] | 0.87 [0.16 to 2.69] | 0.00 [0.00 to 0.92]
  Any, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Any, Week 42 | 0.00 [0.00 to 0.40] | 0.24 [0.00 to 1.97] | 0.00 [0.00 to 1.52]
  Any, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Any, Week 43 | 0.20 [0.00 to 1.37] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Any, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Any, Week 44 | 0.27 [0.02 to 1.20] | 0.64 [0.01 to 3.72] | 0.00 [0.00 to 0.66]
  Any, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Any, Week 45 | 0.22 [0.00 to 1.58] | 0.00 [0.00 to 0.91] | 0.29 [0.01 to 1.58]
  Any, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Any, Week 46 | 0.29 [0.00 to 2.10] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Any, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Any, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Anaphylactic reactions, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Anaphylactic reactions, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Anaphylactic reactions, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Anaphylactic reactions, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Anaphylactic reactions, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Anaphylactic reactions, Week 37 | 0.61 [0.01 to 4.06] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Anaphylactic reactions, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Anaphylactic reactions, Week 38 | 0.44 [0.01 to 2.53] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Anaphylactic reactions, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Anaphylactic reactions, Week 39 | 0.29 [0.01 to 1.48] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Anaphylactic reactions, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Anaphylactic reactions, Week 40 | 0.19 [0.00 to 1.58] | 0.58 [0.01 to 3.53] | 0.00 [0.00 to 0.63]
  Anaphylactic reactions, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Anaphylactic reactions, Week 41 | 0.00 [0.00 to 0.22] | 0.58 [0.07 to 2.09] | 0.00 [0.00 to 0.92]
  Anaphylactic reactions, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Anaphylactic reactions, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Anaphylactic reactions, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Anaphylactic reactions, Week 43 | 0.20 [0.00 to 1.37] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Anaphylactic reactions, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Anaphylactic reactions, Week 44 | 0.00 [0.00 to 0.49] | 0.64 [0.01 to 3.72] | 0.00 [0.00 to 0.66]
  Anaphylactic reactions, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Anaphylactic reactions, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.29 [0.01 to 1.58]
  Anaphylactic reactions, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Anaphylactic reactions, Week 46 | 0.29 [0.00 to 2.10] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Anaphylactic reactions, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Anaphylactic reactions, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Anaphylactic reactions, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Anaphylactic reactions, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Facial oedema, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Facial oedema, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Facial oedema, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Facial oedema, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Facial oedema, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Facial oedema, Week 37 | 0.04 [0.00 to 0.27] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Facial oedema, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Facial oedema, Week 38 | 0.07 [0.01 to 0.26] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Facial oedema, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Facial oedema, Week 39 | 0.05 [0.00 to 0.20] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Facial oedema, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Facial oedema, Week 40 | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Facial oedema, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Facial oedema, Week 41 | 0.06 [0.00 to 0.45] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Facial oedema, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Facial oedema, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Facial oedema, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Facial oedema, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Facial oedema, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Facial oedema, Week 44 | 0.13 [0.00 to 0.74] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Facial oedema, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Facial oedema, Week 45 | 0.22 [0.00 to 1.58] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Facial oedema, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Facial oedema, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Facial oedema, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Facial oedema, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Facial oedema, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Facial oedema, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Hypersensitivity reactions, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Hypersensitivity reactions, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Hypersensitivity reactions, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Hypersensitivity reactions, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Hypersensitivity reactions, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Hypersensitivity reactions, Week 37 | 0.08 [0.01 to 0.29] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Hypersensitivity reactions, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Hypersensitivity reactions, Week 38 | 0.11 [0.02 to 0.36] | 0.00 [0.00 to 30.85] | 0.18 [0.00 to 1.06]
  Hypersensitivity reactions, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Hypersensitivity reactions, Week 39 | 0.07 [0.02 to 0.21] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Hypersensitivity reactions, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Hypersensitivity reactions, Week 40 | 0.24 [0.08 to 0.57] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Hypersensitivity reactions, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Hypersensitivity reactions, Week 41 | 0.24 [0.05 to 0.69] | 0.29 [0.01 to 1.61] | 0.00 [0.00 to 0.92]
  Hypersensitivity reactions, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Hypersensitivity reactions, Week 42 | 0.00 [0.00 to 0.40] | 0.24 [0.00 to 1.97] | 0.00 [0.00 to 1.52]
  Hypersensitivity reactions, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Hypersensitivity reactions, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Hypersensitivity reactions, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Hypersensitivity reactions, Week 44 | 0.13 [0.00 to 0.74] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Hypersensitivity reactions, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Hypersensitivity reactions, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Hypersensitivity reactions, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Hypersensitivity reactions, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Hypersensitivity reactions, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Hypersensitivity reactions, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Hypersensitivity reactions, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Hypersensitivity reactions, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]

74. Secondary Outcome: Weekly Incidence Rates of Rash Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Any, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Any, Week 37 | 0.77 [0.46 to 1.20] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Any, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Any, Week 38 | 0.54 [0.24 to 1.06] | 0.00 [0.00 to 30.85] | 0.37 [0.04 to 1.40]
  Any, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Any, Week 39 | 0.36 [0.20 to 0.60] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Any, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Any, Week 40 | 0.58 [0.30 to 1.02] | 0.29 [0.01 to 1.62] | 0.17 [0.00 to 0.95]
  Any, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Any, Week 41 | 0.12 [0.01 to 0.43] | 0.58 [0.07 to 2.09] | 0.00 [0.00 to 0.92]
  Any, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Any, Week 42 | 0.11 [0.00 to 0.80] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Any, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Any, Week 43 | 0.60 [0.11 to 1.87] | 0.52 [0.06 to 1.88] | 0.00 [0.00 to 2.22]
  Any, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Any, Week 44 | 0.53 [0.11 to 1.53] | 0.21 [0.00 to 1.27] | 0.00 [0.00 to 0.66]
  Any, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Any, Week 45 | 0.22 [0.00 to 1.53] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Any, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Any, Week 46 | 0.57 [0.05 to 2.30] | 0.17 [0.00 to 1.59] | 0.00 [0.00 to 3.73]
  Any, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Any, Week 47 | 0.00 [0.00 to 1.42] | 0.63 [0.02 to 3.48] | 0.00 [0.00 to 1.84]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Any, Week 48 | 0.00 [0.00 to 2.51] | 1.00 [0.01 to 6.22] | 0.00 [0.00 to 8.41]

75. Secondary Outcome: Weekly Incidence Rates of Musculoskeletal Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Musculoskeletal adverse events include any musculoskeletal adverse events, arthropathy, and muscle aches/myalgia. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Any, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Any, Week 37 | 4.26 [3.33 to 5.34] | 0.00 [0.00 to 52.18] | 0.43 [0.05 to 1.53]
  Any, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Any, Week 38 | 3.37 [2.47 to 4.50] | 0.00 [0.00 to 30.85] | 0.37 [0.04 to 1.33]
  Any, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Any, Week 39 | 3.33 [2.78 to 3.95] | 0.00 [0.00 to 3.42] | 0.82 [0.22 to 2.09]
  Any, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Any, Week 40 | 2.63 [1.91 to 3.52] | 1.17 [0.02 to 6.99] | 0.51 [0.06 to 1.86]
  Any, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Any, Week 41 | 2.52 [1.82 to 3.39] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Any, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Any, Week 42 | 1.97 [0.86 to 3.84] | 0.49 [0.06 to 1.74] | 0.00 [0.00 to 1.52]
  Any, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Any, Week 43 | 3.21 [1.38 to 6.25] | 0.26 [0.00 to 1.67] | 1.22 [0.15 to 4.34]
  Any, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Any, Week 44 | 1.87 [0.67 to 4.07] | 1.27 [0.02 to 7.37] | 0.00 [0.00 to 0.66]
  Any, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Any, Week 45 | 2.64 [1.12 to 5.21] | 0.50 [0.06 to 1.78] | 0.29 [0.01 to 1.58]
  Any, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Any, Week 46 | 1.43 [0.47 to 3.30] | 0.17 [0.00 to 1.61] | 2.06 [0.24 to 7.40]
  Any, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Any, Week 47 | 1.94 [0.49 to 5.06] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Any, Week 48 | 0.00 [0.00 to 2.51] | 2.00 [0.24 to 7.04] | 0.00 [0.00 to 8.41]
  Arthropathy, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Arthropathy, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Arthropathy, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Arthropathy, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Arthropathy, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Arthropathy, Week 37 | 1.42 [0.99 to 1.97] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Arthropathy, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Arthropathy, Week 38 | 1.05 [0.62 to 1.67] | 0.00 [0.00 to 30.85] | 0.18 [0.00 to 1.06]
  Arthropathy, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Arthropathy, Week 39 | 0.90 [0.55 to 1.38] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Arthropathy, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Arthropathy, Week 40 | 0.78 [0.24 to 1.86] | 0.88 [0.01 to 5.27] | 0.00 [0.00 to 0.63]
  Arthropathy, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Arthropathy, Week 41 | 0.60 [0.28 to 1.11] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Arthropathy, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Arthropathy, Week 42 | 0.33 [0.06 to 0.99] | 0.24 [0.01 to 1.34] | 0.00 [0.00 to 1.52]
  Arthropathy, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Arthropathy, Week 43 | 1.00 [0.26 to 2.61] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Arthropathy, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Arthropathy, Week 44 | 0.67 [0.12 to 2.05] | 0.64 [0.01 to 3.72] | 0.00 [0.00 to 0.66]
  Arthropathy, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Arthropathy, Week 45 | 0.66 [0.04 to 2.96] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Arthropathy, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Arthropathy, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Arthropathy, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Arthropathy, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Arthropathy, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Arthropathy, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Muscle aches / myalgia, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Muscle aches / myalgia, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Muscle aches / myalgia, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Muscle aches / myalgia, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Muscle aches / myalgia, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Muscle aches / myalgia, Week 37 | 3.77 [2.67 to 5.16] | 0.00 [0.00 to 52.18] | 0.43 [0.05 to 1.53]
  Muscle aches / myalgia, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Muscle aches / myalgia, Week 38 | 3.08 [2.31 to 4.03] | 0.00 [0.00 to 30.85] | 0.18 [0.00 to 1.14]
  Muscle aches / myalgia, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Muscle aches / myalgia, Week 39 | 2.96 [2.47 to 3.53] | 0.00 [0.00 to 3.42] | 0.82 [0.22 to 2.09]
  Muscle aches / myalgia, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Muscle aches / myalgia, Week 40 | 2.43 [1.74 to 3.29] | 1.17 [0.02 to 6.99] | 0.51 [0.06 to 1.86]
  Muscle aches / myalgia, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Muscle aches / myalgia, Week 41 | 2.34 [1.64 to 3.23] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Muscle aches / myalgia, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Muscle aches / myalgia, Week 42 | 1.86 [0.75 to 3.80] | 0.49 [0.06 to 1.74] | 0.00 [0.00 to 1.52]
  Muscle aches / myalgia, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Muscle aches / myalgia, Week 43 | 3.01 [1.18 to 6.20] | 0.26 [0.00 to 1.67] | 1.22 [0.15 to 4.34]
  Muscle aches / myalgia, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Muscle aches / myalgia, Week 44 | 1.60 [0.66 to 3.22] | 1.27 [0.02 to 7.37] | 0.00 [0.00 to 0.66]
  Muscle aches / myalgia, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Muscle aches / myalgia, Week 45 | 2.42 [1.04 to 4.74] | 0.50 [0.06 to 1.78] | 0.29 [0.01 to 1.58]
  Muscle aches / myalgia, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Muscle aches / myalgia, Week 46 | 1.43 [0.47 to 3.30] | 0.17 [0.00 to 1.61] | 2.06 [0.24 to 7.40]
  Muscle aches / myalgia, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Muscle aches / myalgia, Week 47 | 1.94 [0.49 to 5.06] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Muscle aches / myalgia, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Muscle aches / myalgia, Week 48 | 0.00 [0.00 to 2.51] | 2.00 [0.24 to 7.04] | 0.00 [0.00 to 8.41]

76. Secondary Outcome: Weekly Incidence Rates of Neurological Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Neurological adverse events include any neurological adverse events, Bell's palsy, Guillain-Barre Syndrome, peripheral tremor and seizure/febrile convulsions. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Any, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Any, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Any, Week 37 | 0.28 [0.11 to 0.58] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Any, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Any, Week 38 | 0.29 [0.13 to 0.57] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Any, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Any, Week 39 | 0.22 [0.06 to 0.57] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Any, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Any, Week 40 | 0.00 [0.00 to 0.18] | 0.29 [0.00 to 1.78] | 0.00 [0.00 to 0.63]
  Any, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Any, Week 41 | 0.18 [0.03 to 0.59] | 0.29 [0.01 to 1.61] | 0.25 [0.00 to 1.69]
  Any, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Any, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Any, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Any, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Any, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Any, Week 44 | 0.13 [0.00 to 1.05] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Any, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Any, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Any, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Any, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Any, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Any, Week 47 | 0.00 [0.00 to 1.42] | 0.63 [0.01 to 4.02] | 0.00 [0.00 to 1.84]
  Any, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Any, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Bell's palsy, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Bell's palsy, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Bell's palsy, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Bell's palsy, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Bell's palsy, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Bell's palsy, Week 37 | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Bell's palsy, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Bell's palsy, Week 38 | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Bell's palsy, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Bell's palsy, Week 39 | 0.02 [0.00 to 0.18] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Bell's palsy, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Bell's palsy, Week 40 | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Bell's palsy, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Bell's palsy, Week 41 | 0.00 [0.00 to 0.22] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Bell's palsy, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Bell's palsy, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Bell's palsy, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Bell's palsy, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Bell's palsy, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Bell's palsy, Week 44 | 0.00 [0.00 to 0.49] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Bell's palsy, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Bell's palsy, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Bell's palsy, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Bell's palsy, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Bell's palsy, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Bell's palsy, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Bell's palsy, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Bell's palsy, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Guillain-Barre Syndrome, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Guillain-Barre Syndrome, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Guillain-Barre Syndrome, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Guillain-Barre Syndrome, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Guillain-Barre Syndrome, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Guillain-Barre Syndrome, Week 37 | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Guillain-Barre Syndrome, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Guillain-Barre Syndrome, Week 38 | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Guillain-Barre Syndrome, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Guillain-Barre Syndrome, Week 39 | 0.00 [0.00 to 0.09] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Guillain-Barre Syndrome, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Guillain-Barre Syndrome, Week 40 | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Guillain-Barre Syndrome, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Guillain-Barre Syndrome, Week 41 | 0.00 [0.00 to 0.22] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.92]
  Guillain-Barre Syndrome, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Guillain-Barre Syndrome, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Guillain-Barre Syndrome, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Guillain-Barre Syndrome, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Guillain-Barre Syndrome, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Guillain-Barre Syndrome, Week 44 | 0.00 [0.00 to 0.49] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Guillain-Barre Syndrome, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Guillain-Barre Syndrome, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Guillain-Barre Syndrome, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Guillain-Barre Syndrome, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Guillain-Barre Syndrome, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Guillain-Barre Syndrome, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Guillain-Barre Syndrome, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Guillain-Barre Syndrome, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Peripheral tremor, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Peripheral tremor, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Peripheral tremor, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Peripheral tremor, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Peripheral tremor, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Peripheral tremor, Week 37 | 0.24 [0.09 to 0.53] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Peripheral tremor, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Peripheral tremor, Week 38 | 0.29 [0.13 to 0.57] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Peripheral tremor, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Peripheral tremor, Week 39 | 0.19 [0.04 to 0.56] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Peripheral tremor, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Peripheral tremor, Week 40 | 0.00 [0.00 to 0.18] | 0.29 [0.00 to 1.78] | 0.00 [0.00 to 0.63]
  Peripheral tremor, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Peripheral tremor, Week 41 | 0.18 [0.03 to 0.59] | 0.29 [0.01 to 1.61] | 0.00 [0.00 to 0.92]
  Peripheral tremor, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Peripheral tremor, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Peripheral tremor, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Peripheral tremor, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Peripheral tremor, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Peripheral tremor, Week 44 | 0.13 [0.00 to 1.05] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Peripheral tremor, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Peripheral tremor, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Peripheral tremor, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Peripheral tremor, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Peripheral tremor, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Peripheral tremor, Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.00 [0.00 to 1.84]
  Peripheral tremor, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Peripheral tremor, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]
  Seizure/Febrile convulsions, Week 35: number analyzed (Participants) | 0 | 0 | 1
  Seizure/Febrile convulsions, Week 35 |  |  | 0.00 [0.00 to 97.50]
  Seizure/Febrile convulsions, Week 36: number analyzed (Participants) | 1 | 1 | 61
  Seizure/Febrile convulsions, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  Seizure/Febrile convulsions, Week 37: number analyzed (Participants) | 2467 | 5 | 470
  Seizure/Febrile convulsions, Week 37 | 0.04 [0.00 to 0.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.78]
  Seizure/Febrile convulsions, Week 38: number analyzed (Participants) | 2756 | 10 | 541
  Seizure/Febrile convulsions, Week 38 | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.68]
  Seizure/Febrile convulsions, Week 39: number analyzed (Participants) | 4117 | 106 | 486
  Seizure/Febrile convulsions, Week 39 | 0.00 [0.00 to 0.09] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  Seizure/Febrile convulsions, Week 40: number analyzed (Participants) | 2057 | 342 | 585
  Seizure/Febrile convulsions, Week 40 | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 1.07] | 0.00 [0.00 to 0.63]
  Seizure/Febrile convulsions, Week 41: number analyzed (Participants) | 1666 | 343 | 398
  Seizure/Febrile convulsions, Week 41 | 0.00 [0.00 to 0.22] | 0.00 [0.00 to 1.07] | 0.25 [0.00 to 1.69]
  Seizure/Febrile convulsions, Week 42: number analyzed (Participants) | 912 | 412 | 241
  Seizure/Febrile convulsions, Week 42 | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 0.89] | 0.00 [0.00 to 1.52]
  Seizure/Febrile convulsions, Week 43: number analyzed (Participants) | 499 | 382 | 164
  Seizure/Febrile convulsions, Week 43 | 0.00 [0.00 to 0.74] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  Seizure/Febrile convulsions, Week 44: number analyzed (Participants) | 750 | 471 | 561
  Seizure/Febrile convulsions, Week 44 | 0.00 [0.00 to 0.49] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 0.66]
  Seizure/Febrile convulsions, Week 45: number analyzed (Participants) | 455 | 403 | 350
  Seizure/Febrile convulsions, Week 45 | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 1.05]
  Seizure/Febrile convulsions, Week 46: number analyzed (Participants) | 350 | 577 | 97
  Seizure/Febrile convulsions, Week 46 | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.64] | 0.00 [0.00 to 3.73]
  Seizure/Febrile convulsions, Week 47: number analyzed (Participants) | 258 | 158 | 199
  Seizure/Febrile convulsions, Week 47 | 0.00 [0.00 to 1.42] | 0.63 [0.01 to 4.02] | 0.00 [0.00 to 1.84]
  Seizure/Febrile convulsions, Week 48: number analyzed (Participants) | 145 | 100 | 42
  Seizure/Febrile convulsions, Week 48 | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]

77. Secondary Outcome: Weekly Incidence Rates of SAEs Recorded in EHR, by Vaccine Group
Description: SAEs reported here are derived from 2 sources of data - ADR cards and SAE routinely collected from GPs. The weekly incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any SAEs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At Week 35: number analyzed (Participants) | 0 | 0 | 1
  At Week 35 |  |  | 0.00 [0.00 to 97.50]
  At Week 36: number analyzed (Participants) | 1 | 1 | 61
  At Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.87]
  At Week 37: number analyzed (Participants) | 2467 | 5 | 470
  At Week 37 | 0.12 [0.02 to 0.37] | 0.00 [0.00 to 52.18] | 0.21 [0.00 to 1.71]
  At Week 38: number analyzed (Participants) | 2756 | 10 | 541
  At Week 38 | 0.18 [0.04 to 0.52] | 0.00 [0.00 to 30.85] | 0.37 [0.04 to 1.33]
  At Week 39: number analyzed (Participants) | 4117 | 106 | 486
  At Week 39 | 0.07 [0.01 to 0.22] | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 0.76]
  At Week 40: number analyzed (Participants) | 2057 | 342 | 585
  At Week 40 | 0.19 [0.04 to 0.60] | 0.00 [0.00 to 1.07] | 0.17 [0.00 to 1.29]
  At Week 41: number analyzed (Participants) | 1666 | 343 | 398
  At Week 41 | 0.12 [0.01 to 0.55] | 0.00 [0.00 to 1.07] | 0.50 [0.04 to 2.05]
  At Week 42: number analyzed (Participants) | 912 | 412 | 241
  At Week 42 | 0.00 [0.00 to 0.40] | 0.24 [0.01 to 1.34] | 0.00 [0.00 to 1.52]
  At Week 43: number analyzed (Participants) | 499 | 382 | 164
  At Week 43 | 0.40 [0.01 to 2.45] | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 2.22]
  At Week 44: number analyzed (Participants) | 750 | 471 | 561
  At Week 44 | 0.27 [0.00 to 1.90] | 0.21 [0.00 to 1.46] | 0.36 [0.00 to 2.77]
  At Week 45: number analyzed (Participants) | 455 | 403 | 350
  At Week 45 | 0.22 [0.00 to 1.60] | 0.25 [0.00 to 1.77] | 0.00 [0.00 to 1.05]
  At Week 46: number analyzed (Participants) | 350 | 577 | 97
  At Week 46 | 0.57 [0.07 to 2.05] | 0.00 [0.00 to 0.64] | 1.03 [0.01 to 6.91]
  At Week 47: number analyzed (Participants) | 258 | 158 | 199
  At Week 47 | 0.00 [0.00 to 1.42] | 0.00 [0.00 to 2.31] | 0.50 [0.00 to 4.16]
  At Week 48: number analyzed (Participants) | 145 | 100 | 42
  At Week 48 | 0.69 [0.01 to 4.21] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 8.41]

78. Secondary Outcome: Cumulative Incidence Rates of Any AEIs Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on the Cumulative vaccinated cohort which included all subjects who were vaccinated with a seasonal influenza vaccine at any point from study start up to end of the week of interest and were registered in EHR (routine data collection & card-based ADR reporting) during FU period (from vaccination up to 7 days post-vaccination)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Vaccinated_Unknown Brand Group: Volunteered subjects who received influenza vaccination (GSK or non-GSK not known) in 10 volunteer GP practices between 01 September and 30 November 2017
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.61 [0.00 to 14.32]
  Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Week 35-37 | 11.63 [9.72 to 13.76] | 0.00 [0.00 to 45.93] | 1.32 [0.47 to 2.90]
  Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Week 35-38 | 10.78 [8.92 to 12.86] | 6.25 [0.12 to 31.55] | 1.40 [0.78 to 2.30]
  Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Week 35-39 | 10.45 [8.95 to 12.11] | 2.46 [0.33 to 8.32] | 1.67 [0.92 to 2.78]
  Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Week 35-40 | 10.36 [8.58 to 12.37] | 6.03 [3.98 to 8.72] | 1.63 [0.82 to 2.89]
  Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Week 35-41 | 10.13 [8.31 to 12.21] | 5.82 [3.69 to 8.68] | 1.46 [0.72 to 2.61]
  Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Week 35-42 | 9.82 [7.97 to 11.93] | 4.59 [2.92 to 6.85] | 1.47 [0.74 to 2.61]
  Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Week 35-43 | 9.69 [7.84 to 11.79] | 4.56 [2.86 to 6.86] | 1.49 [0.74 to 2.67]
  Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Week 35-44 | 9.50 [7.65 to 11.63] | 4.87 [2.74 to 7.93] | 1.31 [0.69 to 2.24]
  Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Week 35-45 | 9.42 [7.60 to 11.50] | 4.61 [2.45 to 7.80] | 1.56 [0.85 to 2.60]
  Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Week 35-46 | 9.38 [7.54 to 11.48] | 4.03 [1.72 to 7.88] | 1.59 [0.92 to 2.56]
  Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Week 35-47 | 9.30 [7.46 to 11.41] | 3.99 [1.72 to 7.76] | 1.59 [0.90 to 2.59]
  Week 35-48 | 9.21 [7.37 to 11.34] | 4.02 [1.73 to 7.82] | 1.57 [0.89 to 2.56]

79. Secondary Outcome: Cumulative Incidence Rates of Fever/Pyrexia Adverse Events Recorded in EHR, by Vaccine Group
Description: "subjects with a fever/pyrexia read code recorded were considered as having fever/pyrexia, regardless of what temperature had been recorded. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Week 35-37 | 0.45 [0.20 to 0.85] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Week 35-38 | 0.50 [0.29 to 0.80] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Week 35-39 | 0.50 [0.26 to 0.87] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.46]
  Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Week 35-40 | 0.49 [0.29 to 0.79] | 1.08 [0.17 to 3.52] | 0.05 [0.00 to 0.34]
  Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Week 35-41 | 0.47 [0.29 to 0.73] | 0.87 [0.27 to 2.05] | 0.04 [0.00 to 0.29]
  Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Week 35-42 | 0.44 [0.26 to 0.70] | 0.57 [0.14 to 1.52] | 0.04 [0.00 to 0.26]
  Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Week 35-43 | 0.44 [0.26 to 0.69] | 0.44 [0.09 to 1.27] | 0.03 [0.00 to 0.25]
  Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Week 35-44 | 0.43 [0.26 to 0.68] | 0.43 [0.13 to 1.06] | 0.03 [0.00 to 0.21]
  Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Week 35-45 | 0.43 [0.25 to 0.67] | 0.36 [0.10 to 0.94] | 0.05 [0.01 to 0.19]
  Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Week 35-46 | 0.43 [0.25 to 0.69] | 0.33 [0.09 to 0.84] | 0.05 [0.01 to 0.18]
  Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Week 35-47 | 0.43 [0.25 to 0.68] | 0.34 [0.12 to 0.77] | 0.05 [0.01 to 0.18]
  Week 35-48 | 0.43 [0.25 to 0.67] | 0.33 [0.11 to 0.75] | 0.05 [0.01 to 0.18]

80. Secondary Outcome: Cumulative Incidence Rates of Local Symptoms Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Local symptoms include local erythema. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Week 35-37 | 1.90 [0.82 to 3.74] | 0.00 [0.00 to 45.93] | 0.19 [0.00 to 1.04]
  Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Week 35-38 | 1.76 [1.04 to 2.79] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.53]
  Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Week 35-39 | 1.84 [1.20 to 2.69] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.38]
  Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Week 35-40 | 1.86 [1.23 to 2.70] | 0.22 [0.01 to 1.19] | 0.05 [0.00 to 0.30]
  Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Week 35-41 | 1.81 [1.24 to 2.53] | 0.50 [0.05 to 1.94] | 0.04 [0.00 to 0.25]
  Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Week 35-42 | 1.72 [1.23 to 2.35] | 0.49 [0.06 to 1.81] | 0.04 [0.00 to 0.24]
  Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Week 35-43 | 1.68 [1.20 to 2.27] | 0.56 [0.06 to 2.09] | 0.03 [0.00 to 0.22]
  Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Week 35-44 | 1.66 [1.21 to 2.21] | 0.58 [0.08 to 1.99] | 0.03 [0.00 to 0.19]
  Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Week 35-45 | 1.63 [1.20 to 2.17] | 0.57 [0.12 to 1.61] | 0.03 [0.00 to 0.18]
  Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Week 35-46 | 1.63 [1.21 to 2.14] | 0.56 [0.09 to 1.76] | 0.03 [0.00 to 0.18]
  Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Week 35-47 | 1.62 [1.21 to 2.13] | 0.53 [0.09 to 1.68] | 0.02 [0.00 to 0.17]
  Week 35-48 | 1.61 [1.20 to 2.11] | 0.51 [0.09 to 1.63] | 0.02 [0.00 to 0.17]

81. Secondary Outcome: Cumulative Incidence Rates of General Non-specific Symptoms Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, headache, irritability, and malaise. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Any, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Any, Week 35-37 | 4.01 [3.23 to 4.92] | 0.00 [0.00 to 45.93] | 0.19 [0.00 to 1.60]
  Any, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Any, Week 35-38 | 3.58 [2.78 to 4.53] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.77]
  Any, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Any, Week 35-39 | 3.46 [2.70 to 4.35] | 0.82 [0.02 to 4.48] | 0.19 [0.04 to 0.57]
  Any, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Any, Week 35-40 | 3.33 [2.63 to 4.15] | 1.94 [0.67 to 4.31] | 0.14 [0.03 to 0.41]
  Any, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Any, Week 35-41 | 3.15 [2.48 to 3.95] | 1.61 [0.55 to 3.63] | 0.12 [0.02 to 0.34]
  Any, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Any, Week 35-42 | 3.06 [2.37 to 3.88] | 1.23 [0.41 to 2.83] | 0.11 [0.02 to 0.31]
  Any, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Any, Week 35-43 | 3.02 [2.32 to 3.85] | 1.19 [0.31 to 3.08] | 0.10 [0.02 to 0.30]
  Any, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Any, Week 35-44 | 2.96 [2.26 to 3.81] | 1.30 [0.30 to 3.57] | 0.09 [0.02 to 0.25]
  Any, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Any, Week 35-45 | 2.92 [2.23 to 3.75] | 1.33 [0.40 to 3.21] | 0.21 [0.02 to 0.75]
  Any, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Any, Week 35-46 | 2.88 [2.18 to 3.73] | 1.15 [0.24 to 3.32] | 0.20 [0.02 to 0.73]
  Any, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Any, Week 35-47 | 2.84 [2.15 to 3.68] | 1.09 [0.22 to 3.17] | 0.19 [0.02 to 0.70]
  Any, Week 35-48 | 2.82 [2.13 to 3.66] | 1.06 [0.22 to 3.07] | 0.19 [0.02 to 0.70]
  Drowsiness, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Drowsiness, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Drowsiness, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Drowsiness, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Drowsiness, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Drowsiness, Week 35-37 | 1.05 [0.62 to 1.68] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Drowsiness, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Drowsiness, Week 35-38 | 0.92 [0.48 to 1.59] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Drowsiness, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Drowsiness, Week 35-39 | 0.79 [0.42 to 1.36] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Drowsiness, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Drowsiness, Week 35-40 | 0.77 [0.43 to 1.28] | 0.22 [0.01 to 1.19] | 0.00 [0.00 to 0.17]
  Drowsiness, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Drowsiness, Week 35-41 | 0.74 [0.41 to 1.23] | 0.37 [0.08 to 1.08] | 0.00 [0.00 to 0.15]
  Drowsiness, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Drowsiness, Week 35-42 | 0.72 [0.38 to 1.21] | 0.25 [0.05 to 0.72] | 0.00 [0.00 to 0.13]
  Drowsiness, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Drowsiness, Week 35-43 | 0.72 [0.37 to 1.26] | 0.25 [0.07 to 0.64] | 0.00 [0.00 to 0.13]
  Drowsiness, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Drowsiness, Week 35-44 | 0.70 [0.35 to 1.24] | 0.29 [0.06 to 0.86] | 0.00 [0.00 to 0.11]
  Drowsiness, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Drowsiness, Week 35-45 | 0.68 [0.34 to 1.21] | 0.24 [0.04 to 0.76] | 0.00 [0.00 to 0.10]
  Drowsiness, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Drowsiness, Week 35-46 | 0.67 [0.34 to 1.19] | 0.23 [0.03 to 0.85] | 0.00 [0.00 to 0.09]
  Drowsiness, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Drowsiness, Week 35-47 | 0.66 [0.33 to 1.17] | 0.22 [0.02 to 0.82] | 0.00 [0.00 to 0.09]
  Drowsiness, Week 35-48 | 0.65 [0.33 to 1.16] | 0.21 [0.02 to 0.79] | 0.00 [0.00 to 0.09]
  Fatigue, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Fatigue, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Fatigue, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Fatigue, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Fatigue, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Fatigue, Week 35-37 | 2.19 [1.65 to 2.85] | 0.00 [0.00 to 45.93] | 0.19 [0.00 to 1.60]
  Fatigue, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Fatigue, Week 35-38 | 2.03 [1.57 to 2.58] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.77]
  Fatigue, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Fatigue, Week 35-39 | 1.93 [1.50 to 2.44] | 0.00 [0.00 to 2.98] | 0.13 [0.01 to 0.50]
  Fatigue, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Fatigue, Week 35-40 | 1.79 [1.40 to 2.26] | 0.43 [0.02 to 2.14] | 0.09 [0.01 to 0.38]
  Fatigue, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Fatigue, Week 35-41 | 1.71 [1.33 to 2.17] | 0.37 [0.04 to 1.45] | 0.08 [0.01 to 0.31]
  Fatigue, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Fatigue, Week 35-42 | 1.65 [1.26 to 2.13] | 0.25 [0.03 to 0.91] | 0.07 [0.01 to 0.28]
  Fatigue, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Fatigue, Week 35-43 | 1.62 [1.24 to 2.09] | 0.31 [0.03 to 0.31] | 0.07 [0.01 to 0.27]
  Fatigue, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Fatigue, Week 35-44 | 1.58 [1.20 to 2.04] | 0.39 [0.03 to 1.26] | 0.06 [0.01 to 0.21]
  Fatigue, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Fatigue, Week 35-45 | 1.56 [1.20 to 2.00] | 0.40 [0.13 to 0.93] | 0.08 [0.01 to 0.26]
  Fatigue, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Fatigue, Week 35-46 | 1.55 [1.18 to 2.01] | 0.33 [0.08 to 0.88] | 0.08 [0.01 to 0.26]
  Fatigue, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Fatigue, Week 35-47 | 1.53 [1.16 to 1.98] | 0.31 [0.08 to 0.84] | 0.07 [0.01 to 0.25]
  Fatigue, Week 35-48 | 1.52 [1.14 to 1.97] | 0.30 [0.07 to 0.81] | 0.07 [0.01 to 0.24]
  Headache, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Headache, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Headache, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Headache, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Headache, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Headache, Week 35-37 | 2.27 [1.61 to 3.11] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Headache, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Headache, Week 35-38 | 2.09 [1.36 to 3.06] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Headache, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Headache, Week 35-39 | 2.01 [1.34 to 2.89] | 0.82 [0.02 to 4.48] | 0.06 [0.00 to 0.46]
  Headache, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Headache, Week 35-40 | 1.94 [1.34 to 2.71] | 1.29 [0.12 to 4.96] | 0.05 [0.00 to 0.28]
  Headache, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Headache, Week 35-41 | 1.81 [1.25 to 2.54] | 1.12 [0.18 to 3.56] | 0.04 [0.00 to 0.25]
  Headache, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Headache, Week 35-42 | 1.75 [1.20 to 2.46] | 0.82 [0.15 to 2.48] | 0.04 [0.00 to 0.23]
  Headache, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Headache, Week 35-43 | 1.74 [1.19 to 2.45] | 0.81 [0.14 to 2.56] | 0.03 [0.00 to 0.21]
  Headache, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Headache, Week 35-44 | 1.73 [1.19 to 2.42] | 0.87 [0.18 to 2.52] | 0.03 [0.00 to 0.19]
  Headache, Week 35-45: number analyzed (Participants) | 15225 | 2475 | 3858
  Headache, Week 35-45 | 1.72 [1.19 to 2.39] | 0.89 [0.21 to 2.41] | 0.16 [0.01 to 0.68]
  Headache, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Headache, Week 35-46 | 1.68 [1.16 to 2.36] | 0.75 [0.13 to 2.40] | 0.15 [0.01 to 0.66]
  Headache, Week 35-47: number analyzed (Participants) | 16288 | 3052 | 4154
  Headache, Week 35-47 | 1.66 [1.15 to 2.33] | 0.72 [0.12 to 2.29] | 0.14 [0.01 to 0.64]
  Headache, Week 35-48 | 1.65 [1.14 to 2.31] | 0.69 [0.12 to 2.21] | 0.14 [0.01 to 0.63]
  Irritability, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Irritability, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Irritability, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Irritability, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Irritability, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Irritability, Week 35-37 | 0.41 [0.19 to 0.74] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Irritability, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Irritability, Week 35-38 | 0.33 [0.15 to 0.61] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Irritability, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Irritability, Week 35-39 | 0.34 [0.16 to 0.63] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Irritability, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Irritability, Week 35-40 | 0.31 [0.16 to 0.53] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 0.17]
  Irritability, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Irritability, Week 35-41 | 0.28 [0.14 to 0.50] | 0.00 [0.00 to 0.46] | 0.00 [0.00 to 0.15]
  Irritability, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Irritability, Week 35-42 | 0.27 [0.13 to 0.50] | 0.08 [0.00 to 0.46] | 0.00 [0.00 to 0.13]
  Irritability, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Irritability, Week 35-43 | 0.27 [0.13 to 0.50] | 0.12 [0.01 to 0.47] | 0.00 [0.00 to 0.13]
  Irritability, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Irritability, Week 35-44 | 0.26 [0.12 to 0.48] | 0.19 [0.02 to 0.79] | 0.00 [0.00 to 0.11]
  Irritability, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Irritability, Week 35-45 | 0.26 [0.13 to 0.47] | 0.16 [0.01 to 0.69] | 0.00 [0.00 to 0.10]
  Irritability, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Irritability, Week 35-46 | 0.26 [0.13 to 0.46] | 0.13 [0.01 to 0.63] | 0.00 [0.00 to 0.09]
  Irritability, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Irritability, Week 35-47 | 0.25 [0.13 to 0.45] | 0.12 [0.01 to 0.60] | 0.00 [0.00 to 0.09]
  Irritability, Week 35-48 | 0.25 [0.12 to 0.45] | 0.12 [0.01 to 0.58] | 0.00 [0.00 to 0.09]
  Malaise, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Malaise, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Malaise, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Malaise, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Malaise, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Malaise, Week 35-37 | 0.04 [0.00 to 0.25] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Malaise, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Malaise, Week 35-38 | 0.02 [0.00 to 0.11] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Malaise, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Malaise, Week 35-39 | 0.01 [0.00 to 0.07] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Malaise, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Malaise, Week 35-40 | 0.02 [0.00 to 0.07] | 0.22 [0.01 to 1.19] | 0.00 [0.00 to 0.17]
  Malaise, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Malaise, Week 35-41 | 0.02 [0.00 to 0.07] | 0.12 [0.00 to 0.81] | 0.00 [0.00 to 0.15]
  Malaise, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Malaise, Week 35-42 | 0.02 [0.00 to 0.06] | 0.16 [0.02 to 0.59] | 0.00 [0.00 to 0.13]
  Malaise, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Malaise, Week 35-43 | 0.02 [0.00 to 0.06] | 0.12 [0.02 to 0.45] | 0.00 [0.00 to 0.13]
  Malaise, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Malaise, Week 35-44 | 0.02 [0.00 to 0.06] | 0.10 [0.01 to 0.35] | 0.00 [0.00 to 0.11]
  Malaise, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Malaise, Week 35-45 | 0.02 [0.00 to 0.06] | 0.12 [0.03 to 0.35] | 0.00 [0.00 to 0.10]
  Malaise, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Malaise, Week 35-46 | 0.02 [0.00 to 0.05] | 0.10 [0.02 to 0.29] | 0.00 [0.00 to 0.09]
  Malaise, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Malaise, Week 35-47 | 0.02 [0.00 to 0.05] | 0.09 [0.02 to 0.27] | 0.00 [0.00 to 0.09]
  Malaise, Week 35-48 | 0.02 [0.00 to 0.05] | 0.09 [0.02 to 0.26] | 0.00 [0.00 to 0.09]

82. Secondary Outcome: Cumulative Incidence Rates of Respiratory/Miscellaneous Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Respiratory/miscellaneous adverse events include any respiratory/miscellaneous adverse events, conjunctivitis, coryza, cough, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhoea and wheezing. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.61 [0.00 to 14.32]
  Any, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Any, Week 35-37 | 6.44 [5.26 to 7.80] | 0.00 [0.00 to 45.93] | 0.75 [0.10 to 2.64]
  Any, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Any, Week 35-38 | 5.61 [4.75 to 6.57] | 6.25 [0.12 to 31.55] | 0.65 [0.12 to 1.96]
  Any, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Any, Week 35-39 | 5.33 [4.65 to 6.08] | 1.64 [0.20 to 5.80] | 0.83 [0.21 to 2.21]
  Any, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Any, Week 35-40 | 5.33 [4.50 to 6.26] | 3.45 [1.92 to 5.68] | 0.89 [0.25 to 2.22]
  Any, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Any, Week 35-41 | 5.24 [4.42 to 6.17] | 3.59 [2.39 to 5.17] | 0.79 [0.24 to 1.89]
  Any, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Any, Week 35-42 | 5.07 [4.22 to 6.02] | 2.63 [1.70 to 3.86] | 0.86 [0.30 to 1.93]
  Any, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Any, Week 35-43 | 4.99 [4.13 to 5.96] | 2.69 [1.78 to 3.87] | 0.81 [0.29 to 1.80]
  Any, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Any, Week 35-44 | 4.89 [4.03 to 5.88] | 2.90 [1.86 to 4.29] | 0.74 [0.30 to 1.53]
  Any, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Any, Week 35-45 | 4.82 [3.95 to 5.81] | 2.63 [1.49 to 4.26] | 0.88 [0.41 to 1.66]
  Any, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Any, Week 35-46 | 4.77 [3.88 to 5.79] | 2.26 [1.08 to 4.15] | 0.86 [0.40 to 1.62]
  Any, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Any, Week 35-47 | 4.74 [3.85 to 5.76] | 2.21 [1.08 to 4.00] | 0.89 [0.42 to 1.66]
  Any, Week 35-48 | 4.70 [3.81 to 5.73] | 2.21 [1.07 to 4.00] | 0.88 [0.41 to 1.64]
  Conjunctivitis, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Conjunctivitis, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Conjunctivitis, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Conjunctivitis, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Conjunctivitis, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Conjunctivitis, Week 35-37 | 0.24 [0.09 to 0.53] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Conjunctivitis, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Conjunctivitis, Week 35-38 | 0.38 [0.16 to 0.77] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Conjunctivitis, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Conjunctivitis, Week 35-39 | 0.35 [0.21 to 0.56] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.52]
  Conjunctivitis, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Conjunctivitis, Week 35-40 | 0.35 [0.21 to 0.54] | 0.00 [0.00 to 0.79] | 0.05 [0.00 to 0.38]
  Conjunctivitis, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Conjunctivitis, Week 35-41 | 0.36 [0.24 to 0.52] | 0.00 [0.00 to 0.46] | 0.04 [0.00 to 0.31]
  Conjunctivitis, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Conjunctivitis, Week 35-42 | 0.34 [0.22 to 0.51] | 0.08 [0.00 to 0.46] | 0.07 [0.00 to 0.36]
  Conjunctivitis, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Conjunctivitis, Week 35-43 | 0.34 [0.21 to 0.52] | 0.12 [0.01 to 0.47] | 0.07 [0.00 to 0.34]
  Conjunctivitis, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Conjunctivitis, Week 35-44 | 0.35 [0.22 to 0.52] | 0.14 [0.03 to 0.42] | 0.09 [0.01 to 0.37]
  Conjunctivitis, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Conjunctivitis, Week 35-45 | 0.34 [0.21 to 0.51] | 0.12 [0.03 to 0.35] | 0.13 [0.01 to 0.57]
  Conjunctivitis, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Conjunctivitis, Week 35-46 | 0.33 [0.21 to 0.50] | 0.10 [0.02 to 0.29] | 0.13 [0.01 to 0.56]
  Conjunctivitis, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Conjunctivitis, Week 35-47 | 0.33 [0.20 to 0.50] | 0.09 [0.02 to 0.27] | 0.12 [0.01 to 0.54]
  Conjunctivitis, Week 35-48 | 0.32 [0.20 to 0.49] | 0.09 [0.02 to 0.26] | 0.12 [0.01 to 0.53]
  Coryza, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Coryza, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Coryza, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Coryza, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Coryza, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Coryza, Week 35-37 | 1.38 [0.75 to 2.32] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Coryza, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Coryza, Week 35-38 | 1.15 [0.82 to 1.56] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.74]
  Coryza, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Coryza, Week 35-39 | 1.19 [0.91 to 1.53] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.46]
  Coryza, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Coryza, Week 35-40 | 1.16 [0.88 to 1.50] | 1.08 [0.34 to 2.54] | 0.05 [0.00 to 0.28]
  Coryza, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Coryza, Week 35-41 | 1.17 [0.91 to 1.49] | 0.74 [0.27 to 1.61] | 0.04 [0.00 to 0.25]
  Coryza, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Coryza, Week 35-42 | 1.12 [0.87 to 1.42] | 0.49 [0.15 to 1.19] | 0.04 [0.00 to 0.23]
  Coryza, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Coryza, Week 35-43 | 1.11 [0.85 to 1.42] | 0.56 [0.20 to 1.25] | 0.03 [0.00 to 0.21]
  Coryza, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Coryza, Week 35-44 | 1.08 [0.83 to 1.40] | 0.53 [0.25 to 0.99] | 0.03 [0.00 to 0.19]
  Coryza, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Coryza, Week 35-45 | 1.07 [0.80 to 1.39] | 0.48 [0.20 to 1.00] | 0.05 [0.01 to 0.19]
  Coryza, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Coryza, Week 35-46 | 1.06 [0.80 to 1.38] | 0.39 [0.14 to 0.87] | 0.05 [0.01 to 0.18]
  Coryza, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Coryza, Week 35-47 | 1.06 [0.81 to 1.36] | 0.37 [0.13 to 0.83] | 0.05 [0.01 to 0.17]
  Coryza, Week 35-48 | 1.05 [0.80 to 1.35] | 0.36 [0.13 to 0.80] | 0.05 [0.01 to 0.17]
  Cough, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Cough, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Cough, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Cough, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.61 [0.00 to 14.32]
  Cough, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Cough, Week 35-37 | 2.31 [1.64 to 3.15] | 0.00 [0.00 to 45.93] | 0.75 [0.10 to 2.64]
  Cough, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Cough, Week 35-38 | 2.12 [1.61 to 2.76] | 0.00 [0.00 to 20.59] | 0.47 [0.10 to 1.32]
  Cough, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Cough, Week 35-39 | 2.21 [1.88 to 2.57] | 0.82 [0.02 to 4.48] | 0.64 [0.16 to 1.71]
  Cough, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Cough, Week 35-40 | 2.11 [1.71 to 2.57] | 2.16 [0.85 to 4.44] | 0.70 [0.17 to 1.89]
  Cough, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Cough, Week 35-41 | 2.10 [1.73 to 2.52] | 2.11 [1.18 to 3.45] | 0.63 [0.17 to 1.63]
  Cough, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Cough, Week 35-42 | 2.03 [1.66 to 2.46] | 1.48 [0.73 to 2.65] | 0.61 [0.18 to 1.49]
  Cough, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Cough, Week 35-43 | 2.00 [1.62 to 2.45] | 1.56 [0.97 to 2.37] | 0.58 [0.18 to 1.39]
  Cough, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Cough, Week 35-44 | 1.97 [1.59 to 2.41] | 1.69 [1.00 to 2.67] | 0.48 [0.13 to 1.23]
  Cough, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Cough, Week 35-45 | 1.95 [1.57 to 2.39] | 1.58 [0.84 to 2.67] | 0.52 [0.19 to 1.13]
  Cough, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Cough, Week 35-46 | 1.96 [1.58 to 2.40] | 1.34 [0.63 to 2.50] | 0.51 [0.18 to 1.11]
  Cough, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Cough, Week 35-47 | 1.95 [1.56 to 2.41] | 1.28 [0.60 to 2.36] | 0.53 [0.20 to 1.15]
  Cough, Week 35-48 | 1.94 [1.54 to 2.39] | 1.30 [0.61 to 2.41] | 0.52 [0.19 to 1.14]
  Epistaxis, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Epistaxis, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Epistaxis, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Epistaxis, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Epistaxis, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Epistaxis, Week 35-37 | 0.08 [0.00 to 0.48] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Epistaxis, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Epistaxis, Week 35-38 | 0.06 [0.00 to 0.37] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Epistaxis, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Epistaxis, Week 35-39 | 0.09 [0.02 to 0.23] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Epistaxis, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Epistaxis, Week 35-40 | 0.10 [0.04 to 0.21] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 0.17]
  Epistaxis, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Epistaxis, Week 35-41 | 0.09 [0.04 to 0.19] | 0.00 [0.00 to 0.46] | 0.00 [0.00 to 0.15]
  Epistaxis, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Epistaxis, Week 35-42 | 0.09 [0.04 to 0.17] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 0.13]
  Epistaxis, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Epistaxis, Week 35-43 | 0.08 [0.04 to 0.16] | 0.00 [0.00 to 0.23] | 0.00 [0.00 to 0.13]
  Epistaxis, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Epistaxis, Week 35-44 | 0.09 [0.04 to 0.18] | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 0.11]
  Epistaxis, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Epistaxis, Week 35-45 | 0.09 [0.04 to 0.18] | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 0.10]
  Epistaxis, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Epistaxis, Week 35-46 | 0.09 [0.04 to 0.18] | 0.00 [0.00 to 0.12] | 0.00 [0.00 to 0.09]
  Epistaxis, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Epistaxis, Week 35-47 | 0.09 [0.04 to 0.17] | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.09]
  Epistaxis, Week 35-48 | 0.09 [0.04 to 0.17] | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.09]
  Hoarseness, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Hoarseness, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Hoarseness, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Hoarseness, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Hoarseness, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Hoarseness, Week 35-37 | 1.09 [0.72 to 1.59] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Hoarseness, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Hoarseness, Week 35-38 | 0.96 [0.71 to 1.26] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Hoarseness, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Hoarseness, Week 35-39 | 0.77 [0.60 to 0.97] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Hoarseness, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Hoarseness, Week 35-40 | 0.72 [0.57 to 0.89] | 0.22 [0.01 to 1.19] | 0.00 [0.00 to 0.17]
  Hoarseness, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Hoarseness, Week 35-41 | 0.70 [0.55 to 0.87] | 0.37 [0.08 to 1.08] | 0.00 [0.00 to 0.15]
  Hoarseness, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Hoarseness, Week 35-42 | 0.67 [0.53 to 0.82] | 0.25 [0.05 to 0.72] | 0.00 [0.00 to 0.13]
  Hoarseness, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Hoarseness, Week 35-43 | 0.67 [0.53 to 0.84] | 0.25 [0.07 to 0.64] | 0.00 [0.00 to 0.13]
  Hoarseness, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Hoarseness, Week 35-44 | 0.65 [0.52 to 0.81] | 0.24 [0.05 to 0.68] | 0.00 [0.00 to 0.11]
  Hoarseness, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Hoarseness, Week 35-45 | 0.65 [0.51 to 0.82] | 0.20 [0.04 to 0.60] | 0.03 [0.00 to 0.15]
  Hoarseness, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Hoarseness, Week 35-46 | 0.64 [0.50 to 0.81] | 0.16 [0.02 to 0.56] | 0.03 [0.00 to 0.15]
  Hoarseness, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Hoarseness, Week 35-47 | 0.64 [0.51 to 0.80] | 0.16 [0.02 to 0.54] | 0.02 [0.00 to 0.14]
  Hoarseness, Week 35-48 | 0.63 [0.50 to 0.79] | 0.15 [0.02 to 0.52] | 0.02 [0.00 to 0.14]
  Nasal congestion, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Nasal congestion, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Nasal congestion, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Nasal congestion, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Nasal congestion, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Nasal congestion, Week 35-37 | 1.34 [0.92 to 1.87] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Nasal congestion, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Nasal congestion, Week 35-38 | 1.11 [0.81 to 1.48] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.74]
  Nasal congestion, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Nasal congestion, Week 35-39 | 1.04 [0.74 to 1.41] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.46]
  Nasal congestion, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Nasal congestion, Week 35-40 | 1.01 [0.72 to 1.37] | 0.43 [0.01 to 2.34] | 0.05 [0.00 to 0.28]
  Nasal congestion, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Nasal congestion, Week 35-41 | 0.94 [0.67 to 1.29] | 0.62 [0.20 to 1.44] | 0.04 [0.00 to 0.25]
  Nasal congestion, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Nasal congestion, Week 35-42 | 0.91 [0.65 to 1.23] | 0.41 [0.13 to 0.95] | 0.07 [0.01 to 0.29]
  Nasal congestion, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Nasal congestion, Week 35-43 | 0.88 [0.63 to 1.20] | 0.50 [0.22 to 0.98] | 0.07 [0.01 to 0.27]
  Nasal congestion, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Nasal congestion, Week 35-44 | 0.85 [0.61 to 1.17] | 0.43 [0.20 to 0.82] | 0.06 [0.00 to 0.24]
  Nasal congestion, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Nasal congestion, Week 35-45 | 0.85 [0.61 to 1.16] | 0.40 [0.18 to 0.79] | 0.08 [0.02 to 0.23]
  Nasal congestion, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Nasal congestion, Week 35-46 | 0.85 [0.62 to 1.15] | 0.33 [0.11 to 0.74] | 0.08 [0.02 to 0.22]
  Nasal congestion, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Nasal congestion, Week 35-47 | 0.85 [0.61 to 1.16] | 0.31 [0.11 to 0.70] | 0.07 [0.01 to 0.21]
  Nasal congestion, Week 35-48 | 0.85 [0.60 to 1.15] | 0.30 [0.10 to 0.68] | 0.07 [0.01 to 0.21]
  Oropharyngeal pain, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Oropharyngeal pain, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Oropharyngeal pain, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Oropharyngeal pain, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Oropharyngeal pain, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Oropharyngeal pain, Week 35-37 | 2.27 [1.64 to 3.06] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Oropharyngeal pain, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Oropharyngeal pain, Week 35-38 | 1.80 [1.29 to 2.44] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.67]
  Oropharyngeal pain, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Oropharyngeal pain, Week 35-39 | 1.70 [1.31 to 2.17] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.46]
  Oropharyngeal pain, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Oropharyngeal pain, Week 35-40 | 1.58 [1.16 to 2.10] | 0.22 [0.01 to 1.19] | 0.09 [0.00 to 0.44]
  Oropharyngeal pain, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Oropharyngeal pain, Week 35-41 | 1.53 [1.15 to 2.00] | 0.50 [0.05 to 1.94] | 0.08 [0.00 to 0.36]
  Oropharyngeal pain, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Oropharyngeal pain, Week 35-42 | 1.46 [1.07 to 1.94] | 0.41 [0.10 to 1.09] | 0.11 [0.02 to 0.34]
  Oropharyngeal pain, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Oropharyngeal pain, Week 35-43 | 1.43 [1.04 to 1.91] | 0.44 [0.09 to 1.27] | 0.10 [0.02 to 0.31]
  Oropharyngeal pain, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Oropharyngeal pain, Week 35-44 | 1.41 [1.02 to 1.88] | 0.48 [0.07 to 1.63] | 0.11 [0.02 to 0.33]
  Oropharyngeal pain, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Oropharyngeal pain, Week 35-45 | 1.39 [1.01 to 1.87] | 0.48 [0.13 to 1.22] | 0.16 [0.02 to 0.51]
  Oropharyngeal pain, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Oropharyngeal pain, Week 35-46 | 1.37 [0.99 to 1.84] | 0.39 [0.08 to 1.15] | 0.15 [0.02 to 0.49]
  Oropharyngeal pain, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Oropharyngeal pain, Week 35-47 | 1.34 [0.97 to 1.82] | 0.37 [0.08 to 1.10] | 0.17 [0.02 to 0.60]
  Oropharyngeal pain, Week 35-48 | 1.33 [0.96 to 1.80] | 0.36 [0.07 to 1.06] | 0.17 [0.02 to 0.59]
  Rhinorrhoea, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Rhinorrhoea, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Rhinorrhoea, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Rhinorrhoea, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Rhinorrhoea, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Rhinorrhoea, Week 35-37 | 3.28 [2.17 to 4.74] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Rhinorrhoea, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Rhinorrhoea, Week 35-38 | 2.83 [2.07 to 3.78] | 6.25 [0.12 to 31.55] | 0.00 [0.00 to 0.34]
  Rhinorrhoea, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Rhinorrhoea, Week 35-39 | 2.58 [1.91 to 3.41] | 0.82 [0.02 to 4.48] | 0.00 [0.00 to 0.24]
  Rhinorrhoea, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Rhinorrhoea, Week 35-40 | 2.55 [1.91 to 3.34] | 1.08 [0.34 to 2.54] | 0.00 [0.00 to 0.17]
  Rhinorrhoea, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Rhinorrhoea, Week 35-41 | 2.47 [1.83 to 3.26] | 1.36 [0.66 to 2.48] | 0.00 [0.00 to 0.15]
  Rhinorrhoea, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Rhinorrhoea, Week 35-42 | 2.38 [1.74 to 3.16] | 1.07 [0.53 to 1.90] | 0.00 [0.00 to 0.13]
  Rhinorrhoea, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Rhinorrhoea, Week 35-43 | 2.36 [1.70 to 3.19] | 1.19 [0.70 to 1.88] | 0.00 [0.00 to 0.13]
  Rhinorrhoea, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Rhinorrhoea, Week 35-44 | 2.32 [1.67 to 3.13] | 1.16 [0.66 to 1.88] | 0.00 [0.00 to 0.11]
  Rhinorrhoea, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Rhinorrhoea, Week 35-45 | 2.29 [1.64 to 3.10] | 1.05 [0.54 to 1.83] | 0.08 [0.00 to 0.46]
  Rhinorrhoea, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Rhinorrhoea, Week 35-46 | 2.26 [1.61 to 3.09] | 0.88 [0.38 to 1.75] | 0.08 [0.00 to 0.45]
  Rhinorrhoea, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Rhinorrhoea, Week 35-47 | 2.25 [1.60 to 3.07] | 0.87 [0.37 to 1.74] | 0.07 [0.00 to 0.43]
  Rhinorrhoea, Week 35-48 | 2.23 [1.58 to 3.05] | 0.85 [0.36 to 1.68] | 0.07 [0.00 to 0.42]
  Wheezing, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Wheezing, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Wheezing, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Wheezing, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Wheezing, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Wheezing, Week 35-37 | 0.93 [0.59 to 1.40] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Wheezing, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Wheezing, Week 35-38 | 0.75 [0.46 to 1.14] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Wheezing, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Wheezing, Week 35-39 | 0.60 [0.35 to 0.95] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Wheezing, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Wheezing, Week 35-40 | 0.61 [0.35 to 0.97] | 0.22 [0.01 to 1.19] | 0.00 [0.00 to 0.17]
  Wheezing, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Wheezing, Week 35-41 | 0.57 [0.31 to 0.94] | 0.37 [0.08 to 1.08] | 0.00 [0.00 to 0.15]
  Wheezing, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Wheezing, Week 35-42 | 0.54 [0.31 to 0.89] | 0.25 [0.05 to 0.72] | 0.00 [0.00 to 0.13]
  Wheezing, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Wheezing, Week 35-43 | 0.53 [0.31 to 0.85] | 0.31 [0.09 to 0.77] | 0.00 [0.00 to 0.13]
  Wheezing, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Wheezing, Week 35-44 | 0.52 [0.31 to 0.81] | 0.48 [0.15 to 1.15] | 0.00 [0.00 to 0.11]
  Wheezing, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Wheezing, Week 35-45 | 0.51 [0.31 to 0.79] | 0.40 [0.11 to 1.02] | 0.00 [0.00 to 0.10]
  Wheezing, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Wheezing, Week 35-46 | 0.50 [0.30 to 0.78] | 0.39 [0.10 to 1.01] | 0.00 [0.00 to 0.09]
  Wheezing, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Wheezing, Week 35-47 | 0.50 [0.30 to 0.78] | 0.40 [0.13 to 0.95] | 0.00 [0.00 to 0.09]
  Wheezing, Week 35-48 | 0.49 [0.30 to 0.77] | 0.39 [0.13 to 0.92] | 0.00 [0.00 to 0.09]

83. Secondary Outcome: Cumulative Incidence Rates of Gastrointestinal Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhoea, nausea, and vomiting. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who received the ADR card
  * The numerator was the number of subjects from the denominator who reported any AEIs on the ADR card within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Any, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Any, Week 35-37 | 2.11 [2.11 to 1.30] | 0.00 [0.00 to 45.93] | 0.19 [0.00 to 1.60]
  Any, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Any, Week 35-38 | 1.95 [1.40 to 2.64] | 6.25 [0.12 to 31.55] | 0.09 [0.00 to 0.77]
  Any, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Any, Week 35-39 | 1.76 [1.23 to 2.42] | 0.82 [0.02 to 4.48] | 0.06 [0.00 to 0.52]
  Any, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Any, Week 35-40 | 1.70 [1.28 to 2.22] | 1.08 [0.35 to 2.50] | 0.05 [0.00 to 0.38]
  Any, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Any, Week 35-41 | 1.65 [1.24 to 2.14] | 0.87 [0.35 to 1.78] | 0.04 [0.00 to 0.31]
  Any, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Any, Week 35-42 | 1.61 [1.22 to 2.08] | 0.57 [0.23 to 1.18] | 0.04 [0.00 to 0.28]
  Any, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Any, Week 35-43 | 1.58 [1.20 to 2.05] | 0.44 [0.15 to 0.98] | 0.07 [0.00 to 0.53]
  Any, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Any, Week 35-44 | 1.54 [1.17 to 1.98] | 0.43 [0.10 to 1.19] | 0.06 [0.00 to 0.37]
  Any, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Any, Week 35-45 | 1.55 [1.21 to 1.96] | 0.53 [0.21 to 1.10] | 0.13 [0.00 to 0.76]
  Any, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Any, Week 35-46 | 1.55 [1.21 to 1.95] | 0.46 [0.17 to 0.99] | 0.15 [0.01 to 0.69]
  Any, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Any, Week 35-47 | 1.52 [1.19 to 1.92] | 0.44 [0.16 to 0.95] | 0.14 [0.01 to 0.66]
  Any, Week 35-48 | 1.51 [1.18 to 1.90] | 0.42 [0.15 to 0.92] | 0.14 [0.01 to 0.66]
  Decreased appetite, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Decreased appetite, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Decreased appetite, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Decreased appetite, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Decreased appetite, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Decreased appetite, Week 35-37 | 0.73 [0.43 to 1.15] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Decreased appetite, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Decreased appetite, Week 35-38 | 0.59 [0.40 to 0.84] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Decreased appetite, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Decreased appetite, Week 35-39 | 0.54 [0.31 to 0.86] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Decreased appetite, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Decreased appetite, Week 35-40 | 0.50 [0.30 to 0.77] | 0.86 [0.24 to 2.19] | 0.00 [0.00 to 0.17]
  Decreased appetite, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Decreased appetite, Week 35-41 | 0.50 [0.32 to 0.75] | 0.62 [0.20 to 1.44] | 0.00 [0.00 to 0.15]
  Decreased appetite, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Decreased appetite, Week 35-42 | 0.48 [0.31 to 0.72] | 0.41 [0.13 to 0.95] | 0.00 [0.00 to 0.13]
  Decreased appetite, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Decreased appetite, Week 35-43 | 0.46 [0.29 to 0.70] | 0.31 [0.10 to 0.73] | 0.00 [0.00 to 0.13]
  Decreased appetite, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Decreased appetite, Week 35-44 | 0.45 [0.28 to 0.68] | 0.24 [0.07 to 0.61] | 0.00 [0.00 to 0.11]
  Decreased appetite, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Decreased appetite, Week 35-45 | 0.45 [0.30 to 0.65] | 0.24 [0.09 to 0.53] | 0.00 [0.00 to 0.10]
  Decreased appetite, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Decreased appetite, Week 35-46 | 0.46 [0.30 to 0.66] | 0.20 [0.06 to 0.47] | 0.00 [0.00 to 0.09]
  Decreased appetite, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Decreased appetite, Week 35-47 | 0.45 [0.30 to 0.65] | 0.19 [0.06 to 0.45] | 0.00 [0.00 to 0.09]
  Decreased appetite, Week 35-48 | 0.44 [0.30 to 0.64] | 0.18 [0.06 to 0.43] | 0.00 [0.00 to 0.09]
  Diarrhoea, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Diarrhoea, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Diarrhoea, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Diarrhoea, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Diarrhoea, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Diarrhoea, Week 35-37 | 0.97 [0.58 to 1.54] | 0.00 [0.00 to 45.93] | 0.19 [0.00 to 1.60]
  Diarrhoea, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Diarrhoea, Week 35-38 | 0.86 [0.63 to 1.15] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.77]
  Diarrhoea, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Diarrhoea, Week 35-39 | 0.78 [0.59 to 1.02] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.52]
  Diarrhoea, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Diarrhoea, Week 35-40 | 0.76 [0.60 to 0.95] | 0.00 [0.00 to 0.79] | 0.05 [0.00 to 0.38]
  Diarrhoea, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Diarrhoea, Week 35-41 | 0.75 [0.60 to 0.93] | 0.00 [0.00 to 0.46] | 0.04 [0.00 to 0.31]
  Diarrhoea, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Diarrhoea, Week 35-42 | 0.73 [0.59 to 0.90] | 0.00 [0.00 to 0.30] | 0.04 [0.00 to 0.28]
  Diarrhoea, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Diarrhoea, Week 35-43 | 0.72 [0.58 to 0.88] | 0.00 [0.00 to 0.23] | 0.07 [0.00 to 0.53]
  Diarrhoea, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Diarrhoea, Week 35-44 | 0.70 [0.56 to 0.85] | 0.05 [0.00 to 0.27] | 0.06 [0.00 to 0.37]
  Diarrhoea, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Diarrhoea, Week 35-45 | 0.70 [0.56 to 0.85] | 0.08 [0.01 to 0.34] | 0.06 [0.00 to 0.46]
  Diarrhoea, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Diarrhoea, Week 35-46 | 0.70 [0.56 to 0.86] | 0.07 [0.00 to 0.31] | 0.10 [0.01 to 0.41]
  Diarrhoea, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Diarrhoea, Week 35-47 | 0.69 [0.55 to 0.85] | 0.06 [0.00 to 0.30] | 0.10 [0.01 to 0.40]
  Diarrhoea, Week 35-48 | 0.68 [0.55 to 0.84] | 0.06 [0.00 to 0.29] | 0.10 [0.01 to 0.39]
  Nausea, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Nausea, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Nausea, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Nausea, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Nausea, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Nausea, Week 35-37 | 0.97 [0.49 to 1.72] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Nausea, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Nausea, Week 35-38 | 1.01 [0.49 to 1.86] | 6.25 [0.12 to 31.55] | 0.00 [0.00 to 0.34]
  Nausea, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Nausea, Week 35-39 | 0.91 [0.46 to 1.61] | 0.82 [0.02 to 4.48] | 0.00 [0.00 to 0.24]
  Nausea, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Nausea, Week 35-40 | 0.84 [0.45 to 1.43] | 0.22 [0.01 to 1.19] | 0.00 [0.00 to 0.17]
  Nausea, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Nausea, Week 35-41 | 0.80 [0.44 to 1.34] | 0.12 [0.00 to 0.69] | 0.00 [0.00 to 0.15]
  Nausea, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Nausea, Week 35-42 | 0.77 [0.42 to 1.29] | 0.08 [0.00 to 0.46] | 0.00 [0.00 to 0.13]
  Nausea, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Nausea, Week 35-43 | 0.76 [0.42 to 1.27] | 0.06 [0.00 to 0.35] | 0.00 [0.00 to 0.13]
  Nausea, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Nausea, Week 35-44 | 0.75 [0.42 to 1.22] | 0.10 [0.01 to 0.40] | 0.00 [0.00 to 0.11]
  Nausea, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Nausea, Week 35-45 | 0.75 [0.44 to 1.19] | 0.16 [0.04 to 0.41] | 0.03 [0.00 to 0.15]
  Nausea, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Nausea, Week 35-46 | 0.74 [0.43 to 1.17] | 0.13 [0.04 to 0.34] | 0.03 [0.00 to 0.15]
  Nausea, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Nausea, Week 35-47 | 0.72 [0.42 to 1.15] | 0.12 [0.03 to 0.32] | 0.03 [0.00 to 0.14]
  Nausea, Week 35-48 | 0.72 [0.42 to 1.14] | 0.12 [0.03 to 0.31] | 0.03 [0.00 to 0.14]
  Vomiting, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Vomiting, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Vomiting, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Vomiting, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Vomiting, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Vomiting, Week 35-37 | 0.12 [0.02 to 0.38] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Vomiting, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Vomiting, Week 35-38 | 0.17 [0.08 to 0.33] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Vomiting, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Vomiting, Week 35-39 | 0.18 [0.11 to 0.29] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Vomiting, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Vomiting, Week 35-40 | 0.16 [0.09 to 0.25] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 0.17]
  Vomiting, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Vomiting, Week 35-41 | 0.18 [0.11 to 0.26] | 0.12 [0.00 to 0.69] | 0.00 [0.00 to 0.15]
  Vomiting, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Vomiting, Week 35-42 | 0.19 [0.12 to 0.27] | 0.08 [0.00 to 0.46] | 0.00 [0.00 to 0.13]
  Vomiting, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Vomiting, Week 35-43 | 0.19 [0.12 to 0.27] | 0.06 [0.00 to 0.35] | 0.00 [0.00 to 0.13]
  Vomiting, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Vomiting, Week 35-44 | 0.18 [0.12 to 0.27] | 0.05 [0.00 to 0.27] | 0.00 [0.00 to 0.11]
  Vomiting, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Vomiting, Week 35-45 | 0.19 [0.12 to 0.28] | 0.04 [0.00 to 0.22] | 0.05 [0.00 to 0.31]
  Vomiting, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Vomiting, Week 35-46 | 0.19 [0.12 to 0.28] | 0.07 [0.01 to 0.24] | 0.05 [0.00 to 0.30]
  Vomiting, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Vomiting, Week 35-47 | 0.18 [0.12 to 0.27] | 0.06 [0.01 to 0.22] | 0.05 [0.00 to 0.29]
  Vomiting, Week 35-48 | 0.18 [0.12 to 0.27] | 0.06 [0.01 to 0.22] | 0.05 [0.00 to 0.28]

84. Secondary Outcome: Cumulative Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial edema, and hypersensitivity reactions. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Any, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Any, Week 35-37 | 0.69 [0.01 to 4.09] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Any, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Any, Week 35-38 | 0.63 [0.04 to 2.86] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.53]
  Any, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Any, Week 35-39 | 0.54 [0.04 to 2.29] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.37]
  Any, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Any, Week 35-40 | 0.52 [0.04 to 2.16] | 0.43 [0.02 to 2.14] | 0.05 [0.00 to 0.29]
  Any, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Any, Week 35-41 | 0.48 [0.04 to 1.91] | 0.62 [0.06 to 2.42] | 0.04 [0.00 to 0.24]
  Any, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Any, Week 35-42 | 0.45 [0.04 to 1.82] | 0.49 [0.12 to 1.34] | 0.04 [0.00 to 0.22]
  Any, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Any, Week 35-43 | 0.44 [0.04 to 1.76] | 0.37 [0.09 to 1.00] | 0.03 [0.00 to 0.20]
  Any, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Any, Week 35-44 | 0.43 [0.04 to 1.68] | 0.43 [0.07 to 1.42] | 0.03 [0.00 to 0.18]
  Any, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Any, Week 35-45 | 0.43 [0.04 to 1.63] | 0.36 [0.05 to 1.23] | 0.05 [0.01 to 0.19]
  Any, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Any, Week 35-46 | 0.42 [0.04 to 1.63] | 0.29 [0.03 to 1.14] | 0.05 [0.01 to 0.18]
  Any, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Any, Week 35-47 | 0.42 [0.04 to 1.61] | 0.28 [0.03 to 1.09] | 0.05 [0.01 to 0.17]
  Any, Week 35-48 | 0.41 [0.04 to 1.59] | 0.27 [0.03 to 1.05] | 0.05 [0.01 to 0.17]
  Anaphylactic reactions, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Anaphylactic reactions, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Anaphylactic reactions, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Anaphylactic reactions, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Anaphylactic reactions, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Anaphylactic reactions, Week 35-37 | 0.61 [0.01 to 4.06] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Anaphylactic reactions, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Anaphylactic reactions, Week 35-38 | 0.52 [0.01 to 3.09] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Anaphylactic reactions, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Anaphylactic reactions, Week 35-39 | 0.42 [0.01 to 2.37] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Anaphylactic reactions, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Anaphylactic reactions, Week 35-40 | 0.38 [0.01 to 2.25] | 0.43 [0.02 to 2.14] | 0.00 [0.00 to 0.17]
  Anaphylactic reactions, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Anaphylactic reactions, Week 35-41 | 0.33 [0.00 to 2.04] | 0.50 [0.05 to 1.94] | 0.00 [0.00 to 0.15]
  Anaphylactic reactions, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Anaphylactic reactions, Week 35-42 | 0.31 [0.00 to 1.93] | 0.33 [0.04 to 1.21] | 0.00 [0.00 to 0.13]
  Anaphylactic reactions, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Anaphylactic reactions, Week 35-43 | 0.30 [0.00 to 1.86] | 0.25 [0.03 to 0.93] | 0.00 [0.00 to 0.13]
  Anaphylactic reactions, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Anaphylactic reactions, Week 35-44 | 0.29 [0.00 to 1.78] | 0.34 [0.03 to 1.39] | 0.00 [0.00 to 0.11]
  Anaphylactic reactions, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Anaphylactic reactions, Week 35-45 | 0.28 [0.00 to 1.74] | 0.28 [0.02 to 1.20] | 0.03 [0.00 to 0.15]
  Anaphylactic reactions, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Anaphylactic reactions, Week 35-46 | 0.28 [0.00 to 1.74] | 0.23 [0.01 to 1.10] | 0.03 [0.00 to 0.15]
  Anaphylactic reactions, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Anaphylactic reactions, Week 35-47 | 0.28 [0.00 to 1.72] | 0.22 [0.01 to 1.05] | 0.02 [0.00 to 0.14]
  Anaphylactic reactions, Week 35-48 | 0.27 [0.00 to 1.70] | 0.21 [0.01 to 1.02] | 0.02 [0.00 to 0.14]
  Facial oedema, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Facial oedema, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Facial oedema, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Facial oedema, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Facial oedema, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Facial oedema, Week 35-37 | 0.04 [0.00 to 0.27] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Facial oedema, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Facial oedema, Week 35-38 | 0.06 [0.01 to 0.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Facial oedema, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Facial oedema, Week 35-39 | 0.05 [0.01 to 0.17] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Facial oedema, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Facial oedema, Week 35-40 | 0.04 [0.01 to 0.15] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 0.17]
  Facial oedema, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Facial oedema, Week 35-41 | 0.05 [0.01 to 0.14] | 0.00 [0.00 to 0.46] | 0.00 [0.00 to 0.15]
  Facial oedema, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Facial oedema, Week 35-42 | 0.04 [0.01 to 0.13] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 0.13]
  Facial oedema, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Facial oedema, Week 35-43 | 0.04 [0.01 to 0.12] | 0.00 [0.00 to 0.23] | 0.00 [0.00 to 0.13]
  Facial oedema, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Facial oedema, Week 35-44 | 0.05 [0.01 to 0.12] | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 0.11]
  Facial oedema, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Facial oedema, Week 35-45 | 0.05 [0.02 to 0.12] | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 0.10]
  Facial oedema, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Facial oedema, Week 35-46 | 0.05 [0.02 to 0.12] | 0.00 [0.00 to 0.12] | 0.00 [0.00 to 0.09]
  Facial oedema, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Facial oedema, Week 35-47 | 0.05 [0.02 to 0.11] | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.09]
  Facial oedema, Week 35-48 | 0.05 [0.02 to 0.11] | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.09]
  Hypersensitivity reactions, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Hypersensitivity reactions, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Hypersensitivity reactions, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Hypersensitivity reactions, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Hypersensitivity reactions, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Hypersensitivity reactions, Week 35-37 | 0.08 [0.01 to 0.29] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Hypersensitivity reactions, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Hypersensitivity reactions, Week 35-38 | 0.10 [0.03 to 0.23] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.53]
  Hypersensitivity reactions, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Hypersensitivity reactions, Week 35-39 | 0.09 [0.03 to 0.18] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.37]
  Hypersensitivity reactions, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Hypersensitivity reactions, Week 35-40 | 0.11 [0.05 to 0.23] | 0.00 [0.00 to 0.79] | 0.05 [0.00 to 0.29]
  Hypersensitivity reactions, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Hypersensitivity reactions, Week 35-41 | 0.13 [0.06 to 0.25] | 0.12 [0.00 to 0.69] | 0.04 [0.00 to 0.24]
  Hypersensitivity reactions, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Hypersensitivity reactions, Week 35-42 | 0.12 [0.06 to 0.23] | 0.16 [0.02 to 0.59] | 0.04 [0.00 to 0.22]
  Hypersensitivity reactions, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Hypersensitivity reactions, Week 35-43 | 0.12 [0.05 to 0.22] | 0.12 [0.02 to 0.45] | 0.03 [0.00 to 0.20]
  Hypersensitivity reactions, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Hypersensitivity reactions, Week 35-44 | 0.12 [0.06 to 0.21] | 0.10 [0.01 to 0.35] | 0.03 [0.00 to 0.18]
  Hypersensitivity reactions, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Hypersensitivity reactions, Week 35-45 | 0.11 [0.06 to 0.20] | 0.08 [0.01 to 0.29] | 0.03 [0.00 to 0.17]
  Hypersensitivity reactions, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Hypersensitivity reactions, Week 35-46 | 0.11 [0.06 to 0.20] | 0.07 [0.01 to 0.24] | 0.03 [0.00 to 0.16]
  Hypersensitivity reactions, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Hypersensitivity reactions, Week 35-47 | 0.11 [0.06 to 0.20] | 0.06 [0.01 to 0.22] | 0.02 [0.00 to 0.16]
  Hypersensitivity reactions, Week 35-48 | 0.11 [0.06 to 0.19] | 0.06 [0.01 to 0.22] | 0.02 [0.00 to 0.15]

85. Secondary Outcome: Cumulative Incidence Rates of Rash Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. The cumulative incidence rates AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Week 35-37 | 0.77 [0.46 to 1.20] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Week 35-38 | 0.65 [0.38 to 1.04] | 0.00 [0.00 to 20.59] | 0.19 [0.02 to 0.69]
  Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Week 35-39 | 0.52 [0.34 to 0.77] | 0.00 [0.00 to 2.98] | 0.13 [0.01 to 0.49]
  Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Week 35-40 | 0.54 [0.38 to 0.73] | 0.22 [0.01 to 1.19] | 0.14 [0.03 to 0.41]
  Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Week 35-41 | 0.48 [0.34 to 0.67] | 0.37 [0.08 to 1.08] | 0.12 [0.02 to 0.34]
  Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Week 35-42 | 0.46 [0.33 to 0.62] | 0.25 [0.05 to 0.72] | 0.11 [0.02 to 0.31]
  Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Week 35-43 | 0.46 [0.33 to 0.63] | 0.31 [0.10 to 0.73] | 0.10 [0.02 to 0.30]
  Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Week 35-44 | 0.47 [0.34 to 0.63] | 0.29 [0.11 to 0.63] | 0.09 [0.02 to 0.26]
  Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Week 35-45 | 0.46 [0.33 to 0.62] | 0.24 [0.09 to 0.53] | 0.08 [0.01 to 0.25]
  Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Week 35-46 | 0.46 [0.33 to 0.63] | 0.23 [0.09 to 0.47] | 0.08 [0.01 to 0.24]
  Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Week 35-47 | 0.45 [0.32 to 0.62] | 0.25 [0.11 to 0.49] | 0.07 [0.01 to 0.23]
  Week 35-48 | 0.45 [0.32 to 0.62] | 0.27 [0.12 to 0.52] | 0.07 [0.01 to 0.23]

86. Secondary Outcome: Cumulative Incidence Rates of Musculoskeletal Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Musculoskeletal adverse events include any musculoskeletal adverse events, arthropathy and muscle aches/myalgia. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50]
  Any, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Any, Week 35-37 | 4.25 [3.33 to 5.34] | 0.00 [0.00 to 45.93] | 0.38 [0.05 to 1.35]
  Any, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Any, Week 35-38 | 3.79 [2.92 to 4.83] | 0.00 [0.00 to 20.59] | 0.37 [0.10 to 0.96]
  Any, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Any, Week 35-39 | 3.59 [2.91 to 4.37] | 0.00 [0.00 to 2.98] | 0.51 [0.22 to 1.01]
  Any, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Any, Week 35-40 | 3.41 [2.80 to 4.12] | 0.86 [0.03 to 4.26] | 0.51 [0.21 to 1.03]
  Any, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Any, Week 35-41 | 3.30 [2.70 to 3.99] | 0.50 [0.05 to 1.94] | 0.43 [0.16 to 0.93]
  Any, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Any, Week 35-42 | 3.21 [2.58 to 3.94] | 0.49 [0.06 to 1.81] | 0.40 [0.15 to 0.86]
  Any, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Any, Week 35-43 | 3.21 [2.57 to 3.97] | 0.44 [0.10 to 1.22] | 0.44 [0.17 to 0.92]
  Any, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Any, Week 35-44 | 3.15 [2.50 to 3.91] | 0.63 [0.08 to 2.19] | 0.37 [0.12 to 0.88]
  Any, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Any, Week 35-45 | 3.13 [2.51 to 3.85] | 0.61 [0.10 to 1.97] | 0.36 [0.13 to 0.81]
  Any, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Any, Week 35-46 | 3.09 [2.48 to 3.81] | 0.52 [0.06 to 1.97] | 0.40 [0.16 to 0.83]
  Any, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Any, Week 35-47 | 3.08 [2.46 to 3.79] | 0.50 [0.05 to 1.89] | 0.39 [0.15 to 0.80]
  Any, Week 35-48 | 3.05 [2.43 to 3.77] | 0.54 [0.07 to 1.91] | 0.38 [0.15 to 0.80]
  Arthropathy, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Arthropathy, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Arthropathy, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Arthropathy, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Arthropathy, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Arthropathy, Week 35-37 | 1.42 [0.99 to 1.97] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Arthropathy, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Arthropathy, Week 35-38 | 1.23 [0.81 to 1.77] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.53]
  Arthropathy, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Arthropathy, Week 35-39 | 1.08 [0.70 to 1.59] | 0.00 [0.00 to 2.98] | 0.06 [0.00 to 0.37]
  Arthropathy, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Arthropathy, Week 35-40 | 1.03 [0.66 to 1.52] | 0.65 [0.03 to 3.20] | 0.05 [0.00 to 0.29]
  Arthropathy, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Arthropathy, Week 35-41 | 0.97 [0.63 to 1.43] | 0.37 [0.04 to 1.45] | 0.04 [0.00 to 0.24]
  Arthropathy, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Arthropathy, Week 35-42 | 0.93 [0.61 to 1.36] | 0.33 [0.04 to 1.21] | 0.04 [0.00 to 0.22]
  Arthropathy, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Arthropathy, Week 35-43 | 0.93 [0.61 to 1.37] | 0.25 [0.03 to 0.93] | 0.03 [0.00 to 0.20]
  Arthropathy, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Arthropathy, Week 35-44 | 0.92 [0.60 to 1.34] | 0.34 [0.03 to 1.39] | 0.03 [0.00 to 0.18]
  Arthropathy, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Arthropathy, Week 35-45 | 0.91 [0.60 to 1.32] | 0.28 [0.02 to 1.20] | 0.03 [0.00 to 0.17]
  Arthropathy, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Arthropathy, Week 35-46 | 0.89 [0.58 to 1.30] | 0.23 [0.01 to 1.10] | 0.03 [0.00 to 0.16]
  Arthropathy, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Arthropathy, Week 35-47 | 0.88 [0.57 to 1.28] | 0.22 [0.01 to 1.05] | 0.02 [0.00 to 0.16]
  Arthropathy, Week 35-48 | 0.87 [0.57 to 1.27] | 0.21 [0.01 to 1.02] | 0.02 [0.00 to 0.15]
  Myalgia, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Myalgia, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Myalgia, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Myalgia, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Myalgia, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Myalgia, Week 35-37 | 3.77 [2.67 to 5.16] | 0.00 [0.00 to 45.93] | 0.38 [0.05 to 1.35]
  Myalgia, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Myalgia, Week 35-38 | 3.41 [2.53 to 4.48] | 0.00 [0.00 to 20.59] | 0.28 [0.06 to 0.83]
  Myalgia, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Myalgia, Week 35-39 | 3.21 [2.60 to 3.92] | 0.00 [0.00 to 2.98] | 0.45 [0.18 to 0.92]
  Myalgia, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Myalgia, Week 35-40 | 3.07 [2.51 to 3.72] | 0.86 [0.03 to 4.26] | 0.47 [0.17 to 1.01]
  Myalgia, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Myalgia, Week 35-41 | 2.98 [2.42 to 3.62] | 0.50 [0.05 to 1.94] | 0.39 [0.13 to 0.90]
  Myalgia, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Myalgia, Week 35-42 | 2.90 [2.33 to 3.58] | 0.49 [0.06 to 1.81] | 0.36 [0.12 to 0.84]
  Myalgia, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Myalgia, Week 35-43 | 2.91 [2.32 to 3.60] | 0.44 [0.10 to 1.22] | 0.41 [0.14 to 0.92]
  Myalgia, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Myalgia, Week 35-44 | 2.84 [2.25 to 3.54] | 0.63 [0.08 to 2.19] | 0.34 [0.09 to 0.87]
  Myalgia, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Myalgia, Week 35-45 | 2.83 [2.27 to 3.49] | 0.61 [0.10 to 1.97] | 0.34 [0.11 to 0.79]
  Myalgia, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Myalgia, Week 35-46 | 2.80 [2.24 to 3.45] | 0.52 [0.06 to 1.97] | 0.38 [0.14 to 0.82]
  Myalgia, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Myalgia, Week 35-47 | 2.79 [2.23 to 3.44] | 0.50 [0.05 to 1.89] | 0.36 [0.13 to 0.79]
  Myalgia, Week 35-48 | 2.76 [2.20 to 3.42] | 0.54 [0.07 to 1.91] | 0.36 [0.13 to 0.78]

87. Secondary Outcome: Cumulative Incidence Rates of Neurological Adverse Events Recorded in EHR, by Vaccine Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Neurological adverse events include any neurological adverse events, Bell's palsy, Guillain-Barre Syndrome, peripheral tremor and seizure/febrile convulsions. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Any, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Any, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Any, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Any, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Any, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Any, Week 35-37 | 0.28 [0.11 to 0.58] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Any, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Any, Week 35-38 | 0.29 [0.16 to 0.47] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Any, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Any, Week 35-39 | 0.26 [0.15 to 0.41] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Any, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Any, Week 35-40 | 0.21 [0.11 to 0.36] | 0.22 [0.01 to 1.19] | 0.00 [0.00 to 0.17]
  Any, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Any, Week 35-41 | 0.21 [0.12 to 0.33] | 0.25 [0.02 to 0.97] | 0.04 [0.00 to 0.31]
  Any, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Any, Week 35-42 | 0.19 [0.11 to 0.32] | 0.16 [0.02 to 0.60] | 0.04 [0.00 to 0.28]
  Any, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Any, Week 35-43 | 0.19 [0.10 to 0.31] | 0.12 [0.01 to 0.47] | 0.03 [0.00 to 0.27]
  Any, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Any, Week 35-44 | 0.18 [0.10 to 0.31] | 0.10 [0.01 to 0.40] | 0.03 [0.00 to 0.18]
  Any, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Any, Week 35-45 | 0.18 [0.10 to 0.30] | 0.08 [0.01 to 0.34] | 0.03 [0.00 to 0.15]
  Any, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Any, Week 35-46 | 0.17 [0.10 to 0.29] | 0.07 [0.00 to 0.31] | 0.03 [0.00 to 0.15]
  Any, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Any, Week 35-47 | 0.17 [0.09 to 0.29] | 0.09 [0.02 to 0.27] | 0.02 [0.00 to 0.14]
  Any, Week 35-48 | 0.17 [0.09 to 0.29] | 0.09 [0.02 to 0.26] | 0.02 [0.00 to 0.14]
  Bell's palsy, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Bell's palsy, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Bell's palsy, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Bell's palsy, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Bell's palsy, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Bell's palsy, Week 35-37 | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Bell's palsy, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Bell's palsy, Week 35-38 | 0.00 [0.00 to 0.07] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Bell's palsy, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Bell's palsy, Week 35-39 | 0.01 [0.00 to 0.08] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Bell's palsy, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Bell's palsy, Week 35-40 | 0.01 [0.00 to 0.06] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 0.17]
  Bell's palsy, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Bell's palsy, Week 35-41 | 0.01 [0.00 to 0.06] | 0.00 [0.00 to 0.46] | 0.00 [0.00 to 0.15]
  Bell's palsy, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Bell's palsy, Week 35-42 | 0.01 [0.00 to 0.05] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 0.13]
  Bell's palsy, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Bell's palsy, Week 35-43 | 0.01 [0.00 to 0.05] | 0.00 [0.00 to 0.23] | 0.00 [0.00 to 0.13]
  Bell's palsy, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Bell's palsy, Week 35-44 | 0.01 [0.00 to 0.05] | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 0.11]
  Bell's palsy, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Bell's palsy, Week 35-45 | 0.01 [0.00 to 0.05] | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 0.10]
  Bell's palsy, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Bell's palsy, Week 35-46 | 0.01 [0.00 to 0.05] | 0.00 [0.00 to 0.12] | 0.00 [0.00 to 0.09]
  Bell's palsy, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Bell's palsy, Week 35-47 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.09]
  Bell's palsy, Week 35-48 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.09]
  Guillain-Barre Syndrome, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Guillain-Barre Syndrome, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Guillain-Barre Syndrome, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Guillain-Barre Syndrome, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Guillain-Barre Syndrome, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Guillain-Barre Syndrome, Week 35-37 | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Guillain-Barre Syndrome, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Guillain-Barre Syndrome, Week 35-38 | 0.00 [0.00 to 0.07] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Guillain-Barre Syndrome, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Guillain-Barre Syndrome, Week 35-39 | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Guillain-Barre Syndrome, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Guillain-Barre Syndrome, Week 35-40 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 0.17]
  Guillain-Barre Syndrome, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Guillain-Barre Syndrome, Week 35-41 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.46] | 0.00 [0.00 to 0.15]
  Guillain-Barre Syndrome, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Guillain-Barre Syndrome, Week 35-42 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 0.13]
  Guillain-Barre Syndrome, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Guillain-Barre Syndrome, Week 35-43 | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.23] | 0.00 [0.00 to 0.13]
  Guillain-Barre Syndrome, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Guillain-Barre Syndrome, Week 35-44 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.18] | 0.00 [0.00 to 0.11]
  Guillain-Barre Syndrome, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Guillain-Barre Syndrome, Week 35-45 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.15] | 0.00 [0.00 to 0.10]
  Guillain-Barre Syndrome, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Guillain-Barre Syndrome, Week 35-46 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.12] | 0.00 [0.00 to 0.09]
  Guillain-Barre Syndrome, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Guillain-Barre Syndrome, Week 35-47 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.09]
  Guillain-Barre Syndrome, Week 35-48 | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.09]
  Peripheral tremor, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Peripheral tremor, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Peripheral tremor, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Peripheral tremor, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Peripheral tremor, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Peripheral tremor, Week 35-37 | 0.24 [0.09 to 0.53] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Peripheral tremor, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Peripheral tremor, Week 35-38 | 0.27 [0.15 to 0.45] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Peripheral tremor, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Peripheral tremor, Week 35-39 | 0.24 [0.12 to 0.41] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Peripheral tremor, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Peripheral tremor, Week 35-40 | 0.19 [0.09 to 0.35] | 0.22 [0.01 to 1.19] | 0.00 [0.00 to 0.17]
  Peripheral tremor, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Peripheral tremor, Week 35-41 | 0.19 [0.10 to 0.32] | 0.25 [0.02 to 0.97] | 0.00 [0.00 to 0.15]
  Peripheral tremor, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Peripheral tremor, Week 35-42 | 0.18 [0.09 to 0.31] | 0.16 [0.02 to 0.60] | 0.00 [0.00 to 0.13]
  Peripheral tremor, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Peripheral tremor, Week 35-43 | 0.17 [0.09 to 0.30] | 0.12 [0.01 to 0.47] | 0.00 [0.00 to 0.13]
  Peripheral tremor, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Peripheral tremor, Week 35-44 | 0.17 [0.09 to 0.30] | 0.10 [0.01 to 0.40] | 0.00 [0.00 to 0.11]
  Peripheral tremor, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Peripheral tremor, Week 35-45 | 0.17 [0.09 to 0.29] | 0.08 [0.01 to 0.34] | 0.00 [0.00 to 0.10]
  Peripheral tremor, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Peripheral tremor, Week 35-46 | 0.16 [0.08 to 0.28] | 0.07 [0.00 to 0.31] | 0.00 [0.00 to 0.09]
  Peripheral tremor, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Peripheral tremor, Week 35-47 | 0.16 [0.08 to 0.28] | 0.06 [0.00 to 0.30] | 0.00 [0.00 to 0.09]
  Peripheral tremor, Week 35-48 | 0.16 [0.08 to 0.28] | 0.06 [0.00 to 0.29] | 0.00 [0.00 to 0.09]
  Seizure / Febrile convulsions, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Seizure / Febrile convulsions, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Seizure / Febrile convulsions, Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Seizure / Febrile convulsions, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Seizure / Febrile convulsions, Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Seizure / Febrile convulsions, Week 35-37 | 0.04 [0.00 to 0.25] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.69]
  Seizure / Febrile convulsions, Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Seizure / Febrile convulsions, Week 35-38 | 0.02 [0.00 to 0.11] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  Seizure / Febrile convulsions, Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Seizure / Febrile convulsions, Week 35-39 | 0.01 [0.00 to 0.07] | 0.00 [0.00 to 2.98] | 0.00 [0.00 to 0.24]
  Seizure / Febrile convulsions, Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Seizure / Febrile convulsions, Week 35-40 | 0.01 [0.00 to 0.06] | 0.00 [0.00 to 0.79] | 0.00 [0.00 to 0.17]
  Seizure / Febrile convulsions, Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Seizure / Febrile convulsions, Week 35-41 | 0.01 [0.00 to 0.05] | 0.00 [0.00 to 0.46] | 0.04 [0.00 to 0.31]
  Seizure / Febrile convulsions, Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Seizure / Febrile convulsions, Week 35-42 | 0.01 [0.00 to 0.05] | 0.00 [0.00 to 0.30] | 0.04 [0.00 to 0.28]
  Seizure / Febrile convulsions, Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Seizure / Febrile convulsions, Week 35-43 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.23] | 0.03 [0.00 to 0.27]
  Seizure / Febrile convulsions, Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Seizure / Febrile convulsions, Week 35-44 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.18] | 0.03 [0.00 to 0.18]
  Seizure / Febrile convulsions, Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Seizure / Febrile convulsions, Week 35-45 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.15] | 0.03 [0.00 to 0.15]
  Seizure / Febrile convulsions, Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Seizure / Febrile convulsions, Week 35-46 | 0.01 [0.00 to 0.04] | 0.00 [0.00 to 0.12] | 0.03 [0.00 to 0.15]
  Seizure / Febrile convulsions, Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Seizure / Febrile convulsions, Week 35-47 | 0.01 [0.00 to 0.04] | 0.03 [0.00 to 0.23] | 0.02 [0.00 to 0.14]
  Seizure / Febrile convulsions, Week 35-48 | 0.01 [0.00 to 0.04] | 0.03 [0.00 to 0.22] | 0.02 [0.00 to 0.14]

88. Secondary Outcome: Cumulative Incidence Rates of SAEs Recorded in EHR, by Vaccine Group
Description: SAEs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. The cumulative incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  Week 35-36: number analyzed (Participants) | 1 | 1 | 62
  Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.78]
  Week 35-37: number analyzed (Participants) | 2468 | 6 | 532
  Week 35-37 | 0.12 [0.02 to 0.37] | 0.00 [0.00 to 45.93] | 0.19 [0.00 to 1.49]
  Week 35-38: number analyzed (Participants) | 5224 | 16 | 1073
  Week 35-38 | 0.15 [0.06 to 0.34] | 0.00 [0.00 to 20.59] | 0.28 [0.06 to 0.81]
  Week 35-39: number analyzed (Participants) | 9341 | 122 | 1559
  Week 35-39 | 0.12 [0.06 to 0.21] | 0.00 [0.00 to 2.98] | 0.19 [0.04 to 0.56]
  Week 35-40: number analyzed (Participants) | 11398 | 464 | 2144
  Week 35-40 | 0.13 [0.07 to 0.22] | 0.00 [0.00 to 0.79] | 0.19 [0.03 to 0.57]
  Week 35-41: number analyzed (Participants) | 13064 | 807 | 2542
  Week 35-41 | 0.13 [0.06 to 0.23] | 0.00 [0.00 to 0.46] | 0.24 [0.04 to 0.73]
  Week 35-42: number analyzed (Participants) | 13976 | 1219 | 2783
  Week 35-42 | 0.12 [0.06 to 0.22] | 0.08 [0.00 to 0.46] | 0.22 [0.04 to 0.65]
  Week 35-43: number analyzed (Participants) | 14475 | 1601 | 2947
  Week 35-43 | 0.13 [0.06 to 0.26] | 0.06 [0.00 to 0.35] | 0.20 [0.04 to 0.61]
  Week 35-44: number analyzed (Participants) | 15225 | 2072 | 3508
  Week 35-44 | 0.14 [0.05 to 0.30] | 0.10 [0.01 to 0.35] | 0.23 [0.06 to 0.62]
  Week 35-45: number analyzed (Participants) | 15680 | 2475 | 3858
  Week 35-45 | 0.14 [0.06 to 0.28] | 0.12 [0.01 to 0.44] | 0.21 [0.04 to 0.60]
  Week 35-46: number analyzed (Participants) | 16030 | 3052 | 3955
  Week 35-46 | 0.15 [0.06 to 0.31] | 0.10 [0.01 to 0.37] | 0.23 [0.06 to 0.59]
  Week 35-47: number analyzed (Participants) | 16288 | 3210 | 4154
  Week 35-47 | 0.15 [0.06 to 0.31] | 0.09 [0.01 to 0.35] | 0.24 [0.07 to 0.61]
  Week 35-48 | 0.15 [0.06 to 0.33] | 0.09 [0.01 to 0.34] | 0.24 [0.07 to 0.60]

89. Secondary Outcome: Weekly Incidence Rates of Any AEIs Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 1.59 [0.04 to 8.53] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 4.83 [2.34 to 8.70] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 4.07 [0.99 to 10.69] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 1.56 [0.29 to 4.72] | 5.88 [0.00 to 69.40]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 2.10 [0.43 to 6.01] | 20.00 [0.00 to 96.43]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 2.94 [0.10 to 14.43] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 50.00 [1.26 to 98.74] | 0.99 [0.04 to 4.97] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 1.39 [0.04 to 7.50] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 33.33 [0.00 to 100] | 19.05 [3.24 to 49.67] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 50.00 [1.26 to 98.74] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 16.67 [0.02 to 81.43] | 2.02 [0.16 to 8.11] | 0.40 [0.01 to 2.22]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.98 [0.00 to 10.39] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 20.00 [0.02 to 88.39] | 0.36 [0.01 to 2.02] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 1.61 [0.00 to 29.53]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 7.14 [0.02 to 44.90] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 11.11 [0.19 to 51.19] | 50.00 [1.26 to 98.74]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 10.00 [0.00 to 71.81] | 5.88 [0.02 to 38.78] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 3.75 [0.78 to 10.57] | 4.39 [2.03 to 8.17]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 11.82 [9.20 to 14.88] | 0.00 [0.00 to 70.76] | 2.63 [0.72 to 6.60]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 10.81 [7.35 to 15.18] | 0.00 [0.00 to 60.24] | 0.61 [0.01 to 3.60]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 11.52 [9.90 to 13.30] | 10.00 [0.11 to 50.09] | 0.68 [0.00 to 4.80]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 10.39 [5.89 to 16.65] | 11.11 [0.19 to 51.15] | 1.54 [0.32 to 4.43]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 7.72 [4.87 to 11.50] | 6.38 [2.38 to 13.38] | 0.91 [0.02 to 5.16]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 5.63 [2.28 to 11.30] | 1.82 [0.22 to 6.41] | 3.70 [0.50 to 12.30]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 5.88 [1.87 to 13.42] | 7.56 [3.52 to 13.87] | 1.16 [0.03 to 6.31]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 5.43 [2.05 to 11.35] | 17.72 [10.04 to 27.94] | 1.27 [0.03 to 7.12]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 6.25 [3.31 to 10.57] | 3.64 [0.00 to 99.60] | 6.02 [1.48 to 15.53]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 7.62 [4.08 to 12.77] | 7.84 [1.88 to 20.13] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 5.48 [1.98 to 11.73] | 7.69 [0.78 to 26.63] | 1.59 [0.01 to 11.07]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 10.34 [2.07 to 27.92] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.96 [0.00 to 18.80]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 11.64 [9.86 to 13.62] | 0.00 [0.00 to 84.19] | 0.63 [0.02 to 3.50]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 9.77 [7.54 to 12.39] | 16.67 [0.00 to 91.51] | 1.86 [0.75 to 3.79]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 9.31 [7.76 to 11.06] | 0.00 [0.00 to 40.96] | 2.97 [0.96 to 6.82]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 9.75 [6.13 to 14.53] | 7.14 [1.50 to 19.48] | 1.37 [0.22 to 4.43]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 9.04 [6.57 to 12.05] | 8.86 [3.64 to 17.41] | 0.65 [0.00 to 4.69]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 5.12 [2.52 to 9.12] | 6.15 [1.70 to 15.01] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 6.20 [2.56 to 12.27] | 6.10 [0.00 to 86.17] | 1.54 [0.01 to 11.02]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 6.28 [1.99 to 14.32] | 9.38 [3.52 to 19.30] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 7.21 [2.71 to 14.98] | 18.92 [0.00 to 100] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 6.14 [1.96 to 13.99] | 5.41 [0.00 to 68.00] | 9.38 [1.29 to 28.96]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 2.83 [0.59 to 8.05] | 3.70 [0.00 to 99.88] | 3.33 [0.08 to 17.37]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 9.09 [0.00 to 100] | 0.00 [0.00 to 30.85]

90. Secondary Outcome: Cumulative Incidence Rates of Any AEIs Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 month to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 month to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 month to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 month to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 month to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 month to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 month to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 month to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 1.59 [0.04 to 8.53] | 0.00 [0.00 to 84.19]
  6 month to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 month to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 4.07 [1.83 to 7.72] | 0.00 [0.00 to 20.59]
  6 month to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 month to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 4.07 [1.86 to 7.64] | 0.00 [0.00 to 5.78]
  6 month to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 month to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 3.25 [1.55 to 5.94] | 1.27 [0.00 to 13.35]
  6 month to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 month to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 3.02 [1.53 to 5.32] | 2.38 [0.02 to 15.91]
  6 month to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 month to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 3.00 [1.44 to 5.47] | 0.87 [0.08 to 3.41]
  6 month to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 month to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 2.64 [1.20 to 4.98] | 0.86 [0.08 to 3.38]
  6 month to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 month to 5 years, Week 35-46 | 10.00 [0.14 to 48.28] | 2.37 [1.12 to 4.39] | 0.82 [0.08 to 3.22]
  6 month to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 month to 5 years, Week 35-47 | 10.00 [0.14 to 48.28] | 2.32 [1.14 to 4.17] | 0.71 [0.06 to 2.91]
  6 month to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 month to 5 years, Week 35-48 | 10.00 [0.14 to 48.28] | 2.27 [1.11 to 4.10] | 0.70 [0.06 to 2.86]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 3.70 [0.00 to 39.49] | 9.52 [0.71 to 34.64] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 6.90 [0.06 to 39.08] | 5.56 [0.29 to 23.48] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 5.88 [0.15 to 28.66] | 4.00 [0.25 to 16.69] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 5.71 [0.17 to 27.21] | 3.20 [0.17 to 14.11] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 7.32 [0.36 to 30.38] | 2.68 [0.32 to 9.40] | 0.29 [0.01 to 1.61]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 7.14 [0.32 to 30.34] | 2.15 [0.11 to 9.76] | 0.29 [0.01 to 1.61]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 8.51 [1.98 to 21.99] | 1.33 [0.10 to 5.51] | 0.28 [0.01 to 1.55]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 8.51 [1.98 to 21.99] | 1.30 [0.10 to 5.37] | 0.48 [0.06 to 1.71]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 8.33 [2.04 to 21.11] | 1.26 [0.09 to 5.27] | 0.48 [0.06 to 1.71]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 2.63 [0.01 to 18.97] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 2.22 [0.02 to 14.79] | 7.14 [0.04 to 41.49] | 33.33 [0.00 to 99.94]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 3.64 [0.02 to 23.48] | 6.45 [0.34 to 26.78] | 2.86 [0.07 to 14.92]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 3.39 [0.03 to 20.78] | 4.17 [0.48 to 14.52] | 2.86 [0.07 to 14.92]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 3.28 [0.03 to 20.21] | 3.28 [0.33 to 12.04] | 2.78 [0.07 to 14.53]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 3.23 [0.03 to 19.93] | 2.33 [0.22 to 8.82] | 2.00 [0.05 to 10.65]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 2.86 [0.03 to 17.61] | 3.01 [0.99 to 6.89] | 3.92 [1.90 to 7.09]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 2.63 [0.02 to 16.58] | 2.81 [0.92 to 6.43] | 3.89 [1.88 to 7.04]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 2.44 [0.02 to 15.79] | 2.73 [0.89 to 6.26] | 3.82 [1.85 to 6.91]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 2.33 [0.02 to 15.01] | 2.72 [0.89 to 6.23] | 3.82 [1.85 to 6.91]
  18 - 65 years, Weeks 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Weeks 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Weeks 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Weeks 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Weeks 35-37 | 11.82 [9.20 to 14.88] | 0.00 [0.00 to 70.76] | 2.47 [0.68 to 6.20]
  18 - 65 years, Weeks 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Weeks 35-38 | 11.27 [8.66 to 14.35] | 0.00 [0.00 to 40.96] | 1.53 [0.50 to 3.54]
  18 - 65 years, Weeks 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Weeks 35-39 | 11.39 [9.78 to 13.16] | 5.88 [0.15 to 28.69] | 1.27 [0.44 to 2.84]
  18 - 65 years, Weeks 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Weeks 35-40 | 11.19 [9.16 to 13.49] | 10.00 [4.42 to 18.76] | 1.35 [0.62 to 2.54]
  18 - 65 years, Weeks 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Weeks 35-41 | 10.69 [8.73 to 12.91] | 8.05 [4.47 to 13.13] | 1.29 [0.62 to 2.35]
  18 - 65 years, Weeks 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Weeks 35-42 | 10.31 [8.26 to 12.66] | 5.63 [3.25 to 8.99] | 1.51 [0.81 to 2.57]
  18 - 65 years, Weeks 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Weeks 35-43 | 10.11 [8.02 to 12.52] | 6.20 [4.05 to 9.02] | 1.48 [0.81 to 2.47]
  18 - 65 years, Weeks 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Weeks 35-44 | 9.83 [7.72 to 12.29] | 8.09 [5.82 to 10.90] | 1.46 [0.73 to 2.61]
  18 - 65 years, Weeks 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Weeks 35-45 | 9.68 [7.60 to 12.11] | 7.64 [5.53 to 10.22] | 1.81 [0.67 to 3.87]
  18 - 65 years, Weeks 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Weeks 35-46 | 9.60 [7.52 to 12.04] | 7.65 [5.64 to 10.11] | 1.74 [0.65 to 3.73]
  18 - 65 years, Weeks 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Weeks 35-47 | 9.50 [7.43 to 11.92] | 7.66 [5.70 to 10.02] | 1.74 [0.70 to 3.55]
  18 - 65 years, Weeks 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Weeks 35-48 | 9.36 [7.29 to 11.78] | 7.77 [5.84 to 10.10] | 1.70 [0.69 to 3.46]
  >65 years, Weeks 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Weeks 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Weeks 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Weeks 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.92 [0.00 to 17.19]
  >65 years, Weeks 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Weeks 35-37 | 11.64 [9.86 to 13.61] | 0.00 [0.00 to 70.76] | 0.81 [0.12 to 2.67]
  >65 years, Weeks 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Weeks 35-38 | 10.67 [8.97 to 12.56] | 11.11 [0.03 to 62.14] | 1.34 [0.59 to 2.60]
  >65 years, Weeks 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Weeks 35-39 | 10.09 [8.50 to 11.87] | 6.25 [0.16 to 30.23] | 1.85 [0.73 to 3.81]
  >65 years, Weeks 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Weeks 35-40 | 10.03 [8.24 to 12.06] | 6.90 [1.91 to 16.73] | 1.73 [0.67 to 3.60]
  >65 years, Weeks 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Weeks 35-41 | 9.91 [8.10 to 11.98] | 8.03 [4.08 to 13.91] | 1.62 [0.67 to 3.28]
  >65 years, Weeks 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Weeks 35-42 | 9.63 [7.80 to 11.71] | 7.43 [4.22 to 11.95] | 1.51 [0.61 to 3.08]
  >65 years, Weeks 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Weeks 35-43 | 9.53 [7.73 to 11.58] | 7.04 [4.35 to 10.67] | 1.51 [0.63 to 3.01]
  >65 years, Weeks 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Weeks 35-44 | 9.39 [7.61 to 11.42] | 7.47 [4.94 to 10.76] | 1.45 [0.61 to 2.89]
  >65 years, Weeks 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Weeks 35-45 | 9.34 [7.58 to 11.34] | 8.57 [5.97 to 11.83] | 1.41 [0.59 to 2.82]
  >65 years, Weeks 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Weeks 35-46 | 9.30 [7.55 to 11.31] | 8.29 [5.84 to 11.35] | 1.54 [0.71 to 2.89]
  >65 years, Weeks 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Weeks 35-47 | 9.24 [7.47 to 11.25] | 8.02 [5.68 to 10.93] | 1.57 [0.75 to 2.86]
  >65 years, Weeks 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Weeks 35-48 | 9.19 [7.42 to 11.22] | 8.07 [5.77 to 10.91] | 1.56 [0.75 to 2.85]

91. Secondary Outcome: Weekly Incidence Rates of Fever/Pyrexia Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 data sources - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years, and >65 years. Fever/pyrexia = all subjects with a fever/pyrexia read code recorded were considered as having fever/pyrexia, regardless of what temperature had been recorded. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with seasonal influenza vaccine
  Vaccination of subjects happened between weeks 35 and 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 1.45 [0.30 to 4.18] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.90] | 0.00 [0.00 to 19.51]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 0.49 [0.01 to 2.70] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.49 [0.00 to 4.44] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 4.76 [0.03 to 29.74] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.66] | 0.00 [0.00 to 1.47]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.78]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.49 [0.01 to 2.69]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 0.56 [0.15 to 1.42] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 2.40]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 0.81 [0.13 to 2.66] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 2.22]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 0.71 [0.28 to 1.46] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 2.48]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 0.81 [0.07 to 3.27] | 1.59 [0.04 to 8.63] | 0.00 [0.00 to 1.87]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 0.31 [0.02 to 1.39] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 3.30]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.03] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 4.45]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 0.45 [0.01 to 2.91] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 4.20]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 0.32 [0.01 to 1.77] | 0.00 [0.00 to 4.56] | 0.00 [0.00 to 4.56]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 0.45 [0.00 to 3.26] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 4.35]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 0.45 [0.00 to 3.36] | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 0.68 [0.00 to 4.94] | 2.56 [0.00 to 25.31] | 0.00 [0.00 to 5.69]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.98]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 0.40 [0.16 to 0.83] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.16]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 0.43 [0.18 to 0.84] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.97]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 0.41 [0.12 to 1.01] | 0.00 [0.00 to 40.96] | 0.30 [0.00 to 2.21]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 0.23 [0.05 to 0.67] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.01]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 0.39 [0.09 to 1.11] | 2.53 [0.31 to 8.85] | 0.00 [0.00 to 2.35]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 0.00 [0.00 to 0.67] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 0.36 [0.00 to 2.44] | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 5.52]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 0.23 [0.01 to 1.29] | 1.56 [0.00 to 64.84] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 0.88 [0.01 to 6.20] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 10.89]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 11.57]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 30.85]

92. Secondary Outcome: Cumulative Incidence Rates of Fever/Pyrexia Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 data sources - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12, 13 to 17, 18 to 65, and >65 years. Fever/pyrexia = all subjects with a fever/pyrexia read code recorded were considered as having fever/pyrexia, regardless of what temperature had been recorded. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between weeks 35 and 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 1.11 [0.14 to 3.88] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.76 [0.06 to 3.15] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.51 [0.02 to 2.44] | 0.00 [0.00 to 4.56]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.41 [0.01 to 2.18] | 0.00 [0.00 to 4.30]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.43 [0.04 to 1.68] | 0.00 [0.00 to 1.58]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.38 [0.03 to 1.53] | 0.00 [0.00 to 1.57]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.40 [0.06 to 1.29] | 0.00 [0.00 to 1.51]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.37 [0.06 to 1.22] | 0.00 [0.00 to 1.30]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.37 [0.06 to 1.19] | 0.00 [0.00 to 1.28]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 2.38 [0.03 to 14.41] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 1.39 [0.01 to 9.21] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 1.00 [0.01 to 6.59] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.80 [0.01 to 5.53] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.45 [0.00 to 3.38] | 0.00 [0.00 to 1.07]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.31 [0.00 to 2.50] | 0.00 [0.00 to 1.06]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.17 [0.00 to 1.44] | 0.00 [0.00 to 1.03]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.16 [0.00 to 1.40] | 0.00 [0.00 to 0.87]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.16 [0.00 to 1.37] | 0.00 [0.00 to 0.87]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 70.76]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 9.74]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 7.11]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.39 [0.01 to 2.17]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.39 [0.01 to 2.15]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.38 [0.01 to 2.11]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.38 [0.01 to 2.11]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 0.56 [0.15 to 1.42] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 2.25]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 0.70 [0.22 to 1.64] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.13]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 0.70 [0.28 to 1.45] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 0.78]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 0.72 [0.33 to 1.37] | 1.25 [0.03 to 6.77] | 0.00 [0.00 to 0.55]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 0.66 [0.33 to 1.18] | 0.57 [0.01 to 3.16] | 0.00 [0.00 to 0.47]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 0.61 [0.30 to 1.12] | 0.35 [0.01 to 1.95] | 0.00 [0.00 to 0.43]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 0.61 [0.29 to 1.13] | 0.25 [0.01 to 1.37] | 0.00 [0.00 to 0.39]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 0.59 [0.28 to 1.08] | 0.21 [0.01 to 1.15] | 0.00 [0.00 to 0.36]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 0.58 [0.28 to 1.07] | 0.19 [0.00 to 1.03] | 0.00 [0.00 to 0.33]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 0.58 [0.26 to 1.10] | 0.17 [0.00 to 0.94] | 0.00 [0.00 to 0.32]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 0.58 [0.28 to 1.06] | 0.32 [0.04 to 1.15] | 0.00 [0.00 to 0.30]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 0.57 [0.28 to 1.05] | 0.30 [0.04 to 1.10] | 0.00 [0.00 to 0.30]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 0.40 [0.16 to 0.83] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 0.99]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 0.42 [0.23 to 0.68] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 0.49]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 0.41 [0.25 to 0.65] | 0.00 [0.00 to 20.59] | 0.09 [0.00 to 0.67]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 0.38 [0.24 to 0.58] | 0.00 [0.00 to 6.16] | 0.07 [0.00 to 0.52]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 0.38 [0.25 to 0.56] | 1.46 [0.18 to 5.17] | 0.06 [0.00 to 0.47]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 0.36 [0.23 to 0.54] | 0.99 [0.12 to 3.53] | 0.06 [0.00 to 0.43]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 0.36 [0.22 to 0.55] | 0.70 [0.09 to 2.52] | 0.06 [0.00 to 0.42]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 0.36 [0.22 to 0.54] | 0.86 [0.18 to 2.50] | 0.05 [0.00 to 0.40]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 0.35 [0.22 to 0.53] | 0.78 [0.16 to 2.26] | 0.05 [0.00 to 0.39]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 0.35 [0.22 to 0.55] | 0.71 [0.15 to 2.06] | 0.05 [0.00 to 0.38]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 0.35 [0.21 to 0.54] | 0.67 [0.14 to 1.94] | 0.05 [0.00 to 0.37]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 0.35 [0.21 to 0.54] | 0.64 [0.13 to 1.85] | 0.05 [0.00 to 0.37]

93. Secondary Outcome: Weekly Incidence Rates of Local Symptoms Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Local symptoms include local erythema. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.90] | 0.00 [0.00 to 19.51]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.66] | 0.00 [0.00 to 1.47]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.78]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 3.06 [1.93 to 4.60] | 0.00 [0.00 to 70.76] | 0.66 [0.02 to 3.61]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 3.14 [1.56 to 5.58] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 2.22]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 2.19 [1.37 to 3.32] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 2.48]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 3.10 [0.67 to 8.64] | 1.59 [0.04 to 8.63] | 0.00 [0.00 to 1.87]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 1.26 [0.55 to 2.47] | 2.13 [0.26 to 7.48] | 0.00 [0.00 to 3.30]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 0.85 [0.06 to 3.51] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 4.45]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 0.45 [0.01 to 2.91] | 1.68 [0.20 to 5.94] | 0.00 [0.00 to 4.20]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 2.24 [0.76 to 5.02] | 1.27 [0.03 to 6.85] | 0.00 [0.00 to 4.56]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 0.45 [0.00 to 3.33] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 4.35]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 2.24 [0.30 to 7.65] | 3.92 [0.48 to 13.46] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 2.05 [0.10 to 9.40] | 0.00 [0.00 to 9.03] | 0.00 [0.00 to 5.69]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.98]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 1.44 [0.34 to 3.90] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.16]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 0.96 [0.52 to 1.62] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.97]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 1.83 [1.25 to 2.59] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.09]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 1.30 [0.44 to 2.97] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.01]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 1.57 [0.90 to 2.54] | 1.27 [0.03 to 6.85] | 0.00 [0.00 to 2.35]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 0.37 [0.00 to 2.81] | 3.08 [0.37 to 10.68] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 0.36 [0.00 to 2.55] | 1.22 [0.00 to 72.65] | 0.00 [0.00 to 5.52]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 0.47 [0.02 to 2.39] | 3.13 [0.00 to 46.96] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 1.35 [0.09 to 5.79] | 5.41 [0.00 to 99.64] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 2.70 [0.00 to 99.94] | 0.00 [0.00 to 10.89]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 11.57]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 30.85]

94. Secondary Outcome: Cumulative Incidence Rates of Local Symptoms Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Local symptoms include local erythema. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 4.56]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 4.30]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 1.58]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 1.57]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 1.51]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.28] | 0.00 [0.00 to 1.30]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.27] | 0.00 [0.00 to 1.28]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 1.07]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 1.06]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.61] | 0.00 [0.00 to 1.03]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.60] | 0.00 [0.00 to 0.87]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 0.87]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 70.76]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 9.74]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 7.11]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.44]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.43]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.40]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.40]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 3.06 [1.93 to 4.60] | 0.00 [0.00 to 70.76] | 0.62 [0.02 to 3.39]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 3.10 [1.96 to 4.65] | 0.00 [0.00 to 40.96] | 0.31 [0.01 to 1.70]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 2.67 [1.74 to 3.92] | 0.00 [0.00 to 19.51] | 0.21 [0.00 to 1.23]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 2.76 [1.61 to 4.38] | 1.25 [0.03 to 6.77] | 0.15 [0.00 to 0.95]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 2.54 [1.56 to 3.90] | 1.72 [0.36 to 4.96] | 0.13 [0.00 to 0.83]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 2.41 [1.50 to 3.66] | 1.06 [0.22 to 3.06] | 0.12 [0.00 to 0.77]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 2.33 [1.45 to 3.52] | 1.24 [0.40 to 2.87] | 0.11 [0.00 to 0.71]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 2.32 [1.50 to 3.42] | 1.24 [0.46 to 2.69] | 0.10 [0.00 to 0.66]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 2.24 [1.46 to 3.28] | 1.12 [0.41 to 2.42] | 0.09 [0.00 to 0.61]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 2.24 [1.48 to 3.25] | 1.36 [0.59 to 2.66] | 0.09 [0.00 to 0.59]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 2.24 [1.50 to 3.20] | 1.28 [0.55 to 2.50] | 0.08 [0.00 to 0.57]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 2.21 [1.48 to 3.16] | 1.22 [0.53 to 2.39] | 0.08 [0.00 to 0.56]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 1.44 [0.34 to 3.89] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 0.99]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 1.19 [0.49 to 2.42] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 0.49]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 1.46 [0.86 to 2.33] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 1.44 [0.91 to 2.16] | 0.00 [0.00 to 6.16] | 0.00 [0.00 to 0.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 1.45 [0.97 to 2.09] | 0.73 [0.02 to 4.00] | 0.00 [0.00 to 0.23]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 1.39 [0.96 to 1.94] | 1.49 [0.31 to 4.28] | 0.00 [0.00 to 0.21]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 1.36 [0.94 to 1.89] | 1.41 [0.39 to 3.57] | 0.00 [0.00 to 0.21]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 1.32 [0.92 to 1.83] | 1.72 [0.64 to 3.71] | 0.00 [0.00 to 0.20]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 1.32 [0.92 to 1.83] | 2.08 [0.90 to 4.05] | 0.00 [0.00 to 0.19]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 1.31 [0.91 to 1.81] | 2.13 [0.98 to 4.01] | 0.00 [0.00 to 0.19]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 1.29 [0.90 to 1.79] | 2.00 [0.92 to 3.77] | 0.00 [0.00 to 0.19]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 1.29 [0.90 to 1.78] | 1.91 [0.88 to 3.60] | 0.00 [0.00 to 0.19]

95. Secondary Outcome: Weekly Incidence Rates of General Non-specific Symptoms Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, headache, irritability, and malaise. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.48 [0.01 to 2.66] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.90] | 0.00 [0.00 to 19.51]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 0.49 [0.01 to 2.70] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 9.52 [1.17 to 30.38] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.66] | 0.00 [0.00 to 1.47]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.98 [0.00 to 10.39] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.78]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 1.25 [0.03 to 6.77] | 1.95 [0.53 to 4.92]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 3.76 [2.09 to 6.18] | 0.00 [0.00 to 70.76] | 0.66 [0.00 to 5.33]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 3.60 [2.41 to 5.17] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 2.22]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 4.45 [3.38 to 5.75] | 10.00 [0.11 to 50.09] | 0.00 [0.00 to 2.48]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 3.10 [1.98 to 4.62] | 4.76 [0.10 to 24.55] | 0.00 [0.00 to 1.87]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 1.57 [0.76 to 2.88] | 2.13 [0.26 to 7.48] | 0.00 [0.00 to 3.30]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 2.82 [0.89 to 6.58] | 0.91 [0.02 to 4.96] | 0.00 [0.00 to 4.45]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 0.45 [0.00 to 3.10] | 1.68 [0.20 to 5.94] | 0.00 [0.00 to 4.20]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 1.92 [0.71 to 4.13] | 7.59 [2.84 to 15.80] | 0.00 [0.00 to 4.56]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 1.79 [0.26 to 5.92] | 1.82 [0.00 to 93.05] | 1.20 [0.03 to 6.53]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 1.35 [0.28 to 3.89] | 3.92 [0.03 to 24.66] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 0.68 [0.02 to 3.78] | 0.00 [0.00 to 9.03] | 0.00 [0.00 to 5.69]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.98]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 4.15 [3.26 to 5.20] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.16]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 3.04 [2.26 to 4.01] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.97]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 2.73 [1.86 to 3.85] | 0.00 [0.00 to 40.96] | 0.59 [0.07 to 2.13]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 2.53 [1.58 to 3.83] | 4.76 [0.58 to 16.16] | 0.00 [0.00 to 1.01]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 2.26 [1.44 to 3.37] | 2.53 [0.31 to 8.85] | 0.00 [0.00 to 2.35]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 0.91 [0.11 to 3.23] | 1.54 [0.04 to 8.28] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 3.28 [1.50 to 6.18] | 2.44 [0.00 to 92.92] | 0.00 [0.00 to 5.52]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 1.86 [0.54 to 4.58] | 1.56 [0.00 to 64.84] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 1.35 [0.11 to 5.51] | 8.11 [0.32 to 34.78] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 0.88 [0.01 to 6.20] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 10.89]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 11.57]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 30.85]

96. Secondary Outcome: Cumulative Incidence Rates of General Non-specific Symptoms Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, headache, irritability, and malaise. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.37 [0.01 to 2.05] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.25 [0.01 to 1.41] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.17 [0.00 to 0.95] | 0.00 [0.00 to 4.56]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.14 [0.00 to 0.76] | 0.00 [0.00 to 4.30]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.21 [0.03 to 0.77] | 0.00 [0.00 to 1.58]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.19 [0.02 to 0.69] | 0.00 [0.00 to 1.57]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.16 [0.02 to 0.60] | 0.00 [0.00 to 1.51]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.15 [0.02 to 0.57] | 0.00 [0.00 to 1.30]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.15 [0.02 to 0.55] | 0.00 [0.00 to 1.28]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 4.76 [0.58 to 16.16] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 2.78 [0.31 to 10.01] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 2.00 [0.24 to 7.04] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 1.60 [0.19 to 5.66] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.89 [0.06 to 3.76] | 0.00 [0.00 to 1.07]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.92 [0.02 to 4.97] | 0.00 [0.00 to 1.06]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.50 [0.01 to 2.97] | 0.00 [0.00 to 1.03]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.49 [0.01 to 2.90] | 0.00 [0.00 to 0.87]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.47 [0.01 to 2.83] | 0.00 [0.00 to 0.87]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 70.76]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 9.74]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 7.11]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.60 [0.02 to 3.31] | 1.57 [0.43 to 3.97]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.56 [0.01 to 3.09] | 1.56 [0.43 to 3.94]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.55 [0.01 to 3.01] | 1.53 [0.42 to 3.86]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.54 [0.01 to 2.99] | 1.53 [0.42 to 3.86]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 3.76 [2.09 to 6.18] | 0.00 [0.00 to 70.76] | 0.62 [0.00 to 5.00]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 3.67 [2.38 to 5.40] | 0.00 [0.00 to 40.96] | 0.31 [0.00 to 2.44]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 4.04 [3.08 to 5.19] | 5.88 [0.15 to 28.69] | 0.21 [0.00 to 1.62]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 3.86 [3.01 to 4.85] | 5.00 [1.38 to 12.31] | 0.15 [0.00 to 1.15]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 3.52 [2.67 to 4.55] | 3.45 [1.28 to 7.35] | 0.13 [0.00 to 0.97]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 3.47 [2.65 to 4.46] | 2.46 [1.00 to 5.01] | 0.12 [0.00 to 0.89]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 3.34 [2.51 to 4.35] | 2.23 [1.03 to 4.20] | 0.11 [0.00 to 0.80]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 3.25 [2.43 to 4.25] | 3.11 [1.75 to 5.08] | 0.10 [0.00 to 0.73]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 3.19 [2.42 to 4.12] | 2.98 [1.71 to 4.79] | 0.18 [0.00 to 1.28]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 3.12 [2.34 to 4.07] | 3.06 [1.82 to 4.80] | 0.17 [0.00 to 1.24]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 3.06 [2.29 to 3.99] | 2.87 [1.71 to 4.50] | 0.17 [0.00 to 1.17]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 3.01 [2.25 to 3.94] | 2.74 [1.63 to 4.30] | 0.16 [0.00 to 1.14]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 4.15 [3.26 to 5.19] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 0.99]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 3.57 [2.89 to 4.37] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 0.49]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 3.22 [2.42 to 4.19] | 0.00 [0.00 to 20.59] | 0.18 [0.02 to 0.67]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 3.10 [2.31 to 4.05] | 3.45 [0.42 to 11.91] | 0.14 [0.02 to 0.50]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 3.00 [2.27 to 3.88] | 2.92 [0.80 to 7.31] | 0.12 [0.02 to 0.45]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 2.87 [2.13 to 3.78] | 2.48 [0.81 to 5.68] | 0.12 [0.01 to 0.42]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 2.89 [2.13 to 3.81] | 2.46 [1.00 to 5.01] | 0.11 [0.01 to 0.40]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 2.84 [2.10 to 3.75] | 2.30 [0.97 to 4.55] | 0.11 [0.01 to 0.39]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 2.81 [2.07 to 3.71] | 2.86 [1.43 to 5.05] | 0.10 [0.01 to 0.38]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 2.79 [2.04 to 3.71] | 2.61 [1.31 to 4.62] | 0.10 [0.01 to 0.37]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 2.76 [2.01 to 3.68] | 2.45 [1.23 to 4.34] | 0.10 [0.01 to 0.36]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 2.74 [2.00 to 3.67] | 2.34 [1.17 to 4.14] | 0.10 [0.01 to 0.36]

97. Secondary Outcome: Weekly Incidence Rates of Respiratory/Miscellaneous Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported are derived from 2 data sources: ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12, 13 to 17, 18 to 65, and >65 years. Respiratory/miscellaneous adverse events include any respiratory/miscellaneous adverse events, conjunctivitis, coryza, cough, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhea, and wheezing. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator = the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator = the number of subjects from the denominator who reported any AEIs in EHR (routine data collection + card-based ADR reporting system) within 7 days following vaccination with seasonal influenza vaccine
  Vaccination happened between weeks 35 and 48, of 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 1.59 [0.04 to 8.53] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 3.38 [1.37 to 6.84] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 3.25 [0.68 to 9.19] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 1.04 [0.07 to 4.40] | 5.88 [0.00 to 69.40]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.70 [0.00 to 5.22] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 2.45 [0.08 to 12.11] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 50.00 [1.26 to 98.74] | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 1.39 [0.04 to 7.50] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 33.33 [0.00 to 100] | 14.29 [3.05 to 36.34] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 50.00 [1.26 to 98.74] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 16.67 [0.02 to 81.43] | 2.02 [0.16 to 8.11] | 0.40 [0.01 to 2.22]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 20.00 [0.02 to 88.39] | 0.36 [0.01 to 2.02] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 1.61 [0.00 to 29.53]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 7.14 [0.02 to 44.90] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 11.11 [0.19 to 51.19] | 50.00 [1.26 to 98.74]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 5.88 [0.02 to 38.78] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 1.25 [0.03 to 6.77] | 1.95 [0.53 to 4.92]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 6.54 [4.34 to 9.38] | 0.00 [0.00 to 70.76] | 1.32 [0.12 to 5.14]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 4.53 [2.66 to 7.17] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 2.22]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 5.72 [4.51 to 7.15] | 0.00 [0.00 to 30.85] | 0.68 [0.00 to 4.80]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 3.78 [2.49 to 5.47] | 1.59 [0.04 to 8.63] | 1.03 [0.12 to 3.66]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 4.25 [2.70 to 6.33] | 4.26 [1.17 to 10.54] | 0.91 [0.02 to 5.16]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 2.25 [0.95 to 4.48] | 0.00 [0.00 to 3.30] | 3.70 [0.50 to 12.30]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 1.81 [0.29 to 5.76] | 6.72 [2.81 to 13.18] | 0.00 [0.00 to 4.20]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 2.56 [0.98 to 5.37] | 6.33 [2.09 to 14.16] | 1.27 [0.03 to 7.12]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 2.68 [0.66 to 7.09] | 1.82 [0.00 to 93.05] | 4.82 [1.32 to 11.92]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 2.24 [0.43 to 6.60] | 5.88 [0.04 to 35.34] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 4.11 [0.70 to 12.51] | 0.00 [0.00 to 9.03] | 1.59 [0.01 to 11.07]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 6.90 [0.00 to 53.09] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.96 [0.00 to 18.80]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 6.46 [4.99 to 8.19] | 0.00 [0.00 to 84.19] | 0.32 [0.01 to 1.76]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 5.07 [3.95 to 6.39] | 16.67 [0.00 to 91.51] | 0.80 [0.05 to 3.59]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 4.60 [3.57 to 5.83] | 0.00 [0.00 to 40.96] | 1.48 [0.27 to 4.53]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 6.14 [3.57 to 9.75] | 4.76 [0.58 to 16.16] | 0.82 [0.13 to 2.66]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 4.91 [3.32 to 6.96] | 5.06 [1.40 to 12.46] | 0.00 [0.00 to 2.35]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 2.74 [1.09 to 5.62] | 1.54 [0.04 to 8.28] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 3.65 [1.37 to 7.71] | 2.44 [0.00 to 92.92] | 0.00 [0.00 to 5.52]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 3.26 [0.66 to 9.32] | 7.81 [0.28 to 34.30] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 1.80 [0.29 to 5.74] | 8.11 [0.00 to 99.99] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 2.63 [0.50 to 7.81] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 10.89]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 0.94 [0.01 to 5.69] | 3.70 [0.00 to 99.88] | 3.33 [0.08 to 17.37]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 30.85]

98. Secondary Outcome: Cumulative Incidence Rates of Respiratory/Miscellaneous Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12, 13 to 17, 18 to 65, and >65 years. Respiratory/miscellaneous adverse events include any respiratory/miscellaneous adverse events, conjunctivitis, coryza, cough, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhea, and wheezing. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (routine data collection + ADR) within 7 days following vaccination with seasonal influenza vaccine
  Vaccination of the subjects happened between weeks 35 and 48, 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 1.59 [0.04 to 8.53] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 2.96 [1.29 to 5.75] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 3.05 [1.58 to 5.28] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 2.39 [1.23 to 4.17] | 1.27 [0.00 to 13.35]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 2.06 [0.98 to 3.79] | 1.19 [0.00 to 12.33]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 2.15 [0.91 to 4.23] | 0.43 [0.00 to 4.99]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 1.89 [0.76 to 3.85] | 0.43 [0.00 to 4.96]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 10.00 [0.14 to 48.28] | 1.58 [0.58 to 3.43] | 0.41 [0.00 to 4.74]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 10.00 [0.14 to 48.28] | 1.57 [0.62 to 3.25] | 0.35 [0.00 to 4.00]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 10.00 [0.14 to 48.28] | 1.54 [0.61 to 3.18] | 0.35 [0.00 to 3.96]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 3.70 [0.00 to 39.49] | 7.14 [0.82 to 24.02] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 6.90 [0.06 to 39.08] | 4.17 [0.33 to 16.27] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 5.88 [0.15 to 28.66] | 3.00 [0.28 to 11.33] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 5.71 [0.17 to 27.21] | 2.40 [0.19 to 9.55] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 7.32 [0.36 to 30.38] | 2.23 [0.34 to 7.26] | 0.29 [0.01 to 1.61]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 7.14 [0.32 to 30.34] | 1.53 [0.12 to 6.28] | 0.29 [0.01 to 1.60]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 8.51 [1.98 to 21.99] | 1.00 [0.12 to 3.53] | 0.28 [0.01 to 1.55]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 8.51 [1.98 to 21.99] | 0.98 [0.12 to 3.44] | 0.48 [0.06 to 1.71]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 8.33 [2.04 to 21.11] | 0.95 [0.11 to 3.40] | 0.48 [0.06 to 1.71]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 2.63 [0.01 to 18.97] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 2.22 [0.02 to 14.79] | 7.14 [0.04 to 41.49] | 33.33 [0.00 to 99.94]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 1.82 [0.01 to 12.25] | 6.45 [0.34 to 26.78] | 2.86 [0.07 to 14.92]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 1.69 [0.02 to 10.77] | 4.17 [0.48 to 14.52] | 2.86 [0.07 to 14.92]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 1.64 [0.02 to 10.46] | 3.28 [0.33 to 12.04] | 2.78 [0.07 to 14.53]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 1.61 [0.02 to 10.31] | 2.33 [0.22 to 8.82] | 2.00 [0.05 to 10.65]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 1.43 [0.02 to 9.07] | 1.81 [0.37 to 5.19] | 1.96 [0.64 to 4.52]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 1.32 [0.01 to 8.53] | 1.69 [0.35 to 4.85] | 1.95 [0.63 to 4.48]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 1.22 [0.01 to 8.11] | 1.64 [0.34 to 4.72] | 1.91 [0.62 to 4.40]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 1.16 [0.01 to 7.70] | 1.63 [0.34 to 4.69] | 1.91 [0.62 to 4.40]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 6.54 [6.54 to 6.54] | 0.00 [0.00 to 70.76] | 1.23 [0.11 to 4.82]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 5.45 [3.66 to 7.76] | 0.00 [0.00 to 40.96] | 0.61 [0.07 to 2.20]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 5.58 [4.62 to 6.66] | 0.00 [0.00 to 19.51] | 0.63 [0.13 to 1.84]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 5.22 [4.42 to 6.12] | 1.25 [0.03 to 6.77] | 0.75 [0.22 to 1.83]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 5.08 [4.40 to 5.83] | 2.87 [0.94 to 6.58] | 0.77 [0.26 to 1.76]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 4.87 [4.12 to 5.71] | 1.76 [0.57 to 4.06] | 1.05 [0.48 to 1.99]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 4.73 [4.00 to 5.55] | 3.23 [1.43 to 6.19] | 0.95 [0.44 to 1.80]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 4.60 [3.87 to 5.43] | 3.73 [1.60 to 7.30] | 0.98 [0.40 to 1.97]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 4.52 [3.84 to 5.29] | 3.54 [1.54 to 6.85] | 1.26 [0.39 to 3.02]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 4.43 [3.81 to 5.13] | 3.74 [2.33 to 5.67] | 1.22 [0.38 to 2.90]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 4.43 [3.79 to 5.13] | 3.51 [2.21 to 5.26] | 1.24 [0.42 to 2.80]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 4.36 [3.73 to 5.06] | 3.66 [2.31 to 5.48] | 1.21 [0.42 to 2.72]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.92 [0.00 to 17.19]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 6.45 [4.99 to 8.19] | 0.00 [0.00 to 70.76] | 0.54 [0.07 to 1.94]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 5.74 [4.95 to 6.61] | 11.11 [0.03 to 62.14] | 0.67 [0.10 to 2.22]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 5.25 [4.38 to 6.23] | 6.25 [0.16 to 30.23] | 0.92 [0.15 to 2.98]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 5.40 [4.33 to 6.66] | 5.17 [1.08 to 14.38] | 0.90 [0.16 to 2.77]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 5.35 [4.25 to 6.63] | 5.11 [2.08 to 10.24] | 0.81 [0.14 to 2.52]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 5.19 [4.07 to 6.51] | 3.96 [1.73 to 7.65] | 0.75 [0.13 to 2.36]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 5.15 [4.02 to 6.47] | 3.52 [1.70 to 6.38] | 0.73 [0.13 to 2.28]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 5.06 [3.96 to 6.37] | 4.31 [2.43 to 7.01] | 0.70 [0.12 to 2.19]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 4.99 [3.89 to 6.29] | 4.68 [2.79 to 7.29] | 0.68 [0.12 to 2.12]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 4.97 [3.85 to 6.28] | 4.27 [2.55 to 6.66] | 0.67 [0.12 to 2.09]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 4.92 [3.81 to 6.24] | 4.23 [2.57 to 6.53] | 0.71 [0.16 to 1.97]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 4.90 [3.79 to 6.22] | 4.03 [2.45 to 6.23] | 0.70 [0.16 to 1.96]

99. Secondary Outcome: Weekly Incidence Rates of Gastrointestinal Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhea, nausea, and vomiting. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 month to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 month to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 month to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 month to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 month to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 month to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 month to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 month to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 month to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.97 [0.12 to 3.45] | 0.00 [0.00 to 23.16]
  6 month to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 month to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 7.71]
  6 month to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 month to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.90] | 0.00 [0.00 to 19.51]
  6 month to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 month to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 20.00 [0.00 to 96.43]
  6 month to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 month to 5 years, Week 44 |  | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.48]
  6 month to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 month to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 month to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 month to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.49 [0.00 to 3.54] | 0.00 [0.00 to 30.85]
  6 month to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 month to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 9.03]
  6 month to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 month to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.66] | 0.00 [0.00 to 1.47]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.98 [0.00 to 10.39] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.78]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 1.25 [0.03 to 6.77] | 1.46 [0.30 to 4.22]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 1.95 [0.56 to 4.80] | 0.00 [0.00 to 70.76] | 0.66 [0.00 to 5.33]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 1.98 [0.89 to 3.76] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 2.22]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 1.98 [0.91 to 3.72] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 2.48]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 1.62 [0.46 to 4.04] | 3.17 [0.07 to 16.81] | 0.00 [0.00 to 1.87]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 1.10 [0.44 to 2.26] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 3.30]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 1.41 [0.30 to 4.02] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 4.45]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 0.45 [0.01 to 2.91] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 4.20]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 0.64 [0.03 to 3.11] | 1.27 [0.03 to 6.85] | 0.00 [0.00 to 4.56]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 1.34 [0.11 to 5.42] | 1.82 [0.00 to 93.05] | 0.00 [0.00 to 4.35]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 9.03] | 0.00 [0.00 to 5.69]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.98]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 2.19 [1.07 to 3.94] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.16]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 1.76 [1.14 to 2.60] | 16.67 [0.00 to 91.51] | 0.00 [0.00 to 0.97]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 1.27 [0.88 to 1.77] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.09]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 1.38 [0.73 to 2.37] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.01]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 1.38 [0.56 to 2.81] | 2.53 [0.31 to 8.85] | 0.00 [0.00 to 2.35]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 0.91 [0.24 to 2.35] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 1.09 [0.21 to 3.24] | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 5.52]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 0.70 [0.11 to 2.27] | 1.56 [0.00 to 64.84] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 2.70 [0.54 to 7.83] | 2.70 [0.00 to 93.12] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 4.39 [0.58 to 14.55] | 0.00 [0.00 to 9.49] | 3.13 [0.08 to 16.22]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 11.57]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 30.85]

100. Secondary Outcome: Cumulative Incidence Rates of Gastrointestinal Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhoea, nausea and vomiting. The cumulative incidence rates of AEIs expressed as a cumulative percentage of subjects, were estimated as follows:
  The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system); The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine.
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.74 [0.09 to 2.65] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.51 [0.04 to 2.11] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.34 [0.02 to 1.63] | 0.00 [0.00 to 4.56]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.27 [0.01 to 1.45] | 1.19 [0.00 to 11.17]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.21 [0.00 to 1.24] | 0.43 [0.01 to 2.39]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.19 [0.00 to 1.12] | 0.43 [0.01 to 2.37]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.24 [0.03 to 0.87] | 0.41 [0.01 to 2.27]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.22 [0.03 to 0.83] | 0.35 [0.01 to 1.96]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.22 [0.02 to 0.82] | 0.35 [0.01 to 1.93]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 1.07]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.31 [0.00 to 2.50] | 0.00 [0.00 to 1.06]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.17 [0.00 to 1.44] | 0.00 [0.00 to 1.03]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.16 [0.00 to 1.40] | 0.00 [0.00 to 0.87]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.16 [0.00 to 1.37] | 0.00 [0.00 to 0.87]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 70.76]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 9.74]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 7.11]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.60 [0.02 to 3.31] | 1.18 [0.24 to 3.40]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.56 [0.01 to 3.09] | 1.17 [0.24 to 3.37]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.55 [0.01 to 3.01] | 1.15 [0.24 to 3.31]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.54 [0.01 to 2.99] | 1.15 [0.24 to 3.31]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 1.95 [0.56 to 4.80] | 0.00 [0.00 to 70.76] | 0.62 [0.00 to 5.00]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 1.96 [0.76 to 4.10] | 0.00 [0.00 to 40.96] | 0.31 [0.00 to 2.44]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 1.97 [1.01 to 3.45] | 0.00 [0.00 to 19.51] | 0.21 [0.00 to 1.62]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 1.90 [1.14 to 2.97] | 2.50 [0.30 to 8.74] | 0.15 [0.00 to 1.15]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 1.78 [1.09 to 2.76] | 1.15 [0.14 to 4.09] | 0.13 [0.00 to 0.97]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 1.76 [1.09 to 2.68] | 0.70 [0.09 to 2.52] | 0.12 [0.00 to 0.89]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 1.70 [1.04 to 2.61] | 0.50 [0.06 to 1.78] | 0.11 [0.00 to 0.80]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 1.64 [0.99 to 2.53] | 0.62 [0.13 to 1.81] | 0.10 [0.00 to 0.73]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 1.62 [1.00 to 2.48] | 0.74 [0.20 to 1.90] | 0.09 [0.00 to 0.64]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 1.56 [0.96 to 2.40] | 0.68 [0.19 to 1.73] | 0.09 [0.00 to 0.62]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 1.52 [0.93 to 2.34] | 0.64 [0.17 to 1.63] | 0.08 [0.00 to 0.59]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 1.50 [0.92 to 2.30] | 0.61 [0.17 to 1.55] | 0.08 [0.00 to 0.57]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 2.19 [1.07 to 3.94] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 0.99]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 1.97 [1.53 to 2.49] | 11.11 [0.03 to 62.14] | 0.00 [0.00 to 0.49]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 1.67 [1.29 to 2.12] | 6.25 [0.16 to 30.23] | 0.00 [0.00 to 0.34]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 1.62 [1.28 to 2.03] | 1.72 [0.04 to 9.24] | 0.00 [0.00 to 0.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 1.59 [1.24 to 2.01] | 2.19 [0.45 to 6.27] | 0.00 [0.00 to 0.23]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 1.55 [1.22 to 1.94] | 1.49 [0.31 to 4.28] | 0.00 [0.00 to 0.21]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 1.54 [1.21 to 1.93] | 1.06 [0.22 to 3.06] | 0.00 [0.00 to 0.21]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 1.50 [1.20 to 1.86] | 1.15 [0.31 to 2.92] | 0.00 [0.00 to 0.20]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 1.53 [1.23 to 1.88] | 1.30 [0.42 to 3.00] | 0.00 [0.00 to 0.19]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 1.56 [1.24 to 1.93] | 1.18 [0.39 to 2.74] | 0.05 [0.00 to 0.38]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 1.54 [1.23 to 1.91] | 1.11 [0.36 to 2.58] | 0.05 [0.00 to 0.37]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 1.54 [1.22 to 1.90] | 1.06 [0.35 to 2.46] | 0.05 [0.00 to 0.37]

101. Secondary Outcome: Weekly Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 data sources: ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial edema, and hypersensitivity reactions. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between weeks 35 and 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.52 [0.01 to 3.43] | 0.00 [0.00 to 19.51]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.66] | 0.00 [0.00 to 1.47]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.78]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 0.70 [0.04 to 3.03] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 2.40]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 0.81 [0.06 to 3.39] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 2.22]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 0.78 [0.08 to 2.91] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 2.48]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 0.27 [0.03 to 0.97] | 3.17 [0.07 to 16.81] | 0.00 [0.00 to 1.87]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 0.31 [0.01 to 1.85] | 1.06 [0.03 to 5.79] | 0.00 [0.00 to 3.30]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.03] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 4.45]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 0.00 [0.00 to 1.66] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 4.20]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 0.00 [0.00 to 1.17] | 3.80 [0.62 to 11.76] | 0.00 [0.00 to 4.56]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 0.45 [0.00 to 3.33] | 0.00 [0.00 to 6.49] | 1.20 [0.03 to 6.53]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 0.45 [0.00 to 3.36] | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 9.03] | 0.00 [0.00 to 5.69]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.98]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 0.69 [0.01 to 4.78] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.16]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 0.48 [0.08 to 1.56] | 0.00 [0.00 to 45.93] | 0.27 [0.01 to 1.51]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 0.22 [0.02 to 0.96] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.09]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 0.54 [0.02 to 2.62] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.01]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 0.20 [0.01 to 0.93] | 2.53 [0.31 to 8.85] | 0.00 [0.00 to 2.35]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 0.00 [0.00 to 0.67] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 0.36 [0.00 to 2.55] | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 5.52]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 0.47 [0.02 to 2.39] | 0.00 [0.00 to 5.60] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 10.89]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 11.57]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 30.85]

102. Secondary Outcome: Cumulative Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 data sources: ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Sensitivity/anaphylaxis adverse events include any sensitivity/anaphylaxis adverse events, anaphylactic reactions, facial edema, and hypersensitivity reactions. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between weeks 35 and 48 of 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.17 [0.00 to 1.26] | 0.00 [0.00 to 4.56]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.14 [0.00 to 1.01] | 0.00 [0.00 to 4.30]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.11 [0.00 to 0.77] | 0.00 [0.00 to 1.58]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.09 [0.00 to 0.68] | 0.00 [0.00 to 1.57]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.08 [0.00 to 0.58] | 0.00 [0.00 to 1.51]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.07 [0.00 to 0.56] | 0.00 [0.00 to 1.30]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.07 [0.00 to 0.54] | 0.00 [0.00 to 1.28]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 1.07]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 1.06]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.61] | 0.00 [0.00 to 1.03]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.60] | 0.00 [0.00 to 0.87]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 0.87]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 70.76]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 9.74]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 7.11]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.44]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.43]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.40]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.40]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 0.70 [0.04 to 3.03] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 2.25]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 0.76 [0.06 to 3.10] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.13]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 0.77 [0.08 to 2.90] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 0.78]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 0.67 [0.08 to 2.42] | 2.50 [0.30 to 8.74] | 0.00 [0.00 to 0.55]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 0.62 [0.08 to 2.13] | 1.72 [0.36 to 4.96] | 0.00 [0.00 to 0.47]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 0.57 [0.07 to 2.02] | 1.06 [0.22 to 3.06] | 0.00 [0.00 to 0.43]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 0.55 [0.07 to 1.95] | 0.74 [0.15 to 2.16] | 0.00 [0.00 to 0.39]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 0.51 [0.06 to 1.87] | 1.24 [0.46 to 2.69] | 0.00 [0.00 to 0.36]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 0.51 [0.07 to 1.79] | 1.12 [0.41 to 2.42] | 0.09 [0.00 to 0.64]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 0.51 [0.06 to 1.83] | 1.02 [0.38 to 2.21] | 0.09 [0.00 to 0.62]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 0.50 [0.06 to 1.78] | 0.96 [0.35 to 2.07] | 0.08 [0.00 to 0.59]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 0.49 [0.06 to 1.76] | 0.91 [0.34 to 1.98] | 0.08 [0.00 to 0.57]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 0.69 [0.01 to 4.77] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 0.99]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 0.58 [0.03 to 2.80] | 0.00 [0.00 to 33.63] | 0.13 [0.00 to 0.74]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 0.43 [0.02 to 2.00] | 2.00 [0.00 to 20.59] | 0.09 [0.00 to 0.52]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 0.45 [0.02 to 2.08] | 0.00 [0.00 to 6.16] | 0.07 [0.00 to 0.41]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 0.42 [0.03 to 1.85] | 1.46 [0.18 to 5.17] | 0.06 [0.00 to 0.37]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 0.39 [0.02 to 1.77] | 0.99 [0.12 to 3.53] | 0.06 [0.00 to 0.34]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 0.39 [0.03 to 1.71] | 0.70 [0.09 to 2.52] | 0.06 [0.00 to 0.33]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 0.40 [0.03 to 1.62] | 0.57 [0.07 to 2.06] | 0.05 [0.00 to 0.32]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 0.39 [0.03 to 1.59] | 0.52 [0.06 to 1.86] | 0.05 [0.00 to 0.31]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 0.38 [0.03 to 1.57] | 0.47 [0.06 to 1.70] | 0.05 [0.00 to 0.31]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 0.38 [0.03 to 1.57] | 0.45 [0.05 to 1.60] | 0.05 [0.00 to 0.30]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 0.38 [0.03 to 1.57] | 0.42 [0.05 to 1.53] | 0.05 [0.00 to 0.30]

103. Secondary Outcome: Weekly Incidence Rates of Rash Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: as for outcome 89
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.48 [0.01 to 2.66] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.81 [0.01 to 5.15] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.90] | 0.00 [0.00 to 19.51]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 1.40 [0.17 to 4.96] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 0.49 [0.01 to 2.70] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.66] | 0.00 [0.00 to 1.47]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.78]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 0.97 [0.30 to 2.34] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 2.40]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 0.93 [0.16 to 2.88] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 2.22]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 0.57 [0.24 to 1.11] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 2.48]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 0.67 [0.22 to 1.57] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 1.87]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 3.30]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.03] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 4.45]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 0.90 [0.08 to 3.62] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 4.20]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 0.64 [0.06 to 2.51] | 0.00 [0.00 to 4.56] | 0.00 [0.00 to 4.56]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 4.35]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 0.90 [0.07 to 3.65] | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 2.56 [0.06 to 13.48] | 0.00 [0.00 to 5.69]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.98]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 0.69 [0.36 to 1.21] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.16]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 0.37 [0.15 to 0.77] | 0.00 [0.00 to 45.93] | 0.53 [0.05 to 2.02]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 0.26 [0.10 to 0.55] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.09]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 0.54 [0.22 to 1.10] | 0.00 [0.00 to 8.41] | 0.27 [0.01 to 1.52]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 0.20 [0.02 to 0.71] | 1.27 [0.03 to 6.85] | 0.00 [0.00 to 2.35]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 0.18 [0.00 to 1.30] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 0.36 [0.00 to 2.68] | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 5.52]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 0.47 [0.06 to 1.67] | 0.00 [0.00 to 5.60] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 0.45 [0.00 to 2.99] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 2.70 [0.00 to 82.29] | 0.00 [0.00 to 10.89]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 11.57]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 4.55 [0.00 to 99.99] | 0.00 [0.00 to 30.85]

104. Secondary Outcome: Cumulative Incidence Rates of Rash Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: as for outcome 90
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.37 [0.01 to 2.05] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.51 [0.06 to 1.83] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.34 [0.04 to 1.23] | 0.00 [0.00 to 4.56]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.55 [0.15 to 1.40] | 0.00 [0.00 to 4.30]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.54 [0.17 to 1.25] | 0.00 [0.00 to 1.58]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.47 [0.15 to 1.10] | 0.00 [0.00 to 1.57]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.40 [0.13 to 0.92] | 0.00 [0.00 to 1.51]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.37 [0.12 to 0.87] | 0.00 [0.00 to 1.30]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.37 [0.12 to 0.87] | 0.00 [0.00 to 1.28]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 1.07]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 1.06]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.61] | 0.00 [0.00 to 1.03]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.60] | 0.00 [0.00 to 0.87]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 0.87]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 70.76]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 9.74]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 7.11]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.44]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.43]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.40]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.40]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 0.97 [0.30 to 2.34] | 0.00 [0.00 to 70.76] | 0.00 [0.0 to 2.25]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 0.95 [0.34 to 2.08] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.13]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 0.77 [0.38 to 1.38] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 0.78]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 0.75 [0.39 to 1.29] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 0.55]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 0.64 [0.35 to 1.07] | 0.00 [0.00 to 2.10] | 0.00 [0.00 to 0.47]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 0.59 [0.33 to 0.98] | 0.00 [0.00 to 1.29] | 0.00 [0.00 to 0.43]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 0.61 [0.36 to 0.96] | 0.00 [0.00 to 0.91] | 0.00 [0.00 to 0.39]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 0.61 [0.37 to 0.95] | 0.00 [0.00 to 0.76] | 0.00 [0.00 to 0.36]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 0.58 [0.35 to 0.91] | 0.00 [0.00 to 0.68] | 0.00 [0.00 to 0.33]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 0.60 [0.36 to 0.92] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 0.32]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 0.58 [0.35 to 0.90] | 0.16 [0.00 to 0.89] | 0.00 [0.00 to 0.30]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 0.57 [0.35 to 0.89] | 0.15 [0.00 to 0.85] | 0.00 [0.00 to 0.30]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 0.69 [0.36 to 1.20] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 0.99]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 0.53 [0.32 to 0.82] | 0.00 [0.00 to 33.63] | 0.27 [0.03 to 1.03]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 0.41 [0.27 to 0.61] | 0.00 [0.00 to 20.59] | 0.18 [0.02 to 0.73]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 0.44 [0.30 to 0.61] | 0.00 [0.00 to 6.16] | 0.21 [0.04 to 0.60]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 0.41 [0.28 to 0.57] | 0.73 [0.02 to 4.00] | 0.19 [0.04 to 0.55]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 0.39 [0.28 to 0.54] | 0.50 [0.01 to 2.73] | 0.17 [0.04 to 0.51]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 0.39 [0.28 to 0.54] | 0.35 [0.01 to 1.95] | 0.17 [0.03 to 0.49]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 0.40 [0.28 to 0.54] | 0.29 [0.01 to 1.59] | 0.16 [0.03 to 0.47]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 0.40 [0.28 to 0.54] | 0.26 [0.01 to 1.44] | 0.16 [0.03 to 0.46]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 0.39 [0.28 to 0.53] | 0.47 [0.06 to 1.70] | 0.15 [0.03 to 0.45]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 0.39 [0.28 to 0.53] | 0.45 [0.05 to 1.60] | 0.15 [0.03 to 0.44]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 0.39 [0.28 to 0.53] | 0.64 [0.05 to 2.56] | 0.15 [0.03 to 0.44]

105. Secondary Outcome: Weekly Incidence Rates of Musculoskeletal Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Musculoskeletal adverse events include any musculoskeletal adverse events, arthropathy, and muscle aches/myalgia. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.90] | 0.00 [0.00 to 19.51]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.66] | 0.00 [0.00 to 1.47]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.78]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 10.00 [0.00 to 71.81] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.49 [0.01 to 2.69]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 5.29 [3.30 to 7.98] | 0.00 [0.00 to 70.76] | 0.66 [0.02 to 3.61]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 3.72 [2.55 to 5.22] | 0.00 [0.00 to 60.24] | 0.61 [0.01 to 3.60]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 3.96 [3.00 to 5.11] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 2.48]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 3.37 [2.11 to 5.10] | 4.76 [0.10 to 24.55] | 0.51 [0.01 to 2.82]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 2.36 [0.99 to 4.70] | 0.00 [0.00 to 3.85] | 0.00 [0.00 to 3.30]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 2.25 [0.62 to 5.66] | 0.91 [0.02 to 4.96] | 0.00 [0.00 to 4.45]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 4.52 [1.78 to 9.28] | 0.00 [0.00 to 3.05] | 1.16 [0.03 to 6.31]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 1.28 [0.25 to 3.78] | 5.06 [0.82 to 15.56] | 0.00 [0.00 to 4.56]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 2.23 [0.47 to 6.33] | 1.82 [0.00 to 93.05] | 0.00 [0.00 to 4.35]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 2.24 [0.73 to 5.15] | 1.96 [0.02 to 12.89] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 2.05 [0.43 to 5.89] | 0.00 [0.00 to 9.03] | 0.00 [0.00 to 5.69]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 3.45 [0.00 to 94.80] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.98]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 3.86 [2.98 to 4.91] | 0.00 [0.00 to 84.19] | 0.32 [0.01 to 1.76]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 3.26 [2.29 to 4.49] | 0.00 [0.00 to 45.93] | 0.27 [0.01 to 1.51]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 3.03 [2.26 to 3.97] | 0.00 [0.00 to 40.96] | 1.19 [0.32 to 3.01]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 2.23 [1.04 to 4.13] | 2.38 [0.06 to 12.57] | 0.55 [0.07 to 1.97]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 2.55 [1.49 to 4.08] | 0.00 [0.00 to 4.56] | 0.00 [0.00 to 2.35]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 1.83 [0.75 to 3.69] | 1.54 [0.04 to 8.28] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 2.19 [0.81 to 4.71] | 1.22 [0.00 to 92.27] | 1.54 [0.01 to 11.02]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 2.33 [0.54 to 6.33] | 3.13 [0.00 to 88.31] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 3.15 [0.79 to 8.23] | 2.70 [0.00 to 99.67] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 9.49] | 6.25 [0.77 to 20.81]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 1.89 [0.14 to 7.77] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 11.57]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 4.55 [0.00 to 99.99] | 0.00 [0.00 to 30.85]

106. Secondary Outcome: Cumulative Incidence Rates of Musculoskeletal Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Musculoskeletal adverse events include any musculoskeletal adverse events, arthropathy and muscle aches/myalgia. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 4.56]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 4.30]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 1.58]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 1.57]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 1.51]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.28] | 0.00 [0.00 to 1.30]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.27] | 0.00 [0.00 to 1.28]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 1.07]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 1.06]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.61] | 0.00 [0.00 to 1.03]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.60] | 0.00 [0.00 to 0.87]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.87]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 70.76]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 1.82 [0.01 to 12.25] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 1.69 [0.02 to 10.77] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 1.64 [0.02 to 10.46] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 9.74]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 1.61 [0.02 to 10.31] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 7.11]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 1.43 [0.02 to 9.07] | 0.00 [0.00 to 2.20] | 0.39 [0.01 to 2.17]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 1.32 [0.01 to 8.53] | 0.00 [0.00 to 2.05] | 0.39 [0.01 to 2.15]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 1.22 [0.01 to 8.11] | 0.00 [0.00 to 2.00] | 0.38 [0.01 to 2.11]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 1.16 [0.01 to 7.70] | 0.00 [0.00 to 1.98] | 0.38 [0.01 to 2.11]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 5.29 [3.30 to 7.98] | 0.00 [0.00 to 70.76] | 0.62 [0.02 to 3.39]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 4.43 [3.14 to 6.06] | 0.00 [0.00 to 40.96] | 0.61 [0.02 to 3.25]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 4.21 [3.48 to 5.04] | 0.00 [0.00 to 19.51] | 0.42 [0.01 to 2.46]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 4.04 [3.42 to 4.74] | 3.75 [0.78 to 10.57] | 0.45 [0.05 to 1.61]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 3.80 [3.16 to 4.53] | 1.72 [0.36 to 4.96] | 0.39 [0.04 to 1.44]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 3.68 [2.98 to 4.50] | 1.41 [0.39 to 3.57] | 0.35 [0.03 to 1.35]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 3.72 [2.96 to 4.61] | 0.99 [0.99 to 2.52] | 0.42 [0.06 to 1.46]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 3.57 [2.77 to 4.54] | 1.66 [0.72 to 3.24] | 0.39 [0.05 to 1.37]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 3.52 [2.78 to 4.40] | 1.68 [0.77 to 3.16] | 0.36 [0.04 to 1.30]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 3.47 [2.74 to 4.33] | 1.70 [0.82 to 3.11] | 0.35 [0.04 to 1.27]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 3.43 [2.70 to 4.30] | 1.59 [0.77 to 2.91] | 0.33 [0.04 to 1.21]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 3.38 [2.66 to 4.24] | 1.68 [0.84 to 2.98] | 0.32 [0.04 to 1.20]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 3.86 [2.98 to 4.91] | 0.00 [0.00 to 70.76] | 0.27 [0.01 to 1.50]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 3.55 [2.79 to 4.44] | 0.00 [0.00 to 33.63] | 0.27 [0.01 to 1.45]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 3.33 [2.59 to 4.20] | 0.00 [0.00 to 20.59] | 0.55 [0.13 to 1.51]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 3.14 [2.47 to 3.93] | 1.72 [0.04 to 9.24] | 0.55 [0.16 to 1.39]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 3.07 [2.43 to 3.82] | 0.73 [0.02 to 4.00] | 0.50 [0.14 to 1.26]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 2.99 [2.36 to 3.74] | 0.99 [0.12 to 3.53] | 0.46 [0.13 to 1.18]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 2.97 [2.33 to 3.73] | 1.06 [0.22 to 3.06] | 0.50 [0.18 to 1.10]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 2.94 [2.33 to 3.66] | 1.44 [0.47 to 3.32] | 0.48 [0.17 to 1.06]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 2.95 [2.35 to 3.65] | 1.56 [0.57 to 3.36] | 0.47 [0.17 to 1.03]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 2.91 [2.31 to 3.62] | 1.42 [0.52 to 3.07] | 0.56 [0.24 to 1.12]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 2.90 [2.30 to 3.61] | 1.34 [0.49 to 2.89] | 0.56 [0.24 to 1.10]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 2.89 [2.29 to 3.60] | 1.49 [0.60 to 3.04] | 0.55 [0.24 to 1.10]

107. Secondary Outcome: Weekly Incidence Rates of Neurological Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Neurological adverse events include any neurological adverse events, Bell's palsy, Guillain-Barre Syndrome, peripheral tremor and seizure/febrile convulsions. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between weeks 35 and 48 of 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.90] | 0.00 [0.00 to 19.51]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.66] | 0.00 [0.00 to 1.47]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.78]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 0.28 [0.03 to 1.00] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 2.40]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 0.35 [0.04 to 1.25] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 2.22]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 0.28 [0.02 to 1.17] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 2.48]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 0.00 [0.00 to 0.50] | 1.59 [0.04 to 8.63] | 0.00 [0.00 to 1.87]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 0.16 [0.00 to 0.93] | 1.06 [0.03 to 5.79] | 0.00 [0.00 to 3.30]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.03] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 4.45]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 0.00 [0.00 to 1.66] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 4.20]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 0.00 [0.00 to 1.17] | 0.00 [0.00 to 4.56] | 0.00 [0.00 to 4.56]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 4.35]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 2.56 [0.00 to 25.31] | 0.00 [0.00 to 5.69]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.98]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 0.29 [0.09 to 0.67] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.16]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 0.27 [0.07 to 0.72] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.97]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 0.19 [0.06 to 0.44] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.09]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 0.00 [0.00 to 0.28] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.01]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 0.20 [0.00 to 1.20] | 0.00 [0.00 to 4.56] | 0.65 [0.00 to 4.69]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 0.00 [0.00 to 0.67] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 5.52]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 0.23 [0.00 to 1.90] | 0.00 [0.00 to 5.60] | 0.00 [0.00 to 4.99]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 10.89]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 11.57]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 30.85]

108. Secondary Outcome: Cumulative Incidence Rates of Neurological Adverse Events Recorded in EHR, by Vaccine and Age Group
Description: AEIs reported here are derived from 2 data sources: ADR cards and AEI routinely collected from GPs. AEI data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. Neurological adverse events include any neurological adverse events, Bell's palsy, Guillain-Barre Syndrome, peripheral tremor and seizure/febrile convulsions. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between weeks 35 and 48 of 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 4.56]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 4.30]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 1.58]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 1.57]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 1.51]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.28] | 0.00 [0.00 to 1.30]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.27] | 0.00 [0.00 to 1.28]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 1.07]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 1.06]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.61] | 0.00 [0.00 to 1.03]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.60] | 0.00 [0.00 to 0.87]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 0.87]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 70.76]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 9.74]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 7.11]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.44]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.43]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.40]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.40]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 0.28 [0.03 to 1.00] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 2.25]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 0.32 [0.07 to 0.88] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.13]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 0.30 [0.11 to 0.67] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 0.78]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 0.24 [0.07 to 0.60] | 1.25 [0.03 to 6.77] | 0.00 [0.00 to 0.55]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 0.23 [0.07 to 0.55] | 1.15 [0.14 to 4.09] | 0.00 [0.00 to 0.47]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 0.21 [0.06 to 0.52] | 0.70 [0.09 to 2.52] | 0.00 [0.00 to 0.43]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 0.20 [0.06 to 0.50] | 0.50 [0.06 to 1.78] | 0.00 [0.00 to 0.39]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 0.19 [0.05 to 0.48] | 0.41 [0.05 to 1.49] | 0.00 [0.00 to 0.36]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 0.18 [0.05 to 0.46] | 0.37 [0.05 to 1.34] | 0.00 [0.00 to 0.33]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 0.18 [0.05 to 0.44] | 0.34 [0.04 to 1.22] | 0.00 [0.00 to 0.32]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 0.17 [0.05 to 0.43] | 0.48 [0.10 to 1.39] | 0.00 [0.00 to 0.30]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 0.17 [0.05 to 0.43] | 0.46 [0.09 to 1.33] | 0.00 [0.00 to 0.30]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 0.29 [0.09 to 0.67] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 0.99]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 0.28 [0.13 to 0.51] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 0.49]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 0.24 [0.13 to 0.40] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 0.34]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 0.20 [0.11 to 0.33] | 0.00 [0.00 to 6.16] | 0.00 [0.00 to 0.25]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 0.20 [0.11 to 0.33] | 0.00 [0.00 to 2.66] | 0.06 [0.00 to 0.51]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 0.19 [0.10 to 0.32] | 0.00 [0.00 to 1.81] | 0.06 [0.00 to 0.47]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 0.18 [0.10 to 0.31] | 0.00 [0.00 to 1.29] | 0.06 [0.00 to 0.46]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 0.18 [0.10 to 0.31] | 0.00 [0.00 to 1.05] | 0.05 [0.00 to 0.43]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 0.18 [0.09 to 0.31] | 0.00 [0.00 to 0.95] | 0.05 [0.00 to 0.42]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 0.18 [0.09 to 0.30] | 0.00 [0.00 to 0.87] | 0.05 [0.00 to 0.41]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 0.17 [0.09 to 0.30] | 0.00 [0.00 to 0.82] | 0.05 [0.00 to 0.40]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 0.17 [0.09 to 0.30] | 0.00 [0.00 to 0.78] | 0.05 [0.00 to 0.40]

109. Secondary Outcome: Weekly Incidence Rates of SAEs Recorded in EHR, by Vaccine and Age Group
Description: "SAEs reported here are derived from 2 sources of data - ADR cards and SAEs routinely collected from GPs. SAE data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. The weekly incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017"
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 39: number analyzed (Participants) | 2 | 63 | 1
  6 months to 5 years, Week 39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 40: number analyzed (Participants) | 3 | 207 | 14
  6 months to 5 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 1.77] | 0.00 [0.00 to 23.16]
  6 months to 5 years, Week 41: number analyzed (Participants) | 1 | 123 | 46
  6 months to 5 years, Week 41 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.95] | 0.00 [0.00 to 7.71]
  6 months to 5 years, Week 42: number analyzed (Participants) | 1 | 192 | 17
  6 months to 5 years, Week 42 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 1.90] | 0.00 [0.00 to 19.51]
  6 months to 5 years, Week 43: number analyzed (Participants) | 1 | 143 | 5
  6 months to 5 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 2.55] | 0.00 [0.00 to 52.18]
  6 months to 5 years, Week 44: number analyzed (Participants) | 0 | 204 | 147
  6 months to 5 years, Week 44 |  | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.48]
  6 months to 5 years, Week 45: number analyzed (Participants) | 0 | 129 | 2
  6 months to 5 years, Week 45 |  | 0.00 [0.00 to 2.82] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 46: number analyzed (Participants) | 2 | 203 | 10
  6 months to 5 years, Week 46 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 1.80] | 0.00 [0.00 to 30.85]
  6 months to 5 years, Week 47: number analyzed (Participants) | 0 | 72 | 39
  6 months to 5 years, Week 47 |  | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 9.03]
  6 months to 5 years, Week 48: number analyzed (Participants) | 0 | 29 | 4
  6 months to 5 years, Week 48 |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 60.24]
  6 - 12 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 38: number analyzed (Participants) | 7 | 0 | 0
  6 - 12 years, Week 38 | 0.00 [0.00 to 40.96] |  |
  6 - 12 years, Week 39: number analyzed (Participants) | 12 | 21 | 0
  6 - 12 years, Week 39 | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 40: number analyzed (Participants) | 3 | 21 | 10
  6 - 12 years, Week 40 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 41: number analyzed (Participants) | 2 | 30 | 55
  6 - 12 years, Week 41 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 11.57] | 0.00 [0.00 to 6.49]
  6 - 12 years, Week 42: number analyzed (Participants) | 5 | 28 | 23
  6 - 12 years, Week 42 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 14.82]
  6 - 12 years, Week 43: number analyzed (Participants) | 1 | 25 | 7
  6 - 12 years, Week 43 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 40.96]
  6 - 12 years, Week 44: number analyzed (Participants) | 6 | 99 | 249
  6 - 12 years, Week 44 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 3.66] | 0.00 [0.00 to 1.47]
  6 - 12 years, Week 45: number analyzed (Participants) | 1 | 102 | 1
  6 - 12 years, Week 45 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 97.50]
  6 - 12 years, Week 46: number analyzed (Participants) | 5 | 274 | 13
  6 - 12 years, Week 46 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.34] | 0.00 [0.00 to 24.71]
  6 - 12 years, Week 47: number analyzed (Participants) | 0 | 15 | 62
  6 - 12 years, Week 47 |  | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.78]
  6 - 12 years, Week 48: number analyzed (Participants) | 1 | 19 | 0
  6 - 12 years, Week 48 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 17.65] |
  13 - 17 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 38: number analyzed (Participants) | 16 | 0 | 0
  13 - 17 years, Week 38 | 0.00 [0.00 to 20.59] |  |
  13 - 17 years, Week 39: number analyzed (Participants) | 14 | 5 | 1
  13 - 17 years, Week 39 | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 40: number analyzed (Participants) | 7 | 9 | 2
  13 - 17 years, Week 40 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 41: number analyzed (Participants) | 10 | 17 | 32
  13 - 17 years, Week 41 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 10.89]
  13 - 17 years, Week 42: number analyzed (Participants) | 4 | 17 | 0
  13 - 17 years, Week 42 | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 19.51] |
  13 - 17 years, Week 43: number analyzed (Participants) | 2 | 13 | 1
  13 - 17 years, Week 43 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 44: number analyzed (Participants) | 1 | 25 | 14
  13 - 17 years, Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 13.72] | 0.00 [0.00 to 23.16]
  13 - 17 years, Week 45: number analyzed (Participants) | 8 | 80 | 205
  13 - 17 years, Week 45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 1.78]
  13 - 17 years, Week 46: number analyzed (Participants) | 6 | 12 | 2
  13 - 17 years, Week 46 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 84.19]
  13 - 17 years, Week 47: number analyzed (Participants) | 6 | 5 | 5
  13 - 17 years, Week 47 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 52.18]
  13 - 17 years, Week 48: number analyzed (Participants) | 4 | 1 | 0
  13 - 17 years, Week 48 | 25.00 [0.63 to 80.59] | 0.00 [0.00 to 97.50] |
  18 - 65 years, Week 35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 37: number analyzed (Participants) | 719 | 3 | 152
  18 - 65 years, Week 37 | 0.14 [0.00 to 0.95] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 2.40]
  18 - 65 years, Week 38: number analyzed (Participants) | 860 | 4 | 164
  18 - 65 years, Week 38 | 0.00 [0.00 to 0.43] | 0.00 [0.00 to 60.24] | 0.61 [0.01 to 3.47]
  18 - 65 years, Week 39: number analyzed (Participants) | 1415 | 10 | 147
  18 - 65 years, Week 39 | 0.00 [0.00 to 0.26] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 2.48]
  18 - 65 years, Week 40: number analyzed (Participants) | 741 | 63 | 195
  18 - 65 years, Week 40 | 0.27 [0.03 to 0.98] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 1.87]
  18 - 65 years, Week 41: number analyzed (Participants) | 635 | 94 | 110
  18 - 65 years, Week 41 | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 3.85] | 1.82 [0.22 to 6.41]
  18 - 65 years, Week 42: number analyzed (Participants) | 355 | 110 | 81
  18 - 65 years, Week 42 | 0.00 [0.00 to 1.03] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 4.45]
  18 - 65 years, Week 43: number analyzed (Participants) | 221 | 119 | 86
  18 - 65 years, Week 43 | 0.00 [0.00 to 1.66] | 0.00 [0.00 to 3.05] | 0.00 [0.00 to 4.20]
  18 - 65 years, Week 44: number analyzed (Participants) | 313 | 79 | 79
  18 - 65 years, Week 44 | 0.00 [0.00 to 1.17] | 1.27 [0.00 to 19.00] | 0.00 [0.00 to 4.56]
  18 - 65 years, Week 45: number analyzed (Participants) | 224 | 55 | 83
  18 - 65 years, Week 45 | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 4.35]
  18 - 65 years, Week 46: number analyzed (Participants) | 223 | 51 | 40
  18 - 65 years, Week 46 | 0.45 [0.01 to 2.58] | 0.00 [0.00 to 6.98] | 0.00 [0.00 to 8.81]
  18 - 65 years, Week 47: number analyzed (Participants) | 146 | 39 | 63
  18 - 65 years, Week 47 | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 9.03] | 0.00 [0.00 to 5.69]
  18 - 65 years, Week 48: number analyzed (Participants) | 88 | 29 | 28
  18 - 65 years, Week 48 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 12.34]
  >65 years, Week 35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 36: number analyzed (Participants) | 1 | 1 | 51
  >65 years, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.98]
  >65 years, Week 37: number analyzed (Participants) | 1735 | 2 | 317
  >65 years, Week 37 | 0.12 [0.01 to 0.42] | 0.00 [0.00 to 84.19] | 0.32 [0.00 to 2.60]
  >65 years, Week 38: number analyzed (Participants) | 1873 | 6 | 377
  >65 years, Week 38 | 0.27 [0.06 to 0.75] | 0.00 [0.00 to 45.93] | 0.27 [0.00 to 1.83]
  >65 years, Week 39: number analyzed (Participants) | 2674 | 7 | 337
  >65 years, Week 39 | 0.11 [0.02 to 0.35] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 1.09]
  >65 years, Week 40: number analyzed (Participants) | 1303 | 42 | 364
  >65 years, Week 40 | 0.15 [0.01 to 0.62] | 0.00 [0.00 to 8.41] | 0.27 [0.00 to 2.12]
  >65 years, Week 41: number analyzed (Participants) | 1018 | 79 | 155
  >65 years, Week 41 | 0.20 [0.01 to 0.94] | 0.00 [0.00 to 4.56] | 0.00 [0.00 to 2.35]
  >65 years, Week 42: number analyzed (Participants) | 547 | 65 | 120
  >65 years, Week 42 | 0.00 [0.00 to 0.67] | 1.54 [0.04 to 8.28] | 0.00 [0.00 to 3.03]
  >65 years, Week 43: number analyzed (Participants) | 274 | 82 | 65
  >65 years, Week 43 | 0.73 [0.01 to 4.84] | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 5.52]
  >65 years, Week 44: number analyzed (Participants) | 430 | 64 | 72
  >65 years, Week 44 | 0.47 [0.00 to 3.34] | 0.00 [0.00 to 5.60] | 2.78 [0.31 to 9.95]
  >65 years, Week 45: number analyzed (Participants) | 222 | 37 | 59
  >65 years, Week 45 | 0.45 [0.00 to 3.24] | 2.70 [0.00 to 93.12] | 0.00 [0.00 to 6.06]
  >65 years, Week 46: number analyzed (Participants) | 114 | 37 | 32
  >65 years, Week 46 | 0.88 [0.01 to 5.78] | 0.00 [0.00 to 9.49] | 3.13 [0.08 to 16.22]
  >65 years, Week 47: number analyzed (Participants) | 106 | 27 | 30
  >65 years, Week 47 | 0.00 [0.00 to 3.42] | 0.00 [0.00 to 12.77] | 3.33 [0.04 to 19.38]
  >65 years, Week 48: number analyzed (Participants) | 52 | 22 | 10
  >65 years, Week 48 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 15.44] | 0.00 [0.00 to 30.85]

110. Secondary Outcome: Cumulative Incidence Rates of SAEs Recorded in EHR, by Vaccine and Age Group
Description: SAEs reported here are derived from 2 sources of data - ADR cards and SAEs routinely collected from GPs. SAE data was presented by age strata: 6 months to 5 years, 6 to 12 years, 13 to 17 years, 18 to 65 years and >65 years. The cumulative incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  6 months to 5 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 months to 5 years, Week 35-37: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-37 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-38: number analyzed (Participants) | 0 | 0 | 1
  6 months to 5 years, Week 35-38 |  |  | 0.00 [0.00 to 97.50]
  6 months to 5 years, Week 35-39: number analyzed (Participants) | 2 | 63 | 2
  6 months to 5 years, Week 35-39 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 84.19]
  6 months to 5 years, Week 35-40: number analyzed (Participants) | 5 | 270 | 16
  6 months to 5 years, Week 35-40 | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 20.59]
  6 months to 5 years, Week 35-41: number analyzed (Participants) | 6 | 393 | 62
  6 months to 5 years, Week 35-41 | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.93] | 0.00 [0.00 to 5.78]
  6 months to 5 years, Week 35-42: number analyzed (Participants) | 7 | 585 | 79
  6 months to 5 years, Week 35-42 | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.63] | 0.00 [0.00 to 4.56]
  6 months to 5 years, Week 35-43: number analyzed (Participants) | 8 | 728 | 84
  6 months to 5 years, Week 35-43 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.51] | 0.00 [0.00 to 4.30]
  6 months to 5 years, Week 35-44: number analyzed (Participants) | 8 | 932 | 231
  6 months to 5 years, Week 35-44 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.40] | 0.00 [0.00 to 1.58]
  6 months to 5 years, Week 35-45: number analyzed (Participants) | 8 | 1061 | 233
  6 months to 5 years, Week 35-45 | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 0.35] | 0.00 [0.00 to 1.57]
  6 months to 5 years, Week 35-46: number analyzed (Participants) | 10 | 1264 | 243
  6 months to 5 years, Week 35-46 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.29] | 0.00 [0.00 to 1.51]
  6 months to 5 years, Week 35-47: number analyzed (Participants) | 10 | 1336 | 282
  6 months to 5 years, Week 35-47 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.28] | 0.00 [0.00 to 1.30]
  6 months to 5 years, Week 35-48: number analyzed (Participants) | 10 | 1365 | 286
  6 months to 5 years, Week 35-48 | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 0.27] | 0.00 [0.00 to 1.28]
  6 - 12 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  6 - 12 years, Week 35-37: number analyzed (Participants) | 5 | 0 | 0
  6 - 12 years, Week 35-37 | 0.00 [0.00 to 52.18] |  |
  6 - 12 years, Week 35-38: number analyzed (Participants) | 12 | 0 | 0
  6 - 12 years, Week 35-38 | 0.00 [0.00 to 26.46] |  |
  6 - 12 years, Week 35-39: number analyzed (Participants) | 24 | 21 | 0
  6 - 12 years, Week 35-39 | 0.00 [0.00 to 14.25] | 0.00 [0.00 to 16.11] |
  6 - 12 years, Week 35-40: number analyzed (Participants) | 27 | 42 | 10
  6 - 12 years, Week 35-40 | 0.00 [0.00 to 12.77] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 30.85]
  6 - 12 years, Week 35-41: number analyzed (Participants) | 29 | 72 | 65
  6 - 12 years, Week 35-41 | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 4.99] | 0.00 [0.00 to 5.52]
  6 - 12 years, Week 35-42: number analyzed (Participants) | 34 | 100 | 88
  6 - 12 years, Week 35-42 | 0.00 [0.00 to 10.28] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 4.11]
  6 - 12 years, Week 35-43: number analyzed (Participants) | 35 | 125 | 95
  6 - 12 years, Week 35-43 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 3.81]
  6 - 12 years, Week 35-44: number analyzed (Participants) | 41 | 224 | 344
  6 - 12 years, Week 35-44 | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 1.07]
  6 - 12 years, Week 35-45: number analyzed (Participants) | 42 | 326 | 345
  6 - 12 years, Week 35-45 | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 1.13] | 0.00 [0.00 to 1.06]
  6 - 12 years, Week 35-46: number analyzed (Participants) | 47 | 600 | 358
  6 - 12 years, Week 35-46 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.61] | 0.00 [0.00 to 1.03]
  6 - 12 years, Week 35-47: number analyzed (Participants) | 47 | 615 | 420
  6 - 12 years, Week 35-47 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 0.60] | 0.00 [0.00 to 0.87]
  6 - 12 years, Week 35-48: number analyzed (Participants) | 48 | 634 | 420
  6 - 12 years, Week 35-48 | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 0.87]
  13 - 17 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 0
  13 - 17 years, Week 35-37: number analyzed (Participants) | 8 | 0 | 0
  13 - 17 years, Week 35-37 | 0.00 [0.00 to 36.94] |  |
  13 - 17 years, Week 35-38: number analyzed (Participants) | 24 | 0 | 0
  13 - 17 years, Week 35-38 | 0.00 [0.00 to 14.25] |  |
  13 - 17 years, Week 35-39: number analyzed (Participants) | 38 | 5 | 1
  13 - 17 years, Week 35-39 | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 97.50]
  13 - 17 years, Week 35-40: number analyzed (Participants) | 45 | 14 | 3
  13 - 17 years, Week 35-40 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 70.76]
  13 - 17 years, Week 35-41: number analyzed (Participants) | 55 | 31 | 35
  13 - 17 years, Week 35-41 | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-42: number analyzed (Participants) | 59 | 48 | 35
  13 - 17 years, Week 35-42 | 0.00 [0.00 to 6.06] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 10.00]
  13 - 17 years, Week 35-43: number analyzed (Participants) | 61 | 61 | 36
  13 - 17 years, Week 35-43 | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 5.87] | 0.00 [0.00 to 9.74]
  13 - 17 years, Week 35-44: number analyzed (Participants) | 62 | 86 | 50
  13 - 17 years, Week 35-44 | 0.00 [0.00 to 5.78] | 0.00 [0.00 to 4.20] | 0.00 [0.00 to 7.11]
  13 - 17 years, Week 35-45: number analyzed (Participants) | 70 | 166 | 255
  13 - 17 years, Week 35-45 | 0.00 [0.00 to 5.13] | 0.00 [0.00 to 2.20] | 0.00 [0.00 to 1.44]
  13 - 17 years, Week 35-46: number analyzed (Participants) | 76 | 178 | 257
  13 - 17 years, Week 35-46 | 0.00 [0.00 to 4.74] | 0.00 [0.00 to 2.05] | 0.00 [0.00 to 1.43]
  13 - 17 years, Week 35-47: number analyzed (Participants) | 82 | 183 | 262
  13 - 17 years, Week 35-47 | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.40]
  13 - 17 years, Week 35-48: number analyzed (Participants) | 86 | 184 | 262
  13 - 17 years, Week 35-48 | 1.16 [0.03 to 6.31] | 0.00 [0.00 to 1.98] | 0.00 [0.00 to 1.40]
  18 - 65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  18 - 65 years, Week 35-36: number analyzed (Participants) | 0 | 0 | 10
  18 - 65 years, Week 35-36 |  |  | 0.00 [0.00 to 30.85]
  18 - 65 years, Week 35-37: number analyzed (Participants) | 719 | 3 | 162
  18 - 65 years, Week 35-37 | 0.14 [0.00 to 0.95] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 2.25]
  18 - 65 years, Week 35-38: number analyzed (Participants) | 1579 | 7 | 326
  18 - 65 years, Week 35-38 | 0.06 [0.00 to 0.45] | 0.00 [0.00 to 40.96] | 0.31 [0.00 to 1.91]
  18 - 65 years, Week 35-39: number analyzed (Participants) | 2994 | 17 | 473
  18 - 65 years, Week 35-39 | 0.03 [0.00 to 0.03] | 0.00 [0.00 to 19.51] | 0.21 [0.00 to 1.31]
  18 - 65 years, Week 35-40: number analyzed (Participants) | 3735 | 80 | 668
  18 - 65 years, Week 35-40 | 0.08 [0.02 to 0.24] | 0.00 [0.00 to 4.51] | 0.15 [0.00 to 0.97]
  18 - 65 years, Week 35-41: number analyzed (Participants) | 4370 | 174 | 778
  18 - 65 years, Week 35-41 | 0.07 [0.01 to 0.21] | 0.00 [0.00 to 2.10] | 0.39 [0.04 to 1.50]
  18 - 65 years, Week 35-42: number analyzed (Participants) | 4725 | 284 | 859
  18 - 65 years, Week 35-42 | 0.06 [0.01 to 0.19] | 0.00 [0.00 to 1.29] | 0.35 [0.04 to 1.33]
  18 - 65 years, Week 35-43: number analyzed (Participants) | 4946 | 403 | 945
  18 - 65 years, Week 35-43 | 0.06 [0.01 to 0.18] | 0.00 [0.00 to 0.91] | 0.32 [0.03 to 1.22]
  18 - 65 years, Week 35-44: number analyzed (Participants) | 5259 | 482 | 1024
  18 - 65 years, Week 35-44 | 0.06 [0.01 to 0.17] | 0.21 [0.00 to 2.26] | 0.29 [0.03 to 1.13]
  18 - 65 years, Week 35-45: number analyzed (Participants) | 5483 | 537 | 1107
  18 - 65 years, Week 35-45 | 0.05 [0.01 to 0.16] | 0.19 [0.00 to 1.89] | 0.27 [0.03 to 1.05]
  18 - 65 years, Week 35-46: number analyzed (Participants) | 5706 | 588 | 1147
  18 - 65 years, Week 35-46 | 0.07 [0.01 to 0.22] | 0.17 [0.00 to 1.64] | 0.26 [0.03 to 1.01]
  18 - 65 years, Week 35-47: number analyzed (Participants) | 5852 | 627 | 1210
  18 - 65 years, Week 35-47 | 0.07 [0.01 to 0.21] | 0.16 [0.00 to 1.51] | 0.25 [0.02 to 0.95]
  18 - 65 years, Week 35-48: number analyzed (Participants) | 5940 | 656 | 1238
  18 - 65 years, Week 35-48 | 0.07 [0.01 to 0.21] | 0.15 [0.00 to 1.42] | 0.24 [0.02 to 0.93]
  >65 years, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  >65 years, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  >65 years, Week 35-36: number analyzed (Participants) | 1 | 1 | 52
  >65 years, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.85]
  >65 years, Week 35-37: number analyzed (Participants) | 1736 | 3 | 369
  >65 years, Week 35-37 | 0.12 [0.01 to 0.42] | 0.00 [0.00 to 70.76] | 0.27 [0.00 to 2.23]
  >65 years, Week 35-38: number analyzed (Participants) | 3609 | 9 | 746
  >65 years, Week 35-38 | 0.19 [0.06 to 0.45] | 0.00 [0.00 to 33.63] | 0.27 [0.02 to 1.22]
  >65 years, Week 35-39: number analyzed (Participants) | 6283 | 16 | 1083
  >65 years, Week 35-39 | 0.16 [0.07 to 0.29] | 0.00 [0.00 to 20.59] | 0.18 [0.01 to 0.85]
  >65 years, Week 35-40: number analyzed (Participants) | 7586 | 58 | 1447
  >65 years, Week 35-40 | 0.16 [0.08 to 0.28] | 0.00 [0.00 to 6.16] | 0.21 [0.04 to 0.64]
  >65 years, Week 35-41: number analyzed (Participants) | 8604 | 137 | 1602
  >65 years, Week 35-41 | 0.16 [0.07 to 0.31] | 0.00 [0.00 to 2.66] | 0.19 [0.03 to 0.58]
  >65 years, Week 35-42: number analyzed (Participants) | 9151 | 202 | 1722
  >65 years, Week 35-42 | 0.14 [0.07 to 0.29] | 0.50 [0.01 to 2.73] | 0.17 [0.03 to 0.53]
  >65 years, Week 35-43: number analyzed (Participants) | 9425 | 284 | 1787
  >65 years, Week 35-43 | 0.17 [0.07 to 0.35] | 0.35 [0.01 to 1.95] | 0.17 [0.03 to 0.51]
  >65 years, Week 35-44: number analyzed (Participants) | 9855 | 348 | 1859
  >65 years, Week 35-44 | 0.18 [0.06 to 0.41] | 0.29 [0.01 to 1.59] | 0.27 [0.07 to 0.68]
  >65 years, Week 35-45: number analyzed (Participants) | 10077 | 385 | 1918
  >65 years, Week 35-45 | 0.19 [0.07 to 0.40] | 0.52 [0.06 to 1.86] | 0.26 [0.07 to 0.66]
  >65 years, Week 35-46: number analyzed (Participants) | 10191 | 422 | 1950
  >65 years, Week 35-46 | 0.20 [0.07 to 0.42] | 0.47 [0.06 to 1.70] | 0.31 [0.11 to 0.68]
  >65 years, Week 35-47: number analyzed (Participants) | 10297 | 449 | 1980
  >65 years, Week 35-47 | 0.19 [0.07 to 0.41] | 0.45 [0.05 to 1.60] | 0.35 [0.12 to 0.81]
  >65 years, Week 35-48: number analyzed (Participants) | 10349 | 471 | 1990
  >65 years, Week 35-48 | 0.19 [0.07 to 0.41] | 0.43 [0.05 to 1.53] | 0.35 [0.12 to 0.81]

111. Secondary Outcome: Weekly Incidence Rates of Any AEIs Recorded in EHR, by Vaccine Group and United Kingdom Chief Medical Officer (UK CMO)-Specified Risk Status
Description: as for outcome 74
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.69 [0.00 to 16.08]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 11.44 [9.28 to 13.90] | 0.00 [0.00 to 52.18] | 0.68 [0.01 to 4.04]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 9.76 [7.27 to 12.76] | 14.29 [0.00 to 90.97] | 1.61 [0.70 to 3.14]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 9.72 [8.38 to 11.18] | 2.06 [0.25 to 7.25] | 2.46 [0.94 to 5.16]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 9.78 [5.87 to 15.06] | 7.35 [4.71 to 10.82] | 1.72 [0.50 to 4.22]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 8.79 [6.62 to 11.38] | 5.96 [2.86 to 10.77] | 0.30 [0.00 to 2.16]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 5.58 [3.15 to 9.07] | 2.53 [1.14 to 4.80] | 1.89 [0.23 to 6.66]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 6.26 [2.99 to 11.35] | 4.28 [1.91 to 8.16] | 1.52 [0.11 to 6.34]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 6.17 [2.44 to 12.51] | 4.80 [1.53 to 11.02] | 0.19 [0.00 to 1.08]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 6.04 [2.99 to 10.69] | 2.97 [0.05 to 16.62] | 2.61 [0.35 to 8.77]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 5.95 [2.73 to 11.05] | 1.07 [0.06 to 4.86] | 3.85 [0.36 to 14.33]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 3.77 [1.30 to 8.36] | 2.19 [0.45 to 6.27] | 1.14 [0.06 to 5.29]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 4.76 [0.38 to 18.41] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 15.04 [9.43 to 22.26] |  | 9.68 [2.04 to 25.75]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 13.94 [9.05 to 20.18] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 13.53 [9.92 to 17.85] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 12.00 [6.25 to 20.24] | 6.90 [0.85 to 22.77] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 6.71 [1.53 to 17.74] | 2.44 [0.06 to 12.86] | 1.56 [0.01 to 10.47]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 2.27 [0.26 to 8.11] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 3.85 [0.33 to 14.73] | 5.45 [0.66 to 18.46] | 3.13 [0.08 to 16.22]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 4.35 [0.91 to 12.18] | 14.81 [3.75 to 35.25] | 2.17 [0.06 to 11.53]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 9.46 [3.89 to 18.52] | 4.00 [1.10 to 9.93] | 4.68 [2.36 to 8.22]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 12.35 [2.91 to 30.79] | 3.70 [0.24 to 15.41] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 6.52 [1.37 to 17.90] | 9.52 [1.17 to 30.38] | 4.17 [0.02 to 27.48]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 6.25 [0.00 to 64.40] | 0.00 [0.00 to 45.93]

112. Secondary Outcome: Cumulative Incidence Rates of Any AEIs Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 78
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.67 [0.00 to 14.74]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 11.43 [9.27 to 13.90] | 0.00 [0.00 to 45.93] | 0.80 [0.08 to 3.04]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 10.56 [8.59 to 12.79] | 7.69 [0.08 to 41.17] | 1.20 [0.59 to 2.19]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 10.19 [8.58 to 11.99] | 2.73 [0.34 to 9.45] | 1.59 [0.75 to 2.95]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 10.12 [8.28 to 12.21] | 6.15 [4.03 to 8.91] | 1.63 [0.71 to 3.15]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 9.95 [8.12 to 12.04] | 6.07 [3.78 to 9.16] | 1.43 [0.61 to 2.85]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 9.67 [7.83 to 11.79] | 4.90 [2.99 to 7.53] | 1.47 [0.64 to 2.88]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 9.56 [7.73 to 11.66] | 4.76 [2.94 to 7.23] | 1.47 [0.66 to 2.82]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 9.40 [7.56 to 11.50] | 4.77 [2.70 to 7.73] | 1.27 [0.60 to 2.34]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 9.31 [7.50 to 11.38] | 4.51 [2.26 to 7.96] | 1.31 [0.67 to 2.32]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 9.25 [7.44 to 11.32] | 3.89 [1.61 to 7.74] | 1.37 [0.73 to 2.33]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 9.17 [7.35 to 11.26] | 3.80 [1.60 to 7.52] | 1.36 [0.73 to 2.31]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 9.10 [7.28 to 11.20] | 3.83 [1.61 to 7.58] | 1.35 [0.72 to 2.29]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 15.04 [9.43 to 22.26] |  | 9.09 [1.92 to 24.33]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 14.43 [10.64 to 18.94] | 0.00 [0.00 to 70.76] | 3.95 [0.82 to 11.11]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 13.95 [10.83 to 17.57] | 0.00 [0.00 to 26.46] | 2.63 [0.55 to 7.50]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 13.53 [10.44 to 17.13] | 4.88 [0.60 to 16.53] | 1.69 [0.30 to 5.19]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 12.38 [9.23 to 16.15] | 3.66 [0.76 to 10.32] | 1.66 [0.45 to 4.19]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 11.55 [8.60 to 15.08] | 2.17 [0.45 to 6.22] | 1.48 [0.41 to 3.75]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 11.19 [8.25 to 14.73] | 3.11 [1.13 to 6.70] | 1.66 [0.54 to 3.82]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 10.79 [7.93 to 14.25] | 5.67 [2.91 to 9.80] | 1.72 [0.64 to 3.71]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 10.71 [8.05 to 13.89] | 5.19 [3.10 to 8.07] | 2.92 [1.21 to 5.82]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 10.81 [8.35 to 13.71] | 4.84 [2.37 to 8.64] | 2.82 [1.13 to 5.77]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 10.67 [8.29 to 13.46] | 5.04 [2.58 to 8.76] | 2.88 [1.27 to 5.53]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 10.44 [8.07 to 13.22] | 5.08 [2.50 to 9.05] | 2.85 [1.25 to 5.51]

113. Secondary Outcome: Weekly Incidence Rates of Fever/Pyrexia Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 68
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.06]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 0.39 [0.16 to 0.76] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.84]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 0.46 [0.18 to 0.99] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.74]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 0.50 [0.21 to 1.02] | 0.00 [0.00 to 3.73] | 0.22 [0.00 to 1.63]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 0.37 [0.13 to 0.84] | 1.28 [0.12 to 4.96] | 0.00 [0.00 to 0.70]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 0.40 [0.15 to 0.87] | 0.66 [0.08 to 2.37] | 0.00 [0.00 to 1.10]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 0.00 [0.00 to 0.45] | 0.00 [0.00 to 1.03] | 0.00 [0.00 to 1.72]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 0.45 [0.05 to 1.62] | 0.00 [0.00 to 1.12] | 0.00 [0.00 to 2.76]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 0.29 [0.02 to 1.34] | 0.48 [0.06 to 1.72] | 0.00 [0.00 to 0.71]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 0.26 [0.00 to 1.93] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 3.16]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 0.37 [0.00 to 2.71] | 0.21 [0.00 to 2.05] | 0.00 [0.00 to 4.62]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 0.47 [0.00 to 3.37] | 0.73 [0.01 to 4.77] | 0.00 [0.00 to 2.09]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 1.50 [0.18 to 5.33] |  | 0.00 [0.00 to 11.22]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 1.82 [0.30 to 5.77] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 0.59 [0.07 to 2.11] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 1.14 [0.02 to 6.55] | 3.45 [0.09 to 17.76] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 0.00 [0.00 to 2.22] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 5.60]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.89]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 6.60] | 0.00 [0.00 to 7.71]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.43 [0.01 to 2.35]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 1.23 [0.00 to 9.48] | 0.00 [0.00 to 3.36] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 14.25]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 45.93]

114. Secondary Outcome: Cumulative Incidence Rates of Fever/Pyrexia Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Fever/pyrexia = all subjects with a fever/pyrexia read code recorded were considered as having fever/pyrexia, regardless of what temperature had been recorded. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.96]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 0.39 [0.16 to 0.76] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.74]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 0.43 [0.26 to 0.65] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 0.37]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 0.46 [0.25 to 0.77] | 0.00 [0.00 to 3.30] | 0.07 [0.00 to 0.50]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 0.44 [0.27 to 0.68] | 0.95 [0.03 to 4.78] | 0.05 [0.00 to 0.38]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 0.44 [0.29 to 0.64] | 0.83 [0.18 to 2.32] | 0.04 [0.00 to 0.32]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 0.41 [0.26 to 0.61] | 0.56 [0.09 to 1.77] | 0.04 [0.00 to 0.29]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 0.41 [0.26 to 0.61] | 0.43 [0.06 to 1.48] | 0.04 [0.00 to 0.28]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 0.41 [0.26 to 0.60] | 0.44 [0.11 to 1.19] | 0.03 [0.00 to 0.23]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 0.40 [0.26 to 0.60] | 0.38 [0.08 to 1.07] | 0.03 [0.00 to 0.23]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 0.40 [0.26 to 0.60] | 0.35 [0.08 to 0.95] | 0.03 [0.00 to 0.22]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 0.40 [0.26 to 0.59] | 0.37 [0.11 to 0.88] | 0.03 [0.00 to 0.21]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 0.40 [0.26 to 0.59] | 0.35 [0.11 to 0.85] | 0.03 [0.00 to 0.21]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 1.50 [0.18 to 5.33] |  | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 1.68 [0.36 to 4.74] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 4.74]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 1.10 [0.32 to 2.70] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.18]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 1.11 [0.34 to 2.63] | 2.44 [0.06 to 12.86] | 0.00 [0.00 to 2.06]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 0.92 [0.27 to 2.25] | 1.22 [0.03 to 6.61] | 0.00 [0.00 to 1.52]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 0.85 [0.24 to 2.11] | 0.72 [0.02 to 3.97] | 0.00 [0.00 to 1.36]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 0.81 [0.22 to 2.05] | 0.52 [0.01 to 2.85] | 0.00 [0.00 to 1.21]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 0.76 [0.20 to 1.98] | 0.40 [0.01 to 2.23] | 0.00 [0.00 to 1.05]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 0.71 [0.18 to 1.87] | 0.29 [0.01 to 1.60] | 0.17 [0.00 to 0.95]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 0.75 [0.16 to 2.11] | 0.22 [0.01 to 1.22] | 0.17 [0.00 to 0.92]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 0.72 [0.16 to 2.03] | 0.21 [0.01 to 1.16] | 0.16 [0.00 to 0.89]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 0.71 [0.15 to 1.99] | 0.20 [0.01 to 1.13] | 0.16 [0.00 to 0.88]

115. Secondary Outcome: Weekly Incidence Rates of Local Symptoms Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 69
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.06]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 1.71 [0.61 to 3.77] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.84]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 1.35 [0.69 to 2.37] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.74]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 1.80 [1.28 to 2.45] | 0.00 [0.00 to 3.73] | 0.00 [0.00 to 0.82]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 1.70 [0.71 to 3.39] | 0.32 [0.00 to 2.10] | 0.00 [0.00 to 0.70]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 1.53 [0.97 to 2.29] | 0.99 [0.14 to 3.38] | 0.00 [0.00 to 1.10]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 0.61 [0.10 to 1.96] | 0.56 [0.06 to 2.06] | 0.00 [0.00 to 1.72]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 0.45 [0.05 to 1.66] | 0.61 [0.04 to 2.64] | 0.00 [0.00 to 2.76]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 0.88 [0.13 to 2.95] | 0.48 [0.06 to 1.72] | 0.00 [0.00 to 0.71]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 1.05 [0.20 to 3.17] | 0.66 [0.00 to 4.55] | 0.00 [0.00 to 3.16]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 0.74 [0.09 to 2.70] | 0.21 [0.00 to 2.00] | 0.00 [0.00 to 4.62]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 0.94 [0.05 to 4.24] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 2.09]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 5.26 [1.54 to 12.59] |  | 3.23 [0.08 to 16.70]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 6.06 [2.82 to 11.16] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 3.53 [1.49 to 6.97] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 4.57 [1.62 to 9.92] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 0.61 [0.00 to 4.32] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 5.60]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 0.00 [0.00 to 6.85] | 1.82 [0.05 to 9.72] | 0.00 [0.00 to 10.89]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 4.35 [0.91 to 12.18] | 1.85 [0.05 to 9.89] | 0.00 [0.00 to 7.71]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 1.56]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 3.70 [0.08 to 19.40] | 1.85 [0.01 to 13.63] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 2.17 [0.01 to 16.04] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 14.25]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 45.93]

116. Secondary Outcome: Cumulative Incidence Rates of Local Symptoms Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 80
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.96]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 1.71 [0.61 to 3.77] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.74]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 1.52 [0.82 to 2.57] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 0.37]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 1.64 [1.07 to 2.42] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 0.25]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 1.65 [1.09 to 2.41] | 0.24 [0.01 to 1.31] | 0.00 [0.00 to 0.19]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 1.64 [1.13 to 2.29] | 0.55 [0.04 to 2.31] | 0.00 [0.00 to 0.16]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 1.57 [1.13 to 2.07] | 0.56 [0.05 to 2.20] | 0.00 [0.00 to 0.15]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 1.53 [1.11 to 2.03] | 0.57 [0.05 to 2.27] | 0.00 [0.00 to 0.14]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 1.50 [1.09 to 2.02] | 0.55 [0.07 to 1.95] | 0.00 [0.00 to 0.12]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 1.49 [1.09 to 1.99] | 0.56 [0.11 to 1.70] | 0.00 [0.00 to 0.11]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 1.48 [1.08 to 1.96] | 0.50 [0.07 to 1.74] | 0.00 [0.00 to 0.11]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 1.47 [1.08 to 1.95] | 0.48 [0.06 to 1.65] | 0.00 [0.00 to 0.10]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 1.46 [1.07 to 1.94] | 0.46 [0.06 to 1.60] | 0.00 [0.00 to 0.10]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 5.26 [1.54 to 12.59] |  | 3.03 [0.08 to 15.76]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 5.70 [2.72 to 10.36] | 0.00 [0.00 to 70.76] | 1.32 [0.03 to 7.11]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 4.55 [2.27 to 8.04] | 0.00 [0.00 to 26.46] | 0.88 [0.01 to 5.49]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 4.55 [2.58 to 7.37] | 0.00 [0.00 to 8.60] | 0.56 [0.00 to 3.91]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 3.89 [2.24 to 6.23] | 0.00 [0.00 to 4.40] | 0.41 [0.00 to 2.93]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 3.57 [2.12 to 5.59] | 0.00 [0.00 to 2.64] | 0.37 [0.00 to 2.63]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 3.40 [2.06 to 5.26] | 0.52 [0.01 to 2.85] | 0.33 [0.00 to 2.35]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 3.46 [2.21 to 5.14] | 0.81 [0.10 to 2.89] | 0.29 [0.00 to 2.09]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 3.25 [2.08 to 4.82] | 0.58 [0.07 to 2.07] | 0.17 [0.00 to 1.48]
  Not at risk, Week 35-46: number analyzed (Participants) | 341 | 455 | 602
  Not at risk, Week 35-46 | 3.28 [2.27 to 4.57] | 0.88 [0.24 to 2.24] | 0.17 [0.00 to 1.42]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 3.24 [2.26 to 4.50] | 0.84 [0.23 to 2.14] | 0.16 [0.00 to 1.37]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 3.17 [2.20 to 4.41] | 0.81 [0.22 to 2.07] | 0.16 [0.00 to 1.35]

117. Secondary Outcome: Weekly Incidence Rates of General Non-specific Symptoms Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 70
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.06]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 3.98 [3.21 to 4.89] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.84]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 3.20 [2.36 to 4.25] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.74]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 3.12 [2.30 to 4.14] | 1.03 [0.03 to 5.61] | 0.45 [0.05 to 1.60]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 2.55 [1.89 to 3.37] | 2.56 [0.56 to 7.10] | 0.00 [0.00 to 0.70]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 2.00 [1.23 to 3.06] | 1.32 [0.18 to 4.50] | 0.00 [0.00 to 1.10]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 1.70 [0.59 to 3.80] | 0.56 [0.06 to 2.06] | 0.00 [0.00 to 1.72]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 2.24 [0.84 to 4.75] | 0.92 [0.06 to 3.95] | 0.00 [0.00 to 2.76]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 2.06 [0.81 to 4.27] | 1.44 [0.23 to 4.65] | 0.00 [0.00 to 0.71]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 1.57 [0.42 to 4.04] | 1.32 [0.06 to 6.37] | 0.00 [0.00 to 3.16]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 0.74 [0.09 to 2.70] | 0.21 [0.00 to 2.00] | 0.00 [0.00 to 4.62]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 2.09]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 4.51 [1.67 to 9.56] |  | 3.23 [0.02 to 21.72]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 3.03 [0.99 to 6.93] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 5.29 [2.04 to 10.94] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 4.57 [1.90 to 9.06] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 1.83 [0.23 to 6.42] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 5.60]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 1.14 [0.01 to 7.02] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 0.00 [0.00 to 6.85] | 1.82 [0.05 to 9.72] | 0.00 [0.00 to 10.89]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 3.70 [0.16 to 16.98] | 0.00 [0.00 to 7.71]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 1.35 [0.01 to 9.52] | 2.00 [0.10 to 9.21] | 2.13 [0.69 to 4.90]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 2.47 [0.12 to 11.36] | 0.93 [0.00 to 9.43] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 2.17 [0.06 to 11.53] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 14.25]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 45.93]

118. Secondary Outcome: Cumulative Incidence Rates of General Non-specific Symptoms Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 81
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.96]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 3.98 [3.21 to 4.89] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.74]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 3.57 [2.77 to 4.53] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 0.37]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 3.38 [2.56 to 4.36] | 0.91 [0.02 to 4.96] | 0.14 [0.02 to 0.50]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 3.23 [2.49 to 4.12] | 2.13 [0.63 to 5.14] | 0.10 [0.01 to 0.37]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 3.08 [2.37 to 3.93] | 1.79 [0.53 to 4.37] | 0.09 [0.01 to 0.31]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 2.99 [2.26 to 3.87] | 1.39 [0.39 to 3.47] | 0.08 [0.01 to 0.29]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 2.96 [2.23 to 3.86] | 1.28 [0.30 to 3.51] | 0.08 [0.01 to 0.27]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 2.92 [2.18 to 3.82] | 1.32 [0.29 to 3.68] | 0.06 [0.01 to 0.23]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 2.88 [2.15 to 3.78] | 1.32 [0.33 to 3.49] | 0.06 [0.01 to 0.22]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 2.85 [2.12 to 3.74] | 1.12 [0.20 to 3.43] | 0.06 [0.01 to 0.22]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 2.81 [2.08 to 3.70] | 1.06 [0.19 to 3.26] | 0.06 [0.01 to 0.20]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 2.78 [2.06 to 3.68] | 1.03 [0.19 to 3.15] | 0.06 [0.01 to 0.20]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 4.51 [1.67 to 9.56] |  | 3.03 [0.01 to 20.77]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 3.69 [1.86 to 6.51] | 0.00 [0.00 to 70.76] | 1.32 [0.01 to 9.66]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 4.55 [2.51 to 7.51] | 0.00 [0.00 to 26.46] | 0.88 [0.01 to 6.17]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 4.55 [2.93 to 6.70] | 0.00 [0.00 to 8.60] | 0.56 [0.00 to 4.02]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 4.09 [2.49 to 6.31] | 0.00 [0.00 to 4.40] | 0.41 [0.00 to 2.67]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 3.85 [2.32 to 5.97] | 0.00 [0.00 to 2.64] | 0.37 [0.00 to 2.46]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 3.67 [2.21 to 5.70] | 0.52 [0.01 to 2.85] | 0.33 [0.00 to 2.19]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 3.46 [2.05 to 5.43] | 1.21 [0.25 to 3.51] | 0.29 [0.00 to 1.77]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 3.33 [2.06 to 5.08] | 1.44 [0.47 to 3.33] | 1.03 [0.14 to 3.49]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 3.28 [2.05 to 4.95] | 1.32 [0.43 to 3.06] | 1.00 [0.13 to 3.44]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 3.24 [2.09 to 4.79] | 1.26 [0.40 to 2.97] | 0.96 [0.12 to 3.36]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 3.17 [2.04 to 4.69] | 1.22 [0.38 to 2.91] | 0.95 [0.12 to 3.35]

119. Secondary Outcome: Weekly Incidence Rates of Respiratory/Miscellaneous Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 71
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.69 [0.00 to 16.08]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 6.34 [5.19 to 7.65] | 0.00 [0.00 to 52.18] | 0.46 [0.01 to 2.71]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 4.86 [3.62 to 6.37] | 14.29 [0.00 to 90.97] | 0.60 [0.03 to 2.75]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 4.71 [3.97 to 5.55] | 1.03 [0.03 to 5.61] | 1.34 [0.35 to 3.48]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 5.47 [3.22 to 8.62] | 4.15 [2.16 to 7.15] | 1.15 [0.41 to 2.55]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 4.79 [3.67 to 6.14] | 3.97 [2.07 to 6.84] | 0.00 [0.00 to 1.10]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 2.79 [1.54 to 4.63] | 0.84 [0.17 to 2.44] | 1.89 [0.23 to 6.66]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 3.13 [1.02 to 7.19] | 2.75 [0.81 to 6.65] | 0.00 [0.00 to 2.76]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 3.23 [1.03 to 7.47] | 3.12 [1.08 to 6.91] | 0.19 [0.00 to 1.08]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 1.57 [0.30 to 4.67] | 1.32 [0.01 to 8.97] | 1.74 [0.21 to 6.14]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 1.86 [0.41 to 5.21] | 0.21 [0.00 to 2.00] | 0.00 [0.00 to 4.62]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 2.36 [0.33 to 7.88] | 1.46 [0.18 to 5.17] | 1.14 [0.06 to 5.29]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 1.19 [0.01 to 7.80] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 8.27 [4.20 to 14.32] |  | 3.23 [0.02 to 21.72]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 4.85 [2.12 to 9.33] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 7.94 [4.20 to 13.40] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 3.43 [1.27 to 7.31] | 3.45 [0.09 to 17.76] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 3.66 [1.33 to 7.88] | 2.44 [0.06 to 12.86] | 1.56 [0.01 to 10.47]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 0.00 [0.00 to 6.85] | 3.64 [0.44 to 12.53] | 0.00 [0.00 to 10.89]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 1.45 [0.01 to 10.55] | 7.41 [2.06 to 17.89] | 2.17 [0.06 to 11.53]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 5.41 [5.41 to 14.52] | 1.00 [0.03 to 5.45] | 2.55 [0.94 to 5.47]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 6.17 [1.50 to 15.96] | 2.78 [0.15 to 12.35] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 4.35 [0.33 to 17.06] | 0.00 [0.00 to 16.11] | 4.17 [0.02 to 27.48]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 6.25 [0.00 to 64.40] | 0.00 [0.00 to 45.93]

120. Secondary Outcome: Cumulative Incidence Rates of Respiratory/Miscellaneous Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 82
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 1.67 [0.00 to 14.74]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 6.34 [5.19 to 7.65] | 0.00 [0.00 to 45.93] | 0.60 [0.08 to 2.12]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 5.56 [4.76 to 6.45] | 7.69 [0.08 to 41.17] | 0.60 [0.13 to 1.73]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 5.19 [4.45 to 6.02] | 1.82 [0.22 to 6.41] | 0.83 [0.21 to 2.21]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 5.24 [4.33 to 6.29] | 3.55 [1.86 to 6.08] | 0.92 [0.25 to 2.34]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 5.19 [4.30 to 6.19] | 3.72 [2.42 to 5.45] | 0.78 [0.20 to 2.05]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 5.03 [4.13 to 6.06] | 2.78 [1.75 to 4.16] | 0.88 [0.26 to 2.15]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 4.97 [4.06 to 6.01] | 2.77 [1.75 to 4.16] | 0.83 [0.25 to 2.02]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 4.89 [3.98 to 5.92] | 2.85 [1.74 to 4.38] | 0.73 [0.24 to 1.67]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 4.80 [3.90 to 5.83] | 2.63 [1.37 to 4.54] | 0.76 [0.29 to 1.61]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 4.75 [3.83 to 5.81] | 2.19 [0.96 to 4.25] | 0.75 [0.29 to 1.57]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 4.71 [3.80 to 5.77] | 2.16 [0.98 to 4.10] | 0.77 [0.32 to 1.55]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 4.68 [3.76 to 5.74] | 2.13 [0.96 to 4.06] | 0.76 [0.31 to 1.53]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 8.27 [4.20 to 14.32] |  | 3.03 [0.01 to 20.77]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 6.38 [3.88 to 9.78] | 0.00 [0.00 to 70.76] | 1.32 [0.01 to 8.76]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 7.21 [5.08 to 9.87] | 0.00 [0.00 to 26.46] | 0.88 [0.01 to 5.83]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 6.40 [4.46 to 8.83] | 2.44 [0.06 to 12.86] | 0.56 [0.00 to 3.88]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 5.94 [4.35 to 7.88] | 2.44 [0.30 to 8.53] | 0.83 [0.08 to 3.19]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 5.45 [3.94 to 7.31] | 1.45 [0.18 to 5.14] | 0.74 [0.08 to 2.76]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 5.19 [3.75 to 6.98] | 2.07 [0.57 to 5.22] | 0.66 [0.07 to 2.52]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 4.97 [3.59 to 6.70] | 3.24 [1.41 to 6.28] | 0.86 [0.18 to 2.50]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 5.00 [3.77 to 6.49] | 2.59 [1.19 to 4.87] | 1.54 [0.57 to 3.34]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 5.07 [3.96 to 6.38] | 2.64 [1.37 to 4.56] | 1.50 [0.53 to 3.30]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 5.05 [3.96 to 6.33] | 2.52 [1.31 to 4.36] | 1.60 [0.64 to 3.28]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 4.94 [3.87 to 6.20] | 2.64 [1.31 to 4.72] | 1.58 [0.63 to 3.25]

121. Secondary Outcome: Weekly Incidence Rates of Gastrointestinal Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhea, nausea, and vomiting. The weekly incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.06]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 2.10 [1.36 to 3.09] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.84]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 1.74 [0.95 to 2.90] | 14.29 [0.00 to 90.97] | 0.00 [0.00 to 0.74]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 1.46 [0.97 to 2.10] | 0.00 [0.00 to 3.73] | 0.00 [0.00 to 0.82]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 1.54 [0.97 to 2.32] | 1.28 [0.35 to 3.24] | 0.00 [0.00 to 0.70]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 1.26 [0.62 to 2.28] | 0.66 [0.08 to 2.37] | 0.00 [0.00 to 1.10]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 1.09 [0.50 to 2.06] | 0.00 [0.00 to 1.03] | 0.00 [0.00 to 1.72]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 0.89 [0.24 to 2.28] | 0.00 [0.00 to 1.12] | 0.76 [0.00 to 5.65]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 0.73 [0.24 to 1.71] | 0.24 [0.00 to 1.48] | 0.00 [0.00 to 0.71]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 2.10 [0.56 to 5.34] | 0.66 [0.00 to 4.55] | 0.87 [0.02 to 4.75]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 1.86 [0.20 to 6.79] | 0.21 [0.00 to 1.71] | 1.28 [0.01 to 8.31]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 2.09]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 2.26 [0.23 to 8.42] |  | 3.23 [0.02 to 21.72]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 3.03 [0.99 to 6.93] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 2.06 [0.68 to 4.71] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 0.57 [0.01 to 3.31] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 1.22 [0.03 to 6.81] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 5.60]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 1.14 [0.01 to 7.91] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.89]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 1.85 [0.05 to 9.89] | 0.00 [0.00 to 7.71]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 1.35 [0.03 to 7.30] | 2.00 [0.10 to 9.21] | 0.85 [0.10 to 3.04]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 3.36] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 14.25]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 45.93]

122. Secondary Outcome: Cumulative Incidence Rates of Gastrointestinal Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Gastrointestinal adverse events include any gastrointestinal adverse events, decreased appetite, diarrhea, nausea, and vomiting. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.96]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 2.10 [1.36 to 3.09] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.74]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 1.91 [1.42 to 2.50] | 7.69 [0.08 to 41.17] | 0.00 [0.00 to 0.37]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 1.71 [1.24 to 2.31] | 0.91 [0.02 to 4.96] | 0.00 [0.00 to 0.25]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 1.68 [1.29 to 2.16] | 1.18 [0.38 to 2.74] | 0.00 [0.00 to 0.19]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 1.63 [1.24 to 2.11] | 0.97 [0.35 to 2.10] | 0.00 [0.00 to 0.16]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 1.60 [1.22 to 2.05] | 0.65 [0.23 to 1.42] | 0.00 [0.00 to 0.15]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 1.57 [1.20 to 2.02] | 0.50 [0.16 to 1.17] | 0.04 [0.00 to 0.30]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 1.53 [1.18 to 1.96] | 0.44 [0.10 to 1.23] | 0.03 [0.00 to 0.20]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 1.55 [1.22 to 1.94] | 0.47 [0.16 to 1.05] | 0.06 [0.00 to 0.39]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 1.55 [1.23 to 1.94] | 0.42 [0.15 to 0.93] | 0.09 [0.01 to 0.37]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 1.53 [1.20 to 1.92] | 0.40 [0.15 to 0.88] | 0.09 [0.01 to 0.36]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 1.52 [1.19 to 1.90] | 0.39 [0.14 to 0.85] | 0.08 [0.01 to 0.35]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 2.26 [0.23 to 8.42] |  | 3.03 [0.01 to 20.77]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 2.68 [0.87 to 6.18] | 0.00 [0.00 to 70.76] | 1.32 [0.01 to 9.66]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 2.35 [0.93 to 4.85] | 0.00 [0.00 to 26.46] | 0.88 [0.01 to 6.17]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 1.97 [0.76 to 4.12] | 0.00 [0.00 to 8.60] | 0.56 [0.00 to 4.02]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 1.84 [0.79 to 3.62] | 0.00 [0.00 to 4.40] | 0.41 [0.00 to 2.67]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 1.78 [0.81 to 3.37] | 0.00 [0.00 to 2.64] | 0.37 [0.00 to 2.46]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 1.70 [0.77 to 3.23] | 0.00 [0.00 to 1.89] | 0.33 [0.00 to 2.19]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 1.60 [0.69 to 3.14] | 0.40 [0.01 to 2.23] | 0.29 [0.00 to 1.77]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 1.59 [0.73 to 2.99] | 0.86 [0.18 to 2.51] | 0.51 [0.07 to 1.75]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 1.49 [0.67 to 2.84] | 0.66 [0.14 to 1.91] | 0.50 [0.07 to 1.73]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 1.44 [0.66 to 2.74] | 0.63 [0.13 to 1.83] | 0.48 [0.06 to 1.69]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 1.41 [0.64 to 2.67] | 0.61 [0.13 to 1.77] | 0.47 [0.06 to 1.68]

123. Secondary Outcome: Weekly Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 73
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.06]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 0.69 [0.01 to 4.05] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.84]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 0.54 [0.05 to 2.13] | 0.00 [0.00 to 40.96] | 0.20 [0.00 to 1.15]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 0.34 [0.03 to 1.39] | 0.00 [0.00 to 3.73] | 0.00 [0.00 to 0.82]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 0.48 [0.06 to 1.75] | 0.64 [0.01 to 4.17] | 0.00 [0.00 to 0.70]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 0.20 [0.04 to 0.60] | 0.99 [0.14 to 3.38] | 0.00 [0.00 to 1.10]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 0.00 [0.00 to 0.45] | 0.28 [0.00 to 2.18] | 0.00 [0.00 to 1.72]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 0.22 [0.00 to 1.51] | 0.00 [0.00 to 1.12] | 0.00 [0.00 to 2.76]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 0.29 [0.02 to 1.34] | 0.24 [0.00 to 1.48] | 0.00 [0.00 to 0.71]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 0.26 [0.00 to 1.87] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 3.16]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 0.37 [0.00 to 2.68] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 4.62]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 2.09]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 0.75 [0.01 to 5.16] |  | 0.00 [0.00 to 11.22]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 1.21 [0.15 to 4.31] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 1.18 [0.17 to 3.93] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 0.00 [0.00 to 2.09] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 0.61 [0.01 to 3.69] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 5.60]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.89]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 3.70 [0.16 to 16.98] | 0.00 [0.00 to 7.71]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.43 [0.01 to 2.35]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 3.36] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 14.25]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 45.93]

124. Secondary Outcome: Cumulative Incidence Rates of Sensitivity/Anaphylaxis Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 84
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.96]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 0.69 [0.01 to 4.05] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.74]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 0.61 [0.03 to 2.87] | 0.00 [0.00 to 24.71] | 0.10 [0.00 to 0.57]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 0.49 [0.03 to 2.21] | 0.00 [0.00 to 3.30] | 0.07 [0.00 to 0.40]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 0.49 [0.03 to 2.11] | 0.47 [0.01 to 2.52] | 0.05 [0.00 to 0.31]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 0.46 [0.04 to 1.88] | 0.69 [0.05 to 2.89] | 0.04 [0.00 to 0.26]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 0.43 [0.03 to 1.79] | 0.56 [0.11 to 1.63] | 0.04 [0.00 to 0.24]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 0.42 [0.03 to 1.73] | 0.43 [0.09 to 1.23] | 0.04 [0.00 to 0.23]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 0.41 [0.04 to 1.64] | 0.38 [0.06 to 1.26] | 0.03 [0.00 to 0.20]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 0.41 [0.04 to 1.59] | 0.33 [0.04 to 1.17] | 0.03 [0.00 to 0.19]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 0.41 [0.04 to 1.61] | 0.27 [0.02 to 1.07] | 0.03 [0.00 to 0.19]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 0.40 [0.04 to 1.59] | 0.26 [0.02 to 1.02] | 0.03 [0.00 to 0.18]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 0.40 [0.04 to 1.57] | 0.25 [0.02 to 0.99] | 0.03 [0.00 to 0.18]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 0.75 [0.01 to 5.16] |  | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 1.01 [0.18 to 3.13] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 4.74]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 1.10 [0.21 to 3.29] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.18]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 0.86 [0.12 to 2.89] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 2.06]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 0.82 [0.15 to 2.52] | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 1.52]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 0.75 [0.12 to 2.39] | 0.00 [0.00 to 2.64] | 0.00 [0.00 to 1.36]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 0.72 [0.11 to 2.31] | 0.00 [0.00 to 1.89] | 0.00 [0.00 to 1.21]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 0.67 [0.10 to 2.22] | 0.81 [0.10 to 2.89] | 0.00 [0.00 to 1.05]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 0.63 [0.09 to 2.11] | 0.58 [0.07 to 2.07] | 0.17 [0.00 to 0.95]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 0.60 [0.09 to 2.01] | 0.44 [0.05 to 1.58] | 0.17 [0.00 to 0.92]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 0.58 [0.08 to 1.93] | 0.42 [0.05 to 1.51] | 0.16 [0.00 to 0.89]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 0.56 [0.08 to 1.89] | 0.41 [0.05 to 1.46] | 0.16 [0.00 to 0.88]

125. Secondary Outcome: Weekly Incidence Rates of Rash Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 74
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.06]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 0.69 [0.39 to 1.11] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.84]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 0.39 [0.19 to 0.71] | 0.00 [0.00 to 40.96] | 0.40 [0.04 to 1.53]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 0.32 [0.16 to 0.55] | 0.00 [0.00 to 3.73] | 0.00 [0.00 to 0.82]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 0.58 [0.29 to 1.04] | 0.32 [0.01 to 1.77] | 0.19 [0.00 to 1.06]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 0.13 [0.02 to 0.48] | 0.66 [0.08 to 2.37] | 0.00 [0.00 to 1.10]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 0.12 [0.00 to 0.89] | 0.00 [0.00 to 1.03] | 0.00 [0.00 to 1.72]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 0.67 [0.12 to 2.07] | 0.61 [0.07 to 2.19] | 0.00 [0.00 to 2.76]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 0.59 [0.12 to 1.70] | 0.24 [0.00 to 1.45] | 0.00 [0.00 to 0.71]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 0.26 [0.00 to 1.82] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 3.16]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 0.37 [0.00 to 2.54] | 0.21 [0.00 to 1.90] | 0.00 [0.00 to 4.62]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 2.09]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 1.19 [0.01 to 7.80] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 2.26 [0.47 to 6.45] |  | 0.00 [0.00 to 11.22]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 3.03 [0.44 to 9.92] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 0.88 [0.13 to 2.92] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 0.57 [0.00 to 3.97] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 0.00 [0.00 to 2.22] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 5.60]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.89]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 6.60] | 0.00 [0.00 to 7.71]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 1.56]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 1.23 [0.01 to 8.69] | 0.00 [0.00 to 3.36] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 14.25]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 45.93]

126. Secondary Outcome: Cumulative Incidence Rates of Rash Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 78
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.96]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 0.69 [0.39 to 1.11] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.74]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 0.53 [0.35 to 0.77] | 0.00 [0.00 to 24.71] | 0.20 [0.02 to 0.74]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 0.44 [0.31 to 0.60] | 0.00 [0.00 to 3.30] | 0.14 [0.01 to 0.53]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 0.46 [0.34 to 0.61] | 0.24 [0.01 to 1.31] | 0.15 [0.03 to 0.45]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 0.42 [0.31 to 0.55] | 0.41 [0.09 to 1.20] | 0.13 [0.03 to 0.38]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 0.40 [0.30 to 0.53] | 0.28 [0.06 to 0.81] | 0.12 [0.02 to 0.35]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 0.41 [0.31 to 0.54] | 0.36 [0.12 to 0.83] | 0.11 [0.02 to 0.33]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 0.42 [0.32 to 0.54] | 0.33 [0.12 to 0.71] | 0.09 [0.02 to 0.29]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 0.42 [0.32 to 0.54] | 0.28 [0.10 to 0.61] | 0.09 [0.02 to 0.28]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 0.42 [0.32 to 0.54] | 0.27 [0.11 to 0.55] | 0.09 [0.02 to 0.27]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 0.41 [0.31 to 0.53] | 0.26 [0.10 to 0.53] | 0.09 [0.02 to 0.26]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 0.41 [0.31 to 0.53] | 0.28 [0.12 to 0.56] | 0.08 [0.02 to 0.26]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 2.26 [0.47 to 6.45] |  | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 2.68 [0.73 to 6.77] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 4.74]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 1.72 [0.47 to 4.35] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.18]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 1.48 [0.48 to 3.42] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 2.06]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 1.23 [0.41 to 2.79] | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 1.52]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 1.13 [0.39 to 2.52] | 0.00 [0.00 to 2.64] | 0.00 [0.00 to 1.36]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 1.07 [0.38 to 2.39] | 0.00 [0.00 to 1.89] | 0.00 [0.00 to 1.21]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 1.01 [0.35 to 2.27] | 0.00 [0.00 to 1.48] | 0.00 [0.00 to 1.05]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 0.95 [0.33 to 2.13] | 0.00 [0.00 to 1.06] | 0.00 [0.00 to 0.63]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 0.97 [0.39 to 1.98] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.61]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 0.94 [0.37 to 1.93] | 0.21 [0.01 to 1.16] | 0.00 [0.00 to 0.59]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 0.92 [0.36 to 1.90] | 0.20 [0.01 to 1.13] | 0.00 [0.00 to 0.58]

127. Secondary Outcome: Weekly Incidence Rates of Musculoskeletal Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 75
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.06]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 4.11 [2.99 to 5.51] | 0.00 [0.00 to 52.18] | 0.23 [0.00 to 1.36]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 3.36 [2.39 to 4.57] | 0.00 [0.00 to 40.96] | 0.40 [0.05 to 1.44]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 3.20 [2.58 to 3.93] | 0.00 [0.00 to 3.73] | 0.89 [0.24 to 2.27]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 2.39 [1.62 to 3.40] | 1.28 [0.01 to 8.23] | 0.57 [0.07 to 2.08]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 2.53 [1.80 to 3.46] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 1.10]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 2.18 [0.95 to 4.26] | 0.56 [0.06 to 2.06] | 0.00 [0.00 to 1.72]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 3.13 [1.44 to 5.87] | 0.31 [0.00 to 1.95] | 0.76 [0.01 to 5.02]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 2.06 [0.73 to 4.52] | 0.96 [0.01 to 5.84] | 0.00 [0.00 to 0.71]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 2.36 [0.70 to 5.70] | 0.66 [0.05 to 2.81] | 0.00 [0.00 to 3.16]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 1.12 [0.23 to 3.22] | 0.00 [0.00 to 0.78] | 2.56 [0.31 to 8.96]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 1.89 [0.28 to 6.18] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 2.09]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 2.38 [0.29 to 8.34] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 6.77 [2.22 to 15.15] |  | 3.23 [0.08 to 16.70]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 3.64 [1.16 to 8.42] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 4.71 [2.21 to 8.64] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 5.14 [1.78 to 11.28] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 2.44 [0.64 to 6.27] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 5.60]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 3.85 [0.33 to 14.73] | 0.00 [0.00 to 6.49] | 3.13 [0.08 to 16.22]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 3.70 [0.16 to 16.98] | 0.00 [0.00 to 7.71]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 4.05 [0.52 to 13.69] | 0.00 [0.00 to 3.62] | 0.43 [0.01 to 2.35]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 2.47 [0.07 to 12.65] | 0.93 [0.00 to 9.43] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 2.17 [0.06 to 11.53] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 14.25]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 45.93]

128. Secondary Outcome: Cumulative Incidence Rates of Musculoskeletal Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: AEIs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. Musculoskeletal adverse events include any musculoskeletal adverse events, arthropathy, and muscle aches/myalgia. The cumulative incidence rates of AEIs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any AEIs in EHR (combining routine data collection and card-based ADR reporting system) within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.96]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 4.11 [2.99 to 5.51] | 0.00 [0.00 to 45.93] | 0.20 [0.00 to 1.12]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 3.71 [2.74 to 4.92] | 0.00 [0.00 to 24.71] | 0.30 [0.06 to 0.88]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 3.49 [2.70 to 4.43] | 0.00 [0.00 to 3.30] | 0.48 [0.18 to 1.03]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 3.30 [2.62 to 4.10] | 0.95 [0.03 to 5.00] | 0.51 [0.17 to 1.16]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 3.20 [2.54 to 3.97] | 0.55 [0.04 to 2.31] | 0.43 [0.13 to 1.04]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 3.14 [2.46 to 3.93] | 0.56 [0.05 to 2.20] | 0.40 [0.12 to 0.96]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 3.14 [2.46 to 3.94] | 0.50 [0.10 to 1.49] | 0.42 [0.16 to 0.88]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 3.08 [2.40 to 3.89] | 0.60 [0.07 to 2.19] | 0.35 [0.11 to 0.84]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 3.07 [2.41 to 3.84] | 0.61 [0.08 to 2.13] | 0.34 [0.10 to 0.81]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 3.03 [2.38 to 3.80] | 0.50 [0.05 to 1.95] | 0.39 [0.14 to 0.85]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 3.01 [2.36 to 3.79] | 0.48 [0.04 to 1.86] | 0.37 [0.13 to 0.82]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 2.99 [2.34 to 3.77] | 0.53 [0.06 to 1.93] | 0.36 [0.13 to 0.81]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 6.77 [2.22 to 15.15] |  | 15.15 [0.08 to 15.76]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 5.03 [2.53 to 8.85] | 0.00 [0.00 to 70.76] | 1.32 [0.03 to 7.11]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 4.86 [2.85 to 7.68] | 0.00 [0.00 to 26.46] | 0.88 [0.01 to 5.49]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 4.92 [3.02 to 7.52] | 0.00 [0.00 to 8.60] | 0.56 [0.00 to 3.91]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 4.50 [2.87 to 6.69] | 0.00 [0.00 to 4.40] | 0.41 [0.00 to 2.93]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 4.13 [2.69 to 6.03] | 0.00 [0.00 to 2.64] | 0.37 [0.00 to 2.63]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 4.12 [2.71 to 5.98] | 0.00 [0.00 to 1.89] | 0.66 [0.08 to 2.37]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 3.88 [2.57 to 5.60] | 0.81 [0.10 to 2.89] | 0.57 [0.06 to 2.16]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 3.89 [2.72 to 5.37] | 0.58 [0.07 to 2.07] | 0.51 [0.11 to 1.50]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 3.80 [2.78 to 5.07] | 0.66 [0.13 to 1.98] | 0.50 [0.10 to 1.45]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 3.75 [2.75 to 4.98] | 0.63 [0.12 to 1.92] | 0.48 [0.10 to 1.39]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 3.67 [2.68 to 4.89] | 0.61 [0.11 to 1.88] | 0.47 [0.10 to 1.38]

129. Secondary Outcome: Weekly Incidence Rates of Neurological Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 76
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.06]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 0.21 [0.07 to 0.50] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 0.84]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 0.27 [0.11 to 0.56] | 0.00 [0.00 to 40.96] | 0.00 [0.00 to 0.74]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 0.21 [0.04 to 0.63] | 0.00 [0.00 to 3.73] | 0.00 [0.00 to 0.82]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 0.00 [0.00 to 0.20] | 0.32 [0.00 to 2.10] | 0.00 [0.00 to 0.70]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 0.20 [0.03 to 0.66] | 0.33 [0.01 to 1.83] | 0.30 [0.00 to 2.16]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 0.00 [0.00 to 0.45] | 0.00 [0.00 to 1.03] | 0.00 [0.00 to 1.72]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 0.00 [0.00 to 0.82] | 0.00 [0.00 to 1.12] | 0.00 [0.00 to 2.76]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 0.15 [0.00 to 1.16] | 0.00 [0.00 to 0.88] | 0.00 [0.00 to 0.71]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 0.00 [0.00 to 0.96] | 0.00 [0.00 to 1.21] | 0.00 [0.00 to 3.16]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 0.00 [0.00 to 1.36] | 0.00 [0.00 to 0.78] | 0.00 [0.00 to 4.62]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.00 [0.00 to 2.09]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 1.50 [0.18 to 5.33] |  | 0.00 [0.00 to 11.22]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 0.61 [0.01 to 4.01] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 0.29 [0.00 to 2.20] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 0.00 [0.00 to 2.09] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 0.00 [0.00 to 2.22] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 5.60]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.89]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 6.60] | 0.00 [0.00 to 7.71]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 1.56]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 3.36] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 14.25]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 45.93]

130. Secondary Outcome: Cumulative Incidence Rates of Neurological Adverse Events Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: as for outcome 87
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.96]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 0.21 [0.07 to 0.50] | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 0.74]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 0.24 [0.13 to 0.43] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 0.25]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 0.23 [0.10 to 0.44] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 0.19]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 0.19 [0.08 to 0.38] | 0.24 [0.01 to 1.31] | 0.00 [0.00 to 0.19]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 0.19 [0.09 to 0.35] | 0.28 [0.02 to 1.16] | 0.04 [0.00 to 0.35]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 0.18 [0.08 to 0.33] | 0.19 [0.02 to 0.74] | 0.04 [0.00 to 0.32]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 0.17 [0.08 to 0.33] | 0.14 [0.01 to 0.57] | 0.04 [0.00 to 0.30]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 0.17 [0.08 to 0.32] | 0.11 [0.01 to 0.48] | 0.03 [0.00 to 0.20]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 0.17 [0.08 to 0.31] | 0.09 [0.00 to 0.44] | 0.03 [0.00 to 0.20]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 0.16 [0.08 to 0.31] | 0.08 [0.00 to 0.40] | 0.03 [0.00 to 0.19]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 0.16 [0.07 to 0.31] | 0.07 [0.00 to 0.38] | 0.03 [0.00 to 0.18]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 0.16 [0.07 to 0.30] | 0.07 [0.00 to 0.37] | 0.03 [0.00 to 0.18]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 1.50 [0.18 to 5.33] |  | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 1.01 [0.13 to 3.49] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 4.74]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 0.63 [0.08 to 2.26] | 0.00 [0.00 to 2.26] | 0.00 [0.00 to 3.18]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 0.49 [0.05 to 1.84] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 2.06]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 0.41 [0.04 to 1.57] | 0.00 [0.00 to 4.40] | 0.00 [0.00 to 1.52]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 0.38 [0.04 to 1.43] | 0.00 [0.00 to 2.64] | 0.00 [0.00 to 1.36]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 0.36 [0.04 to 1.35] | 0.00 [0.00 to 1.89] | 0.00 [0.00 to 1.21]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 0.34 [0.03 to 1.28] | 0.00 [0.00 to 1.48] | 0.00 [0.00 to 1.05]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 0.32 [0.03 to 1.21] | 0.00 [0.00 to 1.06] | 0.00 [0.00 to 0.63]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 0.30 [0.03 to 1.12] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.61]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 0.29 [0.03 to 1.09] | 0.21 [0.00 to 1.78] | 0.00 [0.00 to 0.59]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 0.28 [0.03 to 1.07] | 0.20 [0.00 to 1.69] | 0.00 [0.00 to 0.58]

131. Secondary Outcome: Weekly Incidence Rates of SAEs Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: SAEs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. The weekly incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Weekly vaccinated cohort for the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any SAEs in EHR (combining routine data collection and card-based ADR reporting system)within 7 days following vaccination with the seasonal influenza vaccine
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 36: number analyzed (Participants) | 1 | 1 | 59
  At risk, Week 36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 6.06]
  At risk, Week 37: number analyzed (Participants) | 2334 | 5 | 439
  At risk, Week 37 | 0.13 [0.02 to 0.39] | 0.00 [0.00 to 52.18] | 0.23 [0.00 to 1.85]
  At risk, Week 38: number analyzed (Participants) | 2591 | 7 | 498
  At risk, Week 38 | 0.19 [0.04 to 0.55] | 0.00 [0.00 to 40.96] | 0.40 [0.05 to 1.44]
  At risk, Week 39: number analyzed (Participants) | 3777 | 97 | 448
  At risk, Week 39 | 0.08 [0.01 to 0.24] | 0.00 [0.00 to 3.73] | 0.00 [0.00 to 0.82]
  At risk, Week 40: number analyzed (Participants) | 1882 | 313 | 522
  At risk, Week 40 | 0.16 [0.02 to 0.62] | 0.00 [0.00 to 2.10] | 0.19 [0.00 to 1.43]
  At risk, Week 41: number analyzed (Participants) | 1502 | 302 | 334
  At risk, Week 41 | 0.13 [0.01 to 0.62] | 0.00 [0.00 to 1.83] | 0.30 [0.00 to 2.28]
  At risk, Week 42: number analyzed (Participants) | 824 | 356 | 212
  At risk, Week 42 | 0.00 [0.00 to 0.45] | 0.28 [0.01 to 1.56] | 0.00 [0.00 to 1.72]
  At risk, Week 43: number analyzed (Participants) | 447 | 327 | 132
  At risk, Week 43 | 0.45 [0.01 to 2.83] | 0.00 [0.00 to 1.12] | 0.00 [0.00 to 2.76]
  At risk, Week 44: number analyzed (Participants) | 681 | 417 | 515
  At risk, Week 44 | 0.29 [0.00 to 2.07] | 0.24 [0.00 to 1.63] | 0.39 [0.00 to 3.12]
  At risk, Week 45: number analyzed (Participants) | 381 | 303 | 115
  At risk, Week 45 | 0.26 [0.00 to 1.93] | 0.33 [0.00 to 2.29] | 0.00 [0.00 to 3.16]
  At risk, Week 46: number analyzed (Participants) | 269 | 469 | 78
  At risk, Week 46 | 0.74 [0.09 to 2.66] | 0.00 [0.00 to 0.78] | 1.28 [0.01 to 8.31]
  At risk, Week 47: number analyzed (Participants) | 212 | 137 | 175
  At risk, Week 47 | 0.00 [0.00 to 1.72] | 0.00 [0.00 to 2.66] | 0.57 [0.00 to 4.84]
  At risk, Week 48: number analyzed (Participants) | 114 | 84 | 36
  At risk, Week 48 | 0.88 [0.01 to 5.39] | 0.00 [0.00 to 4.30] | 0.00 [0.00 to 9.74]
  Not at risk, Week 35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 37: number analyzed (Participants) | 133 | 0 | 31
  Not at risk, Week 37 | 0.00 [0.00 to 2.74] |  | 0.00 [0.00 to 11.22]
  Not at risk, Week 38: number analyzed (Participants) | 165 | 3 | 43
  Not at risk, Week 38 | 0.00 [0.00 to 2.21] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.22]
  Not at risk, Week 39: number analyzed (Participants) | 340 | 9 | 38
  Not at risk, Week 39 | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 33.63] | 0.00 [0.00 to 9.25]
  Not at risk, Week 40: number analyzed (Participants) | 175 | 29 | 63
  Not at risk, Week 40 | 0.57 [0.00 to 4.23] | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 5.69]
  Not at risk, Week 41: number analyzed (Participants) | 164 | 41 | 64
  Not at risk, Week 41 | 0.00 [0.00 to 2.22] | 0.00 [0.00 to 8.60] | 1.56 [0.01 to 10.47]
  Not at risk, Week 42: number analyzed (Participants) | 88 | 56 | 29
  Not at risk, Week 42 | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 6.38] | 0.00 [0.00 to 11.94]
  Not at risk, Week 43: number analyzed (Participants) | 52 | 55 | 32
  Not at risk, Week 43 | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.49] | 0.00 [0.00 to 10.89]
  Not at risk, Week 44: number analyzed (Participants) | 69 | 54 | 46
  Not at risk, Week 44 | 0.00 [0.00 to 5.21] | 0.00 [0.00 to 6.60] | 0.00 [0.00 to 7.71]
  Not at risk, Week 45: number analyzed (Participants) | 74 | 100 | 235
  Not at risk, Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 3.62] | 0.00 [0.00 to 1.56]
  Not at risk, Week 46: number analyzed (Participants) | 81 | 108 | 19
  Not at risk, Week 46 | 0.00 [0.00 to 4.45] | 0.00 [0.00 to 3.36] | 0.00 [0.00 to 17.65]
  Not at risk, Week 47: number analyzed (Participants) | 46 | 21 | 24
  Not at risk, Week 47 | 0.00 [0.00 to 7.71] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 14.25]
  Not at risk, Week 48: number analyzed (Participants) | 31 | 16 | 6
  Not at risk, Week 48 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 45.93]

132. Secondary Outcome: Cumulative Incidence Rates of SAEs Recorded in EHR, by Vaccine Group and UK CMO-specified Risk Status
Description: SAEs reported here are derived from 2 sources of data - ADR cards and AEI routinely collected from GPs. The cumulative incidence rates of SAEs expressed as the percentage of subjects, were estimated as follows:
  * The denominator was the number of subjects in the Cumulative vaccinated cohort up to the week of interest who were registered in EHR (combining routine data collection and card-based ADR reporting system)
  * The numerator was the number of subjects from the denominator who reported any SAEs in EHR (combining routine data collection and card-based ADR reporting system)
  Vaccination of the subjects happened between week 35 and week 48 of the year 2017
Time Frame: Within 7 days post vaccination
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
Number analyzed (Participants) | 16433 | 3310 | 4196
Percentage of subjects
  At risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 1
  At risk, Week 35-35 |  |  | 0.00 [0.00 to 97.50]
  At risk, Week 35-36: number analyzed (Participants) | 1 | 1 | 60
  At risk, Week 35-36 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 5.96]
  At risk, Week 35-37: number analyzed (Participants) | 2335 | 6 | 499
  At risk, Week 35-37 | 0.13 [0.02 to 0.39] | 0.00 [0.00 to 45.93] | 0.22 [0.00 to 1.61]
  At risk, Week 35-38: number analyzed (Participants) | 4926 | 13 | 997
  At risk, Week 35-38 | 0.16 [0.06 to 0.35] | 0.00 [0.00 to 24.71] | 0.30 [0.06 to 0.88]
  At risk, Week 35-39: number analyzed (Participants) | 8703 | 110 | 1445
  At risk, Week 35-39 | 0.13 [0.06 to 0.23] | 0.00 [0.00 to 3.30] | 0.21 [0.04 to 0.61]
  At risk, Week 35-40: number analyzed (Participants) | 10585 | 423 | 1967
  At risk, Week 35-40 | 0.13 [0.07 to 0.22] | 0.00 [0.00 to 0.87] | 0.20 [0.04 to 0.62]
  At risk, Week 35-41: number analyzed (Participants) | 12087 | 725 | 2301
  At risk, Week 35-41 | 0.13 [0.07 to 0.23] | 0.00 [0.00 to 0.51] | 0.22 [0.04 to 0.67]
  At risk, Week 35-42: number analyzed (Participants) | 12911 | 1081 | 2513
  At risk, Week 35-42 | 0.12 [0.07 to 0.21] | 0.09 [0.00 to 0.51] | 0.20 [0.04 to 0.59]
  At risk, Week 35-43: number analyzed (Participants) | 13358 | 1408 | 2645
  At risk, Week 35-43 | 0.13 [0.06 to 0.25] | 0.07 [0.00 to 0.40] | 0.19 [0.04 to 0.56]
  At risk, Week 35-44: number analyzed (Participants) | 14039 | 1825 | 3160
  At risk, Week 35-44 | 0.14 [0.06 to 0.29] | 0.08 [0.01 to 0.40] | 0.22 [0.05 to 0.62]
  At risk, Week 35-45: number analyzed (Participants) | 14420 | 2128 | 3275
  At risk, Week 35-45 | 0.15 [0.07 to 0.28] | 0.14 [0.02 to 0.52] | 0.21 [0.05 to 0.60]
  At risk, Week 35-46: number analyzed (Participants) | 14689 | 2597 | 3353
  At risk, Week 35-46 | 0.16 [0.07 to 0.31] | 0.12 [0.01 to 0.44] | 0.24 [0.07 to 0.59]
  At risk, Week 35-47: number analyzed (Participants) | 14901 | 2734 | 3528
  At risk, Week 35-47 | 0.15 [0.07 to 0.31] | 0.11 [0.01 to 0.42] | 0.26 [0.08 to 0.63]
  At risk, Week 35-48: number analyzed (Participants) | 15015 | 2818 | 3564
  At risk, Week 35-48 | 0.16 [0.06 to 0.33] | 0.07 [0.01 to 0.40] | 0.25 [0.07 to 0.62]
  Not at risk, Week 35-35: number analyzed (Participants) | 0 | 0 | 0
  Not at risk, Week 35-36: number analyzed (Participants) | 0 | 0 | 2
  Not at risk, Week 35-36 |  |  | 0.00 [0.00 to 84.19]
  Not at risk, Week 35-37: number analyzed (Participants) | 133 | 0 | 33
  Not at risk, Week 35-37 | 0.00 [0.00 to 2.74] |  | 0.00 [0.00 to 10.58]
  Not at risk, Week 35-38: number analyzed (Participants) | 298 | 3 | 76
  Not at risk, Week 35-38 | 0.00 [0.00 to 1.23] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 4.74]
  Not at risk, Week 35-39: number analyzed (Participants) | 638 | 12 | 114
  Not at risk, Week 35-39 | 0.00 [0.00 to 0.58] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.18]
  Not at risk, Week 35-40: number analyzed (Participants) | 813 | 41 | 177
  Not at risk, Week 35-40 | 0.12 [0.00 to 0.81] | 0.00 [0.00 to 8.60] | 0.00 [0.00 to 2.06]
  Not at risk, Week 35-41: number analyzed (Participants) | 977 | 82 | 241
  Not at risk, Week 35-41 | 0.10 [0.00 to 0.68] | 0.00 [0.00 to 4.40] | 0.41 [0.00 to 2.77]
  Not at risk, Week 35-42: number analyzed (Participants) | 1065 | 138 | 270
  Not at risk, Week 35-42 | 0.09 [0.00 to 0.62] | 0.00 [0.00 to 2.64] | 0.37 [0.00 to 2.41]
  Not at risk, Week 35-43: number analyzed (Participants) | 1117 | 193 | 302
  Not at risk, Week 35-43 | 0.09 [0.00 to 0.58] | 0.00 [0.00 to 1.89] | 0.33 [0.00 to 2.22]
  Not at risk, Week 35-44: number analyzed (Participants) | 1186 | 247 | 348
  Not at risk, Week 35-44 | 0.08 [0.00 to 0.55] | 0.00 [0.00 to 1.48] | 0.29 [0.00 to 1.97]
  Not at risk, Week 35-45: number analyzed (Participants) | 1260 | 347 | 583
  Not at risk, Week 35-45 | 0.08 [0.00 to 0.52] | 0.00 [0.00 to 1.06] | 0.17 [0.00 to 1.43]
  Not at risk, Week 35-46: number analyzed (Participants) | 1341 | 455 | 602
  Not at risk, Week 35-46 | 0.07 [0.00 to 0.49] | 0.00 [0.00 to 0.81] | 0.17 [0.00 to 1.38]
  Not at risk, Week 35-47: number analyzed (Participants) | 1387 | 476 | 626
  Not at risk, Week 35-47 | 0.07 [0.00 to 0.47] | 0.00 [0.00 to 1.78] | 0.16 [0.00 to 1.32]
  Not at risk, Week 35-48: number analyzed (Participants) | 1418 | 492 | 632
  Not at risk, Week 35-48 | 0.07 [0.00 to 0.46] | 0.00 [0.00 to 1.69] | 0.16 [0.00 to 1.30]

ADVERSE EVENTS:
Time Frame: AEs were collected during the 7 days post-vaccination period. Vaccination of the subjects happened between week 35 and week 48 of the year 2017 (i.e.: between 01 September 2017 and 30 November 2017)
Description: Medical coding was not performed according to MedDRA dictionary. AE codes were determined using an iterative ontological approach [de Lusignan, 2015; Liyanage, 2015] based on the EMA surveillance conditions of interest [EMA, 2016]. These conditions were aggregated under broad system categories to facilitate their reporting.
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Brand Group
All-Cause Mortality (participants affected / at risk) | 3/16433 | 0/3310 | 0/4196
Serious Adverse Events (participants affected / at risk) | 25/16433 | 3/3310 | 10/4196
Other Adverse Events (participants affected / at risk) | 1514/16433 | 133/3310 | 66/4196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccinated_Fluarix Tetra Group (N=16433) | Vaccinated_Non GSK Group (N=3310) | Vaccinated_Unknown Brand Group (N=4196)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1 — No MedDRA coding applied to this event
Accidental fall (Injury, poisoning and procedural complications) | 5 | 0 | 1 — No MedDRA coding applied to this event
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — No MedDRA coding applied to this event
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 — No MedDRA coding applied to this event
Blood transfusion (Surgical and medical procedures) | 1 | 0 | 0 — No MedDRA coding applied to this event
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 — No MedDRA coding applied to this event
Chest Pain (General disorders) | 3 | 1 | 0 — No MedDRA coding applied to this event
Chronic Ear Infection (Infections and infestations) | 0 | 0 | 1 — No MedDRA coding applied to this event
COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — No MedDRA coding applied to this event
Fracture of bone (Injury, poisoning and procedural complications) | 1 | 0 | 0 — No MedDRA coding applied to this event
Frail (General disorders) | 1 | 0 | 0 — No MedDRA coding applied to this event
Gynaecological (Reproductive system and breast disorders) | 1 | 0 | 0 — No MedDRA coding applied to this event
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 — No MedDRA coding applied to this event
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 — No MedDRA coding applied to this event
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 — No MedDRA coding applied to this event
Infection of Chronic Wound (Infections and infestations) | 1 | 0 | 1 — No MedDRA coding applied to this event
Pneumonia (Infections and infestations) | 0 | 0 | 1 — No MedDRA coding applied to this event
Self Harm (Psychiatric disorders) | 0 | 0 | 1 — No MedDRA coding applied to this event
Sensitivity Reaction (Immune system disorders) | 1 | 0 | 0 — No MedDRA coding applied to this event
Stroke (Nervous system disorders) | 1 | 0 | 0 — No MedDRA coding applied to this event
Unknown, non-causal (General disorders) | 5 | 0 | 1 — No MedDRA coding applied to this event
Viral gastroenteritis (Infections and infestations) | 0 | 0 | 1 — No MedDRA coding applied to this event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccinated_Fluarix Tetra Group (N=16433) | Vaccinated_Non GSK Group (N=3310) | Vaccinated_Unknown Brand Group (N=4196)
Fever/pyrexia (General disorders) | 70 | 11 | 2 — No MedDRA coding applied to this event
Local symptoms (i.e. local erythema) (General disorders) | 264 | 17 | 1 — No MedDRA coding applied to this event
Drowsiness (General disorders) | 107 | 7 | 0 — No MedDRA coding applied to this event
Fatigue (General disorders) | 249 | 10 | 3 — No MedDRA coding applied to this event
Headache (General disorders) | 271 | 23 | 6 — No MedDRA coding applied to this event
Irritability (General disorders) | 41 | 4 | 0 — No MedDRA coding applied to this event
Malaise (General disorders) | 3 | 3 | 0 — No MedDRA coding applied to this event
Conjunctivitis (Respiratory, thoracic and mediastinal disorders) | 53 | 3 | 5 — No MedDRA coding applied to this event
Coryza (Respiratory, thoracic and mediastinal disorders) | 172 | 12 | 2 — No MedDRA coding applied to this event
Cough (Respiratory, thoracic and mediastinal disorders) | 318 | 43 | 22 — No MedDRA coding applied to this event
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 0 | 0 — No MedDRA coding applied to this event
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 104 | 5 | 1 — No MedDRA coding applied to this event
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 139 | 10 | 3 — No MedDRA coding applied to this event
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 219 | 12 | 7 — No MedDRA coding applied to this event
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 366 | 28 | 3 — No MedDRA coding applied to this event
Wheezing (Respiratory, thoracic and mediastinal disorders) | 81 | 13 | 0 — No MedDRA coding applied to this event
Decreased appetite (Gastrointestinal disorders) | 73 | 6 | 0 — No MedDRA coding applied to this event
Diarrhoea (Gastrointestinal disorders) | 112 | 2 | 4 — No MedDRA coding applied to this event
Nausea (Gastrointestinal disorders) | 118 | 4 | 1 — No MedDRA coding applied to this event
Vomiting (Gastrointestinal disorders) | 30 | 2 | 2 — No MedDRA coding applied to this event
Anaphylactic reactions (Immune system disorders) | 45 | 7 | 1 — No MedDRA coding applied to this event
Facial oedema (Immune system disorders) | 8 | 0 | 0 — No MedDRA coding applied to this event
Hypersensitivity reactions (Immune system disorders) | 18 | 2 | 1 — No MedDRA coding applied to this event
Rash (Skin and subcutaneous tissue disorders) | 74 | 9 | 3 — No MedDRA coding applied to this event
Arthropathy (Musculoskeletal and connective tissue disorders) | 143 | 7 | 1 — No MedDRA coding applied to this event
Muscle aches / myalgia (Musculoskeletal and connective tissue disorders) | 454 | 18 | 15 — No MedDRA coding applied to this event
Bell's palsy (Nervous system disorders) | 1 | 0 | 0 — No MedDRA coding applied to this event
Peripheral tremor (Nervous system disorders) | 26 | 2 | 0 — No MedDRA coding applied to this event
Seizure / Febrile convulsions (Nervous system disorders) | 1 | 1 | 1 — No MedDRA coding applied to this event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03278067/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT03278067/SAP_001.pdf